Official Title: ISIS 304801-CS7 The APPROACH Open Label Study Volanesorsen (ISIS

304801) An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients With Familial Chylomicronemia Syndrome

(FCS)

NCT Number: NCT02658175

**Document Dates:** Protocol Amendment 10 - France: 01 May 2019

Protocol Amendment 9: 25 May 2018

Amendment 8: 10 April 2017

Amendment 7: 3 February 2017 Protocol Amendment 6: 16 September 2016 Protocol Protocol Amendment 5: 19 August 2016 Protocol

Protocol Amendment 4: 6 June 2016 Protocol Amendment 3: 9 May 2016

Amendment 2: 22 April 2016

Protocol Amendment 1: 2 February 2016 Protocol

Original Protocol: 28 August 2015





#### **Sponsor:**

Akcea Therapeutics 22 Boston Wharf Road, 9<sup>th</sup> Floor Boston, MA 02210

#### **Collaborator:**

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

## ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 10 - France - 01 May 2019** 

EudraCT No: 2015-003755-21

#### ISIS 304801-CS7

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

## An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

### Protocol Amendment 10 - France - 01 May 2019

#### **Protocol History:**

Original Protocol: 28 August 2015
Protocol Amendment 1: 2 February 2016
Protocol Amendment 2: 22 April 2016
Protocol Amendment 3: 9 May 2016
Protocol Amendment 4: 6 June 2016
Protocol Amendment 5: 19 August 2016
Protocol Amendment 6: 16 September 2016
Protocol Amendment 7: 3 February 2017
Protocol Amendment 8: 10 April 2017
Protocol Amendment 9: 25 May 2018

#### Approved by:

Akcea Therapeutics, Inc. 22 Boston Wharf Road, 9<sup>th</sup> Floor Boston, MA 02210 Telephone:



Akcea Therapeutics, Inc.

Protocol - France

Protocol Number: ISIS 304801-CS7

**Protocol Amendment 10 - France** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

## An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Akcea Therapeutics, Inc.

22 Boston Wharf Road, 9th Floor

Boston, MA 02210

Telephone:

**Key Sponsor Contact:** 

Akcea Therapeutics, Inc.

22 Boston Wharf Road, 9th Floor

Boston, MA 02210

Phone:

Email:

Collaborator: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010

Date: 01 May 2019

#### **Confidentiality Statement**

This document contains confidential information of Akcea Therapeutics, Inc. and Ionis Pharmaceuticals, Inc. that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Akcea Therapeutics, Inc. and Ionis Pharmaceuticals, Inc.

Protocol - France

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: An Open-Label Study of Volanesorsen Administered Subcutaneously to with Familial Chylomicronemia Syndrome (FCS) | | • |
| Amendment: | Amendment 10 - France | |
| Date: | 01 May 2019 | |
| Label Study of Volan<br>Syndrome (FCS)", Andescribed herein. I agree to comply with<br>Clinical Practice E6 ( | esorsen Administered Subcutaneo<br>mendment 10 – France, dated 01 I<br>th the International Conference on<br>R2). | the attached clinical protocol, entitled "An Open-<br>busly to Patients with Familial Chylomicronemia<br>May 2019, and agree to conduct the study as Harmonization Tripartite Guideline on Good |
| purpose other than the | | ained in this document will not be used for any ical investigation without the prior written consen. Inc. |
| Investigator's Signa | ture | _ |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

## TABLE OF CONTENTS

| | | Page |
|------------------|--------------------------------------|------|
| <b>PRO</b> T | FOCOL AMENDMENT | 10 |
| | TOCOL SYNOPSIS | |
| STUD | DY DESIGN AND TREATMENT SCHEMA | |
| 1. | OBJECTIVES | |
| 2. | BACKGROUND AND RATIONALE | |
| 2.1 | | |
| 2.2 | 1 | |
| 2.3 | | |
| | 2.3.1 Mechanism of Action | |
| | 2.3.2 Chemistry | |
| | 2.3.3 Preclinical Experience | |
| | 2.3.4 Clinical Experience | |
| 2.4 | | |
| 3. | EXPERIMENTAL PLAN | |
| 3.1 | | |
| 3.2 | | |
| 3.3 | | |
| 3.4 | 1 | |
| | 3.4.1 Qualification | |
| _ | 3.4.2 Treatment | |
| | Extended Treatment Period | |
| _ | 3.4.4 Post-Treatment Follow-Up | |
| 3.5 | • | |
| 3.6 | | |
| 4. | PATIENT ENROLLMENT | |
| 4.1 | | |
| 4.2 | | |
| <b>5.</b> 5.1 | PATIENT ELIGIBILITY | |
| 5.1 | | |
| 5.2<br><b>6.</b> | Exclusion Criteria | |
| 6.1 | | |
| | 5.1.1 Qualification | |
| | 5.1.2 Treatment Period | |
| | 5.1.2 Extended Treatment Period | |
| | 5.1.4 Pharmacokinetic (PK) Subgroup | |
| ( | 7.1.7 I narmacokinene (1 K) suogroup | 43 |

| | 6.1. | 5 Post-Treatment Follow-up | 45 |
|---|---|---|---|
| | 6.2 | Additional Study Assessments | 45 |
| | 6.2. | l Laboratory Assessments | 45 |
| | 6.2. | Physical Exams and Vital Signs | 46 |
| | 6 | .2.2.1 Eruptive Xanthoma | 46 |
| | 6 | .2.2.2 Lipemia Retinalis | 46 |
| | 6.2 | B Echocardiography | 46 |
| | 6.2. | 4 ECG | 46 |
| | 6.2.: | 5 MRI | 47 |
| | 6.2. | Quality of Life Assessments | 47 |
| | 6.2. | 7 Disease Symptom Diary | 47 |
| | 6.2. | 8 Diet Monitoring | 47 |
| | 6.2. | 9 Family History | 47 |
| | 6.2. | 10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2) | 47 |
| | 6.3 | Restriction on the Lifestyle of Patients. | 47 |
| | 6.3. | 1 Contraception Requirements | 47 |
| | 6.3. | 2 Other Requirements | 48 |
| <b>7.</b> | S | TUDY DRUG | 49 |
| | 7.1 | Volanesorsen Description | 49 |
| | 7.2 | Packaging and Labeling | 49 |
| | 7.3 | Study Drug Accountability | 49 |
| 8. | T | REATMENT OF PATIENTS | 49 |
| | 8.1 | Volanesorsen Administration | 49 |
| | 8.2 | Other Protocol-Required Drugs | 50 |
| | 8.3 | Other Protocol-Required Treatment Procedures | 50 |
| | 8.4 | Treatment Precautions | 50 |
| | 8.5 | Safety Monitoring Rules. | |
| | 8.5. | Safety Monitoring for Liver Chemistry Tests | 51 |
| | 8.5. | 2 Safety Monitoring for Platelet Count Results | 51 |
| | 8.5. | Safety Monitoring for Minor Bleeding Events | 53 |
| | 8.5.4 | Safety Monitoring for Constitutional Symptoms | 53 |
| | 8.5.: | Safety Monitoring for LDL-C Elevations | 53 |
| | 8.5. | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | 53 |
| | 8.5. | Safety Monitoring for Documented Severe Hypoglycemia | 54 |
| | 8.5. | Safety Monitoring for Hyperglycemia | 55 |
| | 8.5. | Acute Pancreatitis | 55 |
| | 8.6 | Stopping Rules | 56 |
| | 8.6. | Stopping Rules for Liver Chemistry Elevations | 56 |

| | 8.6.2 | Stopping Rules for Renal Function Test Results | 56 |
|---|---|---|---|
| | 8.6.3 | Stopping Rules for Platelet Count Results | 56 |
| | 8.7 A | Adjustment of Dose Frequency | 59 |
| | 8.8 D | Discontinuation of Study Treatment | 59 |
| | 8.8.1 | Follow-up Visits for Early Termination from Treatment Period | 60 |
| | 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Period | 60 |
| | 8.9 V | Vithdrawal of Patients from the Study | 60 |
| | 8.10 C | Concomitant Therapy and Procedures | 61 |
| | 8.10.1 | Concomitant Therapy | 61 |
| | 8.10.2 | Concomitant Procedures. | 61 |
| | 8.11 T | reatment Compliance | 62 |
| 9. | . SEI | RIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 62 |
| | 9.1 S | ponsor Review of Safety Information | 62 |
| | 9.2 R | legulatory Requirements | 62 |
| | 9.3 E | Definitions | 63 |
| | 9.3.1 | Adverse Event | 63 |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 63 |
| | 9.3.3 | Serious Adverse Event (SAE) | 63 |
| | 9.4 N | Monitoring and Recording Adverse Events | 64 |
| | 9.4.1 | Serious Adverse Events | 64 |
| | 9.4.2 | Non-Serious Adverse Events | 64 |
| | 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | 64 |
| | 9.4. | Relationship to the Study Drug | 64 |
| | 9.4. | 3.2 Severity | 65 |
| | 9.4. | 3.3 Action Taken with Volanesorsen | 65 |
| | 9.4. | 3.4 Treatment Given for Adverse Event | 65 |
| | 9.4. | Outcome of the Adverse Event | 65 |
| | 9.4.4 | Adjudication Committees | 66 |
| | 9.5 P | rocedures for Handling Special Situations | 66 |
| | 9.5.1 | Abnormalities of Laboratory Tests | 66 |
| | 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 66 |
| | 9.5.3 | Treatment Errors | 67 |
| | 9.5.4 | Contraception and Pregnancy | 67 |
| 1( | <b>0. ST</b> / | ATISTICAL CONSIDERATIONS | 68 |
| | 10.1 S | tudy Endpoints | 68 |
| | 10.1.1 | Efficacy Endpoints | 68 |
| | 10.1.2 | Safety Endpoints | 68 |
| | 10.2 S | ample Size | 68 |

| 10.3 | Populations | 69 |
|---|---|---|
| 10.4 | Definition of Baseline. | 69 |
| 10.5 | Interim Analysis | 69 |
| 10.6 | Planned Methods of Analysis | 69 |
| 10.6 | 5.1 Demographic and Baseline Characteristics | 70 |
| 10.6 | 5.2 Safety Analysis | 70 |
| 10.6 | 5.3 Efficacy Analysis | 70 |
| 10.6 | 5.4 Pharmacokinetic and Immunogenicity Analysis | 71 |
| 1 | 0.6.4.1 Pharmacokinetic Analysis | 71 |
| 1 | 0.6.4.2 Immunogenicity Analysis | 71 |
| 11. I | NVESTIGATOR'S REGULATORY OBLIGATIONS | 72 |
| 11.1 | Informed Consent | 72 |
| 11.2 | Ethical Conduct of the Study | 72 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 72 |
| 11.4 | Patient Confidentiality | 73 |
| <b>12.</b> A | ADMINISTRATIVE AND LEGAL OBLIGATIONS | 73 |
| 12.1 | Protocol Amendments | 73 |
| 12.2 | Study Termination | 73 |
| 12.3 | Study Documentation and Storage | 73 |
| 12.4 | Study Monitoring | 74 |
| 12.5 | Language | 74 |
| 12.6 | Compensation for Injury | 75 |
| 13. F | REFERENCES | 76 |
| <b>14.</b> A | APPENDICES | 79 |
| Appen | dix A Schedule of Procedures | 79 |
| Appen | dix B List of Laboratory Analytes | 90 |
| Appen | dix C Pharmacokinetic Sampling Schedule | 92 |
| Appen | dix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities | 95 |
| | TABLE OF TABLES | |
| T 11 1 | W. L. (IGIG 204001) Cl. (C. C. C | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 49 |
| Table 2 | Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal ( $\times$ 2) or $< 100,000/\text{mm}^3$ ( $\times$ 1)* | 52 |
| Table 3 | Actions in Patients with Low Platelet Count | |
| Table 4 | Expected Event for the Protocol Defined Population by Preferred Term and the | 50 |
| 14010 1 | Expected Incidence | 62 |

## **TABLE OF FIGURES**

| | | Page |
|---|---|---|
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 33 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volanesorsen is shown | 35 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 37 |

#### PROTOCOL AMENDMENT

**Protocol Number:** ISIS 304801-CS7

Protocol Title: An Open-Label Study of Volanesorsen Administered Subcutaneously to

Patients with Familial Chylomicronemia Syndrome (FCS)

**Amendment Number:** 10 - France **Amendment Date:** 01 May 2019

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 9 - France dated 25 May 2018:

• To add an up to 52 weeks of additional treatment to the Extended Treatment Period, to clarify the option for patients to receive a volanesorsen dose reduction of 300 mg every two weeks, to clarify discontinuation of patients from the treatment period who are on a dose pause for ≥ 3 months, and to remove the references to landmark visits (if patient stops treatment then they enter the follow-up period).

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Section 2.3.4<br>Clinical<br>Experience | Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo). The clinical experience with volanesorsen includes clinical trials in healthy subjects, patients with hypertriglyceridemia, FCS, or familial partial lipodystrophy. Overall, 431 patients and healthy volunteers have taken part in the clinical development program, of whom 325 have received at least 1 dose of volanesorsen. Ninety-five (95) patients with FCS have been enrolled in studies, all showing clinically meaningful reductions in plasma triglyceride. Patients with FCS continue on treatment in the open-label extension (OLE) and triglyceride reductions persist at similar levels as reported in earlier studies. In the completed Phase 1 and Phase 2 studies, volanesorsen was well-tolerated and demonstrated a favorable safety profile. There was no clinical or laboratory evidence of drug-drug interactions despite many patients in the Phase 2 clinical trials receiving | Update language regarding clinical experience in Phase 1 and 2 studies and incidence of AEs in completed Phase 3 studies and update to language regarding safety risks of Study Drug. |

concomitant medications that are known to be associated with elevations in hepatic enzymes, such as fibrates and statins. There were no volanesorsen-associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). There was a reduction (mean reduction < 30%) in platelets in volanesorsen vs. placebo with mean nadirs for all doses remaining above the lower limit of normal (LLN). The most frequently reported adverse events (AEs) were mild, non-progressive events at the injection site. In Phase 2, a single serious adverse event (SAE) of secondary serum sickness-like reaction was reported as related to Study Drug.

...

In the completed pooled Phase 3 studies (ISIS 304801-CS6 (hereafter referred to as CS6) and ISIS 304801-CS16 (hereafter referred to as CS16), the most common AEs associated with volanesorsen administration were tolerability at the injection site and platelet reductions. The majority of the injection site AEs were mild, none were severe, and the incidence appeared to decrease over time. No deaths have been associated with volanesorsen treatment to date. No cardiac toxicity was associated with volanesorsen treatment. There were no abnormal QTc findings and no study-drug related adjudicated major adverse cardiac events (MACE). There is no evident association between volanesorsen treatment and changes in renal or liver functions. In clinical studies conducted to date volanesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

The safety profile of volanesorsen has been welldescribed in this development program, which has identified 3 safety risks: thrombocytopenia (an identified risk), constitutional symptoms (flu-like reactions and influenza-like illness), and injection site reactions (a tolerability signal). Spontaneous, mild to severe thrombocytopenia has been described in the FCS patient population (Gaudet et al. 2017) but is increased by treatment with volanesorsen. Less frequent and less pronounced platelet declines were also observed with volanesorsen treatment in the hypertriglyceridemic (HTG) population of CS16. When fully complied with, frequent monitoring for this effect and appropriate dose adjustments have been successful both in preventing and promptly detecting the occurrence of severe platelet declines and often in retaining patients on treatment. In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine. proteinuria) or hepatic systems (alanine

| | aminotransferase [ALT], aspartate aminotransferase | |
|---|---|---|
| | [AST], bilirubin). In Phase 2 studies, there was a mild | |
| | decrease of platelet count associated with volanesorsen | |
| | administration that recovered in the post-treatment | |
| | period and was not associated with platelet-related | |
| | adverse events (AEs). In the blinded ongoing clinical | |
| | trials of ISIS 304801, 2 patients of 142 dosed (as of | |
| | February 29, 2016) had a decrease in platelet count to | |
| | less than 50,000/mm3 in the absence of major bleeding | |
| | or clinically relevant non major bleeding and had Study | |
| | Drug paused as per the monitoring and stopping rules | |
| | for platelet counts (Section 8.6.3). Platelet counts | |
| | recovered following suspension of dosing. | |
| | The most frequently observed AEs with volanesorsen | |
| | were local reactions at the injection site. Local | |
| | cutaneous reactions at the injection site defined as | |
| | those events presenting as either pain, tenderness, | |
| | erythema, pruritus or swelling occurring on the day of | |
| | injection and persisting for at least 2 days were | |
| | infrequent (~15% of injections), were almost always | |
| | mild, resolved spontaneously, were non progressive, | |
| | and were not associated with systemic sequelae. | |
| | · | |
| Section 2.4 | The dose and schedule selected for this study is 300 | Language added to clarify dose |
| Rationale for | mg per week for 52 weeks, with the option of continuing | reductions as 300 mg every 2 |
| Dose and | dosingtreatment for up to an additional 52104 weeks. | weeks according to patient's |
| Schedule of | The dose of 300 mg per week and dose reduction of | tolerability on the 300 mg weekly |
| Administration | 300 mg every 2 weeks (delivered as a single 300 mg | dose, given similar extents of |
| | dose) are is supported by both the cumulative | triglyceride lowering anticipated |
| | nonclinical data available to date and the Phase 2 clinical data. | based on population |
| | Cililical data. | pharmacokinetic/<br>pharmacodynamic model-based |
| | | simulations. |
| | No and No aliminal finalisms are an extraordism of the | Simulations. |
| | No nonNon clinical findings were not considered to be | |
| | related to the pharmacologic inhibition of apoC-III. | |
| | l | |
| | In addition to the nonclinical and clinical experience of | Undated to reflect data presented |
| | volanesorsen, the dose and schedule of administration | Updated to reflect data presented in source listed. |
| | is supported by the preclinical and clinical safety | iii soulce listeu. |
| | experience of several other 2' MOE-modified ASOs that | |
| | have been <del>safely</del> administered intravenously and | |
| | subcutaneously in multiple clinical studies at doses up | |
| | to <del>1000</del> <u>1200</u> mg and for treatment durations that | |
| | exceed 24 months (Santos et al. 2015). | |
| Oursenais: Otrod | Synopsis | Edited length of Extended |
| Synopsis: Study | • | Treatment Period to allow patients |
| Design, Study | All patients will receive volanesorsen 300 mg once per | in France to continue to receive |
| Visit Schedule | week for 52 weeks. Dietary counseling will be | study drug until commercialization |
| and Procedures | reinforced at intervals throughout the treatment and | of product. |
| | follow-up period. Following the Week 52 visit, patients | 5. p. 6446. |
| | will have the option to continue dosing treatment for up | |
| | to an additional <del>52</del> 104 weeks for a total of <u>up to 156</u> | |
| I | weeks of <del>dosing <u>treatment</u>. Patients not continuing</del> | |

| | dosing-treatment will enter a 26-week post-treatment follow-up period. | |
|---|---|---|
| | Section 3.1 | |
| Section 3.1<br>Study Design | Following the Week 52 visit, patients will have the option to continue dosingtreatment for up to an additional 52104 weeks for a total of 104up to 156 weeks of dosing treatment. Patients not to-continuing dosing treatment will enter a 26-week post-treatment follow-up period. | |
| | Section6.1.3 | |
| Section 6.1.3<br>Extended<br>Treatment Period | After completion of the Week 52 visit assessments, patients will have the option of continuing desing for up to an additional 52 weeks treatment for up to an additional 104 weeks. For patients that have entered the Extended Treatment Periods, study participation will be up to an additional 104 weeks or until commercialization of product, whichever is sooner. | |
| | During the extended treatment period, patients will have assessments and procedures done during Weeks 54-104156 as per the Schedule of Procedures in Appendix A | |
| Section 3.4.3 Extended Treatment Period | Following the Week 52 visit, patients will have the option to continue dosing-treatment for up to an additional 52104 weeks. Patients not to continuing dosing-treatment will enter a 26-week post-treatment follow-up period. For patients that have entered the Extended Treatment Periods, study participation will be up to an additional 104 weeks or until commercialization of product, whichever is sooner | Edited length of Extended Treatment Period to allow patients in France to continue to receive study drug until commercialization of product. |
| Section 3.4.4 | Section 3.4.4 | Added details of follow-up period |
| Post-Treatment<br>Follow-Up | The post-treatment follow-up period is at least 26 weeks and consists of at least 9 Study Center visits. For patients not continuing into the 52-week extended treatment period, the post-treatment follow-up period visits will be conducted on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse). For patients who have entered the first 52-week extended treatment period, but will not continue into the second 52-weeks of the extended treatment period, the post-treatment follow-up period visits will be conducted on Weeks 105, 106, 107, 108, 109, 110, 117, 123 and 130 (Weeks 105, 106, 107, 108, 109, 110 and 123 may be conducted by a home healthcare nurse). | for the first and second Extended Treatment Periods. |
| | For patients who have entered the second 52-week extended treatment period, the post-treatment follow-up period visits will be on Weeks 157, 158, 159, 160, 161, 162, 169, 175 and 182 (Weeks 157, 158, 159, 160, 161, 162 and 175 may be conducted by a home healthcare nurse). | |
| | Section 6.1.5 | |

| Section 6.1.5 | After completion of the Week 52 visit assessments, | |
|---|---|---|
| Post-Treatment | patients will have the option of continuing <del>dosing</del> | |
| Follow-Up | treatment for up to an additional <del>52</del> 104 weeks as | |
| | described in Section 6.1.3. Patients not continuing | |
| | dosing-treatment will enter the 26-week post treatment | |
| | follow-up. The 26For patients not continuing into the | |
| | 52-week extended treatment period, the 26-week post- | |
| | treatment follow-up period consists of at least 9 Study | |
| | Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, | |
| | and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be | |
| | conducted by a home healthcare nurse). <del>An additional</del> | |
| | <del>26</del> | |
| | For patients who enter the first 52-week post-treatment | |
| | follow-up occurs afterextended treatment period, but will | |
| | not continue into the second 52-weeks of the extended | |
| | treatment period with at least 9 Study Center, the post- | |
| | treatment follow-up period visits will be conducted on | |
| | Weeks 105, 106, 107, 108, 109, 110, 117, 118, 123 and | |
| | <del>125</del> 130 (Weeks 105, 106, 107, 108, 109, 110 and | |
| | 118123 may be conducted by a home healthcare | |
| | nurse). | |
| | nares). | |
| | For patients who enter the second 52-week extended | |
| | treatment period, the post-treatment follow-up period | |
| | visits will be on Weeks 157, 158, 159, 160, 161, 162, | |
| | 169, 175 and 182 (Weeks 157, 158, 159, 160, 161, 162 | |
| | and 175 may be conducted by a home healthcare | |
| | nurse). | |
| | <del></del> | Everations to inclusion or |
| Section 5.2 | 14. Use of any of the following: | Exceptions to inclusion or |
| Exclusion Criteria | | exclusion criteria will not be |
| Synopsis, Study | | granted. |
| Population | c. Systemic corticosteroids or anabolic | |
| | steroids within 6 weeks prior to | |
| - | · | |
| | Qualification <del>unless approved by the</del> | |
| | · | |
| | Qualification <del>unless approved by the</del> | |
| | Qualification <del>unless approved by the</del><br><del>Sponsor Medical Monitor</del><br> | |
| | Qualification <del>unless approved by the Sponsor Medical Monitor</del> 16. Known hypersensitivity to any of the excipients | |
| | Qualification <del>unless approved by the</del><br><del>Sponsor Medical Monitor</del><br> | |
| Section 6.1.3 | Qualification <del>unless approved by the Sponsor Medical Monitor</del> 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 <del>or placebo</del> ) | Modified to indicate that blood |
| Section 6.1.3 | Qualification <del>unless approved by the Sponsor Medical Monitor</del> 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 <del>or placebo</del> ) Blood sampling <u>will be conducted weekly</u> at Weeks 53, | Modified to indicate that blood |
| Extended | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, | sampling will occur weekly for |
| | Qualification unless approved by the Spensor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, | sampling will occur weekly for increased clarity and to include an |
| Extended | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of |
| Extended | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home | sampling will occur weekly for increased clarity and to include an |
| Extended | Qualification unless approved by the Spensor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. |
| Extended | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory |
| Extended Treatment Period Section 6.2.1 | Qualification unless approved by the Spensor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. |
| Extended Treatment Period Section 6.2.1 Laboratory | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory |
| Extended Treatment Period Section 6.2.1 Laboratory Assessments | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory assessments permitted for safety |
| Extended Treatment Period Section 6.2.1 Laboratory Assessments Section 8.5.4 | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory assessments permitted for safety |
| Section 6.2.1 Laboratory Assessments Section 8.5.4 Safety Monitoring | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), high- | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory assessments permitted for safety |
| Section 6.2.1 Laboratory Assessments Section 8.5.4 Safety Monitoring for Constitutional | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), highsensitivity C-reactive protein (hsCRP) and for cytokine | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory assessments permitted for safety |
| Section 6.2.1 Laboratory Assessments Section 8.5.4 Safety Monitoring | Qualification unless approved by the Sponsor Medical Monitor 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) Blood sampling will be conducted weekly at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), high- | sampling will occur weekly for increased clarity and to include an up to 104 additional weeks of extended treatment. To add additional laboratory assessments permitted for safety |

| Section 6.2.4<br>ECG<br>Section 6.2.6 | Patients in the Extended Treatment Periods will have ECGs performed in triplicate at Weeks 76 and, 104. and 130. Triplicate ECGs will be performed at Weeks 13 and 26 of each post-treatment follow-up period. Should the patient enter the extended treatment | To detail additional ECG assessments in the post-treatment follow-up period. To detail additional QoL |
|---|---|---|
| Quality of Life<br>Assessments | periods. Aadditional Quality of Life Questionnaires will be collected at Weeks 1713 and 130 26 of each should the patient enter the extended treatment period post-treatment follow- up period. | assessments in the post-treatment follow-up period. |
| Section 8.1<br>Volanesorsen<br>Administration | For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will continue to receive study drug as a single 300 mg/1.5 mL injection once-weekly for Weeks 53-156104 receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients on dose reduction will receive 300 mg/1.5 mL injections every 2 weeks entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen. Patients should receive 1 dose per week, unless on a dose reduction of 300 mg every 2 weeks, with weeks always defined relative to Study Day 1. | Added language clarifying details of dose reduction option as 300 mg every 2 weeks. |
| Section 8.5.2<br>Safety Monitoring<br>for Platelet Count<br>Results | Monitor every 1 week unless otherwise specified. In addition, platelet function may be evaluated at any time during the study by aggregometry, using an approved point-of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers. Due to the 1 to 32-year study duration it is anticipated that patients may undertake travel including vacations, | Additional point-of-care platelet function testing may be conducted on patients at participating study centers. Included an additional blood draw to assess platelet count prior to any travel that would result in |
| | which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing treatment where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a platelet count drawn within 3-5 days prior to departure and with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing treatment. | missing a weekly monitoring visit. |

| | | | e monitored as per the | |
|---|---|---|---|---|
| | | ministration is resu | | |
| Section 8.6.3<br>Stopping Rules | Table 3 Actions in Patients with Low Platelet Count | | | To provide clarification to the platelet safety monitoring rules, |
| for Platelet Count<br>Results | Platelet<br>Count on<br>Rx | Drug Dose | Monitoring | including dose reduction options. |
| | | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing treatment. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified In addition, platelet function may be evaluated during the study by aggregometry, using an approved point- of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers. Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed. Obtain additional lab tests (Table 2) if 2 occurrences (consecutive or non-consecutive) of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count 140K - > 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as | |

| I | | | |
|---|---|---|---|
| | | | per Investigator discretion. |
| | > 100K/mm <sup>3</sup> | Once Wweekly 300 mg Study Drug administration | uisui euuii. |
| | 100K/mm <sup>3</sup> -<br>> 75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks. | |
| | 75K/mm <sup>3</sup> - > 50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks, then permanently discontinue Study Drug, otherwise dose pause. If dose pause is ≥ 3 months then patient must discontinue treatment and enter the follow up period. When platelet count returns to > 100K/mm³ restart-dosing treatment at dose frequency of 300 mg every 2 weeks only if approved by in consultation with the Sponsor Medical Monitor | Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| | ≤ 50K/mm³ or a rate of decline ≥ 50% between two consecutive assessment s, irrespective of the | Permanently discontinue Study Drug and the patient will enter the follow up period. | Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are |

Protocol - France

Amendment 10 01 May 2019

| | | monitor every 1 week Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management Steroids recommended*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline. Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy Discontinue | |
|---|---|---|---|
| | | 1 | |
| Section 8.7<br>Adjustment of<br>Dose Frequency | Other dose adjustments, including and/or decreasing the dose or dose and a 300 mg every 2 weeks will be allowed tolerability. Any proposed adjust schedule must be discussed with Study Medical Monitor prior to initially adjustments in the treatment scheme and the study line of the s | g dose interruptions, use frequency to owed for safety and ment to treatment use, and approved by, the tiation. Up to 2 edule may be allowed. response to AEs after Medical Monitor is used for ≥ 3 months, he ontinued treatment | Clarification of dose reduction option to reduced dose frequency to allow for safety and tolerability Discontinuation of patients from the study who have been on dose pause and off study drug for >3 months. |

| Section 8.8 Discontinuation of Study Treatment | A patient must permanently discontinue study treatment for any of the following: •The patient is dose-paused for ≥ 3 months. | Added new treatment discontinuation criterion consistent with other protocol changes. |
|---|---|---|
| Section 8.8.1 Follow-up Visits for Early Termination from Treatment Period | Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug. in addition to the applicable landmark visits. A patient who discontinues early from treatment with stable platelet counts above the LLN at the time of treatment discontinuation will have platelet counts drawn every 2 weeks after discontinuing Study Drug. A subsequent platelet count should then be taken after an additional 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. | Removal of language around landmark visits as patients who stop treatment now enter a post-treatment follow-up period Provides guidance for platelet monitoring in the post-treatment follow-up period. |
| Section 8.9 Withdrawal of Patient from the Study Section 8.10.2 | Other reasons for withdrawal of patients from the study might include: • At the discretion of the Investigator for medical reasons • At the discretion of the Investigator or Sponsor for noncompliance • Significant protocol deviation • Commercialization of product Section 8.10.2 | Added commercialization of product as an additional reason for withdrawal from study. Updated to include follow-up |
| Concomitant<br>Procedures | A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit. | period for the first and second<br>Extended Treatment Periods. |

| Section 9.4.1<br>Serious Adverse<br>Events | Section 9.4.1 The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit. | |
|---|---|---|
| Section 9.4.2<br>Non-Serious<br>Adverse Events | Section 9.4.2 The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit. | |
| Section 13<br>REFERENCES | Gaudet D, Baass A, Tremblay K, et al. Natural History (up to 15 years) of Platelet Count in 84 Patients with Familial Hyperchylomicronemia Due to Lipoprotein Lipase Deficiency. Journal of Clinical Lipidology 2017; 11(3): 797-798. | Addition of reference |
| Section 14. APPENDICES | Appendix A Schedule of Procedures The following footnotes have been added to the tables for both the qualification through treatment period and the post-treatment follow-up period. g Genetic testing can be conducted for study Qualification (Group 2 ISIS 304801-CS16 roll over patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing. A blood sample for potential gene sequencing may be collected at timepoints other than Screening or Qualification Visits. | Clarification that blood sampling for gene sequencing may occur during the study. |
| | The table for the first 52-week extended treatment period and post-treatment follow-up period have been defined and additional tables added for the second 52-weekextended treatment period and post-treatment follow-up period. | Added an additional year of extended treatment |
| | Also added platelet function analysis to the first extended treatment period. With Footnote <u>g May be done</u> | Indication that platelet function may be assessed. |
| Section 14. APPENDICES | Appendix B List of Laboratory Analytes Platelet Function Platelet aggregation <sup>3</sup> Platelet function <sup>5</sup> | Addition of laboratory analyte to measure platelet function. |
| | Footnote <u>5</u> : May be done using a point-of-care device <u>on site.</u> | |

| Section 14. APPENDICES | Appendix C Pharmacokinetic Sampling Schedule | Addition of PK sampling timepoints for additional year of |
|---|---|---|
| | Expanded PK Sampling Schedule to include timepoint for the First and Second 52-Week Extended Treatment Periods. | extended treatment. |

## PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of treatment and extended treatment with volanesorsen in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option to continue treatment for up to an additional 104 weeks for a total of up to 156 weeks of treatment. Patients not continuing treatment will enter a 26-week post-treatment follow-up period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent<br/>serum (a creamy top layer after ultracentrifugation of a fasting blood<br/>sample) or documentation of fasting TG measurement ≥ 880 mg/dL<br/>(10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: </li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-causing<br/>genes (such as lipoprotein lipase [LPL], apoC-II, GPIHBP1, or lipase<br/>maturation factor [LMF1])</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical<br/>history. Note: testing of LPL activity should not be performed to<br/>confirm eligibility for the study</li> </ul> |
| | c. Fasting TG $\geq$ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study |

#### Study Population Continued

#### Inclusion Criteria: Continued

- Able and willing to participate in a 78-week study5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and follicle stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **Exclusion Criteria:**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of glucagon-like peptide-1 (GLP-1) agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification

#### **Study Population Continued**

Exclusion Criteria: Continued

- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
    - Estimated creatinine clearance calculated according to the formula
      of Cockcroft and Gault < 50 mL/min (MDRD or
      CKD-EPI formulas can be used instead of Cockcroft-Gault for
      estimation of glomerular filtration rate (GFR) in patients with low
      body weight after discussion with Sponsor Medical Monitor)</li>
  - c. Cardiac Troponin I > ULN at Qualification
  - d. LDL-C > 130 mg/dL at Qualification
  - Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria: Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and over-the-counter [OTC]), or<br>fibrates unless on a stable dose for at least 3 months prior to Qualification<br>and dose and regimen expected to remain constant during the treatment<br>period. Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>Qualification</li> </ul> |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification |
| | d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study |
| | e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to Qualification |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban)<br>unless on a stable dose for at least 4 weeks prior to Qualification and regular<br>clinical monitoring is performed |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | <ul> <li>Plasma apheresis within 4 weeks prior to Qualification or planned during the<br/>study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to Qualification<br/>(Occasional or intermittent use of over-the-counter medications will be<br/>allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule<br>Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the Sponsor).</li> <li>Please refer to Section 4.1 and Appendix A</li> </ul> |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | <ul> <li>Option to participate in an extended treatment period (up to an<br/>additional 104 weeks)</li> </ul> |
| | o A 26-week post-treatment follow-up period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), electrocardiograms (ECGs), echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option to continue treatment for up to an additional 104 weeks. Patients not to continuing treatment will enter a 26-week post-treatment follow-up period. |
| Safety and Tolerability Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |

| Planned Analyses | Safety Endpoints: |
|---|---|
| | Adverse events including adjudicated events of acute pancreatitis and MACE |
| | Vital signs and weight |
| | Physical examinations |
| | Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) |
| | Echocardiography |
| | • ECGs |
| | Use of concomitant medications |
| | • MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high- density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Change in blood viscosity (may be evaluated) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Akcea Therapeutics, Inc. |
| Collaborator | Ionis Pharmaceuticals, Inc. |

#### STUDY DESIGN AND TREATMENT SCHEMA



# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 10 Protocol - France 01 May 2019

## STUDY GLOSSARY

| Abbreviation/Acronym | <u>Definition</u> |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| ароЕ | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| FSH | follicle stimulating hormone |
| FPG | fasting plasma glucose |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |

#### ISIS 304801-CS7 **CONFIDENTIAL** Amendment 10 01 May 2019

Protocol - France

**Definition** Abbreviation/Acronym

**Independent Ethics Committee IEC** 

IM immunogenicity

ISIS 304801-CS6 and ISIS 304801-CS16 **Index Studies** 

International Normalized Ratio **INR** Institutional Review Board **IRB** 

Interactive Voice/Web-Response System **IXRS** 

LDL Low-Density Lipoprotein LLN Lower Limit of Normal

Low-Density Lipoprotein-Cholesterol LDL-C

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

**MACE** Major Acute Cardiovascular Event

MedDRA Medical Dictionary for Regulatory Activities

**MOE** 2'-O-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid **NCS** not clinically-significant

**NOAEL** No-Observed-Adverse-Effect Level

Non-High-Density Lipoprotein-Cholesterol non-HDL-C

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

**SMPG** self-monitored plasma glucose

suspected unexpected serious adverse reaction **SUSAR** 

T2DM type 2 diabetes mellitus

time to maximal concentration  $T_{\text{max}}$ 

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

**TRL** Triglyceride-Rich Lipoproteins

ULN upper limit of normal

|-------------------|--------------|
| Protocol - France | 01 May 2019 |

| Abbreviation/Acronym | <b>Definition</b> |
|----------------------|------------------------------------------|
| VLDL | Very-Low-Density Lipoprotein |
| VLDL-C | Very-Low-Density Lipoprotein-Cholesterol |
| VLDL-TG | Lipoprotein-Triglyceride |
| WMA | World Medical Association |

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of treatment and extended treatment with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V (APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored high-density lipoprotein (HDL)-binding protein 1 (GPIHBP1), a

Amendment 10

capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apolipoprotein E (apoE)-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL,

apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower low-density lipoprotein-cholesterol (LDL-C), increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volanesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing. The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volunesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volanesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown.

### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and
mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

The clinical experience with volanesorsen includes clinical trials in healthy subjects, patients with hypertriglyceridemia, FCS, or familial partial lipodystrophy. Overall, 431 patients and healthy volunteers have taken part in the clinical development program, of whom 325 have received at least 1 dose of volanesorsen. Ninety-five (95) patients with FCS have been enrolled in studies, all showing clinically meaningful reductions in plasma triglyceride. Patients with FCS continue on treatment in the open-label extension (OLE) and triglyceride reductions persist at similar levels as reported in earlier studies.

In the completed Phase 1 and Phase 2 studies, volanesorsen was well-tolerated and demonstrated a favorable safety profile. There was no clinical or laboratory evidence of drug-drug interactions despite many patients in the Phase 2 clinical trials receiving concomitant medications that are known to be associated with elevations in hepatic enzymes, such as fibrates and statins. There were no volanesorsen-associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). There

was a reduction (mean reduction < 30%) in platelets in volunesorsen vs. placebo with mean nadirs for all doses remaining above the lower limit of normal (LLN). The most frequently reported adverse events (AEs) were mild, non-progressive events at the injection site. In Phase 2, a single serious adverse event (SAE) of secondary serum sickness-like reaction was reported as related to Study Drug.

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM. In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the treatment period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In the completed pooled Phase 3 studies (ISIS 304801-CS6 (hereafter referred to as CS6) and ISIS 304801-CS16 (hereafter referred to as CS16), the most common AEs associated with volunesorsen administration were tolerability at the injection site and platelet reductions. The majority of the injection site AEs were mild, none were severe, and the incidence appeared to decrease over time. No deaths have been associated with volanesorsen treatment to date. No cardiac toxicity was associated with volanesorsen treatment. There were no abnormal QTc findings and no study-drug related adjudicated major adverse cardiac events (MACE). There is no evident association between volunesorsen treatment and changes in renal or liver functions.

The safety profile of volanesorsen has been well-described in this development program, which has identified 3 safety risks: thrombocytopenia (an identified risk), constitutional symptoms (flu-like reactions and influenza-like illness), and injection site reactions (a tolerability signal). Spontaneous, mild-to-severe thrombocytopenia has been described in the FCS patient population (Gaudet et al. 2017) but is increased by treatment with volanesorsen. Less frequent and less pronounced platelet declines were also observed with volanesorsen treatment in the hypertriglyceridemic (HTG) population of CS16. When fully complied with, frequent monitoring for this effect and appropriate dose adjustments have been successful both in preventing and promptly detecting the occurrence of severe platelet declines and often in retaining patients on treatment.

### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks, with the option of continuing treatment for up to an additional 104 weeks. The dose of 300 mg per week and dose reduction of 300 mg every 2 weeks (delivered as a single 300 mg dose) are supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. Non clinical findings were not considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been administered intravenously and subcutaneously in multiple clinical studies at doses up to 1200 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

### 3. EXPERIMENTAL PLAN

### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Up to approximately 70 patients will receive 300 mg once weekly volunesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option to continue treatment for up to an additional 104 weeks for a total of up to 156 weeks of treatment. Patients not continuing treatment will enter a 26-week post-treatment follow-up period.

# 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

# 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Qualification

A qualification period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volanesorsen is administered by subcutaneous (SC) injection once weekly.

#### 3.4.3 Extended Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of continuing treatment for up to an additional 104 weeks. Patients not continuing treatment will enter the 26-week post-treatment follow-up. For patients that have entered the Extended Treatment Periods, study participation will be up to an additional 104 weeks or until commercialization of product, whichever is sooner.

# 3.4.4 Post-Treatment Follow-Up

The post-treatment follow-up period is at least 26 weeks and consists of at least 9 Study Center visits. For patients not continuing into the 52-week extended treatment period, the post-treatment follow-up period visits will be conducted on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse).

For patients who have entered the first 52-week extended treatment period, but will not continue into the second 52-weeks of the extended treatment period, the post-treatment follow-up period visits will be conducted on Weeks 105, 106, 107, 108, 109, 110, 117, 123 and 130 (Weeks 105, 106, 107, 108, 109, 110 and 123 may be conducted by a home healthcare nurse).

For patients who have entered the second 52-week extended treatment period, the post-treatment follow-up period visits will be on Weeks 157, 158, 159, 160, 161, 162, 169, 175 and 182 (Weeks 157, 158, 159, 160, 161, 162 and 175 may be conducted by a home healthcare nurse).

# Protocol - France

#### 3.5 **End-of-Study**

The End-of-Study is last patient, last visit.

#### 3.6 **Data and Safety Monitoring Board**

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 **Enrollment**

Patients will be enrolled into the treatment phase of the study after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 **Inclusion Criteria**

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent

- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.
  Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label Study:
  - a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
  - b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
    - Confirmed homozygote, compound heterozygote or double heterozygote for known lossof-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
    - Post heparin plasma LPL activity of  $\leq 20\%$  of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study.
  - c. Fasting  $TG \ge 750 \text{ mg/dL}$  (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
- 4. Able and willing to participate in a 78-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause <u>and</u> follicle stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# **5.2** Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification

- c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])
- d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
- e. Current use of glucagon-like peptide-1 (GLP-1) agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification
- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST  $> 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of glomerular filtration rate (GFR) in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II

- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and over-the-counter [OTC]), or fibrates unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to Qualification
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to Qualification
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to Qualification and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to Qualification or planned during the study
  - j. Prior exposure to ISIS 304801
  - k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801)
- 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

### 6.1 Study Schedule

6.

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

STUDY PROCEDURES

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), electrocardiograms (ECGs), echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

### 6.1.3 Extended Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of continuing treatment for up to an additional 104 weeks. For patients that have entered the Extended Treatment Periods, study participation will be up to an additional 104 weeks or until commercialization of product, whichever is sooner.

During the extended treatment period, patients will have assessments and procedures done during Weeks 54-156 as per the Schedule of Procedures in Appendix A. Assessments and procedures may be conducted by either a home healthcare service or the Study Center, however the patient will be required to visit the study center approximately every 3 months. Study Drug will be administered once weekly unless the patient is on a biweekly treatment schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis),

AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling will be conducted weekly and may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Treatment instructions and training will be provided to the patient where applicable.

#### 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volunesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after treatment on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.5 Post-Treatment Follow-up

After completion of the Week 52 visit assessments, patients will have the option of continuing treatment for up to an additional 104 weeks as described in Section 6.1.3. Patients not continuing treatment will enter the 26-week post-treatment follow-up. For patients not continuing into the 52-week extended treatment period, the 26-week post-treatment follow-up period consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse).

For patients who enter the first 52-week extended treatment period, but will not continue into the second 52-weeks of the extended treatment period, the post-treatment follow-up period visits will be conducted on Weeks 105, 106, 107, 108, 109, 110, 117, 123 and 130 (Weeks 105, 106, 107, 108, 109, 110 and 123 may be conducted by a home healthcare nurse).

For patients who enter the second 52-week extended treatment period, the post-treatment follow-up period visits will be on Weeks 157, 158, 159, 160, 161, 162, 169, 175 and 182 (Weeks 157, 158, 159, 160, 161, 162 and 175 may be conducted by a home healthcare nurse).

These visits are outlined in the Schedule of Procedures in Appendix A.

#### 6.2 **Additional Study Assessments**

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Protocol - France

Each time a hematology lab is drawn and sent to the central laboratory for analysis, an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples), another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm<sup>3</sup>, or the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), high-sensitivity C-reactive protein (hsCRP) and for cytokine analysis.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 **Echocardiography**

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 **ECG**

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52. During the posttreatment follow-up, ECGs will be performed in triplicate at Weeks 65 and 78 for patients not opting to participate in the Extended Treatment Period. Patients in the Extended Treatment Periods will have ECGs performed in triplicate at Weeks 76 and 104. Triplicate ECGs will be performed at Weeks 13 and 26 of each post-treatment follow-up period.

#### 6.2.5 **MRI**

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, and Week 52. During the post-treatment follow-up, patients will complete an EQ-5D and SF-36 during Weeks 65 and 78. Should the patient enter the extended treatment periods, additional Quality of Life Questionnaires will be collected at Weeks 13 and 26 of each post-treatment follow-up period.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 **Diet Monitoring**

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52. During the post-treatment follow-up, patients will complete a 7-day food diary prior to Weeks 65 and 78.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2) 6.2.10

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

#### 6.3 **Restriction on the Lifestyle of Patients**

#### 6.3.1 **Contraception Requirements**

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females < 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

# For male patients:

Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

### For female patients:

- Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.
- \* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.
- † Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

### 7. STUDY DRUG

### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 °C to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

# 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

# 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volunesorsen provided by the Sponsor. The Study Center must return all unused volunesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

# **8.1** Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will continue to receive Study Drug as a single 300 mg/1.5 mL injection once-weekly for Weeks 53-156 as outlined in Sections 8.5 and 8.6. Patients on dose reduction will receive 300 mg/1.5 mL injections every 2 weeks.

Patients should receive 1 dose per week, unless on a dose reduction of 300 mg every 2 weeks, with weeks always defined relative to Study Day 1. For example, if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if treatment

on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 **Other Protocol-Required Drugs**

There are no other protocol-required drugs.

#### 8.3 **Other Protocol-Required Treatment Procedures**

There are no other protocol required treatment procedures for this study.

#### 8.4 **Treatment Precautions**

There are no specific treatment precautions required for this study.

#### 8.5 **Safety Monitoring Rules**

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

Confirmation Guidance: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be** confirmed by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest must be available prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-treatment Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue treatment. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee and will be followed up in accordance with Section 8.8 of the protocol.

### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified. In addition, platelet function may be evaluated at any time during the study by aggregometry, using an approved point-of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers.

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to treatment. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 3-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and treatment where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a platelet count drawn within 3-5 days prior to departure and with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming treatment.

Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (×2) or < 100,000/mm<sup>3</sup> (×1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |

| Auto-antibody screen: |
|--------------------------------------------|
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), hsCRP and for cytokine analysis.

#### Safety Monitoring for LDL-C Elevations 8.5.5

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a lowdensity lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

The Investigator or delegate will review the glucometer reading or printout at every clinic visit to evaluate if fasting pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for Hyperglycemia below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event case report form (CRF). Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as one in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

# 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory fasting plasma glucose (FPG) measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, treatment with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued treatment and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, treatment of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\ge 2$  weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, treatment of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq$  0.3 mg/dL (26.5  $\mu$ mol/L) and  $\geq$  40% above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24 hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible treatment re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

# 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), treatment of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, or a platelet count less than  $75,000/\text{mm}^3$  that

occurs while the patient is on treatment at 300 mg every 2 weeks, then treatment of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (**note:** may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), treatment of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm³. If treatment is continued it should be at a reduced dose frequency of 300 mg every 2 weeks (refer to Section 8.7). The suitability of the patient for continued treatment will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of treatment.

If after the first treatment rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then treatment of the patient with Study Drug will be stopped permanently.

### Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

# Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma > 25 cm<sup>2</sup>
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

 Table 3
 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to treatment. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified In addition, platelet function may be evaluated during the study by aggregometry, using an approved point- of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers. Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed. Obtain additional lab tests (Table 2) if 2 occurrences consecutive or non-consecutive of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. |
| > 100K/mm <sup>3</sup> | Once weekly 300 mg Study Drug administration | |
| 100K/mm <sup>3</sup> - >75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks. | |
| 75K/mm <sup>3</sup> - >50K/mm <sup>3</sup> | <ul> <li>If occurs while on dose of 300 mg every 2 weeks, then permanently discontinue Study Drug, otherwise dose pause. If dose pause is ≥ 3 months then patient must discontinue treatment and enter the follow up period.</li> <li>When platelet count returns to &gt; 100K/mm³ restart treatment at dose frequency of 300 mg every 2 weeks in consultation with the Sponsor Medical Monitor</li> </ul> | Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| < 50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug and the patient will enter the follow up period. | Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management Steroids recommended *. It is strongly recommended that, unless |

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | | the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline. • Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy • Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is< 50K/mm³ if possible. |

# Legend:

\* Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after Methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

# 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose frequency to 300 mg every 2 weeks will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs, and the Study Medical Monitor is informed. If a patient is dose paused for  $\geq 3$  months, he or she is considered to have discontinued treatment and should enter the 26-week post-treatment follow-up period.

### 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6
- The patient is dose paused for  $\geq 3$  months

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug.

A patient who discontinues early from treatment with stable platelet counts above the LLN at the time of treatment discontinuation will have platelet counts drawn every 2 weeks after discontinuing Study Drug for the first 6 weeks after the last dose of Study Drug. A subsequent platelet count should then be taken after an additional 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

# 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 78, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

# 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation
- Commercialization of product

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

# 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), GLP-1 agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline Qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipidaltering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of

informed consent and Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit.

### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

# **8.11** Treatment Compliance

Compliance with treatment is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a treatment diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

# 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

# 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6 (R2). Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

### 9.3 Definitions

### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

# 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment,

they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

# 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 (or Week 130 or 182 if the patient enters the first or second extended treatment period, respectively) visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

# 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

• **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test

- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

# *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- Mild: The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Treatment was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Treatment frequency was reduced

### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

# 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

• **AE Persists:** Patient terminates from the trial and the AE continues

- Recovered: Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- **Persists (as non-serious AE):** Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE electronic Case Report Form (eCRF) (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

### 9.5 **Procedures for Handling Special Situations**

### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was
on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the
study

- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Treatment Errors

Volanesorsen treatment errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Treatment details should be captured on the Treatment Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

# 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, **the Study Center and Sponsor may request access to the** 

mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

### 10. STATISTICAL CONSIDERATIONS

### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

# 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs
- Platelet aggregation (may be evaluated)

# 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 **Populations**

Full Analysis Set (FAS): All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

Per Protocol Set (PPS): Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

PK Population: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### 10.4 **Definition of Baseline**

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline will be the last non-missing assessment prior to the first dose of Study Drug. Details will be provided in the SAP.

#### 10.5 **Interim Analysis**

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 **Planned Methods of Analysis**

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active Study Drug in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naïve group which includes patients on placebo in index studies. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by Medical Dictionary for Regulatory Activities (MedDRA) system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

# 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volunesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

# 10.6.4 Pharmacokinetic and Immunogenicity Analysis

### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration  $(C_{max})$  and the time taken to reach  $C_{max}$   $(T_{max})$  will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0</sub>- $_{24h}/F$ ) will be calculated from  $CL_{0.24h}/F = Actual Dose/AUC_{0.24h}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation, MRT<sub>0-24h</sub> = AUMC<sub>0-24h</sub> /AUC<sub>0-24h</sub>, where AUMC<sub>0-24h</sub> is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

# 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.
Protocol - France

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

## 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

## 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

# 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH E6 (R2) Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

# 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH E6 (R2) Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

# 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

### 12.3 Study Documentation and Storage

An eCRF utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines E6 (R2), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of prestudy documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

# 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH E6 (R2) and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH E6 (R2), and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

# 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Gaudet D, Baass A, Tremblay K, et al. Natural History (up to 15 years) of Platelet Count in 84 Patients with Familial Hyperchylomicronemia Due to Lipoprotein Lipase Deficiency. Journal of Clinical Lipidology 2017; 11(3): 797-798.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Protocol - France

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-α expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PC, Voshol PJ, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

Qualification through Treatment Period

Post-Treatment Follow-up (For patients not opting to participate in the Extended Treatment Period)

First 52-Week Extended Treatment Period

First 52-Week Extended Treatment Period Post-Treatment Follow-Up (For patients not opting to participate in the second 52-Week Extended Treatment Period)

Second 52-Week Extended Treatment Period
Second 52-Week Extended Treatment Period Post-Treatment Follow-Up

Appendix A Schedule of Procedures – Qualification through Treatment Period

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | Treat | ment 1 | Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | -2 to<br>-1 | | /k<br>1 | Wk<br>4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | Mor<br>Wk<br>12 | Wk<br>13 | Wk<br>15<br>&<br>17 | Wk<br>19 | Wk<br>21<br>&<br>23 | Wk<br>25 | Wk<br>26 | Wk<br>28<br>&<br>30 | Wk<br>32 | Wk<br>34<br>&<br>36 | Wk<br>38 | Wk<br>40<br>&<br>42 | Wk<br>44 | Wk<br>46<br>&<br>48 | Mo<br>Wk<br>50 | Wk 52<br>or ET |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Info | rmed Consent | X | | | | | | | | | | | | | | | | | | | | | | |
| Out | patient Visit | X | X | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | X | $X^{j}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | X | $X^{j}$ | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | X | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | $X^{j}$ | X | $X^{j}$ | $X^{j}$ | $X^{j}$ | $\mathbf{X}^{\mathrm{j}}$ | X |
| Incl | usion/Exclusion Criteria | X | | | | | | | | | | | | | | | | | | | | | | |
| Med | lical History <sup>q</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Vita | ll Signs + body weight (+ height on Day 1 only) | X | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Phy | sical Examination | X | X | | | | | | | X | | | | | X | | | | X | | | | | X |
| 12- | lead ECG (triplicate) | X | | | | | | | | X | | | | | X | | | | X | | | | | X |
| MR | I (liver/spleen) | X | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Ech | ocardiography | X | | | | | | | | | | | | | $X^k$ | | | | | | | | | $X^k$ |
| | Chemistry Panel | X | X | | X | | X | | | X | | X | | | X | | X | | X | | X | | | X |
| | CBC with Differential <sup>b</sup> | X | <b>◆</b> | Platele | ts are | asses | ssed | each | caler | ıdar w | eek, | visits | do no | X<br>ot hav | e spec | ified w | indo | ws to | allow | / flexi | bility | of sc | heduli | ing. |
| | Serum Lipid Panel | X | X | | X | | X | | X | X | | | | X | X | | | | X | | | | X | X |
| | Blood viscosity <sup>r</sup> | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| | Platelet aggregation <sup>r</sup> | X | X | | | | | | | X | | | | | X | | | | | | | | | X |
| )c | Coagulation (aPTT, PT, INR) | X | | | | | X | | | X | | | | | X | | | | X | | | | | X |
| ting | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | Xn | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Fas | Sedimentation Rate | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| ⊗ | Complement (C5a, Bb) | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| )ra | Plasma PK - Volanesorsen | | X <sup>1</sup> | X | X | | X | | | X | | | | | X | | | | X | | | | | X |
| l pc | Anti-Volanesorsen Antibodies | | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Blood Draw (Fasting)° | FSH (women only, if applicable) | X | | | | | | | | | | | | | | | | | | | | | | |
| 1 | Serum Pregnancy Test <sup>d</sup> | X | | | X | | X | | | X | | X | | | X | | X | | X | | X | | | X |
| | Archived Serum & Plasma Samples <sup>c</sup> | | X | | | | X | | | X | | | | | X | | | | | | | | | X |
| | Troponin Iº | X | | | | | | | | | | | | | | | | | | | | | | |
| | Platelet Bound Autoantibodies <sup>r</sup> | | X | | | | | | | | | | | | | | | | | | | | | |
| | Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study) <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | |

Appendix A Schedule of Procedures - Qualification through Treatment Period Continued

| Study Period | Quala | | | | | | | | | | , | Treatn | nent P | eriod | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| C. I. W. I. | 2. 1 | W | k | W | Wk | Wk | Wk | | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Moi | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Mo | onth 12 |
| Study Week | -2 to -1 | 1 | | k<br>4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | | Wk 52<br>or ET |
| Study Day | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Urinalysis <sup>c</sup> | X | $X^{m}$ | | X | | X | | | $X^{m}$ | | $X^{m}$ | | | $X^{m}$ | | $X^{m}$ | | $X^{m}$ | | X <sup>m</sup> | | | $X^{m}$ |
| Fundus Photography <sup>f</sup> | X | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Symptom Diary (weekly) | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Quality of Life Assessment(s) | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Food/Drink Diary (quarterly)h | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Diet/Alcohol Counselingi | X | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Adverse Events | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medication | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Appendix A Schedule of Procedures – Post-Treatment Follow-up (for patients not opting to participate in the Extended Treatment Period)

| | Study Period | | P | ost Tre | eatment | Follow-up <sup>p</sup> |
|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| | Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Outpatie | | $X^{j}$ | $X^{j}$ | X | $X^{j}$ | X |
| | ns + body weight<br>on Day 1 only) | | | X | | X |
| Physical | Examination | | | X | | X |
| 12- lead | ECG (triplicate) | | | X | | X |
| | Chemistry Panel | | X | X | X | X |
| <b>5</b> ( | CBC with Differential <sup>b</sup> | Xs | X | X | X | X |
| ing | Serum Lipid Panel | | | X | | X |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | | X | | X |
| × (I | Sedimentation Rate | | | X | | X |
| )ra | Complement (C5a, Bb) | | | X | | X |
| Ιp | Plasma PK - Volanesorsen | | | X | | X |
| 100 | Anti-Volanesorsen Antibodies | | | X | | X |
| ш | Serum Pregnancy Test <sup>d</sup> | | X | X | X | X |
| | Archived Serum & Plasma Samples <sup>e</sup> | | | X | | X |
| Urinalysi | is <sup>c</sup> | | $X^{m}$ | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> |
| Sympton | n Diary (weekly) | X | X | X | X | X |
| Quality o | of Life Assessment(s) | | | X | | X |
| Food/Dri | ink Diary (quarterly) <sup>h</sup> | | | X | | X |
| Diet/Alco | ohol Counseling <sup>i</sup> | | X | X | X | X |
| Adverse | Events | X | X | X | X | X |
| Concomi | tant Medication | X | X | X | X | X |

- Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw.
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 ISIS 304801-CS16 roll over patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)

- g Genetic testing can be conducted for study Qualification (Group 2 ISIS 304801-CS16 roll over patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing. A blood sample for potential gene sequencing may be collected at timepoints other than Screening or Qualification Visits.
- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A  $\pm$  7-day window is allowed for MRI, echocardiography procedures and fundus photography
- 1 Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)
- n HbA1c only
- o All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- p If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- r May be done. Blood viscosity and platelet aggregation in volunesorsen-treatment naïve patients only
- s Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling

Appendix A Schedule of Procedures – First 52-Week Extended Treatment Period

| | Study Period | | | | | | | Ext | ended Tre | eatment P | eriod | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | Wk 60<br>& 62 | Mo 15<br>Wk 64 | Wk 66<br>& 68 | Wk<br>70 | Wk 72<br>& 74 | Mo 18<br>Wk 76 | Wk 78<br>& 80 | Wk<br>82 | Wk 84, 86,<br>& 88 | Mo 21<br>Wk 90 | Wk 92<br>& 94 | Wk<br>96 | Wk 98,<br>100 &<br>102 | Mo 24<br>Wk 104 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 568 | 582, 596 &<br>610 | 624 | 638 &<br>652 | 666 | 680, 694<br>& 708 | 722 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Outp | patient Visit | $X^{f}$ | $X^{f}$ | X <sup>f</sup> | X | $X^{f}$ | Xf | X <sup>f</sup> | X | $X^{f}$ | Xf | $X^{f}$ | X | $X^{f}$ | $X^{f}$ | $X^{f}$ | X |
| Vita | l Signs (+ body weight) | | | | X | | | | X | | | | X | | | | X |
| Phys | sical Examination | | | | | | | | X | | | | | | | | X |
| 12- | lead ECG (triplicate) | | | | | | | | X | | | | | | | | X |
| Urin | alysis (including P/C ratio) | | X | | X | | X | | X | | X | | X | | X | | X |
| | Chemistry Panel | | X | | X | | X | | X | | X | | X | | X | | X |
| | CBC with Differential <sup>a</sup> | <b>+</b> | | Platelets | are assess | sed each ca | alendar | week, visi | - | X – nave speci | fied w | vindows to all | ow flexibi | lity of sch | eduling | <u>, </u> | |
| ıg) <sup>b</sup> | Serum Lipid Panel | | | | X | | | | X | | | | X | | | | X |
| (Fasting) <sup>b</sup> | Coagulation (aPTT, PT, INR) | | | | X | | | | X | | | | X | | | | X |
| lw (I | Troponin I | | | | X | | | | X | | | | X | | | | X |
| Blood Draw | Plasma PK - ISIS 304801° | | | | | | | | X | | | | | | | | X |
| lood | Anti-ISIS 304801 Antibodies | | | | | | | | X | | | | | | | | X |
| Щ | Serum Pregnancy Test <sup>d</sup> | | X | | X | | X | | X | | X | | X | | X | | X |
| | Platelet Function <sup>g</sup> | <b>←</b> | | May be | e assessed | at various | timepo | oints, visits | X do not ha | ve specifi | ed wii | ndows to allo | w flexibili | ty of sched | duling. | | <b>—</b> |
| Wee | kly Study Drug: SC Injection | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Diet | /Alcohol Counseling <sup>e</sup> | | | | X | | | | X | | | | X | | | | X |
| Adv | erse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Con | comitant Medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- g May be done

Appendix A Schedule of Procedures – First 52-Week Extended Treatment Period Post-Treatment Follow-Up (For patients not opting to participate in the second 52 Week Extended Treatment Period)

| | Study Period | | Post Treat | ment Fo | llow-up <sup>a</sup> | |
|---|---|---|---|---|---|---|
| | Study Week | Wk 106<br>&<br>108 | Wk<br>110 | Wk<br>117 | Wk<br>123 | Wk<br>130 |
| | Study Day | 736<br>&<br>750 | 764 | 813 | 855 | 904 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Outpatient | | $X^{b}$ | $X^b$ | X | $X^{b}$ | X |
| (+ height o | s + body weight<br>on Day 1 only) | | | X | | X |
| | xamination | | | X | | X |
| 12- lead E | CG (triplicate) | | | X | | X |
| | Chemistry Panel | **1 | X | X | X | X |
| g)e | CBC with Differential <sup>c</sup> | X <sup>d</sup> | X | X | X | X |
| Blood Draw (Fasting) <sup>e</sup> | Serum Lipid Panel<br>hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | | X | | X |
| (Fа | Sedimentation Rate | | | X | | X |
| aw | Complement (C5a, Bb) | | | X | | X |
| D | Plasma PK - Volanesorsen | | | X | | X |
| poo | Anti-Volanesorsen Antibodies | | | X | | X |
| BI | Serum Pregnancy Test <sup>f</sup> | | X | X | X | X |
| | Archived Serum & Plasma Samples <sup>g</sup> | | | X | | X |
| Urinalysis | | | $X^h$ | Xh | Xh | X <sup>h</sup> |
| Symptom | Diary (weekly) | X | X | X | X | X |
| Quality of | Life Assessment(s) | | | X | | X |
| Diet/Alcoh | nol Counseling <sup>i</sup> | | X | X | X | X |
| Adverse E | vents | X | X | X | X | X |
| Concomita | ant Medication | X | X | X | X | X |

- a If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- b Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- d Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling
- e Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours.
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volunesorsen
- h Expanded urinalysis (see Appendix B)

i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel

Appendix A Schedule of Procedures – Second 52-Week Extended Treatment Period

| | Study Period | | Extended Trea | ntment Period | |
|---|---|---|---|---|---|
| | Study Week | Wk 116 | Mo 30<br>Wk 128 | Mo 33<br>Wk 142 | Wk 156 |
| | Study Day | 806 | 890 | 988 | 1086 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 |
| Outpatio | ent Visit | X | X | X | X |
| Vital Si | gns (+ body weight) | X | X | X | X |
| Physica | 1 Examination | | X | | X |
| Urinaly | sis (including P/C ratio) | X | X | X | X |
| 9 ( | Chemistry Panel | X | X | X | X |
| Blood Draw (Fasting) <sup>b</sup> | CBC with Differential <sup>a</sup> | | assessed each calc<br>windows to allow | endar week, visi | |
| Draw | Serum Lipid Panel | X | X | X | X |
| [ poc | Serum Pregnancy Test <sup>c</sup> | X | X | X | X |
| Ble | Anti-ISIS 304801 Antibodies | | | | X |
| Weekly | Study Drug: SC Injection | 4 | | | <b>—</b> |
| Diet/Ale | cohol Counseling <sup>d</sup> | X | X | X | X |
| Adverse | e Events | X | X | X | X |
| Concon | nitant Medication | X | X | X | X |

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Females of childbearing potential only
- d To reinforce compliance to the diet and alcohol restrictions
- e Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

Appendix A Schedule of Procedures – Second 52-Week Extended Treatment Period Post-Treatment Follow-Up

| | Study Period | | Post Trea | atment Foll | ow-up <sup>a</sup> | |
|---|---|---|---|---|---|---|
| | Study Week | Wk 158 &<br>160 | Wk 162 | Wk 169 | Wk 175 | Wk 182 |
| | Study Day | 1100 &<br>1114 | 1128 | 1177 | 1219 | 1268 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| | ntient Visit | $X^{b}$ | $X^{b}$ | X | $X^{b}$ | X |
| | Signs + body weight | | | X | | Х |
| (+ hei | ight on Day 1 only) | | | Λ | | Λ |
| | cal Examination | | | X | | X |
| 12- le | ad ECG (triplicate) | | | X | | X |
| | Chemistry Panel | | X | X | X | X |
| | CBC with Differential <sup>c</sup> | $X^d$ | X | X | X | X |
| ng) | Serum Lipid Panel | | | X | | X |
| Blood Draw (Fasting) <sup>e</sup> | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | | | X | | X |
| )<br>M | Sedimentation Rate | | | X | | X |
| Drz | Complement (C5a, Bb) | | | X | | X |
| po | Plasma PK - Volanesorsen | | | X | | X |
| Blo | Anti-Volanesorsen Antibodies | | | X | | X |
| | Serum Pregnancy Test <sup>f</sup> | | X | X | X | X |
| | Archived Serum & Plasma Samples <sup>g</sup> | | | X | | X |
| Urina | lysis | | $X^h$ | $X^h$ | $X^h$ | $X^h$ |
| Symp | tom Diary (weekly) | X | X | X | X | X |
| Quali | ty of Life Assessment(s) | | | X | | X |
| Diet/A | Alcohol Counselingi | | X | X | X | X |
| Adve | rse Events | X | X | X | X | X |
| Conce | omitant Medication | X | X | X | X | X |

- a If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- b Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- d Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling
- e Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volunesorsen
- h Expanded urinalysis (see Appendix B)
- To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel

# **Appendix B** List of Laboratory Analytes

## Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volanesorsen or other similar oligonucleotides.

| Clinic | cal Chemistry Panel | Coag | <u>ulation</u> | Hem | atology | Urina | <u>alysis</u> |
|---|---|---|---|---|---|---|---|
| • | Sodium | • | aPTT (sec) | • | Red blood cells | • | Color |
| • | Potassium | • | PT (sec) | • | Hemoglobin | • | Appearance |
| • | Chloride | • | INR | • | Hematocrit | • | Specific gravity |
| • | Bicarbonate | | | • | MCV, MCH, MCHC | • | pН |
| • | Total protein | Lipid | Panel | • | Platelets | • | Protein |
| • | Albumin | • | Total Cholesterol | • | White blood cells | • | Blood |
| • | Calcium | • | LDL-C | • | WBC Differential | • | Ketones |
| • | Magnesium | • | HDL-C | | (% and absolute) | • | Urobilinogen |
| • | Phosphorus | • | Triglycerides | | <ul> <li>Neutrophils</li> </ul> | • | Glucose |
| • | Glucose | • | Non-HDL-C | | <ul> <li>Eosinophils</li> </ul> | • | Bilirubin |
| • | BUN | • | VLDL-C | | <ul> <li>Basophils</li> </ul> | • | Leukocyte esterase |
| • | Creatinine | • | apoA-1 | | <ul> <li>Lymphocytes</li> </ul> | • | Nitrate |
| • | Uric Acid | • | apoB | | <ul> <li>Monocytes</li> </ul> | • | Microscopic |
| • | Total bilirubin | • | apoC-III | | | | examination <sup>4</sup> |
| • | Direct (conjugated) bilirubin | | | | macokinetics <sup>1</sup><br>munogenicity | | tional Measures for |
| • | Indirect (unconjugated)<br>bilirubin<br>ALT<br>AST | | | • | Volanesorsen levels in<br>plasma<br>Anti-volanesorsen<br>antibodies in plasma | <u>Expa</u> • | nded Urinalysis Total protein (quantitative) Microalbumin |
| • | Alkaline phosphatase | | | <u>Othe</u> | r Assessments | • | β2-microglobulin |
| | | | | • | hsCRP | Plate | let Function |
| | | | | • | Sedimentation Rate | • | Platelet aggregation <sup>3</sup> |
| | | | | • | C5a, Bb | • | Platelet function <sup>5</sup> |
| | | | | • | Troponin I <sup>2</sup> | | |
| | | | | • | CK-MB <sup>2</sup> | | |
| | | | | • | Platelet Bound<br>Autoantibodies <sup>3</sup> | | |
| | | | | • | De-lipidated free glycerol | | |
| | | | | • | HbA1c, FPG | | |
| | | | | • | Blood viscosity <sup>3</sup> | | |
| 1 P | lasma DV samulas may al | laa <b>1</b> .a. | and for munifiling of dur | مناه منا م | o proteins bioanalytical n | athad. | 1: 4-4: |

- Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified
- 5 May be done using a point-of-care device on site

# Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to treatment, and at various times throughout the treatment and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime | Anytime |

# PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>Post-dose | Pre-dose | Pre-dose | Pre-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# PK Sampling Schedule - First 52-Week Extended Treatment Period

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 | Wk<br>130 |
|--------------------------|----------|-----------|-----------|-----------|
| Study Day | D526 | D722 | D813 | D904 |
| Visit Window<br>+/- Days | 2 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Anytime | Anytime |

# PK Sampling Schedule – Second 52-Week Extended Treatment Period

| Week | Wk<br>169 | Wk<br>182 |
|--------------------------|-----------|-----------|
| Study Day | D1177 | D1268 |
| Visit Window +/-<br>Days | 7 | 7 |
| Time Point | Anytime | Anytime |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm³ | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm <sup>3</sup> ;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities *Continued*

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>Ionized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - , | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Urine | | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142



#### **Collaborator:**

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

# ISIS 304801-CS7

# The APPROACH Open-Label Study Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 9 - France - 25 May 2018

EudraCT No: 2015-003755-21

# ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

# Protocol Amendment 9 - France - 25 May 2018

# **Protocol History:**

Original Protocol: 28 August 2015
Protocol Amendment 1: 2 February 2016
Protocol Amendment 2: 22 April 2016
Protocol Amendment 3: 9 May 2016
Protocol Amendment 4: 6 June 2016
Protocol Amendment 5: 19 August 2016
Protocol Amendment 6: 16 September 2016
Protocol Amendment 7: 3 February 2017
Protocol Amendment 8: 10 April 2017

Approved by:

MB B,Ch. BAO, FRCP(C)

Akcea Therapeutics, Inc. 55 Cambridge Parkway, Suite 100

Cambridge, MA 02142 Telephone: (617) 207-0202

# **Protocol Number: ISIS 304801-CS7**

**Protocol Amendment 9 - France** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Akcea Therapeutics, Inc.

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Key Sponsor Contact:

Akcea Therapeutics, Inc.

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Phone:

Email:

Collaborator: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010

Date: 25 May 2018

### **Confidentiality Statement**

This document contains confidential information of Akcea Therapeutics, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Akcea Therapeutics, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Volan with Familial Chylomicronemia | esorsen Administered Subcutaneously to Patients<br>a Syndrome (FCS) |
| Amendment: | Amendment 9 - France | |
| Date: | 25 May 2018 | |
| Label Study of Volan | | ne attached clinical protocol, entitled "An Openasly to Patients with Familial Chylomicronemia duct the study as described herein. |
| I agree to comply wit<br>Clinical Practice E6 ( | | Harmonization Tripartite Guideline on Good |
| - | e evaluation or conduct of the clini | ned in this document will not be used for any cal investigation without the prior written consen |
| Investigator's Signa | ture | <del>-</del> |
| Investigator's Name | c (please print) | Date (DD Month YYYY) |

# TABLE OF CONTENTS

| | | | Page |
|---|---|---|---|
| PR | OTO | COL AMENDMENT | 9 |
| PR | OTO | COL SYNOPSIS | 14 |
| | | DESIGN AND TREATMENT SCHEMA | |
| STU | U <b>DY</b> | GLOSSARY | 21 |
| 1. | ( | OBJECTIVES | 23 |
| 2. | P | BACKGROUND AND RATIONALE | 23 |
| 2 | 2.1 | Overview of Disease | |
| 2 | 2.2 | Therapeutic Rationale | 24 |
| 2 | 2.3 | Volanesorsen | 25 |
| | 2.3. | 1 Mechanism of Action | 25 |
| | 2.3. | 2 Chemistry | 26 |
| | 2.3. | - I | |
| | 2.3. | 1 | |
| | 2.4 | Rationale for Dose and Schedule of Administration | 28 |
| 3. | F | EXPERIMENTAL PLAN | |
| 3 | 3.1 | Study Design | |
| 3 | 3.2 | Number of Study Centers | |
| 3 | 3.3 | Number of Patients | |
| 3 | 3.4 | Overall Study Duration and Follow-up | |
| | 3.4. | 1 Qualification | 29 |
| | 3.4. | | |
| | 3.4. | | |
| | 3.4. | 1 | |
| | 3.5 | End-of-Study | |
| | 3.6 | Data and Safety Monitoring Board | |
| 4. | P | PATIENT ENROLLMENT | |
| 4 | 1.1 | Qualification | 30 |
| | 1.2 | Enrollment | |
| <b>5.</b> | | PATIENT ELIGIBILITY | |
| | 5.1 | Inclusion Criteria | |
| 5 | 5.2 | Exclusion Criteria | |
| 6. | | TUDY PROCEDURES | |
| 6 | 5.1 | Study Schedule | |
| | 6.1. | · | |
| | 6.1. | | |
| | 6.1. | | |
| | 6.1. | ( ) & 1 | |
| | 6.1. | 5 Post-Treatment Follow-up | 35 |

| | 6.2 | Additional Study Assessments | 36 |
|---|---|---|---|
| | 6.2.1 | Laboratory Assessments | 36 |
| | 6.2.2 | Physical Exams and Vital Signs | 36 |
| | 6. | 2.2.1 Eruptive Xanthoma | 36 |
| | 6. | 2.2.2 Lipemia Retinalis | 36 |
| | 6.2.3 | Echocardiography | 36 |
| | 6.2.4 | ECG | 36 |
| | 6.2.5 | MRI | 37 |
| | 6.2.6 | Quality of Life Assessments | 37 |
| | 6.2.7 | Disease Symptom Diary | 37 |
| | 6.2.8 | Diet Monitoring | 37 |
| | 6.2.9 | Family History | 37 |
| | 6.2.1 | O Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2) | 37 |
| | 6.3 | Restriction on the Lifestyle of Patients | 37 |
| | 6.3.1 | Contraception Requirements | 37 |
| | 6.3.2 | Other Requirements | 38 |
| <b>7.</b> | S' | TUDY DRUG | 39 |
| | 7.1 | Volanesorsen Description | 39 |
| | 7.2 | Packaging and Labeling | 39 |
| | 7.3 | Study Drug Accountability | 39 |
| 8. | T | REATMENT OF PATIENTS | 39 |
| | 8.1 | Volanesorsen Administration | 39 |
| | 8.2 | Other Protocol-Required Drugs | 40 |
| | 8.3 | Other Protocol-Required Treatment Procedures | 40 |
| | 8.4 | Treatment Precautions | 40 |
| | 8.5 | Safety Monitoring Rules | 40 |
| | 8.5.1 | Safety Monitoring for Liver Chemistry Tests | 40 |
| | 8.5.2 | Safety Monitoring for Platelet Count Results | 41 |
| | 8.5.3 | Safety Monitoring for Minor Bleeding Events | 43 |
| | 8.5.4 | Safety Monitoring for Constitutional Symptoms | 43 |
| | 8.5.5 | Safety Monitoring for LDL-C Elevations | 43 |
| | 8.5.6 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | 43 |
| | 8.5.7 | Safety Monitoring for Documented Severe Hypoglycemia | 44 |
| | 8.5.8 | Safety Monitoring for Hyperglycemia | 44 |
| | 8.5.9 | Acute Pancreatitis | 45 |
| | 8.6 | Stopping Rules | 45 |
| | 8.6.1 | Stopping Rules for Liver Chemistry Elevations | 45 |
| | 8.6.2 | Stopping Rules for Renal Function Test Results | 46 |
| | 8.6.3 | Stopping Rules for Platelet Count Results | 46 |
| | 8.7 | Adjustment of Dose Frequency | 48 |
| | 8.8 | Discontinuation of Study Treatment | 49 |

| | 8.8.1 | Follow-up Visits for Early Termination from Treatment Period | 49 |
|---|---|---|---|
| | 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Period | 49 |
| | 8.9 | Withdrawal of Patients from the Study | 49 |
| | 8.10 | Concomitant Therapy and Procedures | 50 |
| | 8.10. | 1 Concomitant Therapy | 50 |
| | 8.10. | 2 Concomitant Procedures | 51 |
| | 8.11 | Treatment Compliance | 51 |
| 9. | . SI | ERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 51 |
| | 9.1 | Sponsor Review of Safety Information | 51 |
| | 9.2 | Regulatory Requirements | 51 |
| | 9.3 | Definitions | 52 |
| | 9.3.1 | Adverse Event | 52 |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 52 |
| | 9.3.3 | Serious Adverse Event (SAE) | 52 |
| | 9.4 | Monitoring and Recording Adverse Events | 53 |
| | 9.4.1 | Serious Adverse Events | 53 |
| | 9.4.2 | Non-Serious Adverse Events | 53 |
| | 9.4.3 | , | |
| | 9.4 | 4.3.1 Relationship to the Study Drug | 53 |
| | 9.4 | 4.3.2 Severity | 54 |
| | 9.4 | 4.3.3 Action Taken with Volanesorsen | 54 |
| | 9.4 | Treatment Given for Adverse Event | |
| | 9.4 | 4.3.5 Outcome of the Adverse Event | |
| | 9.4.4 | • | |
| | 9.5 | Procedures for Handling Special Situations | |
| | 9.5.1 | Abnormalities of Laboratory Tests | |
| | 9.5.2 | | |
| | 9.5.3 | $\varepsilon$ | |
| | 9.5.4 | | |
| 1 | | TATISTICAL CONSIDERATIONS | |
| | 10.1 | Study Endpoints | |
| | 10.1. | | |
| | 10.1. | ÿ 1 | |
| | 10.2 | Sample Size | |
| | 10.3 | Populations | |
| | 10.4 | Definition of Baseline | |
| | 10.5 | Interim Analysis | |
| | 10.6 | Planned Methods of Analysis | |
| | 10.6. | | |
| | 10.6. | | |
| | 10.6. | 3 Efficacy Analysis | 59 |

| 10 | 0.6.4 | Pharmacokinetic and Immunogenicity Analysis | 60 |
|---|---|---|---|
| | 10.6.4.1 | Pharmacokinetic Analysis | 60 |
| | 10.6.4.2 | Immunogenicity Analysis | 60 |
| 11. | <b>INVES</b> | TIGATOR'S REGULATORY OBLIGATIONS | 61 |
| 11.1 | Infor | med Consent | 61 |
| 11.2 | | al Conduct of the Study | |
| 11.3 | Inde | pendent Ethics Committee/Institutional Review Board | 61 |
| 11.4 | | nt Confidentiality | |
| 12. | | NISTRATIVE AND LEGAL OBLIGATIONS | |
| 12.1 | | ocol Amendments | |
| 12.2 | • | y Termination | |
| 12.3 | • | y Documentation and Storage | |
| 12.4 | • | y Monitoring | |
| 12.5 | _ | uage | |
| 12.6 | | pensation for Injury | |
| 13. | | RENCES | |
| 14. | | IDICES | |
| | endix A | Schedule of Procedures | |
| | endix B | List of Laboratory Analytes | |
| | endix C | Pharmacokinetic Sampling Schedule | |
| Appe | endix D | Grading Scale for Adverse Events Relating to Laboratory Abnormalities | 79 |
| | | TABLE OF TABLES | |
| | | | Page |
| Table 1 | | Volanesorsen (ISIS 304801) Characteristics | 39 |
| Table 2 | | Labs to Be Performed in the Event of a Platelet Count Less than the Lower | 40 |
| T.1.1. 2 | | Limit of Normal (x2) or < 100,000/mm <sup>3</sup> (x1)* | |
| Table 3 Table 4 | | Actions in Patients with Low Platelet Count | 4/ |
| Table 4 | • | Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence | 51 |
| | | TABLE OF FIGURES | |
| | | IADLE OF FIGURES | |
| | | | Page |
| Figure | 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 24 |
| Figure 2 | 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | | (MOE-Gapmer). The sequence of volanesorsen is shown | |
| Figure 3 | 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 28 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 9 - France

**Amendment Date:** 25 May 2018

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 8 dated 10 April 2017:

1. To prolong the extended treatment period an additional 52 weeks.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| <b>Protocol Section</b> | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Design and<br>Study Visit<br>Schedule and<br>Procedures<br>3.1 Study Design<br>3.4.3 Extended<br>Treatment Period | Following the Week 52 visit, patients will enter an at least 26 week post treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. have the option to continue dosing for up to an additional 52 weeks for a total of 104 weeks of dosing. Patients not continuing dosing will enter a 26-week post-treatment follow-up period. | To allow patients the option of continuing treatment with volanesorsen after completion of the 52-week open-label treatment period. |
| Protocol Synopsis:<br>Study Visit<br>Schedule and<br>Procedures | <ul> <li>An at least 26-week post-treatment evaluation period Option to participate in an extended treatment period (up to an additional 52 weeks)</li> <li>A 26-week post-treatment follow-up period</li> </ul> | To allow patients the option of continuing treatment with volanesorsen after completion of the 52-week open-label treatment period. For patients continuing |
| | | treatment up to 104 weeks, the 26-<br>week post-treatment follow-up<br>period has been added for those<br>patients also. |
|---|---|---|
| Section 6.1.3<br>Extended<br>Treatment Period | After completion of the Week 52 visit assessments, patients will have the option of continuing dosing for up to an additional 52 weeks. During the extended treatment period, patients will have assessments and procedures done during Weeks 54-104 as per the Schedule of Procedures in Appendix A. Assessments and procedures may be conducted by either a home healthcare service or the Study Center, however the patient will be required to visit the study center approximately every 3 months. Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable. | To outline the procedures to be performed during the extended treatment period and 26-week post follow up treatment period. The extended treatment period provides additional volanesorsen dose exposure and patient safety evaluations. |
| Section 6.1.5 | After completion of the Week 52 visit assessments, patients will have the option of continuing dosing for up to an additional 52 weeks as described in Section 6.1.3. Patients not continuing dosing will enter the 26-week post-treatment follow-up. After completion of the Week 52 visit assessments, patients will enter the at least 26 week post treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. The 26-week period post-treatment follow-up consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse). An additional 26-week post-treatment follow-up occurs after the extended treatment period with at least 9 Study Center visits on Weeks 105, 106, 107, 108, 109, 110, 117, 118, and 125 (Weeks 105, 106, 107, 108, 109, 110, and 118 may be conducted by a home healthcare nurse. These visits, as are outlined in the Schedule of Procedures in Appendix A. | To outline the procedures to be performed during the extended treatment period and 26-week post follow up treatment period. |

| | Study Period | | | | | tmen | t Follow-up <sup>p</sup> | |
|---|---|---|---|---|---|---|---|---|
| | | Study Week | Wk<br>54<br>&<br>56 | | Wk<br>65 | W<br>k<br>71 | Wk<br>78 | |
| | | Study Day | 372<br>&<br>386 | 400 | 449 | 49<br>1 | 540 | |
| | | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 | |
| | Inform | ed Consent | | | | | | |
| | Outpat | ient Visit | X | X<br>j | X | $X^{j}$ | X | |
| | | on/Exclusion Criteria | | | | | | |
| | (+ heig | igns + body weight<br>ht on Day 1 only) | | | X | | X | |
| | | al Examination | | | X | | X | |
| | 12- lea | d ECG (triplicate) | | | X | | X | |
| Appendix A | | iver/spleen) | | | | | | |
| Schedule of | <u>Echocardiography</u> | | | | ** | ** | ** | Removed assessments that were not |
| Procedures—Post-<br>Treatment Follow- | <b>S</b> _ | Chemistry Panel CBC with Differential <sup>b</sup> | X | X | X | X | X<br>X | conducted during the post-<br>treatment follow-up. |
| Up | Blood Draw (Fasting)° | Serum Lipid Panel | | | X | | X | |
| | Fast | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | | X | | X | |
| | M (] | Sedimentation Rate | | | X | | X | |
| | Dra | Complement (C5a, Bb) | | | X | | X | |
| | ро | Plasma PK - Volanesorsen | | | X | | X | |
| | Blo | Anti-Volanesorsen Antibodies | | | X | | X | |
| | | Serum Pregnancy Test <sup>d</sup> | | X | X | X | X | |
| | | Archived Serum & Plasma Samples <sup>e</sup> | 1 | | X | | X | |
| | Urinaly | /sis <sup>c</sup> | | X | X | $X^{m}$ | $X^{m}$ | |
| | Fundus | <del>: Photography <sup>f</sup></del> | | | | | | |
| | Genetic | e testing for FCS diagnosis (if not available in medical history)* | | | | | | |
| | Weekly Study Drug: SC Injection | | | | | | | |
| | | om Diary (weekly) | X | X | X | X | X | |
| | Quality | v of Life Assessment(s) | | | X | | X | |
| | Food/D | Orink Diary (quarterly) <sup>h</sup> | | | X | | X | |

| | Diet/Alcohol Cor | unselingi | | | X | X X | | X | |
|---|---|---|---|---|---|---|---|---|---|
| | Adverse Events | | | | X | X X | | X | |
| | Concomitant Me | dication | | X | X | X X | | X | |
| Appendix A:<br>Schedule of<br>Procedures—<br>Extended<br>Treatment Period | A S | he 52 week | extende | ed trea | tment p | eriod. | | Schedule of procedures table added for the 52-week extended treatment period. | |
| | | Study Period | Pos | t Treat | ment l | Follow- | up <sup>a</sup> | | |
| | | Study Week | Wk 106<br>&<br>108 | Wk<br>110 | Wk<br>117 | | Wk<br>130 | | |
| | | Study Day | 736<br>&<br>750 | 764 | 813 | 855 | 904 | | |
| | | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 | ] | |
| | Vital Si | ient Visit<br>igns + body weight<br>ht on Day 1 only) | Xb | Xb | X | Xb | X | | |
| Appendix A: | Physical Examination | | | | X | | X | | |
| Schedule of<br>Procedures— | 12- lead ECG (triplicate) | | | | X | | X | 1 | Schedule of procedures table added |
| Extended | | Chemistry Panel | | X | X | X | X | | for 26 week post treatment follow-<br>up subsequent to the 52 week |
| Treatment Period | | CBC with Differential <sup>c</sup> | $X^{d}$ | X | X | X | X | | extended treatment period. |
| Post-Treatment<br>Follow-Up | Blood Draw (Fasting)° | Serum Lipid Panel<br>hsCRP, HbA1c, FPG, and de-lipidated | | | X | - | X | | |
| | (Fas | free glycerol | | | X | | X | | |
| | aw | Sedimentation Rate | | | X | | X | | |
| | Dr | Complement (C5a, Bb) | 1 1 | | X | | X | 1 | |
| | <u> </u> | Plasma PK - Volanesorsen | + | | X | 1 | X | 4 | |
| | l Ia | Anti-Volanesorsen Antibodies Serum Pregnancy Test <sup>f</sup> | + + | X | X | X | X | 1 | |
| | | Archived Serum & Plasma Samples <sup>g</sup> | + + | Λ | X | Λ | X | | |
| | Urinalysis | | | Xi | Xi | Xi | X <sup>i</sup> | 1 | |
| | Sympto | om Diary (weekly) | X | X | X | X | X | 1 | |
| | Quality | of Life Assessment(s) | | | X | | X | 1 | |
| | Diet/Al | cohol Counselingi | | X | X | X | X | | |

| | | Adverse Events | | | X | X | X | X | X | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Concomitant Medication | | Concomitant Medication | | X | X | X | X | X | |
| | | | Week | Wk<br>76 | | /k<br>)4 | Wk<br>117 | | | | |
| Appen | ndix C: | | Study Day | D526 | D7 | 22 | D813 | | | | |
| | nacokinetic<br>ling | | Visit<br>Window +/-<br>Days | 2 | 2 | 2 | 7 | | | | A PK sampling scheduled was added for the 52 week extended treatment period. |
| | | | Time Point | Pre-dose | | re-<br>ose | Anytim | e | | | |

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option to continue dosing for up to an additional 52 weeks for a total of 104 weeks of dosing. Patients not continuing dosing will enter a 26-week post-treatment follow-up period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| Study Population Continued | 2. Age ≥ 18 years at time of informed consent |
| , , | <ol> <li>Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 30480<br/>CS16 (index studies) with an acceptable safety profile, per Sponsor and<br/>Investigator judgement.</li> </ol> |
| | Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: |
| | a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L) |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: </li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-causing<br/>genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical<br/>history. Note: testing of LPL activity should not be performed to<br/>confirm eligibility for the study</li> </ul> |
| | c. Fasting TG $\geq$ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study |
| | 4. Able and willing to participate in a 78-week study |
| | Inclusion Criteria: Continued |

#### Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **Exclusion Criteria:**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification

# Study Population Continued

Exclusion Criteria: Continued

- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
    - Estimated creatinine clearance calculated according to the formula
      of Cockcroft and Gault < 50 mL/min (MDRD or
      CKD-EPI formulas can be used instead of Cockcroft-Gault for
      estimation of GFR in patients with low body weight after
      discussion with Sponsor Medical Monitor)</li>
  - c. Cardiac Troponin I > ULN at Qualification
  - d. LDL-C > 130 mg/dL at Qualification
  - e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria: Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study |
| | Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to Qualification |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor |
| | d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study |
| | Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to Qualification |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to Qualification and regular clinical monitoring is performed |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | Plasma apheresis within 4 weeks prior to Qualification or planned during the study |
| | j. Prior exposure to ISIS 304801 |
| | k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion) |
| | 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule<br>Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the Sponsor).</li> <li>Please refer to Section 4.1 and Appendix A</li> </ul> |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | <ul> <li>Option to participate in an extended treatment period (up to an<br/>additional 52 weeks)</li> </ul> |
| | <ul> <li>A 26-week post-treatment follow-up period</li> </ul> |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option to continue dosing for up to an additional 52 weeks. Patients not to continuing dosing will enter a 26-week post-treatment follow-up period. |
| Safety and Tolerability Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |

| Planned Analyses | Safety Endpoints: |
|---|---|
| | Adverse events including adjudicated events of acute pancreatitis and MACE |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | Frequency and severity of patient reported abdominal pain during the treatment period |
| | <ul> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high- density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Change in blood viscosity (may be evaluated) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Akcea Therapeutics, Inc. |
| Collaborator | Ionis Pharmaceuticals, Inc. |

#### STUDY DESIGN AND TREATMENT SCHEMA



# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 9 Protocol - France 25 May 2018

# STUDY GLOSSARY

Index Studies

| STUDY GLOSSARY | |
|---|---|
| Abbreviation/Acronym | <b>Definition</b> |
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |

ISIS 304801-CS6 and ISIS 304801-CS16

#### ISIS 304801-CS7 CONFIDENTIAL Amendment 9

Protocol - France 25 May 2018

Abbreviation/Acronym **Definition** 

International Normalized Ratio **INR IRB** Institutional Review Board

**IXRS** Interactive Voice/Web-Response System

Low-Density Lipoprotein LDL

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

Major Acute Cardiovascular Event **MACE** 

MOE 2'-O-(2-methoxyethyl) MRI magnetic resonance imaging mRNA messenger ribonucleic acid not clinically-significant **NCS** 

**NOAEL** No-Observed-Adverse-Effect Level

Non-High-Density Lipoprotein-Cholesterol non-HDL-C

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic PPS per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

**SUSAR** suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

 $T_{\text{max}}$ time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

**TRL** Triglyceride-Rich Lipoproteins

ULN upper limit of normal

**VLDL** Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

**VLDL-TG** Lipoprotein-Triglyceride **WMA** World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

# 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V (APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009);

Amendment 9 25 May 2018

glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

# 2.2 Therapeutic Rationale

Protocol - France

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL,

by steric inhibition of the interaction of apoE with these receptors.

Protocol - France 25 May 2018

apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volanesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

# 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing. The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

# 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volanesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volanesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

# 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and

mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

# 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved

TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks, with the option of continuing dosing for an additional 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in

tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

# 3. EXPERIMENTAL PLAN

# 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option to continue dosing for up to an additional 52 weeks for a total of 104 weeks of dosing. Patients not to continuing dosing will enter a 26-week post-treatment follow-up period.

# 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

# 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Qualification

A qualification period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

# 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volanesorsen is administered by SC injection once weekly.

#### 3.4.3 Extended Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of continuing dosing for up to an additional 52 weeks. Patients not continuing dosing will enter the 26-week post-treatment follow-up.

# 3.4.4 Post-Treatment Follow-Up

The post-treatment follow-up period is at least 26 weeks and consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse).

# 3.5 End-of-Study

The End-of-Study is last patient, last visit.

# 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

# 4. PATIENT ENROLLMENT

# 4.1 Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

# 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

# 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

# 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known lossof-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of  $\leq 20\%$  of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study.
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
- 4. Able and willing to participate in a 78-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause <u>and</u> FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

\* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **5.2** Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification
- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$
    - AST  $> 2.0 \times ULN$
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field

 Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)

Amendment 9

25 May 2018

- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm<sup>3</sup>) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to Qualification
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to Qualification
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to Qualification and regular clinical monitoring is performed

- h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period
- i. Plasma apheresis within 4 weeks prior to Qualification or planned during the study
- j. Prior exposure to ISIS 304801
- k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

# 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

Amendment 9 25 May 2018

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

# 6.1.3 Extended Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of continuing dosing for up to an additional 52 weeks.

During the extended treatment period, patients will have assessments and procedures done during Weeks 54-104 as per the Schedule of Procedures in Appendix A. Assessments and procedures may be conducted by either a home healthcare service or the Study Center, however the patient will be required to visit the study center approximately every 3 months. Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

# 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.5 Post-Treatment Follow-up

After completion of the Week 52 visit assessments, patients will have the option of continuing dosing for up to an additional 52 weeks as described in Section 6.1.3. Patients not continuing dosing will enter the 26-week post-treatment follow-up. The 26-week post-treatment follow-up consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse). An additional 26-week post-treatment follow-up occurs after the extended treatment period with at least 9 Study Center visits on Weeks 105, 106, 107, 108, 109, 110, 117, 118, and 125 (Weeks 105, 106, 107, 108, 109, 110, and 118 may be conducted by a home healthcare nurse. These visits are outlined in the Schedule of Procedures in Appendix A.

# 6.2 Additional Study Assessments

# 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm<sup>3</sup>, or the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

# 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

# 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

# 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

# 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

# 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52. During the post-treatment follow-up, ECGs will be performed in triplicate at Weeks 65 and 78 for patients not opting to participate in the Extended Treatment Period. Patients in the Extended Treatment Period will have ECGs performed in triplicate at Weeks 76, 104 and 130.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, and Week 52. During the post-treatment follow-up, patients will complete an EQ-5D and SF-36 during Weeks 65 and 78. Additional Quality of Life Questionnaires will be collected at Weeks 117 and 130 should the patient enter the extended treatment period post-treatment follow-up.

# 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

# 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52. During the post-treatment follow-up, patients will complete a 7-day food diary prior to Weeks 65 and 78.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

# 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

# 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

# 6.3 Restriction on the Lifestyle of Patients

# 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

# For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

# For female patients:

- Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.
- \* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.
- † Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that

Amendment 9

serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

# 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 °C to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength 200 mg/mL | |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

# 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

# 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

# 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example, if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

Amendment 9

25 May 2018

# 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs.

# 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

# 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be redosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee and will be followed up in accordance with Section 8.8 of the protocol.

# 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food

Protocol - France

and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

# 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified.

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption

of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm<sup>3</sup> (x1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

# 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

# 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

# 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

# 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as one in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

# 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

Protocol - France

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control

Amendment 9

25 May 2018

- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq$  0.3 mg/dL (26.5  $\mu$ mol/L) and  $\geq$  40% above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24 hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator **in consultation with** the Sponsor Medical Monitor or designee.

## 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, or a platelet count less than  $75,000/\text{mm}^3$  that occurs while the patient is on dosing at 300 mg every 2 weeks, then dosing of a patient with volunesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days

(**note:** may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks (refer to Section 8.7). The

suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

#### Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

## Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

 Table 3
 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or non-consecutive of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. |
| > 100K/mm <sup>3</sup> | Weekly 300 mg Study Drug administration | |
| 100K/mm <sup>3</sup> - >75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks | |

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| 75K/mm³ - >50K/mm³ | If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor Medical Monitor | Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| < 50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | <ul> <li>Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are &gt; 75K/mm³ then monitor every 1 week</li> <li>Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management</li> <li>Steroids recommended *. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline.</li> <li>Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy</li> <li>Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is&lt; 50K/mm³ if possible</li> </ul> |

#### Legend:

\* Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after Methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

#### 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

## 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

## 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 78, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

# 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Protocol - France

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline Qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 78 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

# 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

# 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6 (R2). Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines. Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

# 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

# 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

## 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

• **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test

- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

# *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

# 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

• AE Persists: Patient terminates from the trial and the AE continues

- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

# 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 **Dosing Errors**

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volanesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

Should an overdose occur, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the

mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

## 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs
- Platelet aggregation (may be evaluated)

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline will be the last non-missing assessment prior to the first dose of Study Drug. Details will be provided in the SAP.

# 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active Study Drug in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naïve group which includes patients on placebo in index studies. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

## 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

# 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volunesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration  $(C_{max})$  and the time taken to reach  $C_{max}$   $(T_{max})$  will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0.74h</sub> /F) will be calculated from  $CL_{0-24h}$  /F = Actual Dose/AUC<sub>0-24h</sub>. Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation, MRT<sub>0-24h</sub> = AUMC<sub>0-24h</sub> /AUC<sub>0-24h</sub>, where AUMC<sub>0-24h</sub> is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., %change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g.,  $C_{trough}$ ) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

## 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

## 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

## 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH

Guidelines E6 (R2), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of prestudy documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

## 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

## 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Protocol - France

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354-357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-α expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008: 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PC, Voshol PJ, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 9 Protocol - France 25 May 2018

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

Qualification through Treatment Period

Post-Treatment Follow-up

Extended Treatment Period

Extended Treatment Period Post-Treatment Follow-Up

Appendix A Schedule of Procedures – Qualification through Treatment Period

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | Treat | ment l | Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | C. I. W. I | -2 to | W | /k | Wk | Wk | Wk | Wk | Moi | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Moi | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Mo | onth 12 |
| | Study Week | -1 | 1 | 1 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Inf | ormed Consent | X | | | | | | | | | | | | | | | | | | | | | | |
| Ou | patient Visit | X | X | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | X<br>j | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | X | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | X | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | X | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | X |
| Inc | usion/Exclusion Criteria | X | | | | | | | | | | | | | | | | | | | | | | |
| | dical History <sup>q</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Vit | al Signs + body weight (+ height on Day 1 only) | X | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Ph | sical Examination | X | X | | | | | | | X | | | | | X | | | | X | | | | | X |
| | lead ECG (triplicate) | X | | | | | | | | X | | | | | X | | | | X | | | | | X |
| MF | I (liver/spleen) | X | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Ecl | ocardiography | X | | | | | | | | | | | | | $X^k$ | | | | | | | | | $X^k$ |
| | Chemistry Panel | X | X | | X | | X | | | X | | X | | | X | | X | | X | | X | | | X |
| | CBC with Differential <sup>b</sup> | X | <b>←</b> I | Platele | ts are | asse | ssed | each | calen | dar w | eek, | visits | do no | – X<br>ot hav | e spec | ified w | indo | ws to | allov | / flexi | ibility | of sc | heduli | ing. |
| | Serum Lipid Panel | X | X | | X | | X | | X | X | | | | X | X | | | | X | | <u> </u> | | X | X |
| | Blood viscosity <sup>r</sup> | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| | Platelet aggregation <sup>r</sup> | X | X | | | | | | | X | | | | | X | | | | | | | | | X |
| °( | Coagulation (aPTT, PT, INR) | X | | | | | X | | | X | | | | | X | | | | X | | | | | X |
| ing | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | Xn | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Fast | Sedimentation Rate | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| № | Complement (C5a, Bb) | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| )ra | Plasma PK - Volanesorsen | | $X^{l}$ | X | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Ιþα | Anti-Volanesorsen Antibodies | | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Blood Draw (Fasting) <sup>c</sup> | FSH (women only, if applicable) | X | | | | | | | | | | | | | | | | | | | | | | |
| Ι – | Serum Pregnancy Test <sup>d</sup> | X | | | X | | X | | | X | | X | | | X | | X | | X | | X | | | X |
| | Archived Serum & Plasma Samples <sup>e</sup> | | X | | | | X | | | X | | | | | X | | | | | | | | | X |
| 1 | Troponin I° | X | | | <u> </u> | | | | | | | | | | | | | | | | | | | |
| 1 | Platelet Bound Autoantibodies <sup>r</sup> | | X | | <u> </u> | | | | | | | | | | | | | | | | | | | |
| | Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study) <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | |

Appendix A Schedule of Procedures - Qualification through Treatment Period Continued

| Study Period | Qual <sup>a</sup> | | Treatment Period | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| C. I.W. I | 24 1 | w | k | w | Wk | Wk | Wk | | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Mo | onth 12 |
| Study Week | -2 to -1 | 1 | | k<br>4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | | Wk 52<br>or ET |
| Study Day | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Urinalysis <sup>c</sup> | X | $X^{m}$ | | X | | X | | | $X^{m}$ | | $X^{m}$ | | | X <sup>m</sup> | | $X^{m}$ | | $X^{m}$ | | $X^{m}$ | | | $X^{m}$ |
| Fundus Photography <sup>f</sup> | X | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Symptom Diary (weekly) | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Quality of Life Assessment(s) | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Food/Drink Diary (quarterly)h | | X | | | | | | | X | | | | | X | | | | | | | | | X |
| Diet/Alcohol Counselingi | X | X | | X | | X | | | X | | | | | X | | | | X | | | | | X |
| Adverse Events | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medication | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Protocol - France

#### **Appendix A** Schedule of Procedures – Post-Treatment Follow-up

| | Study Period | | P | ost Tre | eatment | Follow-up <sup>p</sup> |
|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| | Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Outpatier | | $X^{j}$ | $X^{j}$ | X | $X^{j}$ | X |
| | ns + body weight<br>on Day 1 only) | | | X | | X |
| | Examination | | | X | | X |
| | ECG (triplicate) | i | | X | | X |
| | Chemistry Panel | | X | X | X | X |
| ٥( | CBC with Differential <sup>b</sup> | Xs | X | X | X | X |
| ing. | Serum Lipid Panel | | | X | | X |
| Blood Draw (Fasting)° | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | | X | | X |
| v (F | Sedimentation Rate | | | X | | X |
| )rav | Complement (C5a, Bb) | | | X | | X |
| Ιþ | Plasma PK - Volanesorsen | | | X | | X |
| 001 | Anti-Volanesorsen Antibodies | | | X | | X |
| ш | Serum Pregnancy Test <sup>d</sup> | | X | X | X | X |
| | Archived Serum & Plasma Samples <sup>e</sup> | | | X | | X |
| Urinalysi | S <sup>c</sup> | | $X^{m}$ | X <sup>m</sup> | $\mathbf{X}^{\mathrm{m}}$ | $X^{m}$ |
| Symptom | Diary (weekly) | X | X | X | X | X |
| Quality o | f Life Assessment(s) | | | X | | X |
| Food/Dri | nk Diary (quarterly) <sup>h</sup> | | | X | | X |
| Diet/Alco | hol Counseling <sup>i</sup> | | X | X | X | X |
| Adverse l | Events | X | X | X | X | X |
| Concomi | ant Medication | X | X | X | X | X |

# Legend:

- Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 ISIS 304801-CS16 roll over patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study Qualification (Group 2 ISIS 304801-CS16 roll over patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing

- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- 1 Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)
- n HbA1c only
- o All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- p If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- r May be done. Blood viscosity and platelet aggregation in volunesorsen-treatment naïve patients only
- s Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling

Protocol - France 25 May 2018

Appendix A Schedule of Procedures – Extended Treatment Period

| | Study Period | | | | | | | Ext | ended Tre | eatment P | eriod | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | Wk 60<br>& 62 | Mo 15<br>Wk 64 | Wk 66<br>& 68 | Wk<br>70 | Wk 72<br>& 74 | Mo 18<br>Wk 76 | Wk 78<br>& 80 | Wk<br>82 | Wk 84, 86,<br>& 88 | Mo 21<br>Wk 90 | Wk 92<br>& 94 | Wk<br>96 | Wk 98,<br>100 &<br>102 | Mo 24<br>Wk 104 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 568 | 582, 596 &<br>610 | 624 | 638 &<br>652 | 666 | 680, 694<br>& 708 | 722 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Outp | patient Visit | $X^{f}$ | $X^{f}$ | $X^{f}$ | X | $X^{f}$ | $X^{f}$ | $X^{f}$ | X | $X^{f}$ | $X^{f}$ | Xf | X | $X^{f}$ | $X^{f}$ | $X^{f}$ | X |
| Vital | l Signs (+ body weight) | | | | X | | | | X | | | | X | | | | X |
| Phys | sical Examination | | | | | | | | X | | | | | | | | X |
| 12-1 | ead ECG (triplicate) | | | | | | | | X | | | | | | | | X |
| Urin | alysis (including P/C ratio) | | X | | X | | X | | X | | X | | X | | X | | X |
| | Chemistry Panel | | X | | X | | X | | X | | X | | X | | X | | X |
| (Fasting) <sup>b</sup> | CBC with Differential <sup>a</sup> | <b>+</b> | | Platelets | are assess | sed each ca | alendar | week, vis | - | X<br>nave speci | fied w | vindows to all | ow flexibi | lity of sch | eduling | 5. | |
| astii | Serum Lipid Panel | | | | X | | | | X | | | | X | | | | X |
| w (F | Coagulation (aPTT, PT, INR) | | | | X | | | | X | | | | X | | | | X |
| Dra | Troponin I | | | | X | | | | X | | | | X | | | | X |
| Blood Draw | Plasma PK - ISIS 304801° | | | | | | | | X | | | | | | | | X |
| В | Anti-ISIS 304801 Antibodies | | | | | | | | X | | | | | | | | X |
| | Serum Pregnancy Test <sup>d</sup> | | X | | X | | X | | X | | X | | X | | X | | X |
| Wee | kly Study Drug: SC Injection | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Diet | Alcohol Counseling <sup>e</sup> | | | | X | | | | X | | | | X | | | | X |
| Adv | erse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Cond | comitant Medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

#### Legend:

a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine

# ISIS 304801-CS7 CONFIDENTIAL Amendment 9 Protocol - France 25 May 2018

if the count has met a stopping rule, or the dose reduction rule of  $100,000/\text{mm}^3$ , or the dose pause rule of  $75,000/\text{mm}^3$ . Any case of a platelet count  $< 50,000/\text{mm}^3$  should be reported in an expedited fashion to the Sponsor

- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

Appendix A Schedule of Procedures – Extended Treatment Period (Post-Treatment Follow-Up)

| | Study Period | | Post Treat | ment Fol | llow-up <sup>a</sup> | |
|---|---|---|---|---|---|---|
| | Study Week | Wk 106<br>&<br>108 | Wk<br>110 | Wk<br>117 | Wk<br>123 | Wk<br>130 |
| | Study Day | 736<br>&<br>750 | 764 | 813 | 855 | 904 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Outpatient | | $X^{b}$ | $X^b$ | X | $X^b$ | X |
| | s + body weight<br>n Day 1 only) | | | X | | X |
| | xamination | | | X | | X |
| 12- lead E | CG (triplicate) | | | X | | X |
| | Chemistry Panel | | X | X | X | X |
| | CBC with Differential <sup>c</sup> | $X^d$ | X | X | X | X |
| Blood Draw (Fasting) <sup>e</sup> | Serum Lipid Panel | | | X | | X |
| ast | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | | X | | X |
| D ≫ | Sedimentation Rate | | | X | | X |
| )ra | Complement (C5a, Bb) | | | X | | X |
| I pc | Plasma PK - Volanesorsen | | | X | | X |
| 3loc | Anti-Volanesorsen Antibodies | | | X | | X |
| | Serum Pregnancy Test <sup>f</sup> | | X | X | X | X |
| | Archived Serum & Plasma Samples <sup>g</sup> | | | X | | X |
| Urinalysis | | | $X^h$ | $X^h$ | $X^h$ | $X^h$ |
| Symptom | Diary (weekly) | X | X | X | X | X |
| Quality of | Life Assessment(s) | | | X | | X |
| Diet/Alcoh | ol Counseling <sup>i</sup> | | X | X | X | X |
| Adverse E | vents | X | X | X | X | X |
| Concomita | nt Medication | X | X | X | X | X |

#### Legend:

- a If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- b Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- d Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling
- e Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volunesorsen
- h Expanded urinalysis (see Appendix B)

i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volanesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | Coagulation | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| • Sodium | • aPTT (sec) | <ul> <li>Red blood cells</li> </ul> | • Color |
| • Potassium | • PT (sec) | <ul> <li>Hemoglobin</li> </ul> | • Appearance |
| • Chloride | • INR | • Hematocrit | <ul> <li>Specific gravity</li> </ul> |
| Bicarbonate | | • MCV, MCH, MCHC | • pH |
| Total protein | Lipid Panel | • Platelets | • Protein |
| • Albumin | <ul> <li>Total Cholesterol</li> </ul> | <ul> <li>White blood cells</li> </ul> | • Blood |
| Calcium | • LDL-C | <ul> <li>WBC Differential (% and</li> </ul> | • Ketones |
| Magnesium | • HDL-C | absolute) | • Urobilinogen |
| <ul> <li>Phosphorus</li> </ul> | <ul> <li>Triglycerides</li> </ul> | <ul> <li>Neutrophils</li> </ul> | • Glucose |
| • Glucose | • Non-HDL-C | <ul> <li>Eosinophils</li> </ul> | • Bilirubin |
| • BUN | • VLDL-C | <ul> <li>Basophils</li> </ul> | Leukocyte esterase |
| Creatinine | • apoA-1 | • Lymphocytes | • Nitrate |
| Uric Acid | <ul> <li>apoB</li> </ul> | <ul> <li>Monocytes</li> </ul> | • Microscopic examination <sup>4</sup> |
| Total bilirubin | <ul> <li>apoC-III</li> </ul> | | |
| Direct (conjugated) bilirubin | | Pharmacokinetics <sup>1</sup> & Immunogenicity | Additional Measures for Expanded |
| • Indirect (unconjugated) | | Volanesorsen levels in plasma | <u>Urinalysis</u> |
| bilirubin | | Anti-volanesorsen antibodies | Total protein (quantitative) |
| • ALT | | in plasma | Microalbumin |
| • AST | | - | • β2-microglobulin |
| Alkaline phosphatase | | Other Assessments | Platelet Function |
| | | • hsCRP | • Platelet aggregation <sup>3</sup> |
| | | • Sedimentation Rate | Tracelet aggregation |
| | | • C5a, Bb | |
| | | • Troponin I <sup>2</sup> | |
| | | • CK-MB <sup>2</sup> | |
| | | <ul> <li>Platelet Bound<br/>Autoantibodies<sup>3</sup></li> </ul> | |
| | | De-lipidated free glycerol | |
| | | • HbA1c, FPG | |
| | | • Blood viscosity <sup>3</sup> | |
| 1 Dl DV1. | 1 1 1 0 01 | f drug hinding proteins, biognalytical method | 11.1.2 |

- Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

# **Appendix C** Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime | Anytime |

## PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>Post-dose | Pre-dose | Pre-dose | Pre-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# **PK Sampling Schedule (Extended Treatment Period)**

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Anytime |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Hematology | | | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | ÷ | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Urine | | | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)




**Sponsor:** 

Akcea Therapeutics, Inc. 22 Boston Wharf Road, 9<sup>th</sup> Floor, Boston, MA 02210 Collaborator:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

## ISIS 304801-CS7

# The APPROACH Open-Label Study Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 8 – 21 November 2018

EudraCT No: 2015-003755-21

## ISIS 304801-CS7

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

## Protocol Amendment 8 – 21 November 2018

## Protocol History:

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

Protocol Amendment 3: 9 May 2016

Protocol Amendment 4: 6 June 2016

Protocol Amendment 5: 6 July 2016

Protocol Amendment 6: 18 November 2016

Protocol Amendment 7: 7 April 2017

## Approved by:

Akcea Therapeutics, Inc. 22 Boston Wharf Road, 9<sup>th</sup> Floor Boston, MA 02210 Telephone:

Akcea Therapeutics, Inc.

Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 8** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: 22 Boston Wharf Road, ,9<sup>th</sup> Floor

Boston, MA 02210

Telephone:

**Key Sponsor Contact:** 

Akcea Therapeutics, Inc.

22 Boston Wharf Road, 9th Floor

Boston, MA 02210

Telephone:

Email:

Collaborator: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010

Date: 21 November 2018

## **Confidentiality Statement**

This document contains confidential information of Akcea Therapeutics, Inc. and Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Akcea Therapeutics, Inc. and Ionis Pharmaceuticals, Inc.

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | rsen Administered Subcutaneously to Patients<br>ndrome (FCS) | |
| Amendment: | Amendment 8 | |
| Date: | 21 November 2018 | |
| abel Study of Volanes | orsen Administered Subcutaneously | e attached clinical protocol, entitled "An Open<br>of to Patients with Familial Chylomicronemia<br>conduct the study as described herein. |
| agree to comply with Clinical Practice (E6) (R. | | rmonization Tripartite Guideline on Good |
| ourpose other than the | | ned in this document will not be used for any all investigation without the prior written cals, Inc. |
| Investigator's Signatu | re | |
| Investigator's Name ( | please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| PF | ROTO | COL AMENDMENT10 | |
| PF | ROTO | COL SYNOPSIS20 | |
| ST | TUDY 1 | DESIGN AND TREATMENT SCHEMA26 | |
| ST | CUDY | GLOSSARY27 | |
| 1. | C | DBJECTIVES29 | |
| 2. | В | BACKGROUND AND RATIONALE29 | |
| | 2.1 | Overview of Disease | 29 |
| | 2.2 | Therapeutic Rationale | 30 |
| | 2.3 | Volanesorsen | 31 |
| | 2.3. | 1 Mechanism of Action | 31 |
| | 2.3. | 2 Chemistry | 32 |
| | 2.3. | 3 Preclinical Experience | 32 |
| | 2.3. | 4 Clinical Experience | 33 |
| | 2.4 | Rationale for Dose and Schedule of Administration | 35 |
| 3. | E | EXPERIMENTAL PLAN | |
| | 3.1 | Study Design | 36 |
| | 3.2 | Number of Study Centers | 36 |
| | 3.3 | Number of Patients | 36 |
| | 3.4 | Overall Study Duration and Follow-up | 36 |
| | 3.4. | Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801–CS16 index | |
| | | study): Qualification | 36 |
| | 3.4. | Group 3 Patients (did not participate in an index study): Screening/Qualification | 36 |
| | 3.4. | 3 Treatment | 36 |
| | 3.4. | 4 Post-Treatment | 37 |
| | 3.5 | End-of-Study | 37 |
| | 3.6 | Data and Safety Monitoring Board | 37 |
| 4. | P | PATIENT ENROLLMENT | |
| | 4.1 | Screening/Qualification | 37 |
| | 4.2 | Enrollment | 38 |
| 5. | P | PATIENT ELIGIBILITY38 | |
| | 5.1 | Inclusion Criteria | 38 |
| | 5.2 | Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Stu | udy |
| | | Roll-over Patients | 39 |
| 6. | S | TUDY PROCEDURES42 | |
| | 6.1 | Study Schedule | 42 |
| | 6.1 | 1 Qualification (Groups 1 and 2) | 42 |

| | 6.1.2 | Screening and Qualification (Group 3) | 42 |
|---|---|---|---|
| | 6.1.3 | Treatment Period | 42 |
| | 6.1.4 | Extended Treatment Period | 43 |
| | 6.1.5 | Pharmacokinetic (PK) Subgroup | 43 |
| | 6.1.6 | Post-Treatment Period | 43 |
| | 6.2 Add | litional Study Assessments | 44 |
| | 6.2.1 | Laboratory Assessments | 44 |
| | 6.2.2 | Physical Exams and Vital Signs | 44 |
| | 6.2.2.1 | Eruptive Xanthoma | 44 |
| | 6.2.2.2 | 2 Lipemia Retinalis | 44 |
| | 6.2.3 | Echocardiography | 45 |
| | 6.2.4 | ECG | 45 |
| | 6.2.5 | MRI | 45 |
| | 6.2.6 | Quality of Life Assessments | 45 |
| | 6.2.7 | Disease Symptom Diary | 45 |
| | 6.2.8 | Diet Monitoring | 45 |
| | 6.2.9 | Family History | 45 |
| | 6.2.10 | Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2 and 3) | 46 |
| | 6.3 Res | triction on the Lifestyle of Patients | 46 |
| | 6.3.1 | Contraception Requirements | 46 |
| | 6.3.2 | Other Requirements | 47 |
| 7. | STUD | Y DRUG47 | |
| | 7.1 Vol | anesorsen Description | 47 |
| | 7.2 Pac | kaging and Labeling | 47 |
| | 7.3 Stu | dy Drug Accountability | 48 |
| 8. | TREA | ATMENT OF PATIENTS48 | |
| | 8.1 Vola | anesorsen Administration | 48 |
| | 8.2 Oth | er Protocol-Required Drugs | 48 |
| | 8.3 Oth | er Protocol-Required Treatment Procedures | 48 |
| | 8.4 Trea | atment Precautions | 48 |
| | 8.5 Safe | ety Monitoring Rules | 48 |
| | 8.5.1 | Safety Monitoring for Liver Chemistry Tests | 49 |
| | 8.5.2 | Safety Monitoring for Platelet Count Results | 50 |
| | 8.5.3 | Safety Monitoring for Minor Bleeding Events | |
| | 8.5.4 | Safety Monitoring for Constitutional Symptoms | 53 |
| | 8.5.5 | Safety Monitoring for LDL-C Elevations | |
| | 8.5.6 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | 53 |
| | 8.5.7 | Safety Monitoring for Documented Severe Hypoglycemia | |
| | 8.5.8 | Safety Monitoring for Hyperglycemia | 54 |

| | 8.5.9 | | Acute Pancreatitis | |
|---|---|---|---|---|
| | 8.6 | | pping Rules | |
| | 8.6.1 | | Stopping Rules for Liver Chemistry Elevations | |
| | 8.6.2 | | Stopping Rules for Renal Function Test Results | |
| | 8.6.3 | | Stopping Rules for Platelet Count Results | |
| | 8.7 | | istment of Dose Frequency | |
| | 8.8 | | ontinuation of Study Treatment | |
| | 8.8.1 | | Follow-up Visits for Early Termination from Treatment Period | |
| | 8.8.2 | | Follow-up Visits for Early Termination from Post-Treatment Follow-up Period | |
| | 8.9 | | ndrawal of Patients from the Study | |
| | 8.10 | | comitant Therapy and Procedures | |
| | 8.10 | | Concomitant Therapy | |
| | 8.10 | _ | Concomitant Procedures | |
| | 8.11 | | DUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 62 |
| 9. | 9.1 | | nsor Review of Safety Information | 62 |
| | 9.1<br>9.2 | | ulatory Requirements | |
| | 9.2<br>9.3 | | nitions | |
| | 9.3.1 | | Adverse Event | |
| | 9.3.2 | | Adverse Reaction and Suspected Adverse Reaction | |
| | 9.3.3 | | Serious Adverse Event (SAE) | |
| | 9.3.3<br>9.4 | | nitoring and Recording Adverse Events | |
| | 9.4.1 | | Serious Adverse Events | |
| | 9.4.2 | | Non-Serious Adverse Events | |
| | 9.4.3 | | Evaluation of Adverse Events (Serious and Non-Serious) | |
| | | ,<br>4.3.1 | | |
| | | 4.3.1<br>4.3.2 | | |
| | | 4.3.2<br>4.3.3 | • | |
| | | 4.3.4 | | |
| | | 4.3.5 | | |
| | 9.4.4 | | Adjudication Committees | |
| | 9.5 | | redures for Handling Special Situations | |
| | 9.5.1 | | Abnormalities of Laboratory Tests | |
| | 9.5.2 | | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | |
| | 9.5.3 | | Treatment Errors | |
| | 9.5.4 | | Contraception and Pregnancy | |
| 10. | | | ISTICAL CONSIDERATIONS | 07 |
| | 10.1 | | ly Endpoints | 68 |
| | | | Efficacy Endpoints | |

Table 1

Table 2

Table 3

| 10 | ).1.2 S | afety Endpoints | 69 |
|---|---|---|---|
| 10.2 | Sampl | e Size | 69 |
| 10.3 | Popula | ations | 69 |
| 10.4 | Defini | tion of Baseline | 69 |
| 10.5 | Interir | n Analysis | 70 |
| 10.6 | Planne | ed Methods of Analysis | 70 |
| 10 | 0.6.1 | emographic and Baseline Characteristics | 70 |
| 10 | 0.6.2 S | afety Analysis | 70 |
| 10 | 0.6.3 E | fficacy Analysis | 71 |
| 10 | 0.6.4 P | harmacokinetic and Immunogenicity Analysis | 71 |
| | 10.6.4.1 | Pharmacokinetic Analysis | 71 |
| | 10.6.4.2 | Immunogenicity Analysis | 72 |
| 11. | INVEST | IGATOR'S REGULATORY OBLIGATIONS | .72 |
| 11.1 | | ned Consent | |
| 11.2 | Ethica | I Conduct of the Study | 73 |
| 11.3 | • | endent Ethics Committee/Institutional Review Board | |
| 11.4 | Patien | t Confidentiality | 73 |
| | | | 7.4 |
| 12. | | ISTRATIVE AND LEGAL OBLIGATIONS | |
| 12.<br>12.1 | Protoc | col Amendments | 74 |
| | Protoc<br>Study | col Amendments Termination | 74<br>74 |
| 12.1 | Protoc<br>Study<br>Study | Termination | 74<br>74 |
| 12.1<br>12.2 | Protoc<br>Study<br>Study<br>Study | Termination Documentation and Storage Monitoring | 74<br>74<br>74 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5 | Protoc<br>Study<br>Study<br>Study<br>Langu | Termination Documentation and Storage Monitoring age | 74<br>74<br>75 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6 | Study<br>Study<br>Study<br>Study<br>Langu<br>Comp | col Amendments | 74747575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13. | Study<br>Study<br>Study<br>Langu<br>Compo | Termination Documentation and Storage Monitoring age ensation for Injury ENCES | 7474757575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13. | Study Study Study Langu Compo | Termination Documentation and Storage Monitoring age ensation for Injury ENCES | |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13. | Protoc<br>Study<br>Study<br>Study<br>Langu<br>Compo<br>REFERI<br>APPENI | Termination Documentation and Storage Monitoring age ensation for Injury ENCES Schedule of Procedures | 7475757575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13.<br>14.<br>Appe | Protoc<br>Study<br>Study<br>Study<br>Langu<br>Compo<br>REFERI<br>APPENI<br>endix A | Termination Documentation and Storage Monitoring age ensation for Injury ENCES Schedule of Procedures List of Laboratory Analytes | 7475757575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13.<br>14.<br>Appe | Protoc<br>Study<br>Study<br>Study<br>Langu<br>Comp<br>REFERI<br>APPENI<br>endix A<br>endix B | Termination Documentation and Storage Monitoring age ensation for Injury. ENCES Schedule of Procedures List of Laboratory Analytes Pharmacokinetic Sampling Schedule | 7475757575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13.<br>14.<br>Appe | Protoc<br>Study<br>Study<br>Study<br>Langu<br>Compo<br>REFERI<br>APPENI<br>endix A | Termination Documentation and Storage Monitoring age ensation for Injury ENCES Schedule of Procedures List of Laboratory Analytes | 7475757575 |
| 12.1<br>12.2<br>12.3<br>12.4<br>12.5<br>12.6<br>13.<br>14.<br>Appe | Protoc<br>Study<br>Study<br>Study<br>Langu<br>Comp<br>REFERI<br>APPENI<br>endix A<br>endix B | Termination Documentation and Storage Monitoring age ensation for Injury. ENCES Schedule of Procedures List of Laboratory Analytes Pharmacokinetic Sampling Schedule | 7475757575 |

Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit

## **PROTOCOL AMENDMENT**

Protocol Number: ISIS 304801-CS7

Protocol Title: An Open-Label Study of Volanesorsen Administered Subcutaneously to

Patients with Familial Chylomicronemia Syndrome (FCS)

Amendment Number: 8

Amendment Date: 21 November 2018

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 7 dated 7 April 2017:

To add the option for patients to receive a study drug dose reduction as either 300 mg every
two weeks (prefilled syringe) or 150 mg once-weekly (vial presentation), to clarify that
discontinuation from the treatment period will be required for any patients who are on a dose
pause for ≥ 3 months, and to remove the references to landmark visits (if patient stops drug
treatment then they enter the follow-up period).

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 2.3.4<br>Clinical<br>experience | Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebe controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebe). The clinical experience with volanesorsen includes clinical trials in healthy subjects, patients with hypertriglyceridemia, FCS, or familial partial lipodystrophy. Overall, 431 patients and healthy volunteers have taken part in the clinical development program, of whom 325 have received at least 1 dose of volanesorsen. Ninety-five (95) patients with FCS have been enrolled in studies, all showing clinically meaningful reductions in plasma triglyceride. Patients with FCS continue on treatment in the open-label extension (OLE) and triglyceride reductions persist at similar levels as reported in earlier studies. In the completed Phase 1 and Phase 2 studies, volanesorsen was well-tolerated and demonstrated a favorable safety profile. There was no clinical or laboratory evidence of drug-drug interactions despite many patients in the Phase 2 clinical trials receiving | Update to language regarding clinical experience in Phase 1 and 2 studies and incidence of AEs in completed Phase 3 studies and update to language regarding safety risks of Study Drug. |

Drug.

In clinical studies conducted to date volanesorsen has been well tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine. proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50.000/mm3 in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of treatment.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

In the completed pooled Phase 3 studies (ISIS 304801-CS6 (hereafter CS6) and ISIS 304801-CS16 (hereafter CS16), the most common AEs associated with volanesorsen administration were tolerability at the injection site and platelet reductions. The majority of the injection site AEs were mild, none were severe, and the incidence appeared to decrease over time. No deaths have been associated with volanesorsen treatment to date. No cardiac toxicity was associated with volanesorsen treatment. There were no abnormal QTc findings and no study-drug related adjudicated major adverse cardiac events (MACE). There is no evident association between volanesorsen treatment and changes in renal or liver functions.

| In conclusion,t The safety profile of volanesorsen has |
|---------------------------------------------------------------|
| been well-described in this development program, which |
| has identified 3 safety risks: thrombocytopenia (an |
| identified risk), constitutional symptoms (flu-like reactions |
| and influenza-like illness), and injection site reactions (a |
| tolerability signal). Spontaneous, mild to severe |
| thrombocytopenia has been described in the FCS patient |
| population (Gaudet et al. 2017), but is increased by |
| treatment with volanesorsen. Less frequent and less |
| pronounced platelet declines were also observed with |
| volanesorsen treatment in the hypertriglyceridemic (HTG) |
| population of CS16. When fully complied with, frequent |
| monitoring for this effect and appropriate dose |
| adjustments have been successful both in preventing or |
| promptly detecting the occurrence of severe platelet |

## Section 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week and dose reduction to 300 mg every 2 weeks (delivered as either a single 300-mg dose or as 150 mg onceweekly, respectively) are is supported by both the cumulative nonclinical data available to date and the Phase and 3 clinical data.

declines and often in retaining patients on treatment.

Non nonclinical findings were <u>not</u> considered to be related to the pharmacologic inhibition of apoC-III.

Language added to specify dose reductions as either 300 mg every 2 weeks or 150 mg weekly according to patient's tolerability on the 300 mg dose, given similar extents of triglyceride lowering anticipated based on population pharmacokinetic/pharmacodynamic model based simulations.

## Section 3.4.4 Post-Treatment

Patients not participating in the extended treatment period will enter the post-treatment evaluation period-is of 13 weeks and, consists-consisting of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse). Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 (Appendix A).

Language added to specify that patients who discontinue from treatment during treatment period of the study, who previously would have been followed for landmark visits, will now enter into the 13-week follow-up period

## Section 6.1.3 Treatment Period Synopsis, Study Visits and Procedures

Collection and measurement of <u>race and ethnicity</u>, vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A.

To add a specification that race and ethnicity are to be collected.

## Section 6.2.1 Laboratory Assessments

Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), hsCRP and for cytokine analysis.

To add additional laboratory assessments permitted for safety purposes

## Section 7.1 Volanesorsen Description

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS) or in glass vials.

Table 1 Volanesorsen (ISIS 304801) Characteristics

To add details of study drug preparation to be used in the openlabel extension phase

injection

Protocol

| Study Drug | ISIS 304801<br>Prefilled<br>Syringe | <u>ISIS 304801</u><br><u>Vial*</u> |
|---|---|---|
| Strength | <u>300 mg</u> | <u>200 mg</u> |
| Volume /<br>Formulation | 1.5 mL<br>200 mg/mL ISIS<br>304801 | 1.0 mL<br>200 mg/mL ISIS<br>304801 |
| Dose | 300 mg / 1.5 mL | 150 mg / 0.75<br><u>mL</u> |
| Route of | <u>Subcutaneous</u> | <u>Subcutaneous</u> |

Administration

## Section 7.3 Study Drug Accountability

All used syringes <u>or vials</u> must be disposed of as per the site's hazardous waste destruction policy.

injection

Specified disposal of study drug preparation to be used in the openlabel extension phase

### Section 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52, and patients will continue to receive Study Drug as a single 300 mg/1.5 mL injection once-weekly for Weeks 53-104 of the study. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16). will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients on dose reduction will receive either 300 mg/1.5 mL injections every 2 weeks or 150 mg/0.75 mL injections once-weekly. Treatment with a 150 mg dose during the study will use the glass vials containing 200 mg/mL of volanesorsen. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volunesorsen. Treatment Patients should receive 1 dose per week, unless on a dose reduction of 300 mg every 2 weeks, with weeks always defined relative to Study Day 1.

Added language detailing dose reduction options.

## Section 8.5.2 Safety Monitoring for Platelet Count Results

Monitor every 1 week unless otherwise specified. In addition, platelet function may be evaluated at any time during the study by aggregometry, using an approved point-of-care diagnostic device in some patients. This additional functional testing may be performed at selected study centers.

Additional point-of-care platelet function testing may be conducted on patients at participating study centers.

. . .

Due to the 1 to 2-year study duration, it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and treatment where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be

Included an additional blood draw to assess platelet count prior to any travel that would result in missing a weekly monitoring visit.

| | planned with a platelet count drawn within 3-5 days prior to departure and a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming treatment. Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed. | |
|---|---|---|
| 8.5.4 Safety<br>Monitoring for<br>Constitutional<br>Symptoms | Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), hsCRP, and for cytokine analysis. | To add additional laboratory assessments permitted for safety purposes |
| Section 8.6.3<br>Stopping Rules<br>for Platelet<br>Count Results | In the event of any platelet count less than 50,000/mm³, or a platelet count less than 75,000/mm³ that occurs while the patient is treated at 300 mg every 2 weeks or 150 mg once-weekly then treatment of a patient with volanesorsen will be stopped permanently. In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant | To provide clarification to the platelet safety monitoring rules, including dose reduction options. |
| | non-major bleeding (defined below; Schulman et al. 2005), treatment of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to ≥ 100,000/mm³. If desing is continued treatment is reinitiated, it should be at a reduced dose frequency of 300 mg every 2 weeks or 150 mg onceweekly every week(refer to Section 8.7). | |
| | Table 3 Actions in Patients with Low Platelet Count or Drop in Platelet Count | |

| Platelet | | |
|---|---|---|
| Count on | Drug Dose | Monitoring |
| Rx | | |
| | Study Drug | Monitor every 1 |
| | administration is | week unless |
| | contingent on the | otherwise |
| | availability of the | specified |
| | immediately | In addition, |
| | preceding test result. An | platelet function |
| | interpretable | may be evaluated during the study |
| | platelet value | by aggregometry, |
| | must be available | using an |
| | within 7 days prior | approved point- |
| | to treatment. | of-care diagnostic |
| | Only the study | device, in some |
| | doctor or qualified | <u>patients. This</u> |
| | designee can | additional |
| | authorize<br>continued Study | functional testing |
| | Drug | may be<br>performed at |
| | administration | selected study |
| | based on an | centers. |
| | acceptable | Patients on dose |
| | platelet value. | pause should be |
| | Patients should | monitored as per |
| | not administer a | the platelet |
| | dose until they | monitoring rules |
| | have been contacted by their | outlined in |
| | study doctor or | Section 8.8.1 until |
| | designee and told | Study Drug<br>administration is |
| | that it is | resumed. |
| | acceptable to | Obtain additional |
| | dose. | lab tests |
| | Authorization to | (Table 2) if |
| | dose must be | 2 occurrences |
| | documented in | (consecutive or |
| | the patient's medical records. | non-consecutive) |
| | medical records. | of platelet count |
| | | 140K -<br>> 100K/mm <sup>3</sup> or 1 |
| | | occurrence of |
| | | platelet count ≤ |
| | | 100K/mm <sup>3</sup> . Labs |
| | | only need to be |
| | | performed once. |
| | | Labs may be |
| | | collected over |
| | | multiple visits, if |
| | | blood |
| | | requirements are |
| | | a concern, as per<br>Investigator |
| | | discretion. |

| > 100K/mm <sup>3</sup> | Once -weekly 300<br>mg Study Drug<br>administration | |
|---|---|---|
| 100K/mm <sup>3</sup> -<br>> 75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or 150 mg onceweekly. | |
| 75K/mm³ - > 50K/mm³ | weekly. • If occurs | Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| | Medical<br>Monitor | |

| Section 8.7 | ≤ 50K/mm³ | Permanently discontinue Study Drug and the patient will enter the follow up period. | Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management Steroids recommended*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline. Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is < 50K/mm³ if possible ose interruptions, | Addition of dose reduction options |
|---|---|---|---|---|
| Adjustment of Dose Frequency | and/or decreas<br>the dose freque | ing the dose to 150 mency to 300 mg every safety and tolerability. | <u>ig once-weekly</u> or<br><u>2 <del>other</del> weeks</u> will | to allow for safety and tolerability Discontinuation of patients from the |

| Section 8.8 Discontinuation | Patients may be dose paused in response to AEs after consultations with, and the Study Medical Monitor is informed. If a patient is dose paused for ≥ 3 months, he or she is considered to have discontinued treatment and should enter the 13-week post-treatment follow-up period. A patient must permanently discontinue study treatment for any of the following: | study who have been on dose pause and off study drug for >3 months. Added new treatment discontinuation criterion consistent |
|---|---|---|
| of Study<br>Treatment | •The patient is dose-paused for ≥ 3 months then they must discontinue the treatment period and enter the follow-up period. | with other protocol changes. |
| Section 8.8.1<br>Follow-up Visits<br>for Early<br>Termination<br>from Treatment<br>Period | Patients should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26 and 50, 52 of Randomized Treatment period (calculated based on the time elapsed since Day 1) and at Weeks 64, 65, 77, 78 and 102, 104 of OLE period to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits. | Removal of language around landmark visits as patients who stop treatment now enter a post-treatment follow-up period Provides guidance for platelet monitoring in the post-treatment follow-up period. |
| | A patient who discontinues early from treatment with stable platelet counts above the LLN at the time of treatment discontinuation will have platelet counts drawn every 2 weeks after discontinuing Study Drug for the first 6 weeks after the last dose of Study Drug. A subsequent platelet count should then be taken after an additional 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. | |
| Section 13<br>REFERENCES | Gaudet D, Baass A, Tremblay K, et al. Natural History (up to 15 years) of Platelet Count in 84 Patients with Familial Hyperchylomicronemia Due to Lipoprotein Lipase Deficiency. Journal of Clinical Lipidology 2017; 11(3): 797-798. | Addition of reference |
| Section 14<br>APPENDICES | Appendix A Schedule of Procedures Added platelet function analysis to extended treatment period table. Footnote i: Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing. A blood sample for potential gene sequencing may be collected at timepoints other than Screening or Qualification Visits. Footnote g: May be done | Clarification that blood sampling for gene sequencing may occur during the study. Indication that platelet function may be assessed. |
| Section 14 APPENDICES | Appendix B List of Laboratory Analytes Platelet Function Platelet aggregation <sup>3</sup> Platelet function <sup>5</sup> | Addition of laboratory analyte to measure platelet function. |

| Footnote 5: May be done using a point-of-care device on |
|---------------------------------------------------------|
| site. |

## **PROTOCOL SYNOPSIS**

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of treatment and extended treatment with volanesorsen in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing treatment for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical<br/>history. Note: testing of LPL activity should not be performed to<br/>confirm eligibility for the study</li> </ul> |

ISIS 304801-CS7

#### **PROTOCOL SYNOPSIS Continued**

## Study Population Continued

- c. Group 2: Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
  - Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study<u>Inclusion Criteria:</u> Continued
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- Have any new condition or worsening of existing condition which in the opinion
  of the Investigator would make the patient unsuitable for enrollment, or could
  interfere with the patient participating in or completing the study
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)

Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c ≥ 9.0% at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists

#### **PROTOCOL SYNOPSIS Continued**

## Study Population Continued

- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening <u>Exclusion</u> <u>Criteria for Group 3</u> (patients who did not participate in an index study) <u>Continued</u>
- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Platelet count < lower limit of normal (LLN) for the central laboratory (i.e., < 140,000/mm³)
- d. Cardiac Troponin I > ULN at Screening
- e. LDL-C > 130 mg/dL at Screening
- f. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B

| | Malignancy within 5 years, except for basal or squamous cell reinoma of the skin or carcinoma <i>in situ</i> of the cervix that has been excessfully treated |
|---|---|
| with | Treatment with another investigational drug, biological agent, or device hin 1 month of screening, or 5 half-lives of investigational agent, whichever onger |
| | clusion Criteria for Group 3 (patients who did not participate in an index dy) Continued |
| 13. | Unwilling to comply with lifestyle requirements (Section 6.3) |
| 14. | Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to screening and dose and<br>regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>screening</li> </ul> |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor |
| | d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study |
| | e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to screening |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br>apixaban) unless on a stable dose for at least 4 weeks prior to<br>screening and regular clinical monitoring is performed |
| | <ul> <li>Tamoxifen, estrogens or progestins unless on a stable dose for at<br/>least 4 months prior to screening and dose and regimen expected to<br/>remain constant during the treatment period</li> </ul> |
| | i. Plasma apheresis within 4 weeks prior to screening or planned during the study |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>Any other medication unless stable at least 4 weeks prior to screening<br/>(Occasional or intermittent use of over-the-counter medications will be<br/>allowed at Investigator's discretion)</li> </ul> |
| 15. | Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening |
| 16. | Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| 17. | Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |

| Treatment Group | Volanesorsen 300 mg once per week |
|---|---|
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 and 3 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this openlabel study of FCS patients. |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or<br/>ISIS 304801-CS16 index study): A qualification period of up to<br/>2 weeks (unless approved by the Sponsor). Please refer to<br/>Section 4.1 and Appendix A</li> </ul> |
| | Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A |
| | All patients: |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | <ul> <li>Option to participate in an extended treatment period (up to an<br/>additional 52 weeks)</li> </ul> |
| | <ul> <li>A 13-week post-treatment evaluation period or expanded<br/>access program</li> </ul> |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of race and ethnicity, vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option of participating in an expanded |

| | access program or continuing treatment for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. |
|---|---|
| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation,<br/>urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high- density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) </li> </ul> |
| | Change in blood viscosity (may be evaluated) |
| | <ul> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> </ul> |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic |

| | parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
|---|---|
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Akcea Therapeutics, Inc. |
| Collaborator | Ionis Pharmaceuticals, Inc. |

#### STUDY DESIGN AND TREATMENT SCHEMA



# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 8 Protocol 21 November 2018

## **STUDY GLOSSARY**

| Abbreviation/Acronym | <u>Definition</u> |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| ароВ | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | glycosylphosphatidylinositol-anchored hdl-binding protein 1 |
| HAPI | heritability and phenotype intervention |
| HbA1c | glycated hemoglobin |
| HDL | high-density lipoprotein |
| HDL-C | high-density lipoprotein-cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | intermediate density lipoprotein |
| IEC | Independent Ethics Committee |

IM immunogenicity

Index Studies ISIS 304801-CS6 and ISIS 304801-CS16

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL low-density lipoprotein

LDL-C low-density lipoprotein-cholesterol

LMF1 lipase maturation factor 1

LPL lipoprotein lipase

MACE major acute cardiovascular event

MOE 2'-O-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL no-observed-adverse-effect level

non-HDL-C non-high-density lipoprotein-cholesterol

OTC over the counter PFS prefilled syringe PD pharmacodynamic PΚ pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL triglyceride-rich lipoproteins

ULN upper limit of normal

VLDL very-low-density lipoprotein

VLDL-C very-low-density lipoprotein-cholesterol

VLDL-TG lipoprotein-triglyceride
WMA World Medical Association

## 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of treatment and extended treatment with volanesorsen in patients with familial chylomicronemia syndrome.

## 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V (APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1

(LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

## 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

### 2.3 Volanesorsen

## 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing. The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III

mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

## 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volanesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volanesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'alkoxy: RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volanesorsen is shown

## 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species,

including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

## 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure. A summary is included below.

The clinical experience with volanesorsen includes clinical trials in healthy subjects, patients with hypertriglyceridemia, FCS, or familial partial lipodystrophy. Overall, 431 patients and healthy volunteers

have taken part in the clinical development program, of whom 325 have received at least 1 dose of volanesorsen. Ninety-five (95) patients with FCS have been enrolled in studies, all showing clinically meaningful reductions in plasma triglyceride. Patients with FCS continue on treatment in the open-label extension (OLE) and triglyceride reductions persist at similar levels as reported in earlier studies.

In the completed Phase 1 and Phase 2 studies, volanesorsen was well-tolerated and demonstrated a favorable safety profile. There was no clinical or laboratory evidence of drug-drug interactions despite many patients in the Phase 2 clinical trials receiving concomitant medications that are known to be associated with elevations in hepatic enzymes, such as fibrates and statins. There were no volanesorsenassociated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). There was a reduction (mean reduction < 30%) in platelets in volanesorsen vs. placebo with mean nadirs for all doses remaining above the lower limit of normal (LLN). The most frequently reported adverse events (AEs) were mild, non-progressive events at the injection site. In Phase 2, a single serious adverse event (SAE) of secondary serum sickness-like reaction was reported as related to Study Drug. All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the treatment period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In the completed pooled Phase 3 studies (ISIS 304801-CS6 (hereafter referred to as CS6) and ISIS 304801-CS16 (hereafter referred to as CS16), the most common AEs associated with volanesorsen administration were tolerability at the injection site and platelet reductions. The majority of the injection site AEs were mild, none were severe, and the incidence appeared to decrease over time. No deaths have been associated with volanesorsen treatment to date. No cardiac toxicity was associated with volanesorsen treatment. There were no abnormal QTc findings and no study-drug related adjudicated major adverse cardiac events (MACE). There is no evident association between volanesorsen treatment and changes in renal or liver functions.

The safety profile of volanesorsen has been well-described in this development program, which has identified 3 safety risks: thrombocytopenia (an identified risk), constitutional symptoms (flu-like reactions and influenza-like illness), and injection site reactions (a tolerability signal). Spontaneous, mild-to-severe thrombocytopenia has been described in the FCS patient population (Gaudet et al. 2017) but is increased by treatment with volanesorsen. Less frequent and less pronounced platelet declines were also observed with volanesorsen treatment in the hypertriglyceridemic (HTG) population of CS16. When fully complied with, frequent monitoring for this effect and appropriate dose adjustments have been successful both in preventing and promptly detecting the occurrence of severe platelet declines and often in retaining patients on treatment.

## 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week and dose reduction to 300 mg every 2 weeks (delivered as either a single 300 mg dose or as 150 mg once-weekly, respectively) are supported by both the cumulative nonclinical data available to date and the Phase 2 and 3 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. Nonclinical findings were not considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volunesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-

modified ASOs that have been administered intravenously and subcutaneously in multiple clinical studies at doses up to 1200 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

### 3. EXPERIMENTAL PLAN

## 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing treatment for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period.

### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

## 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

## 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

## 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

## 3.4.3 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures
(Appendix A). During the treatment period, volanesorsen is administered by SC injection once weekly.treatmenttreatment

#### 3.4.4 **Post-Treatment**

Patients not participating in the extended treatment period will enter the post-treatment evaluation period of 13 weeks, consisting of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse). Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 (Appendix A).

Amendment 8

#### 3.5 **End-of-Study**

The End-of-Study is last patient, last visit.

#### 3.6 **Data and Safety Monitoring Board**

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. **PATIENT ENROLLMENT**

#### 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is reconsented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

## 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

## 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age ≥ 18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.
  - Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:
  - a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
  - b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
    - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
    - Post heparin plasma LPL activity of ≤ 20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study
  - c. Group 2: Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
    - Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study

# 5. Satisfy 1 of the following:

- a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

# Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c ≥ 9.0% at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening

- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be
       ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN

## b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Platelet count < LLN for the central laboratory (i.e., < 140,000/mm<sup>3</sup>)
- d. Cardiac Troponin I > ULN at Screening
- e. LDL-C > 130 mg/dL at Screening
- f. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1

- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to screening
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to screening or planned during the study
  - j. Prior exposure to ISIS 304801
  - Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)

Amendment 8

Protocol

17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

### 6. STUDY PROCEDURES

# 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

# 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

### 6.1.3 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly treatment schedule for safety reasons (Section 8.1). Collection and measurement of race and ethnicity, vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as AEs. Dietary counseling will be reinforced at intervals throughout the treatment and followup period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Treatment instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

### 6.1.4 Extended Treatment Period

Patients will have the option of continuing treatment for up to an additional 52 weeks until an expanded access program is approved and available in their country.

During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly treatment schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Treatment instructions and training will be provided to the patient where applicable.

# 6.1.5 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after treatment on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

# 6.1.6 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of participating in an expanded access program or continuing treatment for up to an additional 52 weeks until an expanded access program is approved and available in their country as described in Section 6.1.4. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. This 13-week post-treatment evaluation period consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A. Patients who complete, or terminate early from, the extended

treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A.

# 6.2 Additional Study Assessments

# 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), hsCRP and for cytokine analysis.

# 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

# 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll-over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

# 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65. Patients in the Extended Treatment Period will have ECGs performed in triplicate at Week 76 and Week 104.

## 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

## 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period (Week 65).

# 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service. Patients in the Extended Treatment Period will receive diet/alcohol counseling by qualified study personnel at clinic visits only.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet may be conducted randomly during the treatment and post treatment follow-up periods.

## 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

# 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2 and 3)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

# 6.3 Restriction on the Lifestyle of Patients

# 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent<sup>†</sup> or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

# For male patients:

Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or
the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients
must also encourage their female partner to use effective contraception from the time of
signing the informed consent until 3 months after the patient's last dose of study treatment.
Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal
ligation), hormonal contraception, intrauterine contraception/device, or barrier methods
(female condom\*, diaphragm, sponge, cervical cap) together with spermicidal
foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use
condoms to ensure that the fetus is not exposed to the Study Drug.

# For female patients:

- Using 1 or more of the following acceptable methods of contraception: surgical sterilization
  (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any
  2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or
  cervical cap) together with spermicidal foam/gel/film/cream/suppository.
- \* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

† Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq$  20 g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

# 7. STUDY DRUG

# 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS) or in glass vials. Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 to 8°C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Study Drug | ISIS 304801 Prefilled Syringe | ISIS 304801 Vial |
|---|---|---|
| Strength | 300 mg | 200 mg |
| Volume / Formulation | 1.5 mL<br>200 mg/mL ISIS 304801 | 1.0 mL<br>200 mg/mL ISIS 304801 |
| Dose | 300 mg / 1.5 mL | 150 mg / 0.75 mL |
| Route of Administration | Subcutaneous injection | Subcutaneous injection |

# 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

# 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes or vials must be disposed of as per the site's hazardous waste destruction policy.

### 8. TREATMENT OF PATIENTS

## 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52, and patients will continue to receive Study Drug as a single 300 mg/1.5 mL injection once-weekly for Weeks 53-104 of the study. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients on dose reduction will receive either 300 mg/1.5 mL injections every 2 weeks or 150 mg/0.75 mL injections once-weekly. Treatment with a 150 mg dose during the study will use the glass vials containing 200 mg/mL of volanesorsen.

Patients should receive 1 dose per week, unless on a dose reduction of 300 mg every 2 weeks, with weeks always defined relative to Study Day 1. For example, if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if treatment on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

# 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs.

## 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

## 8.4 Treatment Precautions

There are no specific treatment precautions required for this study.

# 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring, baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

Protocol

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

Confirmation Guidance: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below must be confirmed by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest must be available prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-treatment Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon re-test may continue treatment. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

Frequency of Repeat Measurements: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become ≤ 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels  $> 3 \times 10^{-5}$  X ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was  $> 10^{-5}$  ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

# 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified. In addition, platelet function may be evaluated at any time during the study by aggregometry, using an approved point-of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers.

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to treatment. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 2-year study duration, it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and treatment where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a platelet count drawn within 3-5 days prior to departure and a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming treatment.

Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 8 Protocol 21 November 2018

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm³ (x1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

# 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae,

gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

# 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms, should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

Should a patient experience constitutional or flu-like symptoms after Study Drug administration, investigators may consider additional laboratory assessments. For example, plasma and serum samples may be drawn for complement (Total C3, C4, C5a and Bb), hsCRP, and for cytokine analysis.

# 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

<u>All patients on insulin</u> will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to
evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values
as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

<u>All diabetic patients</u> will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).

Protocol

Amendment 8

O Any changes in insulin dose or oral antidiabetic therapy should be captured into the

# 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

Concomitant Medication CRF.

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

# 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c ≥ 8 and < 9%)</li>

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

An FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

# 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, treatment with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued treatment and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

## 8.6 Stopping Rules

For the purposes of stopping rules, baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, treatment of a patient with volunesorsen

will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

1. ALT or AST > 8 x ULN, which is confirmed

Protocol

- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, treatment of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq$  0.3 mg/dL (26.5  $\mu$ mol/L) and  $\geq$  40% above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible treatment re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator **in consultation with** the Sponsor Medical Monitor or designee.

# 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), treatment of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 50,000/mm<sup>3</sup>, or a platelet count less than 75,000/mm<sup>3</sup> that occurs while the patient is treated at 300 mg every 2 weeks or 150 mg once-weekly then treatment of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or

# Methylprednisolone 30 mg/kg/day for 7 days

(**note:** may require continuation with oral steroids after methylprednisolone). Triglyceride levels will be monitored weekly, and AE monitoring will continue, during cortiscosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), treatment of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to > 100,000/mm³. If treatment is reinitiated it should be at a reduced dose frequency of 300 mg every 2 weeks or 150 mg once-weekly (refer to Section 8.7). The suitability of the patient for continued treatment will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of treatment.

If after the first treatment re-challenge the platelet count again falls below 75,000/mm<sup>3</sup>, then treatment of the patient with Study Drug will be stopped permanently.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

# Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma > 25 cm<sup>2</sup>
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

 Table 3
 Actions in Patients with Low Platelet Count or Drop in Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to treatment. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified In addition, platelet function may be evaluated during the study by aggregometry, using an approved point-of-care diagnostic device, in some patients. This additional functional testing may be performed at selected study centers. Patients on dose pause should be monitored as per the platelet monitoring rules outlined in Section 8.8.1 until Study Drug administration is resumed. Obtain additional lab tests (Table 2) if 2 occurrences consecutive or nonconsecutive) of platelet count 140K -> 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. |
| > 100K/mm <sup>3</sup><br>100K/mm <sup>3</sup> - >75K/mm <sup>3</sup> | Once-weekly 300 mg Study Drug administration Permanently reduce dose frequency to 300 mg every 2 weeks or 150 mg | |
| 75K/mm³ - >50K/mm³ | If occurs while on dose of 300 mg every 2 weeks or 150 mg once-weekly then permanently discontinue Study Drug, otherwise dose pause. If dose pause is ≥ 3 months then patient must discontinue treatment and enter the follow up period. When platelet count returns to > 100K/mm³ restart treatment at dose frequency of 300 mg every 2 weeks or 150 mg once-weekly in consultation with the Sponsor Medical Monitor | Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| ≤ 50K/mm³ | Permanently discontinue Study Drug and the patient will enter the follow up period | <ul> <li>Monitor daily until 2 successive values<br/>show improvement then monitor every<br/>2-3 days until 2 successive values are<br/>&gt; 75K/mm³ then monitor every 1 week</li> </ul> |
| | | <ul> <li>Patient should be evaluated by a<br/>hematologist to provide diagnostic and<br/>therapeutic management</li> </ul> |
| | | <ul> <li>Steroids recommended*. It is strongly<br/>recommended that, unless the patient<br/>has a medical contraindication to<br/>receiving glucocorticoids, the patient<br/>receives glucocorticoid therapy to<br/>reverse the platelet decline.</li> </ul> |
| | | <ul> <li>Monitor triglyceride levels weekly and<br/>continue AE monitoring during steroid<br/>therapy</li> </ul> |
| | | Discontinue antiplatelet agents/<br>NSAIDS/ anticoagulant medication while<br>platelet count is < 50K/mm³ if possible |

Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or methylprednisolone 30 mg/kg/day for 7 days (**note**: may require continuation with oral steroids after methylprednisolone)

# 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose to 150 mg once-weekly or the dose frequency to 300 mg every 2 weeks will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs, and the Study Medical Monitor is informed. If a patient is dose paused for  $\geq$  3 months, he or she is considered to have discontinued treatment and should enter the 13-week post-treatment follow-up period.

# 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4.
- The patient withdraws consent.
- The patient experiences an AE that necessitates permanent discontinuation of study treatment.
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6.
- The patient is dose paused for ≥ 3 months.

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

# 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug.

A patient who discontinues early from treatment with stable platelet counts above the LLN at the time of treatment discontinuation will have platelet counts drawn every 2 weeks after discontinuing Study Drug for the first 6 weeks after the last dose of Study Drug. A subsequent platelet count should then be taken after an additional 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

# 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 65 or Week 117 if terminating from the Extended Treatment Follow-Up Period), see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance

# Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent, every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

# 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

# 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

# **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including over-the-counter preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

# 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 (or Week 117 if patient enters the extended treatment period) visit.

## **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

# 8.11 Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volanesorsen. Patients that are self-administering volanesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

## 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

# 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

# 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6 (R2). Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4

Amendment 8

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 **Definitions**

#### 9.3.1 Adverse Event

An adverse event is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

# 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

# 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

# 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

# 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

# 9.4.3.1 Relationship to the Study Drug

The event's relationship to volanesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volanesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- Not Related: The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

# *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- Mild: The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- Moderate: The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in <u>Section 9.3.3</u>).

### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Treatment was temporarily interrupted or delayed due to the AE and restarted at the same dose

• Reduced schedule: Treatment frequency was reduced

# 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

# 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- Recovered: Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

# 9.5 Procedures for Handling Special Situations

## 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying

diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 **Treatment Errors**

Volanesorsen treatment errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Treatment details should be captured on the Treatment Case Report Form. If the patient takes a dose of volanesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

Should an overdose occur, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 **Contraception and Pregnancy**

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24

hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 **Study Endpoints**

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 **Efficacy Endpoints**

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

# 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs
- Platelet aggregation (may be evaluated)

# 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

# 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

### 10.4 Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification). For Group 3 patients, the baseline for fasting lipid measurements is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 in this open-label study.

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study and Group 3 patients, baseline will be the last non-missing assessment prior to the first dose of Study Drug.

## 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

# 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naive group which including patients on placebo in index studies and Group 3 patients. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

# 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

# 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

#### 10.6.3 **Efficacy Analysis**

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG ≥ 40% reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### **Pharmacokinetic Analysis** 10.6.4.1

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volanesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24h</sub> /F) will be calculated from

CL<sub>0-24h</sub>/F = Actual Dose/AUC<sub>0-24h</sub>. Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,

 $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-

time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

# 10.6.4.2 Immunogenicity Analysis

Protocol

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

# 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.
The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH E6 (R2) Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH E6 (R2) Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

Protocol 21 November 2018

Amendment 8

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of ICH E6 (R2), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of prestudy documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

Amendment 8

#### 12.4 **Study Monitoring**

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH E6 (R2) and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH E6 (R2), and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 **Compensation for Injury**

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in

# ISIS 304801-CS7 **CONFIDENTIAL** Amendment 8 Protocol 21 November 2018

accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Gaudet D, Baass A, Tremblay K, et al. Natural History (up to 15 years) of Platelet Count in 84 Patients with Familial Hyperchylomicronemia Due to Lipoprotein Lipase Deficiency. Journal of Clinical Lipidology 2017; 11(3): 797-798.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PC, Voshol PJ, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

# ISIS 304801-CS7 CONFIDENTIAL Amendment 8 Protocol 21 November 2018

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

#### 14. APPENDICES

### Appendix A Schedule of Procedures

Appendix A **Schedule of Procedures** 

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | Trea | ıtmen | t Perio | od | | | | | | | | | Tre | Post<br>atme | ent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <b>.</b> | -8 to | -2 to | W | /k | Wk | Wk | Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| | Study Week | -2 | -1 | <i>'</i> | 1 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | | 65 |
| | Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 44<br>9 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| In | formed Consent | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| | utpatient Visit | Х | Х | Χ | XI | Χ <sup>I</sup> | XI | Χ <sup>I</sup> | Χ <sup>I</sup> | Χ <sup>l</sup> | Х | ΧI | XI | Χ <sup>I</sup> | ΧI | Χ | Χ <sup>I</sup> | Χ <sup>I</sup> | Χ <sup>I</sup> | Χ | Χ <sup>I</sup> | ΧI | ΧI | Χ <sup>I</sup> | Х | Χ <sup>I</sup> | XI | Х |
| | clusion/Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| | edical History <sup>ь</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | tal Signs + body weight<br>height on Day 1 only) | Х | Х | х | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| | nysical Examination | Х | | Х | | | | | | | Х | | | | | Χ | | | | Χ | | | | | Х | | | Х |
| 12 | 2- lead ECG (triplicate) | Х | | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | | Х |
| М | RI (liver/spleen) | Х | | | | | | | | | | | | | | | | | | | | | | | X <sup>m</sup> | | | |
| Ed | chocardiography | Х | | | | | | | | | | | | | | Xm | | | | | | | | | X <sup>m</sup> | | <u> </u> | |
| | Chemistry Panel | Х | Х | Χ | | Χ | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Χ | | Χ | Х |
| | CBC with Differential <sup>c</sup> | Х | х | <b>←</b> | | F | Platel | ets ar | e ass | essec | d each | calen | dar w | eek, v | isits d | — X<br>o not h | nave sp | ecifie | d wind | ows t | o allov | v flexi | bility c | of sche | duling. | | <b>→</b> | х |
| | Serum Lipid Panel | Х | Х | Х | | Χ | | Χ | | Х | Х | | | | Х | Χ | | | | Χ | | | | Х | Х | | | Х |
| ъ. | Blood viscosity <sup>e</sup> | | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | |
| na | Platelet aggregation <sup>e</sup> | | Х | Х | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | |
| (Fastina) <sup>d</sup> | Coagulation (aPTT, PT, INR) | Х | Х | | | | | Χ | | | Х | | | | | Χ | | | | Χ | | | | | Х | | | |
| Ē | Hepatitis B, C, HIV | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Draw | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | HbA1c | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Blood | Sedimentation Rate | | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Ιĕ | Complement (C5a, Bb) | | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| 1 | Troponin I | Х | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| 1 | Platelet Bound Autoantibodiese | | | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| | Plasma PK - Volanesorsen | | | Xn | Х | Х | Ī | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| 1 | Anti-Volanesorsen Antibodies | | | Х | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | Trea | tmen | t Perio | od | | | | | | | | | Tre | Post<br>atme<br>low- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Charles March | -8 to | -2 to | W | /k | Wk | Wk | Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mon | th 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| Study Week | -2 | -1 | 1 | 1 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 44<br>9 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| FSH (women only, if applicable) | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Serum Pregnancy Test <sup>f</sup> | Х | Х | | | Х | | Х | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Χ | | Χ | Х |

### Appendix A Schedule of Procedures Continued

| | Study Period | Screen/<br>Run Inª | Quala | | | | | | | | | | Tre | eatm | ent F | Period | | | | | | | | | | | Treat | ment<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | -8 to<br>-2 | -2 to<br>-1 | V | Vk<br>1 | Wk<br>4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | Mon | th 3 | Wk<br>15<br>&<br>17 | Wk<br>19 | Wk<br>21<br>&<br>23 | | nth 6 | Wk<br>28<br>&<br>30 | Wk<br>32 | Wk<br>34<br>&<br>36 | Wk<br>38 | Wk<br>40<br>&<br>42 | WI<br>44 | | Мо | nth 12 | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 |
| | | | | | | | | | | Wk<br>12 | Wk<br>13 | | | | Wk<br>25 | Wk<br>26 | | | | | | | | Wk<br>50 | Wk 52<br>or ET | | | |
| | Study Day | -56 to<br>-15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 30 | 316<br>2 &<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| ~ ~ | Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 3; Group 2 if not available from index study) | | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| B ( | Archived Serum & Plasma<br>Samples <sup>9</sup> | | | Х | | | | Х | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| | alysis <sup>d</sup> | Х | Χ | Χ° | | Χ | | Χ | | | Χ° | | Χ° | | | Χ° | | Χ° | | Χ° | | X | | | Χ° | | Χ° | Χ° |
| | dus Photography <sup>h</sup> | Х | | | | | | | | | | | | | | | | | | | | 1 | 1_ | | X <sup>m</sup> | | | 1 |
| | etic testing for FCS diagnosis (if<br>available in medical history) <sup>i</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Once | e-weekly Study Drug: SC Injection | | | Х | | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | | | |
| Sym | ptom Diary (weekly) | Х | Χ | Χ | | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | Χ | Χ | Х |

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | Tre | eatm | ent F | Period | | | | | | | | | | | Treat | ment<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | -8 to<br>-2 | -2 to<br>-1 | W | /k<br>1 | Wk<br>4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | | nth 3 | Wk<br>15<br>&<br>17 | Wk<br>19 | Wk<br>21<br>&<br>23 | | nth 6 | Wk<br>28<br>&<br>30 | Wk<br>32 | Wk<br>34<br>&<br>36 | Wk<br>38 | Wk<br>40<br>&<br>42 | Wk<br>44 | Wk<br>46<br>&<br>48 | Mor | nth 12 | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 |
| | | | | | | | | | Wk<br>12 | Wk<br>13 | | | | Wk<br>25 | Wk<br>26 | | | | | | | | Wk<br>50 | Wk 52<br>or ET | | | |
| Study Day | -56 to<br>-15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Quality of Life Assessment(s) | | | Χ | | | | | | | Χ | | | | | Х | | | | | | | | | Χ | | | Х |
| Food/Drink Diary (quarterly) <sup>j</sup> | | | Х | | | | | | | Χ | | | | | Х | | | | | | | | | Χ | | | Х |
| Diet/Alcohol Counseling <sup>k</sup> | Х | Χ | Х | | Х | | Х | | | Χ | | | | | Х | | | | Х | | | | | Χ | | Х | Х |
| Adverse Events | Х | Χ | Χ | | Χ | Χ | Χ | Х | Х | Х | Х | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Х | Х |
| Concomitant Medication | Х | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х |

- a Screening and Qualification (Group 3) procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor

#### Appendix A Schedule of Procedures Continued

#### Legend Text Continued

- d Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- e May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- h If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- i Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing. A blood sample for potential gene sequencing may be collected at timepoints other than Screening or Qualification Visits.
- In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- k To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- I Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- m A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- n Full or abbreviated PK profile (see Appendix C)
- Expanded urinalysis (see Appendix B)

| | Study Period | | | | | | | ٦ | Freatme | ent Perio | od | | | | | | | | -Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | | Mo 15<br>Wk 64 | Wk 66<br>& 68 | Wk<br>70 | | Mo 18<br>Wk 76 | | | Wk 84,<br>86, & 88 | | | Wk<br>96 | Wk<br>98,<br>100 &<br>102 | Mo 24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | Wk<br>110 | Mo 27<br>Wk<br>117 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 56<br>8 | 582, 596<br>& 610 | 624 | 638 &<br>652 | 666 | 680,<br>694 &<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Out | tpatient Visit | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | Х |
| Vita | al Signs (+ body weight) | | | | Χ | | | | Χ | | | | Х | | | | Х | | | Х |
| | sical Examination | | | | | | | | Χ | | | | | | | | Х | | | |
| - | lead ECG (triplicate) | | | | | | | | Х | | | | | | | | Х | | | |
| Uri | nalysis(including P/C ratio) | | Χ | | Х | | Χ | | Χ | | Χ | | Х | | Χ | | Х | | Χ | Х |
| | Chemistry Panel | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | Χ |
| | CBC with Differential <sup>a</sup> | ◀ | Plate | elets are | assess | ed each | caler | ndar wee | ek, visits | — X<br>do not | —<br>have | specified | window | s to allo | w flex | ibility of | schedul | ing. | <b></b> | Х |
| Draw (Fasting) <sup>b</sup> | Serum Lipid Panel | | | | Х | | | | Χ | | | | Х | | | | Х | | | Х |
| -asti | Coagulation (aPTT, PT, INR) | | | | Х | | | | Х | | | | Х | | | | Х | | | |
| ₹ | Troponin I | | | | Х | | | | Х | | | | Х | | | | Х | | | Х |
| Dra | Plasma PK - ISIS 304801° | | | | | | | | Х | | | | | | | | Х | | | Х |
| Blood | Anti-ISIS 304801 Antibodies | | | | | | | | Х | | | | | | | | Х | | | Х |
| B | Serum Pregnancy Test <sup>d</sup> | | Χ | | Х | | Х | | Χ | | Χ | | Х | | Х | | Х | | Х | Х |
| | Platelet Function <sup>g</sup> | • | | May b | e asses | sed at v | arious | s timepo | ints, visi | its do no | • - | ve specifie | d windo | ws to al | low fle | exibility | of sched | uling. | | <b>→</b> |
| | ce-weekly Study Drug: SC | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | |
| Die | t/Alcohol Counseling <sup>e</sup> | | | | Х | | | | Х | | | | Х | | | | Х | | | |
| Ad۱ | erse Events | Х | Χ | Х | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Χ | Х | Х | Χ | Χ | Х |

| Study Period | | | | | | | 7 | Γreatme | ent Perio | od | | | | | | | | t-Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Wk 54<br>& 56 | Wk<br>58 | | | | | | | | | Wk 84,<br>86, & 88 | | | | Wk<br>98,<br>100 &<br>102 | Mo 24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | Wk<br>110 | Mo 27<br>Wk<br>117 |
| Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 56<br>8 | 582, 596<br>& 610 | 624 | 638 &<br>652 | 666 | 680,<br>694 &<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Concomitant Medication | Х | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Χ |

#### Appendix A Schedule of Procedures – Extended Treatment Period Continued

#### Legend Text

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before treatment can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor.
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- g May be done

## **Appendix B** List of Laboratory Analytes

#### Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volanesorsen or other similar oligonucleotides.

| Clinica | al Chemistry Panel | Screening Tests (Group 3) | Hematology | <u>Urinalysis</u> |
|---|---|---|---|---|
| • | Sodium | Hepatitis B surface | <ul> <li>Red blood cells</li> </ul> | • Color |
| • | Potassium | antigen | <ul> <li>Hemoglobin</li> </ul> | <ul> <li>Appearance</li> </ul> |
| • | Chloride | <ul> <li>Hepatitis C antibody</li> </ul> | <ul> <li>Hematocrit</li> </ul> | <ul> <li>Specific gravity</li> </ul> |
| • | Bicarbonate | <ul> <li>HIV antibody</li> </ul> | <ul> <li>MCV, MCH, MCHC</li> </ul> | • pH |
| • | Total protein | <ul> <li>FSH (women only)</li> </ul> | <ul> <li>Platelets</li> </ul> | <ul> <li>Protein</li> </ul> |
| • | Albumin | <ul> <li>Serum βhCG (women</li> </ul> | <ul> <li>White blood cells</li> </ul> | <ul> <li>Blood</li> </ul> |
| • | Calcium | only) | WBC Differential (% and | <ul> <li>Ketones</li> </ul> |
| • | Magnesium | | absolute) | <ul> <li>Urobilinogen</li> </ul> |
| • | Phosphorus | Coagulation | <ul> <li>Neutrophils</li> </ul> | <ul> <li>Glucose</li> </ul> |
| • | Glucose | aPTT (sec) | <ul> <li>Eosinophils</li> </ul> | • Bilirubin |
| • | BUN | PT (sec) | <ul> <li>Basophils</li> </ul> | Leukocyte esterase |
| • | Creatinine | • INR | <ul> <li>Lymphocytes</li> </ul> | <ul> <li>Nitrate</li> </ul> |
| • | Uric Acid | Linial Daniel | <ul> <li>Monocytes</li> </ul> | <ul> <li>Microscopic</li> </ul> |
| • | Total bilirubin | <u>Lipid Panel</u> | | examination <sup>4</sup> |
| • | Direct (conjugated) | <ul><li>Total Cholesterol</li><li>LDL-C</li></ul> | Pharmacokinetics <sup>1</sup> | |
| | bilirubin | HDL-C | & Immunogenicity | Additional Measures for |
| • | Indirect (unconjugated) | Triglycerides | <ul> <li>Volanesorsen levels in<br/>plasma</li> </ul> | Expanded Urinalysis |
| | bilirubin | Non-HDL-C | Anti-volanesorsen | <ul> <li>Total protein<br/>(quantitative)</li> </ul> |
| • | ALT | VLDL-C | antibodies in plasma | Microalbumin |
| • | AST | <ul> <li>apoA-1</li> </ul> | | β2-microglobulin |
| • | Alkaline phosphatase | <ul><li>apoA-1</li><li>apoB</li></ul> | Other Assessments | p2 meroglobami |
| | | apob apoC-III | <ul> <li>hsCRP</li> </ul> | Platelet Function |
| | | Ф арос-пі | Sedimentation Rate | <ul> <li>Platelet aggregation<sup>3</sup></li> </ul> |
| | | | • C5a, Bb | <ul> <li>Platelet Function<sup>5</sup></li> </ul> |
| | | | • Troponin I <sup>2</sup> | |
| | | | • CK-MB <sup>2</sup> | |
| | | | <ul> <li>Platelet Bound</li> </ul> | |
| | | | Autoantibodies <sup>3</sup> | |
| ĺ | | | <ul> <li>De-lipidated free</li> </ul> | |
| | | | glycerol | |
| | | | <ul> <li>HbA1c, FPG</li> </ul> | |
| i | | | <ul> <li>Blood viscosity<sup>3</sup></li> </ul> | |

- Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified
- 5 May be done using a point-of-care device on site

Amendment 8

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to treatment, and at various times throughout the treatment and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

#### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

#### **PK Sampling Schedule (Extended Treatment Period)**

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|-----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose, | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm <sup>3</sup> ;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160<br>mg/dL; Fasting glucose value >ULN -<br>8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | ÷ | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | U | rine | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





A subsidiary of Ionis Pharmaceuticals, Inc.

**Sponsor:** Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

### ISIS 304801-CS7

### The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 8 - France – 10 April 2017** 

EudraCT No: 2015-003755-21

### ISIS 304801-CS7

### The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

### An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

### Protocol Amendment 8 - France - 10 April 2017

#### **Protocol History:**

Original Protocol: 28 August 2015 Protocol Amendment 1: 2 February 2016 Protocol Amendment 2: 22 April 2016 9 May 2016 Protocol Amendment 3: 6 June 2016 Protocol Amendment 4: Protocol Amendment 5: 19 August 2016 Protocol Amendment 6: 16 September 2016 Protocol Amendment 7: 3 February 2017

#### Sponsor:

Ionis Pharmaceuticals, Inc.
2855 Gazelle Court
Carlsbad, CA 92010

MD, MBA

#### **Ionis Protocol Number: ISIS 304801-CS7**

**Protocol Amendment 8 - France** 

**EudraCT No: 2015-003755-21** 

Clinical Phase: 3

### The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

### An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200 Fax:

**Key Sponsor Contact:** 

Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 10 April 2017

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | • | planesorsen Administered Subcutaneously to omicronemia Syndrome (FCS) |
| Amendment: | Amendment 8 - France | |
| Date: | 10 April 2017 | |
| Open-Label Study of | f Volanesorsen Administered | and the attached clinical protocol, entitled "An Subcutaneously to Patients with Familial ril 2017, and agree to conduct the study as |
| I agree to comply wi<br>Good Clinical Practic | | e on Harmonization Tripartite Guideline on |
| any purpose other that | | contained in this document will not be used for f the clinical investigation without the prior |
| | | _ |
| Investigator's Signa | ture | |
| Investigator's Name | : (please print) | Date (DD Month YYYY) |

### **TABLE OF CONTENTS**

| DD O | <b></b> | | Page |
|---|---|---|---|
| | | OL AMENDMENT | |
| | | OL SYNOPSIS | |
| | | ESIGN AND TREATMENT SCHEMA | |
| | | LOSSARY | |
| 1. | | JECTIVES | |
| <b>2.</b> 2.1 | | CKGROUND AND RATIONALE | |
| | | verview of Disease | |
| 2.2 | | herapeutic Rationale | |
| _ | v<br>2.3.1 | Mechanism of Action | |
| | 2.3.1 | Chemistry | |
| | 2.3.2 | Preclinical Experience | |
| | 2.3.4 | Clinical Experience | |
| 2.4 | | ationale for Dose and Schedule of Administration | |
| 3. | | PERIMENTAL PLAN | |
| 3.1 | | tudy Design | |
| 3.2 | | umber of Study Centers | |
| 3.3 | | umber of Patients | |
| 3.4 | | verall Study Duration and Follow-up | |
| | 3.4.1 | Qualification | |
| | 3.4.2 | Treatment | |
| | 3.4.3 | Post-Treatment | 35 |
| 3.5 | E: | nd-of-Study | 35 |
| 3.6 | | ata and Safety Monitoring Board | |
| 4. | PAT | TIENT ENROLLMENT | 36 |
| 4.1 | Q | ualification | 36 |
| 4.2 | 2 E | nrollment | 36 |
| <b>5.</b> | PAT | FIENT ELIGIBILITY | 36 |
| 5.1 | In | clusion Criteria | 36 |
| 5.2 | 2 E | xclusion Criteria | 37 |
| <b>6.</b> | STU | UDY PROCEDURES | 40 |
| 6.1 | . <b>S</b> 1 | tudy Schedule | 40 |
| | 6.1.1 | Qualification | 40 |
| | 6.1.2 | Treatment Period | |
| | 6.1.3 | Pharmacokinetic (PK) Subgroup | |
| ( | 6.1.4 | Post-Treatment Period | 41 |
| 6.2 | | dditional Study Assessments | |
| | 6.2.1 | Laboratory Assessments | 41 |

| | 6.2.2 | Physical Exams and Vital Signs | 41 |
|---|---|---|---|
| | 6. | 2.2.1 Eruptive Xanthoma | 42 |
| | 6. | 2.2.2 Lipemia Retinalis | 42 |
| | 6.2.3 | 3 Echocardiography | 42 |
| | 6.2.4 | 4 ECG | 42 |
| | 6.2. | 5 MRI | 42 |
| | 6.2.0 | 6 Quality of Life Assessments | 42 |
| | 6.2. | 7 Disease Symptom Diary | 42 |
| | 6.2.8 | 8 Diet Monitoring | 42 |
| | 6.2.9 | 9 Family History | 43 |
| | 6.2. | 10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2) | 43 |
| | 6.3 | Restriction on the Lifestyle of Patients | 43 |
| | 6.3. | 1 Contraception Requirements | 43 |
| | 6.3.2 | 2 Other Requirements | 44 |
| 7. | S' | TUDY DRUG | |
| | 7.1 | Volanesorsen Description | 44 |
| | 7.2 | Packaging and Labeling | |
| | 7.3 | Study Drug Accountability | |
| 8. | | REATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , | |
| | 8.5.2 | , | |
| | 8.5.3 | | |
| | 8.5.4 | $\mathcal{F}$ | |
| | 8.5. | | |
| | 8.5.0 | | |
| | 8.5. | , , , | |
| | 8.5.8 | | |
| | 8.5.9 | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | 11 0 | |
| | 8.6.2 | 11 0 | |
| | 8.6.3 | | |
| | 8.7 | Adjustment of Dose Frequency | |
| | 8.8 | Discontinuation of Study Treatment | |
| | 8.8. | 1 Follow-up Visits for Early Termination from Treatment Period | 55 |

| 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Pe | riod .56 |
|---|---|---|
| 8.9 | Withdrawal of Patients from the Study | 56 |
| 8.10 | Concomitant Therapy and Procedures | 57 |
| 8.10 | .1 Concomitant Therapy | 57 |
| 8.10 | .2 Concomitant Procedures | 57 |
| 8.11 | Treatment Compliance | 57 |
| 9. S | ERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 58 |
| 9.1 | Sponsor Review of Safety Information | 58 |
| 9.2 | Regulatory Requirements | 58 |
| 9.3 | Definitions | |
| 9.3. | | |
| 9.3.2 | 1 | |
| 9.3.3 | | |
| 9.4 | Monitoring and Recording Adverse Events | |
| 9.4. | | |
| 9.4.2 | | |
| 9.4.3 | , | |
| - | 4.3.1 Relationship to the Study Drug | |
| | 4.3.2 Severity | |
| | 4.3.3 Action Taken with Volanesorsen | |
| | 4.3.4 Treatment Given for Adverse Event | |
| | 4.3.5 Outcome of the Adverse Event | |
| 9.4.4 | 3 | |
| 9.5 | Procedures for Handling Special Situations | |
| 9.5. | • | |
| 9.5.2 | · | |
| 9.5.3 | $oldsymbol{arepsilon}$ | |
| 9.5.4 | | |
| | TATISTICAL CONSIDERATIONS | |
| 10.1 | Study Endpoints | |
| 10.1<br>10.1 | J 1 | |
| 10.1 | Sample Size | |
| 10.2 | Populations | |
| 10.3 | Definition of Baseline | |
| 10.4 | | |
| 10.5 | Interim Analysis | |
| 10.6 | • | |
| 10.6 | | |
| | 3 Efficacy Analysis | |

| 10.6 | .4 Pharmacokinetic and Immunogenicity Analysis | 67 |
|---|---|---|
| | 0.6.4.1 Pharmacokinetic Analysis | |
| 10 | 0.6.4.2 Immunogenicity Analysis | 68 |
| 11. II | NVESTIGATOR'S REGULATORY OBLIGATIONS | 68 |
| 11.1 | Informed Consent | 68 |
| 11.2 | Ethical Conduct of the Study | 69 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 69 |
| 11.4 | Patient Confidentiality | 69 |
| 12. A | DMINISTRATIVE AND LEGAL OBLIGATIONS | 70 |
| 12.1 | Protocol Amendments | 70 |
| 12.2 | Study Termination | 70 |
| 12.3 | Study Documentation and Storage | 70 |
| 12.4 | Study Monitoring | 71 |
| 12.5 | Language | 71 |
| 12.6 | Compensation for Injury | 71 |
| 13. R | EFERENCES | 72 |
| 14. A | PPENDICES | 74 |
| Appen | dix A Schedule of Procedures | 75 |
| Appen | dix B List of Laboratory Analytes | 81 |
| Appen | dix C Pharmacokinetic Sampling Schedule | 83 |
| Appen | dix D Grading Scale for Adverse Events Relating to Laboratory Abnorma | lities85 |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 45 |
| Table 2 | Labs to Be Performed in the Event of a Platelet Count Less than the | |
| | Lower Limit of Normal (x2) or $< 100,000/\text{mm}^3 (x1)^*$ | |
| Table 3 | Actions in Patients with Low Platelet Count | |
| Table 4 | Expected Event for the Protocol Defined Population by Preferred Term | |
| | and the Expected Incidence | 58 |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms. | 29 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volunesorsen is shown | |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen. | 33 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 8 - France

**Amendment Date:** 10 April 2017

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 7 dated 3 February 2017:

- 1. To update the platelet safety monitoring rules shown in Table 3.
- 2. To assess acute pancreatitis in medical history in Group 2 patients.
- 3. Added archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study).
- 4 Added Troponin I and platelet bound autoantibody testing at baseline (may be done) to provide added patient safety; blood viscosity (may be done) to assess potential benefit of ISIS 304801 administration; and platelet aggregation (may be done) to assess platelet function.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 3.4.3<br>Post-<br>Treatment | The post-treatment evaluation period is at least 26 weeks and consists of at least $\underline{69}$ Study Center visits on Weeks $\underline{53}$ , $54$ , $\underline{55}$ , $56$ , $\underline{57}$ , $58$ , $65$ , $71$ , and $78$ (Weeks $\underline{53}$ , $54$ , $\underline{55}$ , $56$ , $\underline{57}$ , $58$ , and $71$ may be conducted by a home healthcare nurse). | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis<br>Section 5.1<br>Inclusion<br>Criteria | <ul> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: • Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>• Post heparin plasma LPL activity of ≤ 20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study</li> <li>c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study</li> <li>4. Able and willing to participate in a 78-week study</li> </ul> | To clarify that either genetics or LPL activity can be used as an inclusion criteria and that LPL activity should not be performed unless already in medical history |
| 6.1.2<br>Treatment<br>Period | During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |
| 6.1.4 Post-<br>Treatment<br>Period | After completion of the Week 52 visit assessments, patients will enter the at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. The 26-week period consists of at least 69 Study Center visits on Weeks 53, 54,55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse), as outlined in the Schedule of Procedures in Appendix A. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| 6.2.1<br>Laboratory<br>Assessments | Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, and determined not to have met a stopping rule before dosing can continue or the dose pause rule of 75,000/mm³. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |
| 6.2.10 Chart<br>Review for<br>Incidents of<br>Acute<br>Pancreatitis in<br>Medical<br>History<br>(Group 2) | Added 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2) Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication. | To assess acute pancreatitis in medical history in Group 2 patients |
| 8.1<br>Volanesorsen<br>Administration | Removed Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. | Dosing recommendations provided in updated monitoring and drug administration updates |
| 8.5.2 Safety<br>Monitoring for<br>Platelet Count<br>Results | Actions to be taken in the event of reduced platelet count are shown in Table 23 in Section 8.6.3. Monitor every 1 week unless otherwise specified. Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |

| Monitoring for Platelet Count Results Continued | Protocol<br>Section | Description of Change | Rationale |
|---|---|---|---|
| Fibrinogen split products or D-dimer on fresh blood To Be Performed at Central Lab Citrated sample for platelets Coagulation panel (PT/INR, aPTT) CBC with reticulocytes Folate (folic acid) Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | Monitoring for<br>Platelet Count<br>Results | Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3). Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm³ (x1)* *In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes. Added Table 2: To Be Performed at Local Lab Peripheral smear (should be performed locally, fixed and sent to central | regarding platelet<br>count reductions,<br>ISIS 304801<br>dose exposure,<br>and treatment<br>recommendation |
| Citrated sample for platelets Coagulation panel (PT/INR, aPTT) CBC with reticulocytes Folate (folic acid) Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | Fibrinogen split products or D-dimer on fresh blood | |
| Coagulation panel (PT/INR, aPTT) CBC with reticulocytes Folate (folic acid) Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| CBC with reticulocytes Folate (folic acid) Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | · | |
| Folate (folic acid) Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Vitamin B12 Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | - | |
| Fibrinogen von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | ` ' | |
| von Willebrand factor Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Total globulins, total IgA, IgG and IgM Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Complement: total C3, total C4, Bb, C5a hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| hsCRP Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Helicobacter pylori (breath test) Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Rubella CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| CMV EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | , | |
| EBV Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Parvo B19 Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) | | · · · | |
| Anti-thyroid To Be Performed at Specialty Lab(s) | | | |
| To Be Performed at Specialty Lab(s) | | | |
| Anungiejei anunonies and Anu-PE/Lacca// | | Antiplatelet antibodies and Anti-PF4 assay | |
| Anti-ASO antibody | | | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 8.6.3<br>Stopping<br>Rules for<br>Platelet Count<br>Results | Actions to be taken in the event of a low platelet count are summarized in Table 23 below. In the event of a platelet count less than 75,000/mm³ that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor. In the event of any platelet count less than 50,000/mm³, or a rate of decline 2 50% between two consecutive assessments, irrespective of the platelet level, or a platelet count less than 75,000/mm³ that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3. daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable. Administration of steroids is recommended for patients whose platelet count is less than 2650,000/mm³. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period. In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), d | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |
| Protocol<br>Section | Description of Change | | Rationale | |
|---|---|---|---|---|
| Section 8.6.3 | Table 23 Actions in Patients with Low Platelet Count | | To provide added | |
| Stopping<br>Rules for<br>Platelet Count | Platelet Count on Rx | Drug Dose | Monitoring | patient safety regarding platelet count reductions, |
| Results<br>Continued | Normal range, > 140K/mm³ | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or nonconsecutive) of platelet count 140K -> 100K/mm³ or 1 occurrence of platelet count ≤100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion Monitor every 2 weeks | ISIS 304801 dose exposure, and treatment recommendations |
| | ≥ 100K <u>/mm³</u> -<br><del>140K/mm³</del> | Weekly 300 mg Study Drug<br>administration No action | Closer observation Monitor every 1 week until stable* | |
| | 75K-100K/mm <sup>3</sup> -<br>75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1 week | |
| | <del>50K-</del> 75K/mm <sup>3</sup> <u>-</u><br>50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 weekshow improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication | |

| Protocol<br>Section | Description of Change | | Rationale | |
|---|---|---|---|---|
| Section 8.6.3 | Table 23 Actions in Patients with Low Platelet Count <u>Continued</u> | | To provide added | |
| Stopping<br>Rules for<br>Platelet Count | Platelet Count on Rx | Drug Dose | Monitoring | patient safety<br>regarding platelet<br>count reductions, |
| Results Continued | 25K-≤ 50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are > 75K/mm³ then monitor every 1 week platelet count stable Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management Steroids recommended if platelet count is < 50K/mm³*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline. Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy Discontinue antiplatelet agents/NSAIDS/antico agulant medication while platelet count < 50K/mm³ if possible | ISIS 304801 dose exposure, and treatment recommendations |

| Protocol<br>Section | Description of Change | | Rationale | |
|---|---|---|---|---|
| Section 8.6.3 | Table 23 Ac | tions in Patients with Low Pla | atelet Count <u>Continued</u> | To provide added |
| Stopping Rules for Platelet Count Results | Platelet Count on Rx | Drug Dose | Monitoring | patient safety<br>regarding platelet<br>count reductions, |
| Continued | < 25K/mm³ | Permanently discontinue<br>Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoa gulant medication while platelet count < 50K/mm³ if possible | ISIS 304801 dose exposure, and treatment recommendations |
| | * At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³ **Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period. | | | |
| Synopsis<br>10.1.1 Efficacy<br>Endpoints | <ul> <li>Percent change and absolute change from baseline in fasting TG</li> <li>Frequency and severity of patient reported abdominal pain during the treatment period</li> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C</li> <li>Percent change from baseline in fasting total apolipoprotein C-III</li> <li>Change in blood viscosity (may be evaluated)</li> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> <li>Adjudicated acute pancreatitis event rate</li> <li>Other symptoms: eruptive xanthoma, lipemia retinalis</li> </ul> | | To assess potential benefit of ISIS 304801 administration | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis<br>10.1.2 Safety<br>Endpoints | <ul> <li>Adverse events including adjudicated events of pancreatitis and MACE</li> <li>Vital signs and weight</li> <li>Physical examinations</li> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> <li>Echocardiography</li> <li>Electrocardiograms (ECGs)</li> <li>Use of concomitant medications</li> <li>MRIs</li> <li>Platelet aggregation (may be evaluated)</li> </ul> | To assess platelet function following ISIS 304801 administration |
| Appendix A | CBC with Differential c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. In the event of any platelet count less than 50,000/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations Medical history, blood viscosity and potential gene sequencing to assess potential benefit of ISIS 304801 administration Platelet aggregation to assess platelet function following ISIS 304801 administration |
| | Added: Medical History <sup>q</sup> Blood Viscosity <sup>r</sup> Platelet Aggregation <sup>r</sup> Platelet Bound Autoantibodies <sup>r</sup> Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study) <sup>g</sup> X <sup>s</sup> q Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study r May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only s Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Appendix B | Added: Troponin I² CK-MB² Platelet Bound Autoantibodies³ Blood Viscosity³ Platelet Aggregation³ 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB 3 May be done | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations Blood viscosity to assess potential benefit of ISIS 304801 administration Platelet aggregation to assess platelet function following ISIS 304801 administration |

Amendment 8 10 April 2017

Protocol - France

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | <ol> <li>Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or<br/>ISIS 304801-CS16 (index studies) with an acceptable safety profile, per<br/>Sponsor and Investigator judgement.</li> </ol> |
| | Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: </li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical<br/>history. Note: testing of LPL activity should not be performed<br/>to confirm eligibility for the study</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study |
| | 4. Able and willing to participate in a 78-week study |

#### Study Population Continued

#### Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **Exclusion Criteria:**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b. HbA1c ≥ 9.0% at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)
  - e. Current use of GLP-1 agonists
- Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification

#### Study Population Continued

#### Exclusion Criteria: Continued

- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria: Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to Qualification and dose<br>and regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>Qualification</li> </ul> |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to Qualification |
| | <ul> <li>g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br/>apixaban) unless on a stable dose for at least 4 weeks prior to<br/>Qualification and regular clinical monitoring is performed</li> </ul> |
| | <ul> <li>h. Tamoxifen, estrogens or progestins unless on a stable dose for at<br/>least 4 months prior to Qualification and dose and regimen expected<br/>to remain constant during the treatment period</li> </ul> |
| | <ul> <li>Plasma apheresis within 4 weeks prior to Qualification or planned<br/>during the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A</li> </ul> |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | An at least 26-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |
| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |

| Planned Analyses | Safety Endpoints: |
|---|---|
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation,<br/>urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | Change in blood viscosity (may be evaluated) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



#### STUDY GLOSSARY

| STUDY GLOSSARY | |
|---|---|
| Abbreviation/Acronym | <u>Definition</u> |
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| ароЕ | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |

#### STUDY GLOSSARY Continued

Abbreviation/Acronym

| INR | International Normalized Ratio |
|------|--------------------------------|
| IRB | Institutional Review Board |
| IXRS | Interactive Voice/Web-Response |

IXRS Interactive Voice/Web-Response System

**Definition** 

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volunesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

ISIS 304801-CS7 Amendment 8 Protocol - France 10 April 2017

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 **ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** 

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Protocol - France

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volunesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volunesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), in vitro and in vivo genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volunesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (in vitro and in vivo) and was non-genotoxic (in vitro and in vivo). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

Protocol - France

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

#### 3.4.1 Qualification

A qualification period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is at least 26 weeks and consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse).

#### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide

recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of ≤ 20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study.
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
- 4. Able and willing to participate in a 78-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of  $\pm$  10 units of insulin])

- d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
- e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification
- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$
    - $AST > 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests  $\geq$  trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing  $\leq$  5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II

- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to Qualification
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to Qualification
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to Qualification and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to Qualification or planned during the study
  - j. Prior exposure to ISIS 304801
  - k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification

- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. The 26-week period consists of at least 9 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, 65, 71, and 78 (Weeks 53, 54, 55, 56, 57, 58, and 71 may be conducted by a home healthcare nurse), as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

## 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, Week 65, and Week 78.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

# 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.

- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

# 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

## 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent† or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner

includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

- Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.
- \* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.
- † Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 °C to 8 °C and be protected from light.

#### Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

# 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs.

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

## 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above.

Protocol - France

Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

Frequency of Repeat Measurements: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

Further Investigation into Liver Chemistry Elevations: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified.

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw

upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm<sup>3</sup> (x1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

Protocol - France

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

## 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

<u>All patients on insulin</u> will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

<u>All diabetic patients</u> will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as one in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

#### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and < 9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3$  mg/dL (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24 hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, or a platelet count less than  $75,000/\text{mm}^3$  that occurs while the patient is on dosing at 300 mg every 2 weeks, then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm³. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

#### Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

#### <u>Definition of Clinically-Relevant, Non-Major Bleeding Events</u> (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

 Table 3
 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or non-consecutive of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. |
| > 100K/mm <sup>3</sup> | Weekly 300 mg Study Drug administration | |
| 100K/mm <sup>3</sup> - >75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks | |
| 75K/mm <sup>3</sup> - >50K/mm <sup>3</sup> | <ul> <li>If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause.</li> <li>When platelet count returns to &gt; 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor Medical Monitor</li> </ul> | <ul> <li>Monitor every 2-3 days until<br/>2 successive values are<br/>&gt; 75K/mm³ then monitor every<br/>1 week</li> <li>Consider discontinuation of<br/>antiplatelet agents/NSAIDS/<br/>anticoagulant medication</li> </ul> |
| < 50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | <ul> <li>Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are &gt; 75K/mm³ then monitor every 1 week</li> <li>Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management</li> <li>Steroids recommended if platelet count is &lt; 50K/mm³*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline.</li> <li>Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy</li> <li>Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is&lt; 50K/mm³ if possible</li> </ul> |

#### Table 3 Actions in Patients with Low Platelet Count Continued

Legend:

Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

#### 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient

who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 78, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline Qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 78 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### Amendment 8 10 April 2017

#### 9.4 **Monitoring and Recording Adverse Events**

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a single unifying diagnosis if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- Related: There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- Possible: The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration

- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

#### 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE

- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study

physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, **the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth**. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography

- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs
- Platelet aggregation (may be evaluated)

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

<u>Safety Set</u>: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline will be the last non-missing assessment prior to the first dose of Study Drug. Details will be provided in the SAP.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active Study Drug in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naïve group which includes patients on placebo in index studies. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG  $\geq 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volunesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study will receive the first treatment of volunesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration  $(CL_{0-24h}/F)$  will be calculated from  $CL_{0-24h}/F = Actual Dose/AUC_{0-24h}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., %change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed

informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in

transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-α expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PC, Voshol PJ, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

## 14. APPENDICES

# **Appendix A** Schedule of Procedures

Qualification through Treatment Period

Post-Treatment Follow-up

Appendix A Schedule of Procedures – Qualification through Treatment Period

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | 1 | reatn | nent l | Period | t | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -2 to | ١٨ | II. | Wk | Wk | WL | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 |
| | Study Week | | | Wk<br>1 4 | | 6 | 8 | | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| | Study Day | | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Info | ormed Consent | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Ou | tpatient Visit | Х | Х | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | Χ | $X^{j}$ | $\mathbf{X}^{j}$ | $X^{j}$ | $X^{j}$ | Χ | $X^{j}$ | $X^{j}$ | $X^{j}$ | Χ | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | Χ |
| Inc | usion/Exclusion Criteria | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Ме | dical History <sup>q</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Vita | al Signs + body weight (+ height on Day 1 only) | Χ | Х | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | X |
| Ph | Physical Examination | | Х | | | | | | | Χ | | | | | Χ | | | | Х | | | | | Χ |
| 12- | 12- lead ECG (triplicate) | | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х |
| | MRI (liver/spleen) | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> |
| Ecl | nocardiography | Х | | | | | | | | | | | | | $X^k$ | | | | | | | | | X <sup>k</sup> |
| | Chemistry Panel | Х | Χ | | Х | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х |
| | CBC with Differential <sup>b</sup> | Х | ← X — Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling. | | | | | | | | | | | | | | | | | | | | | |
| | Serum Lipid Panel | Х | Х | | Х | | Χ | | Χ | Χ | Γ | | | Χ | Χ | | | | Χ | | | | Χ | Х |
| | Blood viscosity <sup>r</sup> | | Х | | | | | | | Х | | | | | Χ | | | | | | | | | Х |
| | Platelet aggregation <sup>r</sup> | Х | Х | | | | | | | Χ | | | | | Χ | | | | | | | | | Χ |
| asting) <sup>c</sup> | Coagulation (aPTT, PT, INR) | Χ | | | | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | X |
| tin | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | Xn | Х | | | | | | | Χ | | | | | Χ | | | | | | | | | X |
| (Fas | Sedimentation Rate | | Χ | | | | | | | Χ | | | | | Χ | | | | | | | | | X |
| <del>-</del> ≥ | Complement (C5a, Bb) | | Х | | | | | | | Χ | | | | | Χ | | | | | | | | | X |
| raw | Plasma PK - Volanesorsen | | Χ <sup>I</sup> | Х | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | X |
| Ωp | Anti-Volanesorsen Antibodies | | Χ | | Х | | Χ | | | Χ | | | | | Χ | | | | Х | | | | | Х |
| pool | FSH (women only, if applicable) | Х | | | | | | | | | | | | | | | | | | | | | | |
| В | Serum Pregnancy Test <sup>d</sup> | Х | | | Χ | | Х | | | Х | | Х | | | Х | | Х | | Χ | | Χ | | | X |
| 1 | Archived Serum & Plasma Samples <sup>e</sup> | | Х | | | | Х | | | Х | | | | | Χ | | | | | | | | | Х |
| 1 | Troponin I° | Х | ., | | | | | | | | | | | | | | | | | | | | | |
| 1 | Platelet Bound Autoantibodies | | Х | | <b>.</b> | <u> </u> | | _ | | | <u> </u> | | <b>!</b> | | | | | | | | | | | |
| | Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study) <sup>g</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |

**Appendix A** Schedule of Procedures - Qualification through Treatment Period *Continued* 

| Study Period | Qual <sup>a</sup> | | Treatment Period | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | w | 'k | w | Wk | Wk | Wk | | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk<br>38 | Wk<br>40 | Wk | Wk<br>46 | | |
| Study Week | -2 to -1 | 1 | | 4 | 6 | | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | | &<br>42 | 44 | &<br>48 | | Wk 52<br>or ET |
| Study Day | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Urinalysis <sup>c</sup> | Χ | $X^{m}$ | | Х | | Х | | | X <sup>m</sup> | | X <sup>m</sup> | | | X <sup>m</sup> | | $X^{m}$ | | $X^{m}$ | | $X^{m}$ | | | Xm |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Quality of Life Assessment(s) | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | Х | Х | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х |
| Adverse Events | Х | Х | | Χ | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Concomitant Medication | Х | Х | | Χ | Х | Χ | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Х | Χ | Χ |

# ${\bf Appendix} \ {\bf A} \quad {\bf Schedule} \ {\bf of} \ {\bf Procedures-Post-Treatment} \ {\bf Follow-up}$

| | Study Period | Post | Treat | ment | Follow | /-up <sup>p</sup> |
|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| | Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Informe | ed Consent | | | | | |
| | ent Visit | $X^{j}$ | $X^{j}$ | Χ | Χ <sup>j</sup> | Х |
| | on/Exclusion Criteria | | | | | |
| | gns + body weight | | | Х | | Х |
| | ht on Day 1 only) | | | | | · · |
| , | al Examination | | | X | | X |
| | d ECG (triplicate) /er/spleen) | | | X | | X |
| | , , | | | | | |
| ECHOCA | ardiography | | | | | · · |
| | Chemistry Panel | Vs | X | X | X | X |
| | CBC with Differential <sup>b</sup> | Xs | Х | X | Х | X |
| ي | Serum Lipid Panel | | | Λ. | | |
| ing | Coagulation (aPTT, PT, INR)<br>hsCRP, HbA1c, FPG, and | | | | | |
| ast | de-lipidated free glycerol | | | Χ | | Х |
| Ē, | Sedimentation Rate | | | Х | | Χ |
| Blood Draw (Fasting) <sup>¢</sup> | Complement (C5a, Bb) | | | X | | Х |
| ۵ | Plasma PK - Volanesorsen | | | Χ | | Χ |
| po | Anti-Volanesorsen Antibodies | | | Χ | | Χ |
| 읢 | FSH (women only, if applicable) | | | | | |
| _ | Serum Pregnancy Test <sup>d</sup> | | Χ | Х | Χ | Χ |
| | Archived Serum & Plasma Samplese | | | Χ | | Χ |
| | Troponin I° | | | | | |

Appendix A Schedule of Procedures – Post-Treatment Follow-up Continued

| Study Period | Pos | st Trea | tment l | Follow- | up <sup>p</sup> |
|---|---|---|---|---|---|
| Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Urinalysis <sup>c</sup> | | $X^{m}$ | $X^{m}$ | $X^{m}$ | Xm |
| Fundus Photography <sup>f</sup> | | | | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | | | | | |
| Weekly Study Drug: SC Injection | | | | | |
| Symptom Diary (weekly) | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | | Х | | Х |
| Food/Drink Diary (quarterly)h | | | Х | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | | Х | Х | Х | Х |
| Adverse Events | Х | Х | Х | Х | Х |
| Concomitant Medication | Χ | Х | Х | Х | Х |

#### Appendix A Schedule of Procedures Continued

- a Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 ISIS 304801-CS16 roll over patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- Genetic testing can be conducted for study Qualification (Group 2 ISIS 304801-CS16 roll over patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- I Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)
- n HbA1c only
- o All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- p If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values
- Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- r May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only
- s Platelets are assessed each calendar week, visits do not have specified windows to allow flexibility of scheduling

# **Appendix B** List of Laboratory Analytes

#### Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | <b>Coagulation</b> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Chloride Bicarbonate Total protein Albumin Calcium Magnesium Phosphorus Glucose BUN Creatinine Uric Acid Total bilirubin Direct (conjugated) bilirubin ALT AST Alkaline phosphatase | <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb Troponin I² CK-MB² Platelet Bound Autoantibodies³ De-lipidated free glycerol HbA1c, FPG | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>4</sup></li> </ul> Additional Measures for |

- 1 Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

## Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

## PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime | Anytime |

## PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>Post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities
# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm³ | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Urine | | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

### **Collaborator:**

Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

### ISIS 304801-CS7

# The APPROACH Open-Label Study Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 7 – 7 April 2017** 

EudraCT No: 2015-003755-21

### ISIS 304801-CS7

### The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

### An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

### Protocol Amendment 7 - 7 April 2017

### Protocol History:

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

Protocol Amendment 3: 9 May 2016

Protocol Amendment 4: 6 June 2016

Protocol Amendment 5: 6 July 2016

Protocol Amendment 6: 18 November 2016

### Sponsor:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court

Carlsbad, CA 92010

MD, MBA

### Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 7** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

### The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

### An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200 Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010 Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 7 April 2017

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

### Protocol

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Vol-<br>Patients with Familial Chylor | anesorsen Administered Subcutaneously to nicronemia Syndrome (FCS) |
| Amendment: | Amendment 7 | |
| Date: | 7 April 2017 | |
| Open-Label Study of Chylomicronemia Sydescribed herein. I agree to comply wire Good Clinical Praction I agree to ensure that any purpose other that | f Volanesorsen Administered Styndrome (FCS)", dated 7 April th the International Conference (E6). | and the attached clinical protocol, entitled "An abcutaneously to Patients with Familial 2017, and agree to conduct the study as on Harmonization Tripartite Guideline on ontained in this document will not be used for the clinical investigation without the prior |
| Investigator's Signa Investigator's Name | | Date (DD Month YYYY) |
| mivestigator a Ivanii | - (picase prini) | |

### **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| PRO | тосо | L AMENDMENT | 10 |
| | | L SYNOPSIS | |
| STU | DY DE | SIGN AND TREATMENT SCHEMA | 28 |
| STU | | OSSARY | |
| 1. | | ECTIVES | |
| 2. | BAC | CKGROUND AND RATIONALE | 31 |
| 2.1 | | verview of Disease | |
| 2.2 | | nerapeutic Rationale | |
| 2.3 | 3 V | olanesorsen | |
| | 2.3.1 | Mechanism of Action | |
| | 2.3.2 | Chemistry | |
| | 2.3.3 | Preclinical Experience | |
| | 2.3.4 | Clinical Experience | |
| 2.4 | | ationale for Dose and Schedule of Administration | |
| 3. | | ERIMENTAL PLAN | |
| 3.1 | | udy Design | |
| 3.2 | | umber of Study Centers | |
| 3.3 | | umber of Patients | |
| 3.4 | | verall Study Duration and Follow-up | |
| | 3.4.1 | Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-index study): Qualification | |
| | 3.4.2 | Group 3 Patients (did not participate in an index study): Screening/Qualification | 38 |
| | 3.4.3 | Treatment | 38 |
| | 3.4.4 | Post-Treatment | 39 |
| 3.5 | 5 Er | nd-of-Study | 39 |
| 3.6 | 5 Da | ata and Safety Monitoring Board | 39 |
| 4. | PAT | TIENT ENROLLMENT | 39 |
| 4.1 | l Sc | reening/Qualification | 39 |
| 4.2 | 2 Er | nrollment | 40 |
| <b>5.</b> | PAT | TENT ELIGIBILITY | 40 |
| 5.1 | l In | clusion Criteria | 40 |
| 5.2 | | sclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-day Study Poll over Patients | |
| 6 | | dex Study Roll-over Patients | |
| <b>6.</b> 6.1 | | udy Schedule | |
| | ı sı<br>6.1.1 | Qualification (Groups 1 and 2) | |
| | U.I.I | Quantication (Otoups 1 and 4) | 44 |

7 April 2017

Protocol

| 6.1.2 | Screening and Qualification (Group 3) | 44 |
|---|---|---|
| 6.1.3 | Treatment Period | 44 |
| 6.1.4 | Extended Treatment Period | 45 |
| 6.1.5 | Pharmacokinetic (PK) Subgroup | 45 |
| 6.1.6 | Post-Treatment Period | 46 |
| 6.2 Ad | ditional Study Assessments | 46 |
| 6.2.1 | Laboratory Assessments | 46 |
| 6.2.2 | Physical Exams and Vital Signs | 46 |
| 6.2.2 | 1 Eruptive Xanthoma | 46 |
| 6.2.2 | 2 Lipemia Retinalis | 47 |
| 6.2.3 | Echocardiography | 47 |
| 6.2.4 | ECG | 47 |
| 6.2.5 | MRI | 47 |
| 6.2.6 | Quality of Life Assessments | 47 |
| 6.2.7 | Disease Symptom Diary | 47 |
| 6.2.8 | Diet Monitoring | 47 |
| 6.2.9 | Family History | 48 |
| 6.2.10 | Chart Review for Incidents of Acute Pancreatitis in Medical History | |
| | (Group 2 and 3) | |
| | striction on the Lifestyle of Patients | |
| 6.3.1 | Contraception Requirements | |
| 6.3.2 | Other Requirements | |
| | DY DRUG | |
| | lanesorsen Description | |
| | ckaging and Labeling | |
| | dy Drug Accountability | |
| | ATMENT OF PATIENTS | |
| | lanesorsen Administration | |
| | her Protocol-Required Drugs | |
| | her Protocol-Required Treatment Procedures | |
| | eatment Precautions | |
| | fety Monitoring Rules | |
| 8.5.1 | Safety Monitoring for Liver Chemistry Tests | |
| 8.5.2 | Safety Monitoring for Platelet Count Results | |
| 8.5.3 | Safety Monitoring for Minor Bleeding Events | |
| 8.5.4 | Safety Monitoring for Constitutional Symptoms | |
| 8.5.5 | Safety Monitoring for LDL-C Elevations | |
| 8.5.6 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | |
| 8.5.7 | Safety Monitoring for Documented Severe Hypoglycemia | |
| 8.5.8 | Safety Monitoring for Hyperglycemia | 55 |

Protocol

| | 8.5.9 | Acute Pancreatitis | 56 |
|---|---|---|---|
| | 8.6 Sto | pping Rules | 56 |
| | 8.6.1 | Stopping Rules for Liver Chemistry Elevations | 57 |
| | 8.6.2 | Stopping Rules for Renal Function Test Results | 57 |
| | 8.6.3 | Stopping Rules for Platelet Count Results | 57 |
| | 8.7 Adj | ustment of Dose Frequency | 60 |
| | 8.8 Dis | continuation of Study Treatment | |
| | 8.8.1 | Follow-up Visits for Early Termination from Treatment Period | 60 |
| | 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Per | iod .60 |
| | | chdrawal of Patients from the Study | |
| | 8.10 Cor | ncomitant Therapy and Procedures | 61 |
| | 8.10.1 | Concomitant Therapy | 61 |
| | 8.10.2 | Concomitant Procedures. | 62 |
| | | atment Compliance | |
| 9. | | OUS AND NON-SERIOUS ADVERSE EVENT REPORTING | |
| | - | onsor Review of Safety Information | |
| | 9.2 Reg | gulatory Requirements | 62 |
| | 9.3 Def | initions | |
| | 9.3.1 | Adverse Event | |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | |
| | 9.3.3 | Serious Adverse Event (SAE) | |
| | | nitoring and Recording Adverse Events | |
| | 9.4.1 | Serious Adverse Events | |
| | 9.4.2 | Non-Serious Adverse Events | |
| | 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | |
| | 9.4.3. | 1 , 5 | |
| | 9.4.3.2 | • | |
| | 9.4.3.3 | | |
| | 9.4.3.4 | | |
| | 9.4.3. | | |
| | 9.4.4 | Adjudication Committees | |
| | | cedures for Handling Special Situations | |
| | 9.5.1 | Abnormalities of Laboratory Tests | |
| | 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | |
| | 9.5.3 | Dosing Errors | |
| | 9.5.4 | Contraception and Pregnancy | |
| 10 | | TISTICAL CONSIDERATIONS | |
| | | dy Endpoints | |
| | 10.1.1 | Efficacy Endpoints | |
| | 10 1 2 | Safety Endnoints | 69 |

| ISIS 30480 | 01-CS7 CONFIDENTIAL | Amendment 7 |
|---|---|---|
| Protocol | | 7 April 2017 |
| 10.2 | G1. G'- | (0) |
| 10.2 | Sample Size | |
| 10.3 | Populations | |
| 10.4 | Definition of Baseline | |
| 10.5 | Interim Analysis | |
| 10.6 | Planned Methods of Analysis | |
| 10.6 | 8 1 | |
| 10.6 | | |
| 10.6 | | |
| 10.6 | | |
| | 0.6.4.1 Pharmacokinetic Analysis | |
| | 0.6.4.2 Immunogenicity Analysis | |
| | NVESTIGATOR'S REGULATORY OBLIGATIONS | |
| 11.1 | Informed Consent | |
| 11.2 | Ethical Conduct of the Study | |
| 11.3 | Independent Ethics Committee/Institutional Review Board | |
| 11.4 | Patient Confidentiality | |
| | DMINISTRATIVE AND LEGAL OBLIGATIONS | |
| 12.1 | Protocol Amendments | |
| 12.2 | Study Termination | |
| 12.3 | Study Documentation and Storage | |
| 12.4 | Study Monitoring | |
| 12.5 | Language | |
| 12.6 | Compensation for Injury | |
| | REFERENCES | 77 |
| 14. A | APPENDICES | |
| | ndix A Schedule of Procedures | |
| Appen | · | |
| Appen | 1 0 | |
| Appen | ndix D Grading Scale for Adverse Events Relating to Laboratoria | oratory Abnormalities90 |
| | TABLE OF TABLES | |
| | | Page |
| Tol-1- 1 | Valoresparan (ISIS 204901) Characteristics | <u> </u> |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | |
| Table 2 | Labs to Be Performed in the Event of a Platelet Count Lower Limit of Normal (x2) or $< 100,000/\text{mm}^3$ (x1)*. | |
| Table 3 | Actions in Patients with Low Platelet Count or Drop in | |
| Table 4 | Expected Event for the Protocol Defined Population by | |
| 1 4016 4 | and the Expected Incidence | |

### **TABLE OF FIGURES**

| | | Page |
|---|---|---|
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 32 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volunesorsen is shown | 34 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 36 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 7

**Amendment Date:** 7 April 2017

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 6 dated 18 November 2016:

- 1. To update the platelet safety monitoring rules shown in Table 3.
- 2. To add LPL activity of  $\leq 20\%$  of normal in medical history as an inclusion criteria for Group 2 and 3 patients as has been allowed for Group 1 patients.
- 3. To add platelet count < lower limit of normal (LLN) for the central laboratory (i.e., < 140,000/mm<sup>3</sup>) for Group 3 patients.
- 4. To assess acute pancreatitis in medical history in Group 2 patients.
- 5. Added archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 3; Group 2 if not available from index study)
- 6. Added blood viscosity (may be done) to assess potential benefit of ISIS 304801 administration and platelet aggregation (may be done) to assess platelet function.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 3.4.4<br>Post-<br>Treatment | Was The post-treatment evaluation period is 13 weeks and consists of 4 Study Center visits on Weeks 54, 56, 58, and 65 (Weeks 54, 56, and 58 may be conducted by a home healthcare nurse). | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |
| | The post-treatment evaluation period is 13 weeks and consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse). | |

Protocol

| | | <u> </u> |
|---|---|---|
| Protocol<br>Section | Description of Change | Rationale |
| Synopsis<br>Section 5.1<br>Inclusion<br>Criteria | <ul> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study</li> </ul> </li> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study</li> <li>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label study</li> </ul></li></ul> | To add LPL activity of ≤ 20% of normal in medical history as an inclusion criteria for Group 2 and 3 patients as has been allowed for Group 1 patients |
| Synopsis 5.2 Exclusion Criteria for Group 3 | <ul> <li>a. Hepatic: <ul> <li>Total bilirubin &gt; upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL</li> <li>ALT &gt; 2.0 x ULN</li> <li>AST &gt; 2.0 x ULN</li> </ul> </li> <li>b. Renal: <ul> <li>Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of &lt; 500 mg/24 hrs</li> <li>Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field</li> <li>Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault &lt; 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)</li> </ul> </li> <li>c. Platelet count &lt; lower limit of normal (LLN) for the central laboratory (i.e., &lt; 140,000/mm³)</li> </ul> | To provide added patient safety regarding platelet count reductions, and ISIS 304801 dose exposure |

fe. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion

de. Cardiac Troponin I > ULN at Screening ed. LDL-C > 130 mg/dL at Screening

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis 6.1.3 Treatment Period | During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesoren administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |
| 6.14 Extended<br>Treatment<br>Period | During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.—Dosing instructions and training will be provided to the patient where applicable. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |

| Protocol | | |
|---|---|---|
| Section | Description of Change | Rationale |
| 6.1.6<br>Post-Treatment<br>Period | After completion of the Week 52 visit assessments, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country as described in Section 6.1.4. Patients not participating in an expanded access program will enter the 13-week post treatment evaluation period. This 13-week post treatment evaluation period. This 13-week post treatment evaluation period consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A. Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure |
| 6.2.1<br>Laboratory<br>Assessments | Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, and determined not to have met a stopping rule before dosing can continue or the dose pause rule of 75,000/mm³. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |
| 6.2.10 Chart<br>Review for<br>Incidents of<br>Acute<br>Pancreatitis in<br>Medical History | Added 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2 and 3) | To assess acute<br>pancreatitis in<br>medical history in<br>Group 2 patients |
| 8.1<br>Volanesorsen<br>Administration | Removed Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. | Dosing recommendations provided in updated monitoring and drug administration updates |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| 8.5.2 Safety Monitoring for Platelet Count Results | Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3. Monitor every 1 week unless otherwise specified. Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing. The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3). | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| 8.5.2 Safety<br>Monitoring for<br>Platelet Count<br>Results<br>Continued | Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm³ (x1)*< 75,000/mm³ *In patients who have any 2 occurrences (consecutive or nonconsecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |
| | To Be Performed at Local Lab | |
| | Peripheral smear (should be performed locally, fixed and sent to central lab for review) | |
| | Fibrinogen split products or D-dimer on fresh blood | |
| | To Be Performed at Central Lab | |
| | Citrated sample for platelets | |
| | Coagulation panel (PT/INR, aPTT) | |
| | CBC with reticulocytes | |
| | Folate (folic acid) | |
| | Vitamin B12 | |
| | Fibrinogen | |
| | von Willebrand factor | |
| | Total globulins, total IgA, IgG and IgM | |
| | Complement: total C3, total C4, Bb, C5a | |
| | hsCRP | |
| | Helicobacter pylori (breath test) | |
| | Serology for: | |
| | HBV, HCV, HIV (if not done recently for screening) | |
| | Rubella | |
| | CMV | |
| | EBV | |
| | Parvo B19 | |
| | Helicobacter pylori (IgG serum test) | |
| | Auto-antibody screen: | |
| | Antiphospholipid | |
| | Rheumatoid factor | |
| | Anti-dsDNA | |
| | Anti-thyroid | |
| | To Be Performed at Specialty Lab(s) | |
| | Antiplatelet antibodies and Anti-PF4 assay | |
| | Anti-ASO antibody | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 8.6.3<br>Stopping<br>Rules for<br>Platelet<br>Count<br>Results | Actions to be taken in the event of a low platelet count are summarized in Table 3 below. In the event of a platelet count less than 75,000/mm³ that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor. In the event of any platelet count less than 2550,000/mm³, or a platelet count less than 75,000/mm³ that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3. daily until 2 successive values show improvement then monitored overy 2-3 days until platelet count is stable. Administration of steroids is recommended for patients whose platelet count is less than 2650,000/mm³. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5 2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). Triglyceride levels will be monitored weekly, and AE monitoring will continue, during cortiscosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period. In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to > 100,000/mm³. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a r | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations |

| | Rationale | | |
|---|---|---|---|
| Was:<br>Table 3 Actions | To provide added patient safety | | |
| Platelet<br>Count on Rx | Drug Dose | Monitoring | regarding platelet<br>count reductions,<br>ISIS 304801 |
| Normal range,<br>> 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks | dose exposure,<br>and treatment<br>recommendations |
| 100K-<br>140K/mm <sup>3</sup> | No action | Closer observation<br>Monitor every 1 week until<br>stable* | rossimionadasis |
| 75K-<br>100K/mm <sup>3</sup> | Permanently reduce<br>dose frequency to<br>300 mg every 2 weeks<br>or reduce dose to<br>150 mg weekly | Closer observation<br>Monitor every 1 week | |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication | |
| 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible | |

| Protocol<br>Section | Description of Change | | | Rationale |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping<br>Rules for<br>Platelet | Stopping Rules for | | | |
| Count<br>Results<br>Continued | Platelet<br>Count on Rx | Drug Dose | Monitoring | |
| Continued | < 25K/mm <sup>3</sup> | Permanently<br>discontinue<br>Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible | |
| | determined ** Recovery in dose steroic (Provan et a every 2-4 w weeks then | by the Sponsor Medical Management platelet count may be access. Treatment guidelines fal. 2010) recommend Dexageeks for 1-4 cycles; Prednataper; or Methylprednisological. | ed weekly that are stable as lonitor and > 100,000/mm <sup>3</sup> celerated by administration of high for immune thrombocytopenia amethasone 40 mg daily for 4 days is(ol)one 0.5-2 mg/kg/d for 2-4 one 30 mg/kg/day for 7 days ( <b>note</b> : roids after methyl prednisolone) | |

| Protocol<br>Section | | Description of Cha | ange | Rationale |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping<br>Rules for<br>Platelet Count | Table 3 Actions in Patients with Low Platelet Count or Drop in Platelet Count | | | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose |
| Results<br>Continued | Platelet<br>Count on Rx | Drug Dose | Monitoring | exposure, and treatment |
| | | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or non-consecutive) of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. | recommendations |
| | > 100K/mm <sup>3</sup> | Weekly 300 mg Study Drug administration | | |
| | 100K/mm <sup>3</sup> -<br>> 75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks | | |
| | 75K/mm <sup>3</sup> -<br>> 50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor Medical Monitor | <ul> <li>Monitor every 2-3 days until 2 successive values are &gt;75K/mm³ then monitor every 1 week</li> <li>Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication</li> </ul> | |

| Protocol<br>Section | Description of Change | | | Rationale |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping | Table 3 Actions in Patients with Low Platelet Count or Drop in Platelet Count Continued | | | To provide added patient safety |
| Rules for<br>Platelet Count<br>Results | Platelet<br>Count on Rx | Drug Dose | Monitoring | regarding platelet<br>count reductions,<br>ISIS 304801 dose |
| Continued | dose steroic<br>(Provan et a<br>every 2-4 w | ls. Treatment guidelines for i | ethasone 40 mg daily for 4 days<br>ol)one 0.5-2 mg/kg/d for 2- | exposure, and treatment recommendations |
| 9.4.1 Serious | methylpredr | • | o fulfill regulatory requirements, | To provide |
| Adverse<br>Events | all SAEs (regard reported to the S first knowledge of patient signs the follow-up period patient enters the reporting by tele leaving a messa | less of their relationship to vo<br>sponsor or designee within 24<br>of the event. The collection of<br>informed consent form and s<br>which is defined as the Weel<br>e extended treatment period) | planesorsen) should be I hours of the Study Center's If SAEs will begin after the Stop at the end of the patient's If 65 visit (or Week 117 if I When the Investigator is I to someone in person versus I to Event Form should be | consistent SAE reporting rules |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis<br>10.1.1<br>Efficacy<br>Endpoints | <ul> <li>Percent change and absolute change from baseline in fasting TG</li> <li>Frequency and severity of patient reported abdominal pain during the treatment period</li> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C</li> <li>Percent change from baseline in fasting total apolipoprotein C-III</li> <li>Change in blood viscosity (may be evaluated)</li> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> <li>Adjudicated acute pancreatitis event rate</li> <li>Other symptoms: eruptive xanthoma, lipemia retinalis</li> </ul> | To assess<br>potential benefit of<br>ISIS 304801<br>administration |
| Synopsis<br>10.1.2 Safety<br>Endpoints | Adverse events including adjudicated events of pancreatitis and MACE Vital signs and weight Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Platelet aggregation (may be evaluated) | To assess platelet function following ISIS 304801 administration |
| Appendix A | Removed Week 2.5 CBC with Differential c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable and determined not to have met a stopping rule-before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that determine if the count has not-met the a stopping rule, and to determine whether the rate of decline is suggestive that the patient could be approaching the or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor Added: Blood Viscosity and Platelet Aggregation e May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only Added: Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 3; Group 2 if not available from index study) | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations. Blood viscosity and potential gene sequencing to assess potential benefit of ISIS 304801 administration. Platelet aggregation to assess platelet function following ISIS 304801 administration. |
| Appendix B | Added Blood Viscosity and Platelet Aggregation | To assess potential benefit of ISIS 304801 administration To assess platelet function following ISIS 304801 administration |

### PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | <ol> <li>Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or<br/>ISIS 304801-CS16 (index studies) with an acceptable safety profile, per<br/>Sponsor and Investigator judgement.</li> </ol> |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) supported by documentation of at least 1 of<br/>the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medica<br/>history. Note: testing of LPL activity should not be performed to<br/>confirm eligibility for the study</li> </ul> |
| | <ul> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for<br/>the ISIS 304801-CS16 index study</li> <li>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label<br/>study</li> </ul> |
| | 4. Able and willing to participate in a 65-week study |

Protocol

#### PROTOCOL SYNOPSIS Continued

#### Study Population Continued

Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)

Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c ≥ 9.0% at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening

#### PROTOCOL SYNOPSIS Continued

#### Study Population Continued

Protocol

Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued

- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
    - Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
  - c. Platelet count < lower limit of normal (LLN) for the central laboratory (i.e., < 140,000/mm³)
  - d. Cardiac Troponin I > ULN at Screening
  - e. LDL-C > 130 mg/dL at Screening
  - f. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- Treatment with another investigational drug, biological agent, or device within 1 month of screening, or 5 half-lives of investigational agent, whichever is longer

| Study Population Continued | Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued |
|---|---|
| | 13. Unwilling to comply with lifestyle requirements (Section 6.3) |
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to screening and dose and<br>regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>screening</li> </ul> |
| | <ul> <li>Systemic corticosteroids or anabolic steroids within 6 weeks prior to<br/>screening unless approved by the Sponsor Medical Monitor</li> </ul> |
| | d. Atypical antipsychotic medications (e.g., olanzapine and clozapine)<br>unless on a stable dose for at least 3 months prior to screening and<br>dose and regimen expected to remain stable throughout the study |
| | <ul> <li>Antihypertensive medication unless on a stable dose for at least</li> <li>4 weeks prior to screening and dose and regimen expected to remain<br/>constant during the treatment period</li> </ul> |
| | f. Glybera gene therapy within 2 years prior to screening |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br>apixaban) unless on a stable dose for at least 4 weeks prior to<br>screening and regular clinical monitoring is performed |
| | <ul> <li>Tamoxifen, estrogens or progestins unless on a stable dose for at<br/>least 4 months prior to screening and dose and regimen expected to<br/>remain constant during the treatment period</li> </ul> |
| | <ul> <li>Plasma apheresis within 4 weeks prior to screening or planned during<br/>the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>Any other medication unless stable at least 4 weeks prior to screening<br/>(Occasional or intermittent use of over-the-counter medications will be<br/>allowed at Investigator's discretion)</li> </ul> |
| | <ul><li>15. Blood donation of 50 to 499 mL within 30 days of screening or of</li><li>&gt; 499 mL within 60 days of screening</li></ul> |
| | <ol> <li>Known hypersensitivity to any of the excipients of the Study Drug<br/>(ISIS 304801 or placebo)</li> </ol> |
| | 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

#### **Rationale for Dose and Schedule** The dose of 300 mg once weekly was chosen for the double-blinded Selection placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. Study Visit Schedule and The study for an individual patient will generally consist of the following **Procedures** periods: Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A All patients: A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection Option to participate in an extended treatment period (up to an additional 52 weeks) A 13-week post-treatment evaluation period or expanded access program The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period.

### PROTOCOL SYNOPSIS Continued

| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Change in blood viscosity (may be evaluated) |
| | <ul> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> </ul> |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



### STUDY GLOSSARY

**Index Studies** 

| STUDY GLOSSARY | |
|---|---|
| Abbreviation/Acronym | <u>Definition</u> |
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | glycosylphosphatidylinositol-anchored hdl-binding protein 1 |
| HAPI | heritability and phenotype intervention |
| HbA1c | glycated hemoglobin |
| HDL | high-density lipoprotein |
| HDL-C | high-density lipoprotein-cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| T 1 0 1 | 1919 20 1001 697 11919 20 1001 6917 |

ISIS 304801-CS6 and ISIS 304801-CS16

INR International Normalized Ratio IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL low-density lipoprotein

LDL-C low-density lipoprotein-cholesterol

LMF1 lipase maturation factor 1

LPL lipoprotein lipase

MACE major acute cardiovascular event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL no-observed-adverse-effect level

non-HDL-C non-high-density lipoprotein-cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL triglyceride-rich lipoproteins

ULN upper limit of normal

VLDL very-low-density lipoprotein

VLDL-C very-low-density lipoprotein-cholesterol

VLDL-TG lipoprotein-triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volunesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

ISIS 304801-CS7 **CONFIDENTIAL** Amendment 7 Protocol 7 April 2017

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



**ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** Figure 1

From Ooi et al. 2008: ABCA1 = ATP-binding cassette A1, and = apolipoprotein, CE = cholesterol ester. CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.
The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

# 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volunesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volunesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), in vitro and in vivo genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volunesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (in vitro and in vivo) and was non-genotoxic (in vitro and in vivo). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

# 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

# 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

#### 3.4.3 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.4 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse).

#### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

# 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

# 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.
  - Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:
  - a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
  - b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
    - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
    - Post heparin plasma LPL activity of  $\leq 20\%$  of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study
  - c. Group 2: Fasting  $TG \ge 750 \text{ mg/dL}$  (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
    - Group 3: Fasting TG  $\geq$  750 mg/dL at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study

#### 5. Satisfy 1 of the following:

- a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

# Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c  $\geq$  9.0% at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening

- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$
    - AST > 2.0 x ULN

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Platelet count < lower limit of normal (LLN) for the central laboratory (i.e., < 140,000/mm<sup>3</sup>)
- d. Cardiac Troponin I > ULN at Screening
- e. LDL-C > 130 mg/dL at Screening
- f. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP  $\geq$  160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1

- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to screening
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to screening or planned during the study
  - j. Prior exposure to ISIS 304801
  - k. Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening

- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

# 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

#### 6.1.3 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted

by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.4 Extended Treatment Period

Patients will have the option of continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country.

During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volunesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

# 6.1.5 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.6 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country as described in Section 6.1.4. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. This 13-week post-treatment evaluation period consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A. Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A.

# 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

# 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll-over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65. Patients in the Extended Treatment Period will have ECGs performed in triplicate at Week 76 and Week 104.

# 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period (Week 65).

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service. Patients in the Extended Treatment Period will receive diet/alcohol counseling by qualified study personnel at clinic visits only.

3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet may be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2 and 3)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

# 6.3 Restriction on the Lifestyle of Patients

# 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent<sup>†</sup> or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male

patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

# For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

† Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

# 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

## 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs.

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or

assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

Further Investigation into Liver Chemistry Elevations: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified.

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm<sup>3</sup> (x1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

Amendment 7 7 April 2017

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Protocol

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

## 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

## 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

<u>All patients on insulin</u> will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

<u>All diabetic patients</u> will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - o Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).

o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

#### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

# 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

Protocol

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\ge$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

# 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 50,000/mm<sup>3</sup>, or a platelet count less than 75,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Protocol

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). Triglyceride levels will be monitored weekly, and AE monitoring will continue, during cortiscosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm³. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

## Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Table 3 Actions in Patients with Low Platelet Count or Drop in Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or nonconsecutive) of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. |
| > 100K/mm <sup>3</sup> | Weekly 300 mg Study Drug administration | |
| 100K/mm <sup>3</sup> - >75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks | |
| 75K/mm³ - >50K/mm³ | <ul> <li>If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause</li> <li>When platelet count returns to &gt; 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor Medical Monitor</li> </ul> | <ul> <li>Monitor every 2-3 days until<br/>2 successive values are &gt; 75K/mm³<br/>then monitor every 1 week</li> <li>Consider discontinuation of<br/>antiplatelet agents/NSAIDS/<br/>anticoagulant medication</li> </ul> |
| ≤ 50K/mm³ | Permanently discontinue Study Drug | <ul> <li>Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are &gt; 75K/mm³ then monitor every 1 week</li> <li>Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management</li> <li>Steroids recommended*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline.</li> <li>Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy</li> <li>Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is &lt; 50K/mm³ if possible</li> </ul> |

Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or methylprednisolone 30 mg/kg/day for 7 days (**note**: may require continuation with oral steroids after methylprednisolone)

# 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

# 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

# 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in

Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 65 (or Week 117 if terminating from the Extended Treatment Follow-Up Period), see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

# 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be

recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

# **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

# **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 (or Week 117 if patient enters the extended treatment period) visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### 8.11 Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

## 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH

E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

# 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

# 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volunesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will

begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

# 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

#### 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- **Ongoing:** SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)

• Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

# 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

# 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

# 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

## 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs
- Platelet aggregation (may be evaluated)

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.
#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification). For Group 3 patients, the baseline for fasting lipid measurements is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 in this open-label study.

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study and Group 3 patients, baseline will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naive group which including patients on placebo in index studies and Group 3 patients.

Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG  $\ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volunesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index studies had been on volunesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration ( $C_{max}$ ) and the time taken to reach  $C_{max}$  ( $T_{max}$ ) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24h</sub> /F) will be calculated from  $CL_{0-24h}/F = Actual Dose/AUC_{0-24h}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after

treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP)

as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or

the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### **12.2** Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of pre-study documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting

the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-α expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PC, Voshol PJ, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

## 14. APPENDICES

# **Appendix A** Schedule of Procedures

## Appendix A Schedule of Procedures

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | Trea | ıtmen | t Peri | od | | | | | | | | | Tre | Post<br>atme<br>low-u | nt |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -8 to | -2 to | W | 112 | \A/IL | \A/Iz | Wk | WIL | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | \A/k |
| | Study Week | -6 to<br>-2 | -2 to<br>-1 | | 1 1 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | 8<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | 34<br>&<br>36 | 38 | 40<br>&<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | 54<br>&<br>56 | | 65 |
| | Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 44<br>9 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| ln <sup>-</sup> | formed Consent | Χ | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| O | utpatient Visit | Х | Х | Х | ΧI | ΧI | ΧI | Χ <sup>I</sup> | Χ <sup>I</sup> | ΧI | Χ | Χ <sup>I</sup> | ΧI | ΧI | ΧI | Χ | Χ <sup>I</sup> | ΧI | ΧI | Χ | ΧI | ΧI | ΧI | ΧI | Х | ΧI | ΧI | Х |
| | clusion/Exclusion Criteria | Χ | Χ | | | | | | | | | | | | | | | | | | | | | | | | | |
| | edical History <sup>b</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | Ш |
| (+ | tal Signs + body weight<br>height on Day 1 only) | Х | Х | Х | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| | nysical Examination | Χ | | Х | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Χ | | | Х |
| | 2- lead ECG (triplicate) | Х | | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | | Χ |
| | RI (liver/spleen) | X | | | | | | | | | | | | | | | | | | | | | | | Xm | | | |
| Ed | chocardiography | X | | | | | | | | | | | | | | Xm | | | | | | | | | X <sup>m</sup> | | | |
| | Chemistry Panel | Х | Х | Х | | Χ | | Х | | | Χ | | Χ | | | Χ | | Х | | Χ | | Х | | | X | | Х | Х |
| | CBC with Differential <sup>c</sup> | Х | Х | <b>←</b> | | F | Platel | ets ar | e ass | essec | d each | calen | dar w | eek, v | isits d | — X<br>o not I | nave sp | ecifie | d wind | ows to | o allov | v flexi | bility c | f sche | duling. | | <b>→</b> | Х |
| | Serum Lipid Panel | Х | Х | Х | | Х | | Χ | | Χ | Х | | | | Х | Х | | | | Х | | | | Х | Х | | | Х |
| | Blood viscosity <sup>e</sup> | | | Χ | | | | | | | Χ | | | | | Χ | | | | | | | | | Х | | | |
| <u>p</u> | Platelet aggregation <sup>e</sup> | | Χ | Χ | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | |
| astina) <sup>d</sup> | Coagulation (aPTT, PT, INR) | Х | Х | | | | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | | |
| ast | Hepatitis B, C, HIV | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| aw (F | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | HbA1c | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| تّ | Sedimentation Rate | | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| р | Complement (C5a, Bb) | | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Blood | Troponin I | Х | | Х | | | | | | | Х | | | | | Х | | | | | | | | | X | | | Х |
| | Platelet Bound Autoantibodies <sup>e</sup> | | | Х | | | | | 1 | | | | | | | | | | | | | | | | | | | |
| I | Plasma PK - Volanesorsen | | | Xn | Х | Х | | Х | 1 | | Х | | | | | Х | | l | | Х | | | | | Х | | | Х |
| | Anti-Volanesorsen Antibodies | | | X | Ė | Х | | X | | | Х | | | | | X | | | | X | | | | | X | | П | Х |
| | FSH (women only, if applicable) | Х | | | | | | Ė | 1 | | | | | | | | | l | | | | | | | | | | 一 |
| | Serum Pregnancy Test <sup>f</sup> | X | Х | | | Х | | Х | 1 | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | | Х | Х |

#### Appendix A Schedule of Procedures Continued

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual | | | | | | | | | | Tr | eatm | ent F | eriod | | | | | | | | | | | Treat | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | -2 to<br>-1 | W | /k<br>1 | Wk<br>4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | Mor | nth 3 | Wk<br>15<br>&<br>17 | Wk<br>19 | Wk<br>21<br>&<br>23 | | nth 6 | Wk<br>28<br>&<br>30 | Wk<br>32 | Wk<br>34<br>&<br>36 | Wk<br>38 | Wk<br>40<br>&<br>42 | Wk<br>44 | Wk<br>46<br>&<br>48 | | nth 12 | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | |
| | | _ | - | | - | - | | | | Wk<br>12 | Wk<br>13 | | | | Wk<br>25 | Wk<br>26 | | | | | | | | Wk<br>50 | Wk 52<br>or ET | | | |
| | Study Day | -56 to<br>-15 | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Blood Draw<br>(Fasting) <sup>d</sup> | Archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 3; Group 2 if not available from index study) | | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| ш - | Archived Serum & Plasma<br>Samples <sup>g</sup> | | | Х | | | | Х | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Urina | alysis <sup>d</sup> | Χ | Х | Χ° | | Х | | Х | | | Χ° | | Χ° | | | Χ° | | Χ° | | Χ° | | Χ° | | | Χ° | | Χ° | Χ° |
| | dus Photography <sup>h</sup> | X | ( | | | | | | | | | | | | | | | | | | | | | | X <sup>m</sup> | | | |
| Gen<br>not a | etic testing for FCS diagnosis (if available in medical history) <sup>i</sup> | Х | ( | | | | | | | | | | | | | | | | | | | | | | | | | |
| Wee | kly Study Drug: SC Injection | | | Χ | | Χ | Χ | Χ | Х | Χ | Х | Х | Χ | Χ | Х | Х | Χ | Х | Х | Χ | Χ | Х | Х | Χ | Х | | | |
| Sym | ptom Diary (weekly) | Х | Χ | Х | | Χ | Χ | Х | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Χ | Х | Χ | Х | Х | Χ | Х |
| Qua | lity of Life Assessment(s) | | | Χ | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | Х |
| Food | d/Drink Diary (quarterly) <sup>j</sup> | | | Х | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | <u> </u> | Х |
| Diet/ | 'Alcohol Counseling <sup>k</sup> | Х | Χ | Х | | Х | | Х | | | Х | | | | | Χ | | | | Х | | | | | Х | | Х | Х |
| Adve | erse Events | Х | Χ | Х | | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Х |
| Cond | comitant Medication | Χ | Х | Х | | Х | Х | Х | Х | Χ | Χ | Х | Χ | Х | Х | Χ | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Χ | Х | Х |

- a Screening and Qualification (Group 3) procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor

#### Appendix A Schedule of Procedures Continued

#### Legend Text Continued

- d Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- e May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only
- f Females of childbearing potential only
- Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- h If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- i Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- k To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- I Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- m A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- n Full or abbreviated PK profile (see Appendix C)
- Expanded urinalysis (see Appendix B)

**Appendix A** Schedule of Procedures – Extended Treatment Period

| | Study Period | | | | | | | ٦ | reatme | nt Perio | od | | | | | | | | -Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | Wk 60<br>& 62 | Mo 15<br>Wk 64 | | Wk<br>70 | | Mo 18<br>Wk 76 | | | Wk 84,<br>86, & 88 | | | Wk<br>96 | Wk<br>98,<br>100 &<br>102 | Mo 24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | Wk<br>110 | Mo 27<br>Wk<br>117 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 56<br>8 | 582, 596<br>& 610 | 624 | 638 &<br>652 | 666 | 680,<br>694 &<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Οι | utpatient Visit | $X^f$ | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | $X^f$ | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | $X^f$ | Χ | X <sup>f</sup> | X <sup>f</sup> | Х |
| Vi | tal Signs (+ body weight) | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | Χ |
| Ph | ysical Examination | | | | | | | | Χ | | | | | | | | Χ | | | |
| 12 | - lead ECG (triplicate) | | | | | | | | Χ | | | | | | | | Χ | | | |
| Ur | inalysis(including P/C ratio) | | Х | | Х | | Χ | | Х | | Х | | Х | | Х | | Χ | | Χ | Χ |
| | Chemistry Panel | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | Х | | Χ | | Χ | Χ |
| astina) <sup>b</sup> | CBC with Differential <sup>a</sup> | ▼ | Plate | elets are | assess | ed each | caler | ndar wee | ek. visits | do not | | specified | window | s to allo | w flex | ibility of | schedul | lina. | - | Х |
| i to | Serum Lipid Panel | | | | Χ | | | | X | | | | Χ | | | | Χ | | | Χ |
| 1 4 | Coogulation (aDTT_DT_IND) | | | | Χ | | | | Χ | | | | Χ | | | | Χ | | | |
| Draw | Troponin I | | | | Χ | | | | Χ | | | | Χ | | | | Χ | | | Х |
| Blood | Plasma PK - ISIS 304801° | | | | | | | | Χ | | | | | | | | Χ | | | Х |
| <u>8</u> | Anti-ISIS 304801 Antibodies | | | | | | | | Χ | | | | | | | | Χ | | | Χ |
| | Serum Pregnancy Test <sup>d</sup> | | Х | | Χ | | Χ | | Χ | | Χ | | Χ | | Х | | Χ | | Х | Х |
| W | eekly Study Drug: SC Injection | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Χ | Χ | Χ | | | |
| Di | et/Alcohol Counseling <sup>e</sup> | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | |
| Ac | Iverse Events | Х | Χ | Χ | Х | Χ | Χ | Х | Х | Х | Χ | Х | Х | Х | Χ | Χ | Х | Х | Χ | Χ |
| Co | oncomitant Medication | X | Х | Х | Χ | Х | Х | X | X | Χ | Χ | Х | Χ | Х | Х | X | X | Χ | Х | X |

#### Appendix A Schedule of Procedures – Extended Treatment Period Continued

#### Legend Text

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

# **Appendix B** List of Laboratory Analytes

## Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| linical Chemistry Panel | <b>Screening Tests (Group 3)</b> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| <ul> <li>Sodium</li> <li>Potassium</li> <li>Chloride</li> <li>Bicarbonate</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>Phosphorus</li> <li>Glucose</li> <li>BUN</li> <li>Creatinine</li> <li>Uric Acid</li> <li>Total bilirubin</li> </ul> | <ul> <li>Hepatitis B surface antigen</li> <li>Hepatitis C antibody</li> <li>HIV antibody</li> <li>FSH (women only)</li> <li>Serum βhCG (women only)</li> </ul> Coagulation <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> </ul> | <ul> <li>Red blood cells</li> <li>Hemoglobin</li> <li>Hematocrit</li> <li>MCV, MCH, MCHC</li> <li>Platelets</li> <li>White blood cells</li> <li>WBC Differential (% and absolute)</li> <li>Neutrophils</li> <li>Eosinophils</li> <li>Basophils</li> <li>Lymphocytes</li> <li>Monocytes</li> </ul> | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>4</sup></li> </ul> |
| <ul> <li>Direct (conjugated) bilirubin</li> <li>Indirect (unconjugated) bilirubin</li> <li>ALT</li> <li>AST</li> <li>Alkaline phosphatase</li> </ul> | <ul> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | Pharmacokinetics¹ & Immunogenicity • Volanesorsen levels in plasma • Anti-volanesorsen antibodies in plasma Other Assessments • hsCRP • Sedimentation Rate • C5a, Bb • Troponin I² • CK-MB² • Platelet Bound Autoantibodies³ • De-lipidated free glycerol • HbA1c, FPG • Blood viscosity³ | Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin β2-microglobulin Platelet Function Platelet aggregation <sup>3</sup> |

- 1 Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

#### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

#### **PK Sampling Schedule (Extended Treatment Period)**

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|-----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose, | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hem | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 - 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm <sup>3</sup> ;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | | pH >7.5 |
| Aspartate<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>Ionized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | • | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | • | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 -<br/>7.0 mg/dL; &lt;2.0 - 1.75 mmol/L;<br/>lonized calcium &lt;1.0 - 0.9<br/>mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 -<br>7.0 mg/dL; <2.0 - 1.75 mmol/L;<br>lonized calcium <1.0 - 0.9<br>mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td></td><td>&lt;130 mmol/L</td></lln> | | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria | 1 | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





A subsidiary of Ionis Pharmaceuticals, Inc.

**Sponsor:** Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

#### ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 7 - France – 3 February 2017** 

EudraCT No: 2015-003755-21

## ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 7 - France - 3 February 2017

#### Protocol History:

Original Protocol:

28 August 2015

Protocol Amendment 1:

2 February 2016

Protocol Amendment 2:

22 April 2016

Protocol Amendment 3:

9 May 2016

Protocol Amendment 4:

6 June 2016

Protocol Amendment 5:

19 August 2016

Protocol Amendment 6:

16 September 2016

#### Sponsor:

Ionis Pharmaceuticals, Inc.
2855 Gazelle Cc
Carlsbad, CA 92

MD, MBA

#### Protocol - France

Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 7 - France** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200 Fax:

Key Sponsor Contact:

Ph.D.
2855 Gazelle Court

Carlsbad, CA 92010 Phone:

\_\_\_\_\_

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 3 February 2017

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Volanesorsen Administered Subcutaneous<br>Patients with Familial Chylomicronemia Syndrome (FCS) | |
| Amendment: | Amendment 7 - France | |
| Date: | 3 February 2017 | |
| Open-Label Study of | Volanesorsen Administered S | and the attached clinical protocol, entitled "An Subcutaneously to Patients with Familial nary 2017, and agree to conduct the study as |
| I agree to comply wit<br>Good Clinical Praction | | e on Harmonization Tripartite Guideline on |
| any purpose other that | | contained in this document will not be used for fithe clinical investigation without the prior |
| Investigator's Signat | ture | |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| DD ( | OTOGOL AMENDMENT | Page |
|---|---|---|
| | OTOCOL AMENDMENTOTOCOL SYNOPSIS | |
| | UDY DESIGN AND TREATMENT SCHEMA | |
| | UDY GLOSSARYUDY GLOSSARY | |
| 1.<br>2. | OBJECTIVES BACKGROUND AND RATIONALE | |
| | 2.1 Overview of Disease | |
| | 2.2 Therapeutic Rationale | |
| | 2.3 Volanesorsen | |
| _ | 2.3.1 Mechanism of Action | |
| | 2.3.2 Chemistry | |
| | 2.3.3 Preclinical Experience | |
| | 2.3.4 Clinical Experience | |
| 2. | 2.4 Rationale for Dose and Schedule of Administration | |
| 3. | EXPERIMENTAL PLAN | 29 |
| 3 | 3.1 Study Design | 29 |
| 3. | Number of Study Centers | 29 |
| 3 | Number of Patients | 29 |
| 3. | 3.4 Overall Study Duration and Follow-up | 29 |
| | 3.4.1 Qualification | 29 |
| | 3.4.2 Treatment | 29 |
| | 3.4.3 Post-Treatment | |
| 3. | 3.5 End-of-Study | |
| | Data and Safety Monitoring Board | |
| 4. | PATIENT ENROLLMENT | |
| | 4.1 Qualification | |
| | 4.2 Enrollment | |
| 5. | | |
| | 5.1 Inclusion Criteria | |
| | 5.2 Exclusion Criteria | |
| 6. | STUDY PROCEDURES | |
| 6. | 5.1 Study Schedule | |
| | 6.1.1 Qualification | |
| | 6.1.2 Treatment Period | |
| | <ul><li>6.1.3 Pharmacokinetic (PK) Subgroup</li><li>6.1.4 Post-Treatment Period</li></ul> | |
| 6 | 5.2 Additional Study Assessments | |
| U. | 6.2.1 Laboratory Assessments | |
| | 0.2.1 Laboratory Assessments | |

| | 6.2.2 | Physical Exams and Vital Signs | .35 |
|---|---|---|---|
| | 6. | .2.2.1 Eruptive Xanthoma | .36 |
| | 6. | .2.2.2 Lipemia Retinalis | |
| | 6.2.3 | 3 Echocardiography | .36 |
| | 6.2.4 | 4 ECG | .36 |
| | 6.2. | 5 MRI | .36 |
| | 6.2.0 | 6 Quality of Life Assessments | .36 |
| | 6.2. | 7 Disease Symptom Diary | .36 |
| | 6.2.8 | 8 Diet Monitoring | .36 |
| | 6.2.9 | 9 Family History | .37 |
| | 6.3 | Restriction on the Lifestyle of Patients | .37 |
| | 6.3. | 1 Contraception Requirements | .37 |
| | 6.3.2 | 2 Other Requirements | .38 |
| 7. | . S' | TUDY DRUG | 38 |
| | 7.1 | Volanesorsen Description | .38 |
| | 7.2 | Packaging and Labeling. | .39 |
| | 7.3 | Study Drug Accountability | .39 |
| 8. | . <b>T</b> | REATMENT OF PATIENTS | <b>39</b> |
| | 8.1 | Volanesorsen Administration | .39 |
| | 8.2 | Other Protocol-Required Drugs | .39 |
| | 8.3 | Other Protocol-Required Treatment Procedures | .39 |
| | 8.4 | Treatment Precautions | .39 |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , , | |
| | 8.5.2 | , | |
| | 8.5.3 | , | |
| | 8.5.4 | , U | |
| | 8.5.5 | $\mathcal{E}$ | |
| | 8.5.0 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | .42 |
| | 8.5.7 | 7 Safety Monitoring for Documented Severe Hypoglycemia | .42 |
| | 8.5.8 | 8 Safety Monitoring for Hyperglycemia | .43 |
| | 8.5.9 | 9 Acute Pancreatitis | .44 |
| | 8.6 | Stopping Rules | .44 |
| | 8.6. | 11 8 | |
| | 8.6.2 | 2 Stopping Rules for Renal Function Test Results | .45 |
| | 8.6.3 | | |
| | 8.7 | Adjustment of Dose Frequency | |
| | 8.8 | Discontinuation of Study Treatment | |
| | 8.8. | 1 | |
| | 8.8.2 | 2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period | 48 |

| | 8.9 | Withdrawal of Patients from the Study | 49 |
|---|---|---|---|
| | 8.10 | Concomitant Therapy and Procedures | |
| | 8.10 | | |
| | 8.10 | .2 Concomitant Procedures | 50 |
| | 8.11 | Treatment Compliance | 50 |
| 9. | . <b>S</b> | ERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 50 |
| | 9.1 | Sponsor Review of Safety Information | 50 |
| | 9.2 | Regulatory Requirements | 50 |
| | 9.3 | Definitions | 51 |
| | 9.3. | Adverse Event | 51 |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 51 |
| | 9.3.3 | Serious Adverse Event (SAE) | 52 |
| | 9.4 | Monitoring and Recording Adverse Events | 52 |
| | 9.4. | Serious Adverse Events | 52 |
| | 9.4.2 | Non-Serious Adverse Events | 53 |
| | 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | 53 |
| | 9. | 4.3.1 Relationship to the Study Drug | 53 |
| | 9. | 4.3.2 Severity | 53 |
| | 9. | 4.3.3 Action Taken with Volanesorsen | 54 |
| | 9. | 4.3.4 Treatment Given for Adverse Event | 54 |
| | 9. | 4.3.5 Outcome of the Adverse Event | |
| | 9.4.4 | Adjudication Committees | 55 |
| | 9.5 | Procedures for Handling Special Situations | 55 |
| | 9.5. | Abnormalities of Laboratory Tests | 55 |
| | 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 55 |
| | 9.5.3 | B Dosing Errors | 56 |
| | 9.5.4 | Contraception and Pregnancy | 56 |
| 1 | 0. S' | FATISTICAL CONSIDERATIONS | 57 |
| | 10.1 | Study Endpoints | 57 |
| | 10.1 | .1 Efficacy Endpoints | 57 |
| | 10.1 | .2 Safety Endpoints | 57 |
| | 10.2 | Sample Size | |
| | 10.3 | Populations | 57 |
| | 10.4 | Definition of Baseline | |
| | 10.5 | Interim Analysis | |
| | 10.6 | Planned Methods of Analysis | |
| | 10.6 | | |
| | 10.6 | | |
| | 10.6 | | |
| | 10.6 | .4 Pharmacokinetic and Immunogenicity Analysis | 60 |

| 10.6.4.1 | Pharmacokinetic Analysis | 60 |
|---|---|---|
| 10.6.4.2 | Immunogenicity Analysis | |
| 11. INVEST | IGATOR'S REGULATORY OBLIGATIONS | |
| | ed Consent | |
| | Conduct of the Study | |
| | ndent Ethics Committee/Institutional Review Board | |
| | Confidentiality | |
| | STRATIVE AND LEGAL OBLIGATIONS | |
| | ol Amendments | |
| 12.2 Study | Termination | 62 |
| 12.3 Study 1 | Documentation and Storage | 63 |
| • | Monitoring | |
| 12.5 Langua | age | 64 |
| | ensation for Injury | |
| - | ENCES | |
| 14. APPENI | DICES | 67 |
| Appendix A | Schedule of Procedures | 68 |
| Appendix B | List of Laboratory Analytes | 74 |
| Appendix C | Pharmacokinetic Sampling Schedule | 76 |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 V | olanesorsen (ISIS 304801) Characteristics | 38 |
| | ctions in Patients with Low Platelet Count | |
| Table 3 Ex | xpected Event for the Protocol Defined Population by Preferred Term | |
| | nd the Expected Incidence | |
| | TABLE OF FIGURES | |
| | | D |
| Eiguro 1 A | noC III Dagulatas Linanyatain Matakalism ky Multipla Mackanisma | Page |
| | poC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 23 |
| | esign of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | 25 |
| (1) | MOE-Gapmer). The sequence of volunesorsen is shown | / 7 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 7 - France

**Amendment Date:** 3 February 2017

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 6 dated 16 September 2016:

- 1. To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies
- 2. To add post heparin plasma LPL activity of ≤ 20% of normal in medical history as an inclusion criteria for ISIS 304801-CS16 (Group 2) patients as has been allowed for ISIS 304801-CS6 (Group 1) patients

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Design<br>3.1 Study Design | Was This is a multi-center open-label study of: Group 1: ISIS 304801-CS6 (index study) roll over FCS patients Group 2: ISIS 304801-CS16 (index study) roll over FCS patients Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies Is This is a multi-center open-label study of: Group 1: ISIS 304801-CS6 (index study) roll over FCS patients Group 2: ISIS 304801-CS16 (index study) roll over FCS patients | To exclude<br>enrollment of FCS<br>patients who did<br>not participate in<br>an index study<br>from this open<br>label study |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Population<br>5.1 Inclusion Criteria | <ul> <li>Was</li> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> </li> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study Group 1st between</li> </ul></li></ul> | To define the inclusion criteria for each group of patients. To add LPL activity of ≤ 20% of normal in medical history as an inclusion criteria for Group 2 patients as has been allowed for Group 1 patients |
| | <ul> <li>Is</li> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the openlabel study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical history</li> <li>c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study</li> </ul> </li> </ul></li></ul> | |
| Protocol Synopsis:<br>Study Population<br>5.2 Exclusion Criteria | Was (noted throughout Exclusion Criteria) Screening* *(Group 3) or Qualification (Groups 1 and 2) Is (noted throughout Exclusion Criteria) Qualification | To distinguish that patients who are rolling over from an index study will have Qualification assessments |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis: Study Visit Schedule and Procedures 3.4 Overall Study Duration and Follow-up Study Design and Treatment Schema | <ul> <li>Was</li> <li>The study for an individual patient will generally consist of the following periods:</li> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.</li> <li>Group 3 patients (did not participate in an index study): An</li> </ul> | To remove FCS patients who did not participate in an index study from the study schedule |
| Appendix A | up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A. • All patients: | |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection</li> <li>A 13-week post-treatment evaluation period</li> </ul> | |
| | <u>Is</u> The study for an individual patient will generally consist of the following periods: | |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by<br/>the Sponsor). Please refer to Section 4.1 and Appendix A.</li> </ul> | |
| | <ul> <li>A 52-week treatment period during which volanesorsen will<br/>be administered as a once weekly SC injection</li> </ul> | |
| | A 13-week post-treatment evaluation period | |
| 4.1<br>Screening/Qualification | Was Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial. | To remove FCS patients who did not participate in an index study from Screening/ Qualification |
| | Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and rescreened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used. | |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| 4.1<br>Screening/Qualification<br>Continued | Ls During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial. | To remove FCS patients who did not participate in an index study from Screening/ Qualification |
| 6.1.1 Screening 6.1.2 Screening and Qualification (Group 3) | Was 6.1.1 Qualification (Groups 1 and 2) Please refer to Section 4.1 and Appendix A. 6.1.2 Screening and Qualification (Group 3) Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes Is 6.1.1 Qualification Please refer to Section 4.1 and Appendix A. | To remove FCS patients who did not participate in an index study from Screening/ Qualification |
| Section 10.3<br>Populations | Updated: Full Analysis Set (FAS): All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. PK Population: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported. | Modified to include, in the FAS, only those patients that are randomized and dosed and have a baseline TG assessment and clarified the PK Population |
# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) by documentation of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical<br/>history</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study |
| | 4. Able and willing to participate in a 78-week study |

#### Study Population Continued

#### Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **Exclusion Criteria:**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b. HbA1c ≥ 9.0% at Qualification
  - Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)
  - e. Current use of GLP-1 agonists
- Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification

#### Study Population Continued

### Exclusion Criteria: Continued

- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria: Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to Qualification and dose<br>and regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>Qualification</li> </ul> |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to Qualification |
| | <ul> <li>g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br/>apixaban) unless on a stable dose for at least 4 weeks prior to<br/>Qualification and regular clinical monitoring is performed</li> </ul> |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period |
| | <ul> <li>Plasma apheresis within 4 weeks prior to Qualification or planned<br/>during the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A</li> </ul> |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | An at least 26-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |
| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |

| Planned Analyses | Safety Endpoints: |
|---|---|
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation,<br/>urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

# STUDY DESIGN AND TREATMENT SCHEMA



# STUDY GLOSSARY

| Abbraviation/Amonym | Definition |
|---|---|
| Abbreviation/Acronym | Definition |
| ADA | anti-drug antibody |
| ALD | adverse Event |
| ALT | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |
| mach budges | 1010 50 1001 C00 wild 1010 50 1001 C010 |

Amendment 7 3 February 2017 Protocol - France

#### STUDY GLOSSARY Continued

| Abbreviation/Acronym | <u>Definition</u> |
|----------------------|-------------------|

INR International Normalized Ratio **IRB** Institutional Review Board

**IXRS** Interactive Voice/Web-Response System

**LDL** Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

Lipase Maturation Factor 1 LMF1

LPL Lipoprotein Lipase

Major Acute Cardiovascular Event **MACE** 

**MOE** 2'-O-(2-methoxyethyl)

magnetic resonance imaging MRI mRNA messenger ribonucleic acid **NCS** not clinically-significant

No-Observed-Adverse-Effect Level **NOAEL** 

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event Statistical Analysis Plan SAP

SC subcutaneous

**SUSAR** suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

time to maximal concentration  $T_{\text{max}}$ 

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

Triglyceride-Rich Lipoproteins **TRL** 

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride World Medical Association **WMA** 

#### 1. **OBJECTIVES**

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volunesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

Amendment 7

3 February 2017

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 **ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** 

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

# 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

# 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

## 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

# 3. EXPERIMENTAL PLAN

### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities.

# 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

# 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Qualification

A qualification period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is at least 26 weeks and consists of at least 6 Study Center visits on Weeks 54, 56, 58, 65, 71, and 78 (Weeks 54, 56, 58, and 71 may be conducted by a home healthcare nurse).

# 3.5 End-of-Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide

recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

### 4.1 Qualification

Protocol - France

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of  $\leq 20\%$  of normal in medical history
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
- 4. Able and willing to participate in a 78-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of Qualification
  - b.  $HbA1c \ge 9.0\%$  at Qualification
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of Qualification [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)

- e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to Qualification
- 4. History within 6 months of Qualification of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of Qualification
- 5. Any of the following laboratory values at Qualification
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$
    - AST  $> 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests  $\geq$  trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing  $\leq$  5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Qualification
- d. LDL-C > 130 mg/dL at Qualification
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Qualification
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1

- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1 month of Qualification, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to Qualification
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to Qualification unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to Qualification and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to Qualification
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to Qualification and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to Qualification and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to Qualification or planned during the study
  - j. Prior exposure to ISIS 304801
  - k. Any other medication unless stable at least 4 weeks prior to Qualification (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of Qualification or of > 499 mL within 60 days of Qualification
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)

17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, and 50 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

## 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this

subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. The 26-week period consists of at least 6 Study Center visits on Weeks 54, 56, 58, 65, 71, and 78 (Weeks 54, 56, 58, and 71 may be conducted by a home healthcare nurse), as outlined in the Schedule of Procedures in Appendix A.

## 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

## 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

# 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

# 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, Week 65, and Week 78.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.

### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

# 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.

- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.3 **Restriction on the Lifestyle of Patients**

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent<sup>†</sup> or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq$  55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

# For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

† Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 °C to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 **Packaging and Labeling**

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 **Study Drug Accountability**

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### TREATMENT OF PATIENTS 8.

#### 8.1 **Volanesorsen Administration**

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volunesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 **Other Protocol-Required Drugs**

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 **Other Protocol-Required Treatment Procedures**

There are no other protocol required treatment procedures for this study.

#### 8.4 **Treatment Precautions**

There are no specific treatment precautions required for this study.

#### 8.5 **Safety Monitoring Rules**

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

# 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3.

Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

# 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional

symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

# 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

<u>All diabetic patients</u> will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as one in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the

patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

# 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

• Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)

- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\ge 2$  weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5

4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24 hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

# 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 2 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

# <u>Definition of Clinically-Relevant, Non-Major Bleeding Events</u> (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Protocol - France

Table 2 **Actions in Patients with Low Platelet Count** 

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1 week until stable* |
| 75K-100K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1 week |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and  $> 100,000/\text{mm}^3$ 

#### 8.7 **Adjustment of Dose Frequency**

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 2 (above).

Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

## **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

# 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and  $> 100,000/\text{mm}^3$ ), the next platelet count should be taken within at least
6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 78, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline Qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 78 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Protocol - France

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 3 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial

Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

• **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities

- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- **Ongoing:** SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

STATISTICAL CONSIDERATIONS

Protocol - France

10.

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### **10.2** Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

Per Protocol Set (PPS): Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

PK Population: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### 10.4 **Definition of Baseline**

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline will be the last non-missing assessment prior to the first dose of Study Drug. Details will be provided in the SAP.

#### 10.5 **Interim Analysis**

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 **Planned Methods of Analysis**

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active Study Drug in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naïve group which includes patients on placebo in index studies. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG  $\geq 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volunesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study will receive the first treatment of volunesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration  $(CL_{0-24h}/F)$  will be calculated from  $CL_{0-24h}/F = Actual Dose/AUC_{0-24h}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with

positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., %change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of

Amendment 7 3 February 2017

the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 **Patient Confidentiality**

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 **Protocol Amendments**

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 **Study Termination**

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

## 14. APPENDICES

# **Appendix A** Schedule of Procedures

Qualification through Treatment Period

Post-Treatment Follow-up

 $Appendix \ A \quad Schedule \ of \ Procedures - Qualification \ through \ Treatment \ Period$ 

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | | Treatr | nent F | Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | w | /I. | \A/Iz | \A/Iz | \A/Iz | Wk | \A/Iz | Mon | th 3 | Wk<br>15 | Wk | Wk<br>21 | Mon | th 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | onth 12 |
| | Study Week | -2 to -1 | 1 | l<br>I | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| | Study Day | -14 to -7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| | Visit Window+/- Days | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Info | ormed Consent | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| | tpatient Visit | Х | Х | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | Χ | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | Χ | $X^{j}$ | $X^{j}$ | X <sup>j</sup> | Χ | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | $X^{j}$ | Χ |
| | lusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | | | | |
| | al Signs + body weight<br>height on Day 1 only) | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х |
| | ysical Examination | Х | Х | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х |
| 12- | · lead ECG (triplicate) | Х | | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х |
| | RI (liver/spleen) | Х | | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| | hocardiography | Х | | | | | | | | | | | | | | $X^k$ | | | | | | | | | $X^k$ |
| | Chemistry Panel | Х | Х | | | Х | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | | Х | Х | Х | Х | Χ | Χ | Х | Х | Χ | Х | Χ | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х |
| | Serum Lipid Panel | Х | Х | | | Χ | | Χ | | Χ | Χ | | | | Χ | Χ | | | | Χ | | | | Χ | Х |
| ی ا | Coagulation (aPTT, PT, INR) | Χ | | | | | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | X <sup>n</sup> | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Fa | Sedimentation Rate | | Х | | | | | | | | Х | | | | | Χ | | | | | | | | | Х |
| ≥ | Complement (C5a, Bb) | | Х | | | | | | | | Χ | | | | | Χ | | | | | | | | | Х |
| Draw | Plasma PK - Volanesorsen | | Χ¹ | Х | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| l b | Anti-Volanesorsen Antibodies | | Х | | | Χ | | Х | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| Blood | FSH (women only, if applicable) | Х | | | | | | | | | | | | | | | | | | | | | | | |
| B | Serum Pregnancy Test <sup>d</sup> | Χ | | | | Χ | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | X |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | Х | | | | | Х | | | Х | | | | | Х | | | | | | | | | Х |
| 1 | Troponin I° | Х | | | | | | | | | | | | | | | | | | | | | | | |

**Appendix A** Schedule of Procedures - Qualification through Treatment Period *Continued* 

| Study Period | Qual <sup>a</sup> | | | | | | | | | | | Tı | reatmo | ent Pe | riod | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | w | 'k | Wk | Wk | Wk | Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 |
| Study Week | -2 to -1 | "1 | | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| Study Day | -14 to -<br>7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| Visit Window+/- Days | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Urinalysis <sup>c</sup> | Х | $X^{m}$ | | | Х | | Х | | | X <sup>m</sup> | | $X^{m}$ | | | X <sup>m</sup> | | $X^{m}$ | | $X^{m}$ | | X <sup>m</sup> | | | X <sup>m</sup> |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | $X^k$ |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>g</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ |
| Quality of Life Assessment(s) | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х |
| Adverse Events | Х | Χ | | Х | Х | Χ | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х |
| Concomitant Medication | Х | Χ | | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х |

# ${\bf Appendix} \ {\bf A} \quad {\bf Schedule} \ {\bf of} \ {\bf Procedures-Post-Treatment} \ {\bf Follow-up}$

| | Study Period | Post | Treat | ment | Follow | /-up <sup>p</sup> |
|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| | Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Informe | ed Consent | | | | | |
| | ient Visit | X <sup>j</sup> | $X^{j}$ | Χ | X <sup>j</sup> | Х |
| | on/Exclusion Criteria | | | | | |
| | gns + body weight | | | Х | | Х |
| , , | ht on Day 1 only) | | | · · | | · · |
| | al Examination | | | X | | X |
| | d ECG (triplicate) ver/spleen) | | | Λ. | | ^ |
| _ \ | , , | | | | | |
| ECHOCA | ardiography | | | | | · · |
| | Chemistry Panel | Х | X | X | X | X |
| | CBC with Differential <sup>b</sup> Serum Lipid Panel | Λ | | X | Λ | X |
| ی د | Coagulation (aPTT, PT, INR) | | | ^ | | _^_ |
| ing | hsCRP, HbA1c, FPG, and | | | | | |
| ast | de-lipidated free glycerol | | | Χ | | Х |
| Ē, | Sedimentation Rate | | | Х | | Χ |
| a | Complement (C5a, Bb) | | | Χ | | Χ |
| Blood Draw (Fasting) <sup>c</sup> | Plasma PK - Volanesorsen | | | Χ | | Χ |
| poo | Anti-Volanesorsen Antibodies | | | Χ | | Χ |
| 용 | FSH (women only, if applicable) | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | | Χ | Χ | Χ | Χ |
| | Archived Serum & Plasma Samples <sup>e</sup> | | | Χ | | Χ |
| | Troponin I° | | | | | |

# ${\bf Appendix} \ {\bf A} \quad {\bf Schedule} \ {\bf of} \ {\bf Procedures-Post-Treatment} \ {\bf Follow-up} \ {\bf \it Continued}$

| Study Period | Pos | st Treat | tment I | Follow- | up <sup>p</sup> |
|---|---|---|---|---|---|
| Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Urinalysis <sup>c</sup> | | X <sup>m</sup> | X <sup>m</sup> | $X^{m}$ | $X^{m}$ |
| Fundus Photography <sup>f</sup> | | | | | |
| Genetic testing for FCS diagnosis<br>(if not available in medical<br>history) <sup>9</sup> | | | | | |
| Weekly Study Drug: SC Injection | | | | | |
| Symptom Diary (weekly) | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | | Х | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | | Х | Х | Х | Χ |
| Adverse Events | Х | Х | Х | Х | Х |
| Concomitant Medication | Х | Х | Х | Х | Х |

CONFIDENTIAL Amendment 7 Protocol - France 3 February 2017

#### Appendix A Schedule of Procedures Continued

- Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>. In the event of any platelet count less than 50,000/mm<sup>3</sup> or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently. Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor
- Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- Females of childbearing potential only
- Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 ISIS 304801-CS16 roll over patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- Genetic testing can be conducted for study Qualification (Group 2 ISIS 304801-CS16 roll over patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- Full or abbreviated PK profile (see Appendix C)
- Expanded urinalysis (see Appendix B) m
- HbA1c only n
- All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB 0
- If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values

# **Appendix B** List of Laboratory Analytes

## Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| | Hematology | Uringlysis |
|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Potasium P | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Pharmacokinetics¹ KImmunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | Urinalysis Color Appearance Specific gravity pH Protein Blood Ketones Urobilinogen Glucose Bilirubin Leukocyte esterase Nitrate Microscopic examination <sup>2</sup> Additional Measures for Expanded Urinalysis Total protein (quantitative) Microslobulin |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

## PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime | Anytime |

## PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>Post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>Ionized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 -<br/>7.0 mg/dL; &lt;2.0 - 1.75 mmol/L;<br/>Ionized calcium &lt;1.0 - 0.9<br/>mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 -<br>7.0 mg/dL; <2.0 - 1.75 mmol/L;<br>Ionized calcium <1.0 - 0.9<br>mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria | 1 2 2 2 2 2 | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaguist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

#### **Collaborator:**

Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

#### ISIS 304801-CS7

# The APPROACH Open-Label Study Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 6 - Netherlands - 11 April 2017

EudraCT No: 2015-003755-21

## ISIS 304801-CS7

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

## An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

## Protocol Amendment 6 - Netherlands - 11 April 2017

#### **Protocol History:**

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

Protocol Amendment 3: 9 May 2016

Protocol Amendment 4: 6 June 2016

Protocol Amendment 5: 6 July 2016

#### Sponsor:

Ionis Pharmaceuticals, Inc.
2855 Gazelle Court
Carlsbad, CA 92010

MD, MBA

#### **Ionis Protocol Number: ISIS 304801-CS7**

**Protocol Amendment 6 - Netherlands** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200 Fax:

**Key Sponsor Contact:** 

, Ph.D. 2855 Gazelle Court

Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 11 April 2017

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.
# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) | |
| Amendment: | Amendment 6 Netherlands | |
| Date: | 11 April 2017 | |
| Open-Label Study of Chylomicronemia Sydescribed herein. I agree to comply wit Good Clinical Practical Practical agree to ensure that any purpose other that | th the International Conference (E6). the confidential information of an the evaluation or conduct of nis Pharmaceuticals, Inc. | nd the attached clinical protocol, entitled "An ubcutaneously to Patients with Familial 1 2017, and agree to conduct the study as on Harmonization Tripartite Guideline on ontained in this document will not be used for the clinical investigation without the prior |
| Investigator's Name | e (please print) | Date (DD Month YYYY) |

# **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| PRO | госо | L AMENDMENT | 10 |
| <b>PRO</b> | ГОСО | L SYNOPSIS | 28 |
| STUI | OY DE | SIGN AND TREATMENT SCHEMA | 32 |
| STUI | | OSSARY | |
| 1. | OBJ | ECTIVES | 35 |
| 2. | | KGROUND AND RATIONALE | |
| 2.1 | | verview of Disease | |
| 2.2 | | nerapeutic Rationale | |
| 2.3 | Vo | planesorsen | |
| | 2.3.1 | Mechanism of Action | |
| | 2.3.2 | Chemistry | |
| 2 | 2.3.3 | Preclinical Experience | |
| | 2.3.4 | Clinical Experience | |
| 2.4 | | ationale for Dose and Schedule of Administration | |
| 3. | | ERIMENTAL PLAN | |
| 3.1 | | udy Design | |
| 3.2 | | umber of Study Centers | |
| 3.3 | | umber of Patients | |
| 3.4 | | verall Study Duration and Follow-up | |
| 3 | 3.4.1 | Qualification | |
| _ | 3.4.2 | Treatment | |
| _ | 3.4.3 | Post-Treatment | |
| 3.5 | | nd-of-Study | |
| 3.6 | | ata and Safety Monitoring Board | |
| 4. | | IENT ENROLLMENT | |
| 4.1 | | ualification | |
| 4.2 | | rollment | |
| <b>5.</b> | | IENT ELIGIBILITY | |
| 5.1 | | clusion Criteria | |
| 5.2 | | aclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (IS | |
| | | dex Study Roll-over Patients | |
| 6. | | DY PROCEDURES | |
| 6.1 | | udy Schedule | |
| | 5.1.1 | Qualification | |
| | 5.1.2 | Treatment Period | |
| | 5.1.3 | Extended Treatment Period | |
| 6 | 5.1.4 | Pharmacokinetic (PK) Subgroup | 46 |

| | 6.1. | Post-Treatment Period | 46 |
|----|--------------|-----------------------------------------------|----|
| | 6.2 | Additional Study Assessments | 47 |
| | 6.2. | Laboratory Assessments | 47 |
| | 6.2. | Physical Exams and Vital Signs | 47 |
| | 6 | 2.2.1 Eruptive Xanthoma | 47 |
| | 6 | 2.2.2 Lipemia Retinalis | 47 |
| | 6.2. | Echocardiography | 47 |
| | 6.2. | | |
| | 6.2. | | |
| | 6.2. | | |
| | 6.2. | J 1 | |
| | 6.2. | $oldsymbol{arepsilon}$ | |
| | 6.2. | | |
| | 6.2. | J ( 1 ) | |
| | 6.3 | Restriction on the Lifestyle of Patients | |
| | 6.3. | | |
| | 6.3. | 1 | |
| 7. | | TUDY DRUG | |
| | 7.1 | Volanesorsen Description | |
| | 7.2 | Packaging and Labeling | |
| _ | 7.3 | Study Drug Accountability | |
| 8. | | REATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , | |
| | | Safety Monitoring for Platelet Count Results | |
| | 8.5.<br>8.5. | | |
| | 8.5. | | |
| | 8.5. | • | |
| | 8.5. | • | |
| | 8.5. | | |
| | 8.5. | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | Stopping Rules for Liver Chemistry Elevations | |
| | 8.6. | • | |
| | 8.6. | | 58 |

| | 8.7 | Ad | justment of Dose Frequency | 61 |
|---|---|---|---|---|
| | 8.8 | Dis | continuation of Study Treatment | 61 |
| | 8.8. | 1 | Follow-up Visits for Early Termination from Treatment Period | 61 |
| | 8.8.2 | 2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Peri | od .62 |
| | 8.9 | Wi | thdrawal of Patients from the Study | 62 |
| | 8.10 | Con | ncomitant Therapy and Procedures | 62 |
| | 8.10 | ).1 | Concomitant Therapy | 63 |
| | 8.10 | ).2 | Concomitant Procedures | 63 |
| | 8.11 | Tre | atment Compliance | 63 |
| 9. | . <b>S</b> ] | ERI | OUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 64 |
| | 9.1 | Spo | onsor Review of Safety Information | 64 |
| | 9.2 | Reg | gulatory Requirements | 64 |
| | 9.3 | Det | finitions | 65 |
| | 9.3. | 1 | Adverse Event | |
| | 9.3.2 | 2 | Adverse Reaction and Suspected Adverse Reaction | |
| | 9.3.3 | 3 | Serious Adverse Event (SAE) | 65 |
| | 9.4 | Mo | nitoring and Recording Adverse Events | 66 |
| | 9.4. | 1 | Serious Adverse Events | |
| | 9.4.2 | 2 | Non-Serious Adverse Events | |
| | 9.4.3 | 3 | Evaluation of Adverse Events (Serious and Non-Serious) | |
| | 9. | .4.3. | 1 Relationship to the Study Drug | 66 |
| | 9. | .4.3. | • | |
| | 9. | .4.3. | 3 Action Taken with Volanesorsen | 67 |
| | 9. | .4.3. | | |
| | 9. | .4.3 | | |
| | 9.4.4 | 4 | Adjudication Committees | 68 |
| | 9.5 | Pro | cedures for Handling Special Situations | |
| | 9.5. | | Abnormalities of Laboratory Tests | |
| | 9.5.2 | 2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 69 |
| | 9.5.3 | | Dosing Errors | |
| | 9.5.4 | | Contraception and Pregnancy | |
| 10 | 0. S' | | TISTICAL CONSIDERATIONS | |
| | 10.1 | | dy Endpoints | |
| | 10.1 | | Efficacy Endpoints | |
| | 10.1 | | Safety Endpoints | |
| | 10.2 | | nple Size | |
| | 10.3 | _ | pulations | |
| | 10.4 | | finition of Baseline | |
| | 10.5 | | erim Analysis | |
| | 10.6 | Dla: | nned Methods of Analysis | 72 |

| ocol - Netherlands | | 11 April 2017 |
|---|---|---|
| 10.6.1 | Demographic and Baseline Characteristics | 72 |

| .1 Demographic and Baseline Char | acteristics | 2 |
|---|---|---|
| .3 Efficacy Analysis | 7 | 3 |
| .4 Pharmacokinetic and Immunoge | nicity Analysis7 | 3 |
| 0.6.4.1 Pharmacokinetic Analysis | 7 | 3 |
| 0.6.4.2 Immunogenicity Analysis | | 4 |
| NVESTIGATOR'S REGULATORY | OBLIGATIONS74 | 4 |
| Informed Consent | 7- | 4 |
| Ethical Conduct of the Study | 7 | 5 |
| Independent Ethics Committee/Instit | utional Review Board7 | 5 |
| Patient Confidentiality | 7 | 5 |
| DMINISTRATIVE AND LEGAL ( | DBLIGATIONS70 | 6 |
| Protocol Amendments | 70 | 6 |
| Study Termination | 7 | 6 |
| Study Documentation and Storage | 70 | 6 |
| • | | |
| Language | 7′ | 7 |
| Compensation for Injury | 7′ | 7 |
| EFERENCES | | 8 |
| PPENDICES | 8 | 0 |
| dix A Schedule of Procedures | 8 | 1 |
| dix C Pharmacokinetic Sampling S | schedule8 | 9 |
| dix D Grading Scale for Adverse E | vents Relating to Laboratory Abnormalities9 | 1 |
| | 2 Safety Analysis | 2 Safety Analysis 7 3 Efficacy Analysis 7 4 Pharmacokinetic and Immunogenicity Analysis 7 0.6.4.1 Pharmacokinetic Analysis 7 0.6.4.2 Immunogenicity Analysis 7 INVESTIGATOR'S REGULATORY OBLIGATIONS 7 Informed Consent 7 Ethical Conduct of the Study 7 Independent Ethics Committee/Institutional Review Board 7 Patient Confidentiality 7 DMINISTRATIVE AND LEGAL OBLIGATIONS 7 Protocol Amendments 7 Study Termination 7 Study Monitoring 7 Language 7 Compensation for Injury 7 EFFERENCES 7 PPENDICES 8 dix A Schedule of Procedures 8 dix B List of Laboratory Analytes 8 dix C Pharmacokinetic Sampling Schedule 8 |

# **TABLE OF TABLES**

| | | Page |
|---|---|---|
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 50 |
| Table 2 | Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or $< 100,000/\text{mm}^3$ (x1)* | 54 |
| Table 3 | Actions in Patients with Low Platelet Count or Drop in Platelet Count | |
| Table 4 | Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence | 64 |

# **TABLE OF FIGURES**

| | | Page |
|---|---|---|
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 36 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volunesorsen is shown | 38 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 40 |

Amendment 6 11 April 2017


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered Subcutaneously

to Patients with Familial Chylomicronemia Syndrome (FCS)

**Amendment Number:** 6 - Netherlands

**Amendment Date:** 11 April 2017

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 5 dated 6 July 2016:

1. To update the platelet safety monitoring rules shown in Table 3.

- 2. To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies.
- 3. To add post heparin plasma LPL activity of ≤ 20% of normal in medical history as an inclusion criteria for ISIS 304801-CS16 (Group 2) patients as has been allowed for ISIS 304801-CS6 (Group 1) patients.
- 4. To allow patients who complete the 52-week treatment period to participate in an expanded access program or continue dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period.
- 5. Added archive blood sample for potential gene sequencing related to hypertriglyceridemia (Group 2 if not available from index study).
- 6. Added: Troponin I, platelet bound autoantibody testing at baseline (may be done), and Table 2 Labs to be performed in the event of a platelet count Less than the Lower Limit of Normal (x2) or < 100,000/mm³ (x1) to provided added patient safety; blood viscosity (may be done) to assess potential benefit of ISIS 304801 administration; and platelet aggregation (may be done) to assess platelet function.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol, additions are indicated as underline and deletions are indicated as strikethrough:

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis<br>Section 3.1<br>Study Design | This is a multi-center open-label study of: Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |
| Synopsis<br>Section 5.1<br>Inclusion<br>Criteria | <ul> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Groups 2-and 3: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study:</li> <li>c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at ScreeningQualification for the ISIS 304801-CS16 index study Group 3: Fasting TG ≥ 750 mg/dL at Screeningfor this open-label study</li> </ul> | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |
| Synopsis<br>Section 5.1<br>Inclusion<br>Criteria | <ul> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) <u>supported</u> by documentation <u>of at least 1</u> of the following:</li> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤ 20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study</li> </ul> | To add LPL activity of ≤ 20% of normal in medical history as an inclusion criteria for Group 2 patients as has been allowed for Group 1 patients. |
| Synopsis<br>Section 5.2<br>Exclusion<br>Criteria | <ul> <li>Exclusion Criteria for Group 3 (patients who did not participate in an index study)</li> <li>Diabetes mellitus with any of the following: <ul> <li>a. Newly diagnosed within 12 weeks of screening</li> <li>b. HbA1c ≥ 9.0% at Screening</li> <li>c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of ± 10 units of insulin])</li> <li>d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)</li> <li>e. Current use of GLP 1 agonists</li> </ul> </li> <li>Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome</li> <li>Active pancreatitis within 4 weeks prior to screening</li> </ul> | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |

| Synopsis Section 5.2 Exclusion Criteria Continued 14. Use of any of the following: a. Statins, omega 3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to escreening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega 3 fatty acids should make every effort to remain on the same brand throughout the study b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Spensor Medical Monitor d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period f. Cilybera gene therapy within 2 years prior to screening g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed h. Tamexifion, estregens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period i. Plasma apheresis within 4 weeks prior to screening or planned during the study j. Prior exposure to ISIS 304801 k. Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over the counter medications will be allowed at Investigator's discretion) 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) 17. Have any other conditions, which, in the opinion of the Investigator or the Spensor would make the patient uns | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |
|---|---|

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis Study Design and Treatment Schema Section 3.1 Study Design Section 3.4.1 Qualification | The study for an individual patient will generally consist of the following periods: • Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A • Group 3 patients (did not participate in an index study): An up to 8 week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A • All patients: • A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection • Option to participate in an extended treatment period (up to an additional 52 weeks) • A 13-week post-treatment evaluation period or expanded access program The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option of participatin | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. To allow patients who complete the 52-week treatment period to participate in an expanded access program or continue dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. |
| Section 3.4.3<br>Post-<br>Treatment | The post-treatment evaluation period is 13 weeks and consists of 27 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse). | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 4.1<br>Qualification | Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used. | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |
| Section 6.1<br>Study<br>Schedule | 6.1.2 Screening and Qualification (Group 3) Before any study specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |
| Section 6.1.2<br>Treatment<br>Period | During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 5051 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.—Dosing instructions and training will be provided to the patient where applicable. | To provide added patient safety regarding platelet count reductions and ISIS 304801 dose exposure. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 6.1.3 Extended Treatment Period | Patients will have the option of continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable. | To allow patients who complete the 52-week treatment period to participate in an expanded access program or continue dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. |
| Section 6.1.5 Post-Treatment Period | After completion of the Week 52 visit assessments, patients will | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 8.5.2 Safety Monitoring for Platelet Count Results | Actions to be taken in the event of reduced platelet count are shown in Table 23 in Section 8.6.3. Monitor every 1 week unless otherwise specified. Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing. The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3). | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 8.5.2<br>Safety<br>Monitoring for<br>Platelet Count<br>Results<br>Continued | Added Table 2: Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm³ (x1)* *In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion. Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations. |
| | To Be Performed at Local Lab | |
| | Peripheral smear (should be performed locally, fixed and sent to central lab for review) | |
| | Fibrinogen split products or D-dimer on fresh blood | |
| | To Be Performed at Central Lab | |
| | Citrated sample for platelets | |
| | Coagulation panel (PT/INR, aPTT) | |
| | CBC with reticulocytes | |
| | Folate (folic acid) | |
| | Vitamin B12 | |
| | Fibrinogen | |
| | von Willebrand factor | |
| | Total globulins, total IgA, IgG and IgM | |
| | Complement: total C3, total C4, Bb, C5a | |
| | hsCRP | |
| | Helicobacter pylori (breath test) | |
| | Serology for: | |
| | HBV, HCV, HIV (if not done recently for Qualification) | |
| | Rubella | |
| | CMV | |
| | EBV | |
| | Parvo B19 | |
| | Helicobacter pylori (IgG serum test) | |
| | Auto-antibody screen: | |
| | Antiphospholipid | |
| | Rheumatoid factor | |
| | Anti-dsDNA | |
| | Anti-thyroid | |
| | To Be Performed at Specialty Lab(s) | |
| | Antiplatelet antibodies and Anti-PF4 assay | |
| | Anti-ASO antibody | |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Section 8.6.3<br>Stopping<br>Rules for<br>Platelet<br>Count<br>Results | Actions to be taken in the event of a low platelet count are summarized in Table 23 below. In the event of a platelet count less than 75,000/mm³ that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor. In the event of any platelet count less than 2550,000/mm³, or a platelet count less than 75,000/mm³ that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3. daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable. | To provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations. |
| | Administration of steroids is recommended for patients whose platelet count is less than 2550,000/mm³. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5 2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). Triglyceride levels be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from | |
| | an increase of 2,000 to 500 mg/dL during that period. In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to > 100,000/mm³. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing. | |
| | If after the first dosing rechallenge the platelet count again falls below 75,000/mm³, then dosing of the patient with Study Drug will be stopped permanently. Following a rechallenge platelet count should be tested every week until count is stable. Any unreportable platelet count result must be rechecked and determined | |
| | not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. | |

| Protocol<br>Section | | Description of C | hange | Rationale |
|---|---|---|---|---|
| Section<br>8.6.3 | Was: Table 2 Actions in Patients with Low Platelet Count | | | To provide added patient safety |
| Stopping<br>Rules for<br>Platelet | Platelet<br>Count on Rx | Drug Dose | Monitoring | regarding platelet<br>count reductions,<br>ISIS 304801 dose |
| Count<br>Results<br>Continued | Normal range,<br>> 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks | exposure, and treatment recommendations. |
| Communica | 100K-<br>140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1 week until stable* | recommendations. |
| | 75K-<br>100K/mm <sup>3</sup> | Permanently reduce<br>dose frequency to 300<br>mg every 2 weeks or<br>reduce dose to 150 mg<br>weekly | Closer observation<br>Monitor every 1 week | |
| | 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication | |
| | 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible | |

| Protocol<br>Section | | Description of Change | | |
|---|---|---|---|---|
| Section | Table 2 Actions | in Patients with Low P | atelet Count Continued | To provide added |
| 8.6.3<br>Stopping<br>Rules for | Platelet<br>Count on Rx | Drug Dose | Monitoring | patient safety<br>regarding platelet<br>count reductions, |
| | < 25K/mm <sup>3</sup> | Permanently<br>discontinue<br>Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible | ISIS 304801 dose exposure, and treatment recommendations. |
| | determined ** Recovery in dose steroid (Provan et a every 2-4 we 2-4 weeks th | by the Sponsor Medical Management Platelet count may be access. Treatment guidelines for 1. 2010) recommend Dexaged For 1-4 cycles; Prednant aper; or Methylprednarequire continuation with | ed weekly that are stable as donitor and > 100,000/mm <sup>3</sup> celerated by administration of high for immune thrombocytopenia amethasone 40 mg daily for 4 days is(ol)one 0.5-2 mg/kg/d for isolone 30 mg/kg/day for 7 days oral steroids after methyl | |

| Protocol<br>Section | | Description of Cha | ange | Rationale |
|---|---|---|---|---|
| Platelet Co. | ble 3 Actions<br>unt | s in Patients with Low Plate | elet Count or Drop in Platelet | To provide added patient safety regarding platelet count reductions, |
| Platelet Count Results Continued Col Co | | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. Weekly 300 mg Study Drug administration Permanently reduce dose frequency to 300 mg every 2 weeks If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or nonconsecutive) of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per Investigator discretion. • Monitor every 2-3 days until 2 successive values are >75K/mm³ then monitor every 1 week • Consider discontinuation of antiplatelet agents/NSAIDS/anticoagulant medication | |

| Protocol<br>Section | | Description of Ch | ange | Rationale |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping | Table 3 Action Count Continue | | elet Count or Drop in Platelet | To provide added patient safety |
| Rules for<br>Platelet<br>Count | Platelet<br>Count on Rx | Drug Dose | Monitoring | regarding platelet<br>count reductions,<br>ISIS 304801 dose |
| Results Continued | dose steroid<br>(Provan et a<br>every 2-4 w<br>2-4 weeks t | ds. Treatment guidelines for<br>al. 2010) recommend dexame<br>eeks for 1-4 cycles; prednison<br>hen taper; or methylprednison<br>require continuation with ora | ethasone 40 mg daily for 4 days<br>ol)one 0.5-2 mg/kg/d for<br>lone 30 mg/kg/day for 7 days | exposure, and treatment recommendations. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Synopsis<br>Section<br>10.1.1<br>Efficacy<br>Endpoints | <ul> <li>Percent change and absolute change from baseline in fasting TG</li> <li>Frequency and severity of patient reported abdominal pain during the treatment period</li> <li>Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C</li> <li>Percent change from baseline in fasting total apolipoprotein C-III</li> <li>Change in blood viscosity (may be evaluated)</li> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> <li>Adjudicated acute pancreatitis event rate</li> <li>Other symptoms: eruptive xanthoma, lipemia retinalis</li> </ul> | Blood viscosity<br>added to assess<br>potential benefit<br>of ISIS 304801<br>administration. |
| Synopsis<br>Section<br>10.1.2 Safety<br>Endpoints | <ul> <li>Adverse events including adjudicated events of pancreatitis and MACE</li> <li>Vital signs and weight</li> <li>Physical examinations</li> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> <li>Echocardiography</li> <li>Electrocardiograms (ECGs)</li> <li>Use of concomitant medications</li> <li>MRIs</li> <li>Platelet aggregation (may be evaluated)</li> </ul> | Platelet<br>aggregation<br>added to assess<br>platelet function<br>following<br>ISIS 304801<br>administration. |
| Section 10.3<br>Populations | Full Analysis Set (FAS): All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9. Per Protocol Set (PPS): Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock. Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen. PK Population: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 evaluable post first dose PK sample collected, analyzed, and reported. | Modified to include, in the FAS, only those patients that are randomized and dosed and have a baseline TG assessment and clarified the PK Population. |
| Section 10.4<br>Definition of<br>Baseline | Definitions of baseline are given below for the purposes of the final analysis. For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).—For Group 3 patients, the baseline for fasting lipid measurements is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 in this open label study. For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study—and Group 3 patients, baseline will be the last non-missing assessment prior to the first dose of Study Drug. | To exclude enrollment of FCS patients in this open-label study who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Appendix A | Removed Screening period (Group 3) Removed Week 2.5 Added: Medical History b Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study CBC with Differential c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable and determined not to have met a stopping rule-before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that determine if the count has not-met the a stopping rule, and to determine whether the rate of decline is suggestive that the patient could be approaching the or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor Added: Blood Viscosity, Platelet Aggregation, Platelet Bound Autoantibodies e May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only Added: archive blood sample for potential gene sequencing related to | Added troponin, platelet bound autoantibodies, and modified CBC blood draws to provide added patient safety regarding platelet count reductions, ISIS 304801 dose exposure, and treatment recommendations. Added patient chart review, blood viscosity and potential gene sequencing to assess potential benefit of ISIS 304801 administration. Added platelet aggregation to assess platelet function following ISIS 304801 administration. |
| Appendix A | hypertriglyceridemia (Group 2 if not available from index study) Added: Appendix A Schedule of Procedures – Extended Treatment Period Table and Legend. | To allow patients who complete the 52-week treatment period to participate in an expanded access program or continue dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. |

| Protocol<br>Section | Description of Change | Rationale |
|---|---|---|
| Appendix B | Added: Troponin I <sup>2</sup> CK-MB <sup>2</sup> Platelet Bound Autoantibodies <sup>3</sup> Blood Viscosity <sup>3</sup> Platelet Aggregation <sup>3</sup> 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB 3 May be done | Added troponin, CK-MB, and platelet bound autoantibodies, provide added patient safety. Added Blood Viscosity to assess potential benefit of ISIS 304801 administration Added Platelet Aggregation to assess platelet function following ISIS 304801 administration. |
| Appendix C | Added: Appendix C PK Sampling Schedule (Extended Treatment Period) Table. | To collect intermittent PK data in patients who enter the extended treatment period. |

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following: </li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study</li> </ul> |
| | c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Qualification for the ISIS 304801-CS16 index study |
| | 4. Able and willing to participate in a 65-week study |

# PROTOCOL SYNOPSIS Continued

| Study Population Continued | Inclusion Criteria: Continued |
|---|---|
| | 5. Satisfy 1 of the following: |
| | <ul> <li>a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females &gt; 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration</li> <li>b. Males: Surgically sterile, abstinent* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration</li> </ul> |
| | * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients |
| | Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study |
| | Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |

#### PROTOCOL SYNOPSIS Continued

#### Study Visit Schedule and The study for an individual patient will generally consist of the following Procedures A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection Option to participate in an extended treatment period (up to an additional 52 weeks) A 13-week post-treatment evaluation period or expanded access program The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel. blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. Safety and Tolerability Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse **Evaluations** events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters.

# PROTOCOL SYNOPSIS Continued

| Planned Analyses | Safety Endpoints: |
|---|---|
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | MRIs |
| | Platelet aggregation (may be evaluated) |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Change in blood viscosity (may be evaluated) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



#### STUDY GLOSSARY

#### Abbreviation/Acronym **Definition** anti-drug antibody ADA AΕ adverse Event alkaline Phosphatase **ALP** alanine Aminotransferase ALT ANA antinuclear Antibody apoA-1 apolipoprotein A-1 apoB apolipoprotein B apoC-III apolipoprotein C-III apolipoprotein E apoE activated partial thromboplastin time aPTT antisense oligonucleotide ASO **AST** aspartate aminotransferase **AUC** area under the curve body mass index BMI **CBC** complete blood count $C_{max}$ maximum observed drug concentration case report form **CRF** deoxyribonucleic Acid DNA **DSMB** Data and Safety Monitoring Board **ECG** electrocardiogram **eCRF** electronic Case Report Form electronic data capture **EDC** ET early termination full analysis set FAS **FCS** Familial Chylomicronemia Syndrome Good Clinical Practice **GCP** GLP-1 glucagon-like peptide-1 GPIHBP1 glycosylphosphatidylinositol-anchored hdl-binding protein 1 heritability and phenotype intervention **HAPI** glycated hemoglobin HbA1c **HDL** high-density lipoprotein high-density lipoprotein-cholesterol HDL-C

hsCRP High-sensitivity C-reactive protein

ICH International Conference on Harmonization

IDLintermediate density lipoproteinIECIndependent Ethics Committee

IM immunogenicity

Index Studies ISIS 304801-CS6 and ISIS 304801-CS16

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL low-density lipoprotein

LDL-C low-density lipoprotein-cholesterol

LMF1 lipase maturation factor 1

LPL lipoprotein lipase

MACE major acute cardiovascular event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL no-observed-adverse-effect level

non-HDL-C non-high-density lipoprotein-cholesterol

OTC over the counter PFS prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL triglyceride-rich lipoproteins

ULN upper limit of normal

VLDL very-low-density lipoprotein

VLDL-C very-low-density lipoprotein-cholesterol

VLDL-TG lipoprotein-triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volunesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.
# 2.3.4 Clinical Experience

Protocol - Netherlands

Detailed information concerning the clinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies, there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

# 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period.

# 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Qualification

A Qualification period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, 58, and 65 (Weeks 53, 54, 55, 56, 57, and 58 may be conducted by a home healthcare nurse).

# 3.5 End-of-Study

The End-of-Study is last patient, last visit.

# 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 **Qualification**

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent

- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.
  - Group 2: Patients who enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the open-label Study:
  - a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
  - b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) supported by documentation of at least 1 of the following:
    - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
    - Post heparin plasma LPL activity of ≤20% of normal in medical history. Note: testing of LPL activity should not be performed to confirm eligibility for the study
  - c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Qualification for the ISIS 304801-CS16 index study
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \*Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.

2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

### 6. STUDY PROCEDURES

# 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, blood viscosity, volanesorsen plasma concentrations, immunogenicity (IM) testing, platelet aggregation, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 39, 40, 41, 42, 43, 44, 45, 46, 47, 48, 49, 50, and 51 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Extended Treatment Period

Patients will have the option of continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country.

During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volunesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 53, 54, 55, 56, 57, 58, 59, 60, 61, 62,63, 65, 66, 67, 68, 69, 70, 71, 72, 73, 74, 75, 77, 78, 79, 80, 81, 82, 83, 84, 85, 86, 87, 88, 89, 91, 92, 93, 94, 95, 96, 97, 98, 99, 100, 101, 102, and 103 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Dosing instructions and training will be provided to the patient where applicable.

# 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

### 6.1.5 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country as described in Section 6.1.3. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. This 13-week post-treatment evaluation period consists of 7 Study Center visits on Weeks 53, 54, 55, 56, 57, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A. Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 7 Study Center visits on Weeks 105, 106, 107, 108, 109, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A.

# 6.2 Additional Study Assessments

# 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

# 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

# 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll-over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65. Patients in the Extended Treatment Period will have ECGs performed in triplicate at Week 76 and Week 104.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

# 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period (Week 65).

# 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service. Patients in the Extended Treatment Period will receive diet/alcohol counseling by qualified study personnel at clinic visits only.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet may be conducted randomly during the treatment and post treatment follow-up periods.

### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

# 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 2)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to Qualification and information relating to these events will be collected for independent adjudication.

#### 6.3 **Restriction on the Lifestyle of Patients**

#### 6.3.1 Contraception Requirements

Protocol - Netherlands

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent<sup>†</sup> or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq$  55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

# For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

### For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

† Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

# 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example, if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

# 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs.

# 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules,

if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volunesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

# 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel

- Amendment 6 11 April 2017
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

# 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

Monitor every 1 week unless otherwise specified.

Protocol - Netherlands

Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records.

Due to the 1 to 2-year study duration it is anticipated that patients may undertake travel including vacations, which may impede weekly platelet monitoring. In some situations, it may be possible to arrange for local laboratory testing or use of the home healthcare service at their temporary location. The intent is to maintain weekly platelet monitoring and dosing where possible, as well as Investigator site contact with the study patients. However, if the above options are not possible, a temporary interruption of study treatment will be planned with a prompt blood draw upon the patient's return which must be reported and reviewed by the Investigator prior to the patient resuming dosing.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count Less than the Lower Limit of Normal (x2) or < 100,000/mm<sup>3</sup> (x1)\*

\*In patients who have any 2 occurrences (consecutive or non-consecutive) of platelet count less than the lower limit of normal or who have any 1 occurrence of platelets < 100,000/mm<sup>3</sup>. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion.

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Folate (folic acid) |
| Vitamin B12 |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Helicobacter pylori (breath test) |
| Serology for: |
| HBV, HCV, HIV (if not done recently for Qualification) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinicallyrelevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will review the glucometer reading or printout at every clinic visit to evaluate if fasting pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for Hyperglycemia below.

All diabetic patients will note any changes in their insulin dose and /or oral antidiabetic therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - o Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose  $\leq$  70 mg/dL ( $\leq$  3.9 mmol/L).

Protocol - Netherlands 11 April 2017

o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

# 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

# 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volunesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 50,000/mm<sup>3</sup>, or a platelet count less than 75,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored as outlined in Table 3.

Administration of steroids is recommended for patients whose platelet count is less than 50,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). Triglyceride levels be monitored weekly, and AE monitoring will continue, during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

### Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Table 3 Actions in Patients with Low Platelet Count or Drop in Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| | Study Drug administration is contingent on the availability of the immediately preceding test result. An interpretable platelet value must be available within 7 days prior to dosing. Only the study doctor or qualified designee can authorize continued Study Drug administration based on an acceptable platelet value. Patients should not administer a dose until they have been contacted by their study doctor or designee and told that it is acceptable to dose. Authorization to dose must be documented in the patient's medical records. | Monitor every 1 week unless otherwise specified Obtain additional lab tests (Table 2) if 2 occurrences consecutive or non-consecutive) of platelet count 140K - > 100K/mm³ or 1 occurrence of platelet count ≤ 100K/mm³. Labs only need to be performed once. Labs may be collected over multiple visits, if blood requirements are a concern, as per investigator discretion. |
| > 100K/mm <sup>3</sup> | Weekly 300 mg Study Drug administration | |
| 100K/mm <sup>3</sup> - > 75K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks | |
| 75K/mm <sup>3</sup> - > 50K/mm <sup>3</sup> | <ul> <li>If occurs while on dose of 300 mg every 2 weeks then permanently discontinue Study Drug, otherwise dose pause</li> <li>When platelet count returns to &gt; 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks only if approved by Sponsor Medical Monitor</li> </ul> | <ul> <li>Monitor every 2-3 days until<br/>2 successive values are &gt; 75K/mm³<br/>then monitor every 1 week</li> <li>Consider discontinuation of antiplatelet<br/>agents/NSAIDS/ anticoagulant<br/>medication</li> </ul> |
| ≤ 50K/mm³ | Permanently discontinue Study Drug | <ul> <li>Monitor daily until 2 successive values show improvement then monitor every 2-3 days until 2 successive values are &gt;75K/mm³ then monitor every 1 week</li> <li>Patient should be evaluated by a hematologist to provide diagnostic and therapeutic management</li> <li>Steroids recommended*. It is strongly recommended that, unless the patient has a medical contraindication to receiving glucocorticoids, the patient receives glucocorticoid therapy to reverse the platelet decline</li> <li>Monitor triglyceride levels weekly and continue AE monitoring during steroid therapy</li> <li>Discontinue antiplatelet agents/ NSAIDS/ anticoagulant medication while platelet count is&lt; 50K/mm³ if possible</li> </ul> |

<sup>\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone)

# 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

# 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

# 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 65 (or Week 117 if terminating from the Extended Treatment Follow-Up Period), see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 **Concomitant Therapy and Procedures**

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

# 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

# **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

# **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 (or Week 117 if patient enters the extended treatment period) visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

# **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

Protocol - Netherlands

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

# 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

# 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

# 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

# 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

# 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration

• Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)

Amendment 6

11 April 2017

• **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

# 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

# 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

# 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE

- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- **Persists (as non-serious AE):** Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

### 9.5 Procedures for Handling Special Situations

### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

Amendment 6

11 April 2017

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 **Dosing Errors**

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volanesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

Should an overdose occur, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study

physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

# 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

# 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Change in blood viscosity (may be evaluated)
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography

- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

Protocol - Netherlands

• Platelet aggregation (may be evaluated)

#### 10.2 **Sample Size**

No sample size calculations were performed as this is an open-label study.

#### 10.3 **Populations**

Full Analysis Set (FAS): All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

Per Protocol Set (PPS): Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

PK Population: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### 10.4 **Definition of Baseline**

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 **Interim Analysis**

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

Protocol - Netherlands

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naive group which including patients on placebo in index studies. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

# 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

# 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

# 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG  $\geq 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

# 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volunesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study will receive the first treatment of volunesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration  $(CL_{0-24h}/F)$  will be calculated from  $CL_{0-24h}/F$  = Actual Dose/AUC<sub>0-24h</sub>. Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

# 10.6.4.2 Immunogenicity Analysis

Protocol - Netherlands

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

# 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed

informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

# 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.
Protocol - Netherlands

### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

## 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

# 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Protocol - Netherlands

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-α expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

# Appendix A Schedule of Procedures

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | Trea | tmen | t Perio | od | | | | | | | | | Tre | ost<br>atme | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -2 to | w | 112 | Wk | Wk | Wk | VA/Iz | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | ith 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | VA/Ic |
| | Study Week | -2 10 | 1 | | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | | 65 |
| | Study Day | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 44<br>9 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Int | ormed Consent | Χ | | | | | | | | | | | | | | | | | | | | | | | | | |
| | ıtpatient Visit | Х | Χ | ΧI | Χ <sup>I</sup> | ΧI | ΧI | ΧI | ΧI | Χ | Χ <sup>I</sup> | Χ <sup>I</sup> | Χ <sup>I</sup> | ΧI | Χ | Χ <sup>I</sup> | Χ <sup>I</sup> | ΧI | Χ | Χ <sup>I</sup> | ΧI | Χ <sup>I</sup> | ΧI | Х | Χ <sup>I</sup> | ΧI | Χ |
| | clusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| Vi | edical History <sup>b</sup> al Signs + body weight | Х | Х | | X | | X | | | Х | | | | | Х | | | | X | | | | | Х | | | Х |
| | height on Day 1 only) | , , | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical Examination 12- lead ECG (triplicate) | | | Х | | | | | | | X | | | | | X | | | | X | | | | | X | | | X |
| | MRI (liver/spleen) | | | | | | | | | _^ | | | | | ^ | | | | ^ | | | | | Xm | | | ^ |
| | hocardiography | | | | | | | | | | | | | | Xm | | | | | | | | | Xm | | | |
| F | Chemistry Panel | Х | Х | | Х | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | X | | Х | Х |
| | CBC with Differential <sup>c</sup> | Х | • | | | Platel | | e ass | essec | | calen | | eek, v | sits de | X | ave sp | | d wind | | o allov | | oility o | f sche | | | <b>→</b> | Х |
| | Serum Lipid Panel | Х | Х | | Χ | | Х | | Х | Х | | | | Х | Χ | | | | Χ | | | | Χ | Х | | | Х |
| p( | Blood viscosity <sup>e</sup> | | Х | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | |
| astina) <sup>d</sup> | Platelet aggregation <sup>e</sup> | Х | Х | | | | | | | Χ | | | | | Χ | | | | | | | | | Х | | | |
| ast | Coagulation (aPTT, PT, INR) | Χ | | | | | Х | | | Х | | | | | Χ | | | | Χ | | | | | Χ | | | |
| Draw (F | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| ت | Sedimentation Rate | | Х | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | Х |
| Blood | Complement (C5a, Bb) | | Х | | | | | Î | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| 8 | Troponin I | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| 1 " | Platelet Bound Autoantibodies <sup>e</sup> | | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| ĺ | Plasma PK - Volanesorsen | | Xn | Х | Х | | Х | | | Х | | | | | Χ | | | | Χ | | | | | Х | | | Х |
| ĺ | Anti-Volanesorsen Antibodies | | Х | | Х | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | | Х |
| 1 | Serum Pregnancy Test <sup>f</sup> | Χ | | | Х | | Х | | | Х | | Χ | | | Χ | | Х | | Χ | | Х | | | Χ | | Х | Χ |

# Appendix A Schedule of Procedures Continued

| | Study Period | Quala | | | | | | | | | | Tre | eatm | ent P | eriod | | | | | | | | | | | Treati | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | -2 to<br>-1 | W | | Wk<br>4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | Mor | nth 3 | Wk<br>15<br>&<br>17 | Wk<br>19 | Wk<br>21<br>&<br>23 | Моі | nth 6 | Wk<br>28<br>&<br>30 | Wk<br>32 | Wk<br>34<br>&<br>36 | Wk<br>38 | Wk<br>40<br>&<br>42 | Wk<br>44 | Wk<br>46<br>&<br>48 | Mor | nth 12 | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 |
| | | - | | | - | | | | Wk<br>12 | Wk<br>13 | | | | Wk<br>25 | Wk<br>26 | | | | | | | | Wk<br>50 | Wk 52<br>or ET | | | |
| | Study Day | -14 to<br>-7 | 1 | 2 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| V | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | |
| d Draw<br>sting) <sup>d</sup><br>(Gr | chive blood sample for<br>ential gene sequencing<br>ated to hypertriglyceridemia<br>oup 2 if not available from<br>ex study) <sup>i</sup> | × | х | | | | | | | | | | | | | | | | | | | | | | | | |
| AIC | chived Serum & Plasma<br>mples <sup>g</sup> | | Х | | | | Х | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Urinalysis | s <sup>d</sup> | Х | Χ° | | Х | | Х | | | Χ° | | Χ° | | | Χ° | | Χ° | | Χ° | | Χ° | | | Χ° | | Χ° | Χ° |
| | Photography <sup>h</sup> | Х | | | | | | | | | | | | | | | | | | | | | | Xm | | | |
| | testing for FCS diagnosis (if able in medical history) <sup>i</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly S | Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | X | | <u> </u> | |
| Symptom | n Diary (weekly) | Х | Х | | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Χ | Χ | Х | Χ | Х |
| Quality of | Quality of Life Assessment(s) | | Х | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Χ |
| Food/Drin | Food/Drink Diary (quarterly) <sup>j</sup> | | Χ | | | | | | | Х | | | | | Χ | | | | | | | | | Χ | | | Х |
| Diet/Alcohol Counseling <sup>k</sup> | | Χ | Х | | Х | | Х | | | Х | | | | | Χ | | | | Χ | | | | | Х | | Х | Х |
| Adverse | Adverse Events X | | | | Χ | Χ | Х | Χ | Х | Х | Х | Х | Χ | Х | Χ | Х | Χ | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Х |
| Concomi | tant Medication | Х | Х | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х |

- a Qualification procedures performed (Please refer to Sections 3.4.1, 4.1, and 6.1.1)
- b Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor

# Appendix A Schedule of Procedures Continued

#### Legend Text Continued

- d Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- e May be done. Blood viscosity and platelet aggregation in volanesorsen-treatment naïve patients only
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- h If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 roll-over patients]) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- i Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 roll-over patients]); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- k To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- I Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- m A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- n Full or abbreviated PK profile (see Appendix C)
- Expanded urinalysis (see Appendix B)

Appendix A Schedule of Procedures – Extended Treatment Period

| | Study Period | | | | | | | ٦ | reatme | nt Perio | od | | | | | | | | -Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | Wk 60<br>& 62 | Mo 15<br>Wk 64 | | Wk<br>70 | | Mo 18<br>Wk 76 | | | Wk 84,<br>86, & 88 | | | Wk<br>96 | Wk<br>98,<br>100 &<br>102 | Mo 24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | Wk<br>110 | Mo 27<br>Wk<br>117 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 56<br>8 | 582, 596<br>& 610 | 624 | 638 &<br>652 | 666 | 680,<br>694 &<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Οι | utpatient Visit | $X^f$ | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | $X^f$ | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | $X^f$ | Χ | X <sup>f</sup> | X <sup>f</sup> | Х |
| Vi | tal Signs (+ body weight) | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | Χ |
| Ph | ysical Examination | | | | | | | | Χ | | | | | | | | Χ | | | |
| 12 | - lead ECG (triplicate) | | | | | | | | Χ | | | | | | | | Χ | | | |
| Ur | inalysis(including P/C ratio) | | Х | | Х | | Χ | | Х | | Х | | Х | | Х | | Χ | | Χ | Χ |
| | Chemistry Panel | | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | Х | | Χ | | Χ | Χ |
| astina) <sup>b</sup> | CBC with Differential <sup>a</sup> | <b>▼</b> | Plate | elets are | assess | ed each | caler | ndar wee | ek. visits | do not | | specified | window | s to allo | w flex | ibility of | schedul | lina. | - | Х |
| i to | Serum Lipid Panel | | | | Χ | | | | X | | | | Χ | | | | Χ | | | Χ |
| 1 4 | Coogulation (aDTT_DT_IND) | | | | Χ | | | | Χ | | | | Χ | | | | Χ | | | |
| Draw | Troponin I | | | | Χ | | | | Χ | | | | Χ | | | | Χ | | | Х |
| Blood | Plasma PK - ISIS 304801° | | | | | | | | Χ | | | | | | | | Χ | | | Х |
| <u>8</u> | Anti-ISIS 304801 Antibodies | | | | | | | | Χ | | | | | | | | Χ | | | Χ |
| | Serum Pregnancy Test <sup>d</sup> | | Х | | Χ | | Χ | | Χ | | Χ | | Х | | Х | | Χ | | Х | Х |
| W | eekly Study Drug: SC Injection | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Χ | Χ | Χ | | | |
| Di | et/Alcohol Counseling <sup>e</sup> | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | |
| Ac | Iverse Events | Х | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Χ | Χ |
| Co | oncomitant Medication | X | Х | Х | Χ | Х | Х | X | X | Χ | Χ | Х | Χ | Х | Х | X | Х | Χ | Х | X |

### Appendix A Schedule of Procedures – Extended Treatment Period Continued

#### Legend Text

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and the result must be reviewed by the Investigator and confirmed to be acceptable before dosing can continue. All platelet count results will be promptly reviewed by the Investigator to determine if the count has met a stopping rule, or the dose reduction rule of 100,000/mm³, or the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

# **Appendix B** List of Laboratory Analytes

## Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

Amendment 6

11 April 2017

| nical Chemistry Panel | <b>Coagulation</b> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| Sodium | • aPTT (sec) | <ul> <li>Red blood cells</li> </ul> | <ul> <li>Color</li> </ul> |
| Potassium | • PT (sec) | <ul> <li>Hemoglobin</li> </ul> | <ul> <li>Appearance</li> </ul> |
| Chloride | • INR | <ul> <li>Hematocrit</li> </ul> | <ul> <li>Specific gravity</li> </ul> |
| Bicarbonate | | • MCV, MCH, MCHC | • pH |
| Total protein | Lipid Panel | • Platelets | • Protein |
| Albumin | <ul> <li>Total Cholesterol</li> </ul> | <ul> <li>White blood cells</li> </ul> | • Blood |
| Calcium | • LDL-C | • WBC Differential (% | • Ketones |
| Magnesium | • HDL-C | and absolute) | <ul> <li>Urobilinogen</li> </ul> |
| Phosphorus | <ul> <li>Triglycerides</li> </ul> | <ul> <li>Neutrophils</li> </ul> | <ul> <li>Glucose</li> </ul> |
| Glucose | • Non-HDL-C | <ul> <li>Eosinophils</li> </ul> | • Bilirubin |
| BUN | • VLDL-C | <ul> <li>Basophils</li> </ul> | Leukocyte esterase |
| Creatinine | • apoA-1 | <ul> <li>Lymphocytes</li> </ul> | • Nitrate |
| Uric Acid | • apoB | <ul> <li>Monocytes</li> </ul> | <ul> <li>Microscopic</li> </ul> |
| Total bilirubin | <ul> <li>apoC-III</li> </ul> | | examination <sup>4</sup> |
| Direct (conjugated) bilirubin Indirect (unconjugated) bilirubin ALT AST Alkaline phosphatase | ) | Pharmacokinetics & Immunogenicity • Volanesorsen levels in plasma • Anti-volanesorsen antibodies in plasma Other Assessments • hsCRP • Sedimentation Rate • C5a, Bb • Troponin I <sup>2</sup> • CK-MB <sup>2</sup> • Platelet Bound Autoantibodies <sup>3</sup> • De-lipidated free glycerol • HbA1c, FPG • Blood viscosity <sup>3</sup> | Additional Measures for Expanded Urinalvsis • Total protein (quantitative) • Microalbumin • β2-microglobulin Platelet Function • Platelet aggregation |

- 1 Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

### Appendix C Pharmacokinetic Sampling Schedule

Protocol - Netherlands

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65# |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

### **PK Sampling Schedule (Extended Treatment Period)**

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>Ionized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | U | rine | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

# Collaborator:

Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

# ISIS 304801-CS7

# The APPROACH Open-Label Study Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 6 – 18 November 2016

EudraCT No: 2015-003755-21

# ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

### Protocol Amendment 6 – 18 November 2016

# **Protocol History:**

Original Protocol:

28 August 2015

Protocol Amendment 1:

2 February 2016

Protocol Amendment 2:

22 April 2016

Protocol Amendment 3:

9 May 2016

Protocol Amendment 4:

6 June 2016

Protocol Amendment 5:

6 July 2016

### Sponsor:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

MD, MBA

# **Ionis Protocol Number: ISIS 304801-CS7**

**Protocol Amendment 6** 

**EudraCT No: 2015-003755-21** 

**Clinical Phase: 3** 

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200 Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 18 November 2016

### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

Protocol

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Volanesorsen Administered Subcutaneously to<br>Patients with Familial Chylomicronemia Syndrome (FCS) | |
| Amendment: | Amendment 6 | |
| Date: | 18 November 2016 | |
| Open-Label Study of<br>Chylomicronemia Sy<br>as described herein.<br>I agree to comply wi<br>Good Clinical Practi<br>I agree to ensure that<br>any purpose other the | f Volanesorsen Administered yndrome (FCS)", dated 18 No of the International Conference (E6). It the confidential information an the evaluation or conduct comis Pharmaceuticals, Inc. | and the attached clinical protocol, entitled "An Subcutaneously to Patients with Familial vember 2016, and agree to conduct the study re on Harmonization Tripartite Guideline on contained in this document will not be used for of the clinical investigation without the prior |
| Investigator's Name | e (please print) | Date (DD Month YYYY) |

# **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| PRO | госо | L AMENDMENT | 10 |
| <b>PRO</b> | ГОСО | L SYNOPSIS | 15 |
| STUI | Y DE | SIGN AND TREATMENT SCHEMA | 21 |
| STUI | | OSSARY | |
| 1. | | ECTIVES | |
| 2. | BAC | CKGROUND AND RATIONALE | 24 |
| 2.1 | | verview of Disease | |
| 2.2 | | nerapeutic Rationale | |
| 2.3 | V | olanesorsen | |
| | 2.3.1 | Mechanism of Action | |
| 2 | 2.3.2 | Chemistry | |
| | 2.3.3 | Preclinical Experience | |
| | 2.3.4 | Clinical Experience | |
| 2.4 | | ationale for Dose and Schedule of Administration | |
| 3. | | ERIMENTAL PLAN | |
| 3.1 | | udy Design | |
| 3.2 | | umber of Study Centers | |
| 3.3 | | umber of Patients | |
| 3.4 | O | verall Study Duration and Follow-up | |
| 3 | 3.4.1 | Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801 index study): Qualification | |
| 3 | 3.4.2 | Group 3 Patients (did not participate in an index study): Screening/ Qualification | 31 |
| 3 | 3.4.3 | Treatment | 31 |
| 3 | 3.4.4 | Post-Treatment | 32 |
| 3.5 | Er | nd-of-Study | 32 |
| 3.6 | Da | ata and Safety Monitoring Board | 32 |
| 4. | PAT | TENT ENROLLMENT | 32 |
| 4.1 | Sc | reening/Qualification | 32 |
| 4.2 | Er | nrollment | 33 |
| <b>5.</b> | PAT | TENT ELIGIBILITY | 33 |
| 5.1 | In | clusion Criteria | 33 |
| 5.2 | | cclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801 | |
| | | dex Study Roll-over Patients | |
| <b>6.</b> | | DY PROCEDURES | |
| 6.1 | | udy Schedule | |
| 6 | 5.1.1 | Qualification (Groups 1 and 2) | 37 |

| 6. | 1.2 | Screening and Qualification (Group 3) | 37 |
|---|---|---|---|
| 6. | 1.3 | Treatment Period | |
| 6. | 1.4 | Extended Treatment Period | 38 |
| 6. | 1.5 | Pharmacokinetic (PK) Subgroup | 38 |
| 6. | 1.6 | Post-Treatment Period | 38 |
| 6.2 | Ad | ditional Study Assessments | 39 |
| 6. | 2.1 | Laboratory Assessments | 39 |
| 6. | 2.2 | Physical Exams and Vital Signs | 39 |
| | 6.2.2. | 1 Eruptive Xanthoma | 39 |
| | 6.2.2. | 2 Lipemia Retinalis | 39 |
| 6. | 2.3 | Echocardiography | 40 |
| 6. | 2.4 | ECG | 40 |
| 6. | 2.5 | MRI | 40 |
| 6. | 2.6 | Quality of Life Assessments. | 40 |
| 6. | 2.7 | Disease Symptom Diary | 40 |
| 6. | 2.8 | Diet Monitoring | 40 |
| 6. | 2.9 | Family History | 40 |
| 6. | 2.10 | Chart Review for Incidents of Acute Pancreatitis in Medical History (Group | 3)41 |
| 6.3 | Re | striction on the Lifestyle of Patients | 41 |
| 6. | 3.1 | Contraception Requirements | 41 |
| 6. | 3.2 | Other Requirements | 42 |
| <b>7.</b> | | DY DRUG | |
| 7.1 | Vo | lanesorsen Description | 42 |
| 7.2 | | ekaging and Labeling | |
| 7.3 | | dy Drug Accountability | |
| <b>8.</b> | TRE | ATMENT OF PATIENTS | 43 |
| 8.1 | | lanesorsen Administration | |
| 8.2 | | ner Protocol-Required Drugs | |
| 8.3 | | ner Protocol-Required Treatment Procedures | |
| 8.4 | Tre | eatment Precautions | 43 |
| 8.5 | | Tety Monitoring Rules | |
| | 5.1 | Safety Monitoring for Liver Chemistry Tests | |
| | 5.2 | Safety Monitoring for Platelet Count Results | |
| | 5.3 | Safety Monitoring for Minor Bleeding Events | |
| | 5.4 | Safety Monitoring for Constitutional Symptoms | |
| _ | 5.5 | Safety Monitoring for LDL-C Elevations | |
| | 5.6 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | |
| | 5.7 | Safety Monitoring for Documented Severe Hypoglycemia | |
| | 5.8 | Safety Monitoring for Hyperglycemia | |
| 8. | 5.9 | Acute Pancreatitis | 49 |

| | 8.6 St | opping Rules | 49 |
|---|---|---|---|
| | 8.6.1 | Stopping Rules for Liver Chemistry Elevations | 49 |
| | 8.6.2 | Stopping Rules for Renal Function Test Results | 50 |
| | 8.6.3 | Stopping Rules for Platelet Count Results | 50 |
| | 8.7 A | djustment of Dose Frequency | 52 |
| | 8.8 D | scontinuation of Study Treatment | 53 |
| | 8.8.1 | Follow-up Visits for Early Termination from Treatment Period | 53 |
| | 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Per | riod .53 |
| | 8.9 W | ithdrawal of Patients from the Study | 54 |
| | 8.10 C | oncomitant Therapy and Procedures | 54 |
| | 8.10.1 | Concomitant Therapy | 54 |
| | 8.10.2 | Concomitant Procedures | 55 |
| | 8.11 T <sub>1</sub> | eatment Compliance | 55 |
| 9. | SER | IOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 55 |
| | 9.1 S <sub>I</sub> | onsor Review of Safety Information | 55 |
| | 9.2 Re | egulatory Requirements | 55 |
| | 9.3 D | efinitions | 56 |
| | 9.3.1 | Adverse Event | 56 |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 56 |
| | 9.3.3 | Serious Adverse Event (SAE) | 57 |
| | 9.4 M | onitoring and Recording Adverse Events | 57 |
| | 9.4.1 | Serious Adverse Events | 57 |
| | 9.4.2 | Non-Serious Adverse Events | 58 |
| | 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | 58 |
| | 9.4.3 | .1 Relationship to the Study Drug | 58 |
| | 9.4.3 | .2 Severity | 58 |
| | 9.4.3 | .3 Action Taken with Volanesorsen | 59 |
| | 9.4.3 | .4 Treatment Given for Adverse Event | 59 |
| | 9.4.3 | .5 Outcome of the Adverse Event | 59 |
| | 9.4.4 | Adjudication Committees | 60 |
| | 9.5 Pr | ocedures for Handling Special Situations | 60 |
| | 9.5.1 | Abnormalities of Laboratory Tests | 60 |
| | 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 60 |
| | 9.5.3 | Dosing Errors | |
| | 9.5.4 | Contraception and Pregnancy | |
| 1 | 0. STA | TISTICAL CONSIDERATIONS | 62 |
| | 10.1 St | udy Endpoints | |
| | 10.1.1 | Efficacy Endpoints | |
| | 10.1.2 | Safety Endpoints | |
| | 10.2 Sa | mple Size | 62 |

|-----------------|------------------|
| Protocol | 18 November 2016 |

| 10.3 | Populations | 63 |
|---|---|---|
| 10.4 | Definition of Baseline | 63 |
| 10.5 | Interim Analysis | 63 |
| 10.6 | Planned Methods of Analysis | 63 |
| 10.6 | Demographic and Baseline Characteristics | 64 |
| 10.6 | 5.2 Safety Analysis | 64 |
| 10.6 | 5.3 Efficacy Analysis | 64 |
| 10.6 | 5.4 Pharmacokinetic and Immunogenicity Analysis | 65 |
| 10 | 0.6.4.1 Pharmacokinetic Analysis | 65 |
| 10 | 0.6.4.2 Immunogenicity Analysis | 65 |
| 11. II | NVESTIGATOR'S REGULATORY OBLIGATIONS | 66 |
| 11.1 | Informed Consent | 66 |
| 11.2 | Ethical Conduct of the Study | 66 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 67 |
| 11.4 | Patient Confidentiality | 67 |
| 12. A | DMINISTRATIVE AND LEGAL OBLIGATIONS | 67 |
| 12.1 | Protocol Amendments | 67 |
| 12.2 | Study Termination | 68 |
| 12.3 | Study Documentation and Storage | 68 |
| 12.4 | Study Monitoring | 69 |
| 12.5 | Language | 69 |
| 12.6 | Compensation for Injury | 69 |
| 13. R | EFERENCES | <b> 70</b> |
| 14. A | PPENDICES | 72 |
| Appen | dix A Schedule of Procedures | 73 |
| Appen | dix B List of Laboratory Analytes | 79 |
| Appen | dix C Pharmacokinetic Sampling Schedule | 81 |
| Appen | dix D Grading Scale for Adverse Events Relating to Laboratory Abnormaliti | es83 |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 42 |
| Table 2 | Labs to Be Performed in the Event of a Platelet Count < 75,000/mm <sup>3</sup> | 46 |
| Table 3 | Actions in Patients with Low Platelet Count | 52 |
| Table 4 | Expected Event for the Protocol Defined Population by Preferred Term | 56 |
| | and the Expected Incidence | 36 |

# **TABLE OF FIGURES**

| | | Page |
|---|---|---|
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 25 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volunesorsen is shown | 27 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 29 |

### PROTOCOL AMENDMENT

**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 6

**Amendment Date:** 18 November 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 5 dated 6 July 2016:

- 1. To allow patients who complete the 52-week treatment period to participate in an expanded access program or continue dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter the 13-week post treatment evaluation period.
- 2. The following assessments were added: Troponin I; labs to be performed in the event of a platelet count < 75,000/mm<sup>3</sup>; platelet bound autoantibody testing at baseline (may be done); plus medical history, hepatitis B, C, and HIV at Screening (Group 3 patients).

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Design<br>Study Visit Schedule<br>and Procedures<br>3.1 Study Design<br>6.1.6 Post-Treatment<br>Period | Was: Following the Week 52 visit, patients will enter a 13-week post treatment evaluation period. Is: Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period. | To allow patients the option of continuing treatment with volanesorsen after completion of the 52-week open-label treatment period. |

| Protocol Section Description of Change Rationale | Protocol Section | Description of Change Rationale |
|---|---|---|
|---|---|---|

For consistency with the above changes:

appropriate wording was added to the following sections:

Protocol Synopsis: Study Visit Schedule and Procedures Study Design and Treatment Schema

6.2.4 ECG

6.2.7 Disease Symptom Diary6.2.8 Diet Monitoring

8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

8.10.2 Concomitant Procedures

9.4.2 Non-Serious Adverse Events

and the following table and footnotes were added to Appendix A: Schedule of Procedures:

Appendix A Schedule of Procedures - Extended Treatment Period

| Study Period | | | | | | | | Tre | atme | nt Pe | riod | | | | | | | | Treati | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>60<br>&<br>62 | Mo<br>15<br>Wk<br>64 | Wk<br>66<br>&<br>68 | Wk<br>70 | Wk<br>72<br>&<br>74 | Mo<br>18<br>Wk<br>76 | Wk<br>78<br>&<br>80 | Wk<br>82 | Wk<br>84,<br>86<br>&<br>88 | Mo<br>21<br>Wk<br>90 | Wk<br>92<br>&<br>94 | Wk<br>96 | Wk<br>98,<br>100<br>&<br>102 | Mo<br>24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | Wk<br>110 | Mo<br>27<br>Wk<br>117 |
| | Study Day | 372<br>&<br>386 | 400 | 414<br>&<br>428 | 442 | 456<br>&<br>470 | 484 | 498<br>&<br>512 | 526 | 540<br>&<br>554 | 568 | 582,<br>596<br>&<br>610 | 624 | 638<br>&<br>652 | 666 | 680,<br>694<br>&<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| Visit | Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Outpa | tient Visit | $X^f$ | $X^f$ | $X^f$ | Χ | $X^f$ | $X^f$ | X <sup>f</sup> | Х | $X^f$ | $X^f$ | $X^f$ | Х | $X^f$ | $X^f$ | $X^f$ | Χ | $X^f$ | X <sup>f</sup> | Χ |
| Vital S<br>weigh | Signs (+ body<br>t) | | | | Х | | | | Х | | | | Х | | | | Х | | | Х |
| Physic | cal Examination | | | | | | | | Х | | | | | | | | Χ | | | |
| 12- lea | ad ECG (triplicate) | | | | | | | | Х | | | | | | | | Χ | | | |
| Urinal<br>P/C ra | ysis (including<br>atio) | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Χ |
| | Chemistry Panel | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Χ | | Χ | Χ |
| | CBC with<br>Differential <sup>a</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | X | Х |
| ug) <sup>ه</sup> | Serum Lipid<br>Panel | | | | Х | | | | Х | | | | Х | | | | Х | | | Х |
| Blood Draw (Fasting) <sup>b</sup> | Coagulation<br>(aPTT, PT, INR) | | | | Х | | | | Х | | | | Х | | | | Х | | | |
| Draw | Troponin I | | | | Х | | | | Х | | | | Х | | | | Χ | | | Χ |
| l pools | Plasma PK -<br>ISIS 304801° | | | | | | | | Х | | | | | | | | Х | | | Х |
| ш | Anti-ISIS 304801<br>Antibodies | | | | | | | | Х | | | | | | | | Х | | | Х |
| | Serum<br>Pregnancy Test <sup>d</sup> | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Х |
| Week<br>Injecti | ly Study Drug: SC<br>on | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | | | |
| | lcohol<br>seling <sup>e</sup> | | | | Х | | | | Х | | | | Х | | | | Х | | | |
| Adver | se Events | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Χ |
| Conco | omitant Medication | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Х |

Protocol

### Appendix A Schedule of Procedures – Extended Treatment Period Continued

#### **Legend Text**

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>. Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor
- Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

and the following table and footnotes were added to Appendix C: Pharmacokinetic Sampling Schedule:

Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

#### PK Sampling Schedule: Extended Treatment Schedule

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Anytime |

| 6.1.4 | Extended | |
|--------|-------------|---|
| Treati | ment Period | l |

### Added

Patients will have the option of continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country.

During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the schedule of procedures in Appendix A.

To outline the procedures to be performed during the extended treatment period.

**Description of Change** 

Protocol

Period

Rationale

To outline the

period.

procedures to be performed during the

extended treatment

| 6.1.4 Extended |
|------------------|
| Treatment Period |
| Continued |

**Protocol Section** 

Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 54. 56, 58, 60, 62, 66, 68, 70, 72, 74, 78, 80, 82, 84, 86, 88, 92, 94, 96, 98, 100, and 102 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

# 6.1.6 Post-Treatment

#### Added:

Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation period consisting of 4 Study Center visits on Weeks 106, 108, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A.

To describe the follow-up visits for patients that terminate early from the extended treatment period.

### 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 3) Appendix A: Schedule of Procedures

#### Added:

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

To collect acute pancreatitis medical history events on patients that did not participate in an index study (ISIS 304801-CS6 or ISIS 304801-CS16).

### 8.5.2 Safety Monitoring for Platelet Count Results

### Added:

Table 2 Labs to Be Performed in the Event of a Platelet Count  $< 75,000 / \text{mm}^3$ .

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes. To increase platelet count monitoring for safety purposes.

### To Be Performed at Local Lab

Peripheral smear (should be performed locally, fixed and sent to central lab for review)

Fibrinogen split products or D-dimer on fresh blood

### To Be Performed at Central Lab

Citrated sample for platelets Coagulation panel (PT/INR, aPTT) CBC with reticulocytes

Fibrinogen

von Willebrand factor

Total globulins, total IgA, IgG and IgM

Complement: total C3, total C4, Bb, C5a

hsCRP

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| 8.5.2 Safety Monitoring for Platelet Count Results Continued | To Be Performed at Central Lab Continued Serology for: HBV, HCV, HIV (if not done recently for screening) Rubella CMV EBV Parvo B19 Helicobacter pylori (IgG serum test) Auto-antibody screen: Antiphospholipid Rheumatoid factor Anti-dsDNA Anti-thyroid To Be Performed at Specialty Lab(s) Antiplatelet antibodies and Anti-PF4 assay | To increase platelet count monitoring for safety purposes. |
| Section 10.3 Populations Section 10.4 Definition of Baseline | Updated: Full Analysis Set (FAS): All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. PK Population: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported. Added: Enr Croup 3 patients, the baseline for feeting ligid. | Modified to include, in the FAS, only those patients that are randomized and dosed and have a baseline TG assessment and clarified the PK Population. To add the baseline definition for Group 3 |
| Definition of Baseline | For Group 3 patients, the baseline for fasting lipid measurements is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 in this open-label study, and the baseline for other assessments is defined as the last non-missing assessment prior to the first dose of Study Drug. | patients. |
| Appendix A: Schedule of Procedures Appendix B: List of Laboratory Analytes | Added: Troponin I at Screening (Group 3 patients only) and Weeks 13, 26, 52, and 65 (All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB). Platelet bound autoantibody testing at baseline (may be done). Medical history, hepatitis B, C, and HIV at Screening (Group 3 patients only). | To ensure that Troponin I is monitored in patients that did not previously receive volanesorsen (i.e., Group 3 patients and placebo patients from the index studies) consistently with what was done in the ISIS 304801-CS6 index study. To increase platelet count monitoring for safety purposes. To make the eligibility criteria for the Group 3 patients consistent with those for the ISIS 304801-CS6 index study patients. |

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) by documentation of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for<br/>the ISIS 304801-CS16 index study<br/>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label<br/>study</li> </ul> |
| | 4. Able and willing to participate in a 65-week study |

### PROTOCOL SYNOPSIS Continued

#### Study Population Continued

Inclusion Criteria: Continued

- Satisfy 1 of the following:
  - Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years. 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)

Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c ≥ 9.0% at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of ± 10 units of insulin1)
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening

### PROTOCOL SYNOPSIS Continued

### Study Population Continued

Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued

- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
    - Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
  - c. Cardiac Troponin I > ULN at Screening
  - d. LDL-C > 130 mg/dL at Screening
  - e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- Treatment with another investigational drug, biological agent, or device within 1 month of screening, or 5 half-lives of investigational agent, whichever is longer
# PROTOCOL SYNOPSIS Continued

| Study Population Continued | Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued |
|---|---|
| | 13. Unwilling to comply with lifestyle requirements (Section 6.3) |
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study |
| | Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to screening |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br>apixaban) unless on a stable dose for at least 4 weeks prior to<br>screening and regular clinical monitoring is performed |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period |
| | Plasma apheresis within 4 weeks prior to screening or planned during the study |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to screening<br/>(Occasional or intermittent use of over-the-counter medications will be<br/>allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

#### Rationale for Dose and Schedule The dose of 300 mg once weekly was chosen for the double-blinded Selection placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. Study Visit Schedule and The study for an individual patient will generally consist of the following **Procedures** periods: Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A All patients: A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection Option to participate in an extended treatment period (up to an additional 52 weeks) A 13-week post-treatment evaluation period or expanded access program The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will

enter the 13-week post-treatment evaluation period.

| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | <ul><li>Quality of Life questionnaires (EQ-5D, SF-36)</li><li>Adjudicated acute pancreatitis event rate</li></ul> |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



# STUDY GLOSSARY

| Abbreviation/Acronym | <u>Definition</u> |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | glycosylphosphatidylinositol-anchored hdl-binding protein 1 |
| HAPI | heritability and phenotype intervention |
| HbA1c | glycated hemoglobin |
| HDL | high-density lipoprotein |
| HDL-C | high-density lipoprotein-cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL low-density lipoprotein

LDL-C low-density lipoprotein-cholesterol

LMF1 lipase maturation factor 1

LPL lipoprotein lipase

MACE major acute cardiovascular event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL no-observed-adverse-effect level

non-HDL-C non-high-density lipoprotein-cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event Statistical Analysis Plan SAP

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL triglyceride-rich lipoproteins

ULN upper limit of normal

VLDL very-low-density lipoprotein

VLDL-C very-low-density lipoprotein-cholesterol

VLDL-TG lipoprotein-triglyceride WMA World Medical Association

#### 1. **OBJECTIVES**

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

Amendment 6 18 November 2016 Protocol

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



**ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** Figure 1

From Ooi et al. 2008: ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester. CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Amendment 6

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volunesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volanesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing. The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll-over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll-over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country. Patients not participating in an expanded access program will enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

#### 3.4.3 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

Amendment 6

#### 3.4.4 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 4 Study Center visits on Weeks 54, 56, 58, and 65 (Weeks 54, 56, and 58 may be conducted by a home healthcare nurse).

#### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

#### 4.2 **Enrollment**

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 **Inclusion Criteria**

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.
  - Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:
  - a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement  $\geq$  880 mg/dL (10 mmol/L)
  - b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following:
    - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - c. Group 2: Fasting  $TG \ge 750 \text{ mg/dL}$  (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
    - Group 3: Fasting  $TG \ge 750 \text{ mg/dL}$  at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq$  55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory

- involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

# Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b.  $HbA1c \ge 9.0\%$  at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening
- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:

- Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
- ALT > 2.0 x ULN
- AST  $> 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Screening
- d. LDL-C > 130 mg/dL at Screening
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP  $\geq$  160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

#### 14. Use of any of the following:

- a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
- b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening
- c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor
- d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study
- e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period
- f. Glybera gene therapy within 2 years prior to screening
- g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed
- h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period
- i. Plasma apheresis within 4 weeks prior to screening or planned during the study
- j. Prior exposure to ISIS 304801
- k. Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

# 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

#### 6.1.3 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, and 50 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

Patients will have the option of continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country.

During the extended treatment period, patients will report to the study center for clinic visits during Weeks 54-104 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly unless the patient is on a biweekly dosing schedule for safety reasons (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volunesorsen plasma concentrations, IM testing, ECGs, and physical examinations will be performed according to the Schedule of Procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the extended treatment period. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 54, 56, 58, 60, 62, 66, 68, 70, 72, 74, 78, 80, 82, 84, 86, 88, 92, 94, 96, 98, 100, and 102 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

#### 6.1.5 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

## 6.1.6 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will have the option of participating in an expanded access program or continuing dosing for up to an additional 52 weeks until an expanded access program is approved and available in their country as described in Section 6.1.4. Patients not participating in an expanded access program will enter the 13-week post-treatment evaluation period. This 13-week post-treatment evaluation period consists of 4 Study Center visits on Weeks 54, 56, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A. Patients who complete, or terminate early from, the extended treatment period without subsequently participating in an expanded access program will enter a 13-week post-treatment evaluation

period consisting of 4 Study Center visits on Weeks 106, 108, and 110 (which may be conducted by a home healthcare nurse), and Week 117 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

## 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 roll-over patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65. Patients in the Extended Treatment Period will have ECGs performed in triplicate at Week 76 and Week 104.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

# 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period (Week 65).

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service. Patients in the Extended Treatment Period will receive diet/alcohol counseling by qualified study personnel at clinic visits only.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet may be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

Amendment 6

#### 6.2.10 Chart Review for Incidents of Acute Pancreatitis in Medical History (Group 3)

Patient records will be reviewed for incidents of acute pancreatitis occurring up to 5 years prior to screening and information relating to these events will be collected for independent adjudication.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent<sup>†</sup> or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

## For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female

condom\* with diaphragm, sponge, or cervical cap) <u>together with spermicidal</u> <u>foam/gel/film/cream/suppository</u>.

\* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

† Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

## 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2 to 8 °C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

## 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

## 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

# 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

Amendment 6 18 November 2016

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

## 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

Frequency of Repeat Measurements: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 3 in Section 8.6.3.

The tests outlined in Table 2 should also be performed as soon as possible. Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

# Table 2 Labs to Be Performed in the Event of a Platelet Count < 75,000/mm<sup>3</sup>

Note: The following labs may change as additional data is assessed, and sites will be updated regarding any changes.

| To Be Performed at Local Lab |
|---|
| Peripheral smear (should be performed locally, fixed and sent to central lab for review) |
| Fibrinogen split products or D-dimer on fresh blood |
| To Be Performed at Central Lab |
| Citrated sample for platelets |
| Coagulation panel (PT/INR, aPTT) |
| CBC with reticulocytes |
| Fibrinogen |
| von Willebrand factor |
| Total globulins, total IgA, IgG and IgM |
| Complement: total C3, total C4, Bb, C5a |
| hsCRP |
| Serology for: |
| HBV, HCV, HIV (if not done recently for screening) |
| Rubella |
| CMV |
| EBV |
| Parvo B19 |
| Helicobacter pylori (IgG serum test) |
| Auto-antibody screen: |
| Antiphospholipid |
| Rheumatoid factor |
| Anti-dsDNA |
| Anti-thyroid |
| To Be Performed at Specialty Lab(s) |
| Antiplatelet antibodies and Anti-PF4 assay |
| Anti-ASO antibody |

# 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

## 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level

Protocol

 $\leq$  70 mg/dL ( $\leq$  3.9 mmol/L). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

#### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

# 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

## 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 3 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 25,000/mm<sup>3</sup>, or a platelet count less than 75,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one

0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (**note:** may require continuation with oral steroids after methylprednisolone).

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

## <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

# <u>Definition of Clinically-Relevant, Non-Major Bleeding Events</u> (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Table 3 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1 week until stable* |
| 75K-100K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1 week |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>

#### 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 3 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment

<sup>\*\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone)

schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Amendment 6 18 November 2016

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 3 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and  $> 100,000/\text{mm}^3$ ), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.
Patients should also be encouraged to undergo a final follow-up visit (Week 65 (or Week 117 if terminating from the Extended Treatment Follow-Up Period), see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 (or Week 117 if patient enters the extended treatment period) visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

Amendment 6 18 November 2016

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 4 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's

follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit (or Week 117 if patient enters the extended treatment period). The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

## 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volunesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- Mild: The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)

Amendment 6

Protocol

- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

# 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment

Protocol

• The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and received at least 1 dose of active Study Drug and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

<u>Safety Set</u>: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 post first dose PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification). For Group 3 patients, the baseline for fasting lipid measurements is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 in this open-label study.

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study and Group 3 patients, baseline will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group of the index studies for patients on active in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies, and pooled treatment naive group which including patients on placebo in index studies and Group 3 patients.

Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

TG related endpoints will be assessed in the FAS and PPS, and all other efficacy endpoints will be assessed in the FAS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group and overall. The patient disposition will be summarized by treatment group and overall. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group and overall.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting TG  $\geq 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volunesorsen plasma concentrations will be summarized using descriptive statistics by treatment group and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index studies had been on volunesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24h</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24h</sub>/F) will be calculated from  $CL_{0.24h}/F = Actual Dose/AUC_{0.24h}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24h} = AUMC_{0-24h}/AUC_{0-24h}$ , where  $AUMC_{0-24h}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics by treatment group and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after

treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by treatment group. Furthermore, onset and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP)

as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or

the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### **12.2** Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of pre-study documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

Amendment 6

#### 12.4 Study Monitoring

Protocol

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

# **Appendix A** Schedule of Procedures

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | - | Treatr | nent I | Period | I | | | | | | | | | Post<br>Treatment<br>Follow-up | | ent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 240 | W | n, | Wk | VA/Iz | Wk | \A/Iz | \A/Iz | Mor | ıth 3 | Wk<br>15 | Wk | Wk | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| | Study Week | -8 to -2 | -2 to<br>-1 | 1 | | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | 4<br>17 | 19 | 21<br>&<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | 34<br>&<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | %<br>56 | 58 | 65 |
| | Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| | med Consent | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | atient Visit | Х | Х | Х | X | X | Χ <sup>l</sup> | Χ <sup>I</sup> | Χ <sup>l</sup> | Χ <sup>I</sup> | XI | Χ | Χ¹ | Χ <sup>l</sup> | Χ <sup>l</sup> | Χ <sup>I</sup> | Χ | Χ <sup>I</sup> | Χ <sup>l</sup> | XI | Χ | Χ <sup>l</sup> | Χ <sup>I</sup> | Χ¹ | XI | Х | Χ¹ | Χ <sup>l</sup> | Х |
| | ısion/Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | ical History⁵ | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| (+ h | Signs + body weight<br>eight on Day 1 only) | X | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| | sical Examination | Х | | Х | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | | Х |
| | ead ECG (triplicate) | Χ | | | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Χ | | | Х |
| | (liver/spleen) | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>m</sup> | | | |
| Ech | ocardiography | X | | | | | | | | | | | | | | | X <sup>m</sup> | | | | | | | | | X <sup>m</sup> | | | |
| | Chemistry Panel | Χ | Х | Х | | | Χ | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Х | | Χ | Χ |
| | CBC with Differential <sup>c</sup> | Χ | Х | Х | | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| | Serum Lipid Panel | Χ | Х | Х | | | Χ | | Χ | | Χ | Χ | | | | Χ | Χ | | | | Χ | | | | Χ | Χ | | | Х |
| | Coagulation (aPTT, PT, INR) | Χ | Х | | | | | | Х | | | Χ | | | | | Χ | | | | Х | | | | | Χ | | | |
| | Hepatitis B, C, HIV | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Blood Draw (Fasting) <sup>d</sup> | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| ast | Sedimentation Rate | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Ë | Complement (C5a, Bb) | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | X | | | Х |
| ak | Troponin I | Χ | | Х | | | | | | | | X | | | | | X | | | | | | | | | X | | | Х |
| ă | Platelet Bound Autoantibodies <sup>e</sup> | | | Х | | | | | | | | | | | | | | | | | | | | | | | | | |
| poc | Plasma PK - Volanesorsen | | | Xn | Х | | Х | | Х | | | Х | | | | | Х | | | | Х | | | 1 | | Х | | | Х |
| Ħ | Anti-Volanesorsen Antibodies | | | Х | | | Х | | X | | | X | | | | | Х | | | | Х | | | | | X | | | Х |
| | FSH (women only, if applicable) | Х | | | | | | | | | | | | | | | | | | | | | | Ì | | | | | |
| | Serum Pregnancy Test <sup>f</sup> | Х | Х | | | | Х | 1 | Х | t | | Х | 1 | Х | | | Х | | Х | | Х | | Х | 1 | | Х | 1 | Х | Х |
| | Archived Serum & Plasma<br>Samples <sup>9</sup> | | | Х | | | | | Х | | | Х | | | | | Х | | | | | | | | | X | | | Х |

### Appendix A Schedule of Procedures Continued

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | Treatment Period | | | | | | | | Post<br>Treatment<br>Follow-up | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -2 to - | W | IV. | WL | Wk | WL | Wk | WL | | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk 28 | WL | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | WL | Wk |
| Study Week | -8 to -2 | 1 | " | I | 2.5 | | 6 | 8 | 10 | | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>d</sup> | Х | Х | Χ° | | | Х | | Х | | | Χ° | | Χ° | | | Χ° | | Χ° | | Χ° | | Χ° | | | Χ° | | Χ° | Χ° |
| Fundus Photography <sup>h</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>m</sup> | | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>i</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | |
| Symptom Diary (weekly) | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Food/Drink Diary (quarterly) <sup>j</sup> | | | Х | | | | | | | | Χ | | | | | Х | | | | | | | | | Х | | | Х |
| Diet/Alcohol Counseling <sup>k</sup> | Х | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | Х | Х |
| Adverse Events | Х | Х | Х | | Х | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Х | Х |
| Concomitant Medication | Х | Χ | Х | | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ |

- a Screening and Qualification (Group 3) procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Patient charts will be reviewed in order to collect data for events of acute pancreatitis or suspected pancreatitis in the patient's medical history. Chart review may be conducted at any time during the study. These events will be adjudicated in the same manner as for events of pancreatitis during the study
- c Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>. Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor

#### Appendix A Schedule of Procedures Continued

#### Legend Text Continued

- d Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- e May be done
- f Females of childbearing potential only
- g Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- h If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- i Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 roll-over patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- j In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- k To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- I Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- m A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- n Full or abbreviated PK profile (see Appendix C)
- Expanded urinalysis (see Appendix B)

Appendix A Schedule of Procedures – Extended Treatment Period

| | Study Period | | | | | | | - | Freatme | nt Perio | od | | | | | | | | t-Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Study Week | Wk 54<br>& 56 | Wk<br>58 | Wk 60<br>& 62 | Mo 15<br>Wk 64 | | Wk<br>70 | Wk 72<br>& 74 | Mo 18<br>Wk 76 | Wk 78<br>& 80 | | Wk 84,<br>86, & 88 | | | Wk<br>96 | Wk 98,<br>100 &<br>102 | Mo 24<br>Wk<br>104 | Wk<br>106<br>&<br>108 | | Mo 27<br>Wk 117 |
| | Study Day | 372 &<br>386 | 400 | 414 &<br>428 | 442 | 456 &<br>470 | 484 | 498 &<br>512 | 526 | 540 &<br>554 | 200 | 582, 596<br>& 610 | 624 | 638 &<br>652 | 666 | 680,<br>694 &<br>708 | 722 | 736<br>&<br>750 | 764 | 813 |
| | Visit Window+/- Days | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Ou | tpatient Visit | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Х | X <sup>f</sup> | X <sup>f</sup> | X <sup>f</sup> | Χ | X <sup>f</sup> | X <sup>f</sup> | Х |
| Vit | al Signs (+ body weight) | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | Х |
| Ph | ysical Examination | | | | | | | | Χ | | | | | | | | Χ | | | |
| 12 | lead ECG (triplicate) | | | | | | | | Χ | | | | | | | | Χ | | | |
| Uri | nalysis(including P/C ratio) | | Χ | | Χ | | Χ | | Χ | | Χ | | Х | | Χ | | Χ | | Х | X |
| | Chemistry Panel | | Х | | Χ | | Х | | Χ | | Χ | | Х | | Х | | Χ | | Х | Х |
| asting) <sup>b</sup> | CBC with Differential <sup>a</sup> | Χ | Х | Х | Х | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Χ | Χ | Х | Х | X |
| astir | Serum Lipid Panel | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | X |
| 1 🖺 | Coagulation (aPTT, PT, INR) | | | | Χ | | | | Χ | | | | Х | | | | Χ | | | |
| Draw | Troponin I | | | | Х | | | | Χ | | | | Х | | | | Χ | | | X |
| ] pc | Plasma PK - ISIS 304801° | | | | | | | | Χ | | | | | | | | Χ | | | X |
| Blood | Anti-ISIS 304801 Antibodies | | | | | | | | Χ | | | | | | | | Χ | | | X |
| | Serum Pregnancy Test <sup>d</sup> | | Х | | Χ | | Х | | Χ | | Χ | | Х | | Х | | Χ | | Χ | X |
| We | ekly Study Drug: SC Injection | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Χ | Х | Χ | Χ | Χ | | | |
| Die | t/Alcohol Counseling <sup>e</sup> | | | | Х | | | | Х | | | | Х | | | | Х | | | |
| Ad | verse Events | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х |
| Со | ncomitant Medication | Х | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Х | Χ | Х | Χ | Χ | Х | Х |

#### Appendix A Schedule of Procedures – Extended Treatment Period Continued

#### Legend Text

- a Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1 week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>. Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor
- b Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration.
- c Abbreviated PK collection (see Appendix C)
- d Females of childbearing potential only
- e To reinforce compliance to the diet and alcohol restrictions
- f Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | Screening Tests (Group 3) | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| <ul> <li>Sodium</li> <li>Potassium</li> <li>Chloride</li> <li>Bicarbonate</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>Phosphorus</li> <li>Glucose</li> <li>BUN</li> <li>Creatinine</li> <li>Uric Acid</li> <li>Total bilirubin</li> <li>Direct (conjugated) bilirubin</li> <li>Indirect (unconjugated) bilirubin</li> <li>ALT</li> <li>AST</li> <li>Alkaline phosphatase</li> </ul> | <ul> <li>Hepatitis B surface antigen</li> <li>Hepatitis C antibody</li> <li>HIV antibody</li> <li>FSH (women only)</li> <li>Serum βhCG (women only)</li> </ul> Coagulation <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | <ul> <li>Red blood cells</li> <li>Hemoglobin</li> <li>Hematocrit</li> <li>MCV, MCH, MCHC</li> <li>Platelets</li> <li>White blood cells</li> <li>WBC Differential (% and absolute)</li> <li>Neutrophils</li> <li>Eosinophils</li> <li>Basophils</li> <li>Lymphocytes</li> <li>Monocytes</li> </ul> Pharmacokinetics¹ <ul> <li>Immunogenicity</li> <li>Volanesorsen levels in plasma</li> <li>Anti-volanesorsen antibodies in plasma</li> </ul> Other Assessments <ul> <li>hsCRP</li> <li>Sedimentation Rate</li> <li>C5a, Bb</li> <li>Troponin I²</li> <li>CK-MB²</li> <li>Platelet Bound Autoantibodies³</li> <li>De-lipidated free glycerol</li> <li>HbA1c, FPG</li> </ul> | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>4</sup></li> </ul> Additional Measures for Expanded Urinalysis <ul> <li>Total protein (quantitative)</li> <li>Microalbumin</li> <li>β2-microglobulin</li> </ul> |

- 1 Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents
- 2 All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- 3 May be done
- 4 Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

Amendment 6

## **Appendix C** Pharmacokinetic Sampling Schedule

Protocol

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 <sup>#</sup> |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 <sup>#</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

#### **PK Sampling Schedule (Extended Treatment Period)**

| Week | Wk<br>76 | Wk<br>104 | Wk<br>117 |
|--------------------------|-----------|-----------|-----------|
| Study Day | D526 | D722 | D813 |
| Visit Window<br>+/- Days | 2 | 2 | 7 |
| Time Point | Pre-dose, | Pre-dose | Anytime |

<sup>#</sup> Week 65 PK collection will be omitted for patients continuing to receive volanesorsen beyond Week 52

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm³ | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I and below the level of myocardial increased infarction as defined by the manufacturer | | - | Levels consistent with myocardial infarction as defined by the manufacturer |

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>ī</td><td>&lt;130 mmol/L</td></lln> | ī | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria<br>Adults | 1+ proteinuria; | 2+ proteinuria; | Urinary protein ≥3.5 g/24 hrs; |
| Children | urinary protein <1.0 g/24 hrs | urinary protein 1.0 - 3.4 g/24 hrs;<br>Urine P/C (Protein/Creatinine) | Urine P/C >1.9 |
| | | ratio 0.5 - 1.9 | Gross hematuria; transfusion, |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or<br>bladder irrigation indicated | IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





A subsidiary of Ionis Pharmaceuticals, Inc.

**Sponsor:** Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

## ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 6 - France – 16 September 2016** 

EudraCT No: 2015-003755-21

# ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

# Protocol Amendment 6 - France - 16 September 2016

#### **Protocol History:**

Original Protocol:

28 August 2015

Protocol Amendment 1:

2 February 2016

Protocol Amendment 2:

22 April 2016

Protocol Amendment 3:

9 May 2016

Protocol Amendment 4:

6 June 2016

Protocol Amendment 5:

19 August 2016

#### Sponsor:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

MD, MBA

#### Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 6 - France** 

EudraCT No: 2015-003755-21

**Clinical Phase: 3** 

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 16 September 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.
# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | anesorsen Administered Subcutaneously to<br>micronemia Syndrome (FCS) | |
| Amendment: | Amendment 6 - France | |
| Date: | 16 September 2016 | |
| Open-Label Study of Chylomicronemia Sy as described herein. I agree to comply wit Good Clinical Practical Practical agree to ensure that any purpose other that | Nolanesorsen Administered Stradrome (FCS)", dated 16 September (FCS)", dated 16 September (FCS). The International Conference (FCS). The confidential information of the evaluation or conduct of this Pharmaceuticals, Inc. | nd the attached clinical protocol, entitled "Ar ubcutaneously to Patients with Familial tember 2016, and agree to conduct the study on Harmonization Tripartite Guideline on contained in this document will not be used for the clinical investigation without the prior |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

# **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| | | DL AMENDMENT | |
| | | OL SYNOPSIS | |
| | | ESIGN AND TREATMENT SCHEMA | |
| | | LOSSARY | |
| | | CTIVES | |
| | | KGROUND AND RATIONALE | |
| 2.1 | | verview of Disease | |
| 2.2 | | herapeutic Rationale | |
| 2.3 | | olanesorsen | |
| | .3.1 | Mechanism of Action | |
| | .3.2 | Chemistry | |
| 2. | .3.3 | Preclinical Experience | |
| 2. | .3.4 | Clinical Experience | |
| 2.4 | | ationale for Dose and Schedule of Administration | |
| 3. I | EXPE | RIMENTAL PLAN | 29 |
| 3.1 | St | udy Design | 29 |
| 3.2 | N | umber of Study Centers | 29 |
| 3.3 | N | umber of Patients | 29 |
| 3.4 | O. | verall Study Duration and Follow-up | 29 |
| 3. | .4.1 | Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304 index study): Qualification | |
| 3. | .4.2 | Group 3 Patients (did not participate in an index study): Screening/Q | |
| 3. | .4.3 | Treatment | |
| 3. | .4.4 | Post-Treatment | 30 |
| 3.5 | Eı | nd-of-Study | 30 |
| 3.6 | D | ata and Safety Monitoring Board | 30 |
| 4. I | | ENT ENROLLMENT | |
| 4.1 | So | creening/Qualification | 30 |
| 4.2 | | nrollment | |
| 5. I | PATI | ENT ELIGIBILITY | 31 |
| 5.1 | | clusion Criteria | |
| 5.2 | E | xclusion Criteria | 32 |
| 6. 8 | | OY PROCEDURES | |
| 6.1 | | udy Schedule | |
| _ | .1.1 | Qualification (Groups 1 and 2) | |
| | .1.2 | Screening and Qualification (Group 3) | |
| | .1.3 | Treatment Period | |
| | .1.4 | Pharmacokinetic (PK) Subgroup | |

| | 6.1.5 | 5 Post-Treatment Period | 36 |
|----|-------|----------------------------------------------|----|
| | 6.2 | Additional Study Assessments | 36 |
| | 6.2. | 1 Laboratory Assessments | 36 |
| | 6.2.2 | Physical Exams and Vital Signs | 36 |
| | 6. | .2.2.1 Eruptive Xanthoma | 37 |
| | 6. | .2.2.2 Lipemia Retinalis | 37 |
| | 6.2.3 | 3 Echocardiography | 37 |
| | 6.2.4 | 4 ECG | 37 |
| | 6.2.5 | 5 MRI | 37 |
| | 6.2.6 | 6 Quality of Life Assessments | 37 |
| | 6.2.7 | 7 Disease Symptom Diary | 37 |
| | 6.2.8 | 8 Diet Monitoring | 37 |
| | 6.2.9 | 9 Family History | 38 |
| | 6.3 | Restriction on the Lifestyle of Patients | |
| | 6.3. | 1 Contraception Requirements | 38 |
| | 6.3.2 | 2 Other Requirements | 39 |
| 7. | ST | UDY DRUG | 39 |
| | 7.1 | Volanesorsen Description | |
| | 7.2 | Packaging and Labeling | |
| | 7.3 | Study Drug Accountability | |
| 8. | | EATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , 8 | |
| | 8.5.2 | , 8 | |
| | 8.5.3 | , & | |
| | 8.5.4 | <i>y y</i> 1 | |
| | 8.5.5 | $\boldsymbol{\mathcal{C}}$ | |
| | 8.5.6 | 5 | |
| | 8.5.7 | J C J | |
| | 8.5.8 | | |
| | 8.5.9 | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | 11 8 | |
| | 8.6.2 | 11 & | |
| | 8.6.3 | | |
| | 8.7 | Adjustment of Dose Frequency | 49 |

| | 8.8 | Discontinuation of Study Treatment | 49 |
|----|------|-------------------------------------------------|-----|
| | 8.8. | · | |
| | 8.8. | | |
| | 8.9 | Withdrawal of Patients from the Study | |
| | 8.10 | Concomitant Therapy and Procedures | 50 |
| | 8.10 | | |
| | 8.10 | 0.2 Concomitant Procedures | 51 |
| | 8.11 | Treatment Compliance | 51 |
| 9. | SE | RIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 51 |
| | 9.1 | Sponsor Review of Safety Information | 51 |
| | 9.2 | Regulatory Requirements | 52 |
| | 9.3 | Definitions | 52 |
| | 9.3. | 1 Adverse Event | 52 |
| | 9.3. | Adverse Reaction and Suspected Adverse Reaction | 53 |
| | 9.3. | | |
| | 9.4 | Monitoring and Recording Adverse Events | |
| | 9.4. | | |
| | 9.4. | | |
| | 9.4. | , | |
| | | .4.3.1 Relationship to the Study Drug | |
| | | .4.3.2 Severity | |
| | | .4.3.3 Action Taken with Volanesorsen | |
| | | .4.3.4 Treatment Given for Adverse Event | |
| | | .4.3.5 Outcome of the Adverse Event | |
| | 9.4. | <b>3</b> | |
| | 9.5 | Procedures for Handling Special Situations | |
| | 9.5. | · | |
| | 9.5. | • | |
| | 9.5. | | |
| | 9.5. | | |
| 1( | | ATISTICAL CONSIDERATIONS | |
| | 10.1 | Study Endpoints | |
| | 10.1 | y 1 | |
| | 10.1 | J 1 | |
| | 10.2 | Sample Size | |
| | 10.3 | Populations | |
| | 10.4 | Definition of Baseline | |
| | 10.5 | Interim Analysis | |
| | 10.6 | Planned Methods of Analysis | |
| | 106 | LI Demographic and Baseline Unaracteristics | n l |

Protocol - France

| 10.0 | 5.2 Sa | fety Analysis | 60 |
|---|---|---|---|
| 10.0 | | ficacy Analysis | |
| 10.0 | | armacokinetic and Immunogenicity Analysis | |
| | 0.6.4.1 | Pharmacokinetic Analysis | |
| | 0.6.4.2 | Immunogenicity Analysis | |
| | | GATOR'S REGULATORY OBLIGATIONS | |
| 11.1 | | ed Consent | |
| 11.2 | | Conduct of the Study | |
| 11.3 | | ndent Ethics Committee/Institutional Review Board | |
| 11.4 | | Confidentiality | |
| | | FRATIVE AND LEGAL OBLIGATIONS | |
| 12.1 | | ol Amendments | |
| 12.2 | Study 7 | Fermination | 64 |
| 12.3 | • | Documentation and Storage | |
| 12.4 | - | Monitoring | |
| 12.5 | • | ige | |
| 12.6 | | nsation for Injury | |
| 13. RE | EFEREN | ICES | 66 |
| 14. AP | PENDI | CES | 68 |
| Apper | ndix A | Schedule of Procedures | 69 |
| Apper | ndix B | List of Laboratory Analytes | 75 |
| Apper | ndix C | Pharmacokinetic Sampling Schedule | 77 |
| Apper | ndix D | Grading Scale for Adverse Events Relating to Laboratory Abnormaliti | es79 |
| | | TABLE OF TABLES | |
| | | | Page |
| Table 1 | Volane | sorsen (ISIS 304801) Characteristics | 40 |
| Table 2 | Actions | s in Patients With Low Platelet Count | 48 |
| Table 3 | Expect | ed Event for the Protocol Defined Population by Preferred Term and | |
| | the Exp | pected Incidence | 52 |
| | | TABLE OF FIGURES | |
| | | | Page |
| Figure 1 | - | poC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 23 |
| Figure 2 | | esign of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | _ |
| | | MOE-Gapmer). The sequence of volunesorsen is shown | |
| Figure 3 | Fa | sting Triglycerides in Patients with FCS Treated with Volanesorsen | 27 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 6 - France

**Amendment Date:** 16 September 2016

The purpose of this protocol amendment is to incorporate changes requested by ANSM as part of the conditional approval of the study, dated 7 September 2016. As such, the following modifications to Protocol ISIS 304801-CS7 Amendment 5 dated 19 August 2016 have been made:

- 1. In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from 2,000 to 500 mg/dL during this period.
- 2. To increase the post-treatment follow-up period from 13 weeks to 26 weeks or longer, if needed, until apoC-III levels return to baseline values.

In addition, language was added to indicate that after completion of the Week 52 visit assessments, patients will enter the at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Design<br>Protocol Synopsis:<br>Study Visit<br>Schedule and<br>Procedures<br>3.1 Study Design | Was: Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. Is: Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. | To follow guidance provided by the ANSM to extend the post-treatment follow-up period until apoC-III levels return to baseline values To provide an expanded access program as an option for patients that may be benefiting from active drug treatment |
| Protocol Synopsis:<br>Study Population<br>5.1 Inclusion<br>Criteria | Was: 4. Able and willing to participate in a 65-week study Is: 4. Able and willing to participate in a 78-week study | To follow guidance provided<br>by the ANSM to extend the<br>post-treatment follow-up<br>period until apoC-III levels<br>return to baseline values |

| Protocol Section | Description of Change | | | | | Rationale | |
|---|---|---|---|---|---|---|---|
| Study Design and | Was: | | | | | | To follow guidance provided |
| Treatment Schema Appendix A Schedule of | | | Study Period | Post Fo | Treat | | by the ANSM to extend the post-treatment follow-up period until apoC-III levels |
| Procedures | | | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | return to baseline values |
| | | | Study Day | 372<br>&<br>386 | 400 | | |
| | | ١ ١ | /isit Window+/- Days | 2 | 7 | 7 | |
| | | | rmed Consent | | | | |
| | | | patient Visit | X <sup>j</sup> | X <sup>j</sup> | Χ | |
| | | Vita | usion/Exclusion Criteria<br>I Signs + body weight | | | | |
| | | | eight on Day 1 only) | | | Χ | |
| | | | sical Examination | | | Χ | |
| | | | lead ECG (triplicate) | | | Χ | |
| | | MR | (liver/spleen) | | | | |
| | | Ech | ocardiography | | | | |
| | | | Chemistry Panel | | Χ | Χ | |
| | | | CBC with Differential <sup>b</sup> | Χ | Х | Х | |
| | | | Serum Lipid Panel | | | Χ | |
| | | | Coagulation (aPTT, PT, INR) | | | | |
| | | ing) <sup>c</sup> | hsCRP, HbA1c, FPG,<br>and de-lipidated free<br>glycerol | | | Х | |
| | | ast | Sedimentation Rate | | | Х | |
| | | )<br> <br> | Complement (C5a, Bb) | | | Χ | |
| | | Dra∖ | Plasma PK -<br>Volanesorsen | | | Х | |
| | | Blood Draw (Fasting) <sup>c</sup> | Anti-Volanesorsen<br>Antibodies | | | Х | |
| | | | FSH (women only, if applicable) | | | | |
| | | | Serum Pregnancy Test <sup>d</sup> | | Х | Х | |
| | | | Archived Serum & | | | | |
| | | | Plasma Samples <sup>e</sup> | | | Х | |
| | | <u> </u> | Troponin I° | | | | |
| | | Urir | alysis <sup>c</sup> | | X | X | |
| | | Fun | dus Photography <sup>f</sup> | | | | |
| | | Ger | netic testing for FCS | | | | |
| | | | nosis (if not available in | | | | |
| | | med | dical history) <sup>g</sup><br>ekly Study Drug: SC | | | | |
| | | | ction | | | | |
| | | Syn | nptom Diary (weekly) | Х | Х | Х | |
| | | Qua | lity of Life | | | Χ | |
| | | | essment(s) | | | | |
| | | | d/Drink Diary<br>arterly) <sup>h</sup> | | | Χ | |
| | | Die | :/Alcohol Counseling <sup>i</sup> | | Х | Х | |
| | | Adv | erse Events | Χ | Χ | Χ | |
| | | Cor | comitant Medication | Χ | Χ | Χ | |

| Protocol Section | Description of Change | | | | | | Rationale | 9 | |
|---|---|---|---|---|---|---|---|---|---|
| Study Design and | ls: | | | | | | | To follow guidance | provided |
| Treatment Schema | | Study Period | Post | Treat | ment l | Follov | v-up <sup>p</sup> | by the ANSM to expost-treatment follo | tend the |
| Appendix A<br>Schedule of<br>Procedures<br>Continued | | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 | period until apoC-II<br>return to baseline v | l levels |
| | | Study Day | 372<br>&<br>386 | 400 | 449 | 49<br>1 | 540 | | |
| | \ | /isit Window+/- Days | 2 | 7 | 7 | 7 | 7 | | |
| | | rmed Consent | | | | | | | |
| | | patient Visit | X <sup>J</sup> | X <sup>J</sup> | Χ | X <sup>J</sup> | Χ | | |
| | | usion/Exclusion Criteria | | | | | | | |
| | | al Signs + body weight<br>neight on Day 1 only) | | | Х | | Х | | |
| | | sical Examination | | | Х | | Х | | |
| | | lead ECG (triplicate) | | | X | | X | | |
| | | I (liver/spleen) | | | | | | | |
| | Ech | nocardiography | | | | | | | |
| | | Chemistry Panel | | Х | Х | Х | Χ | | |
| | | CBC with Differential <sup>b</sup> | Χ | Χ | Х | Χ | Χ | | |
| | | Serum Lipid Panel | | | Χ | | Χ | | |
| | | Coagulation (aPTT, PT, INR) | | | | | | | |
| | Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG,<br>and de-lipidated free<br>glycerol | | | х | | х | | |
| | asti | Sedimentation Rate | | | Х | | Х | | |
| | , (F | Complement (C5a, Bb) | | | Х | | Χ | | |
| | Oraw | Plasma PK - | | | Х | | Х | | |
| | ] pc | Volanesorsen Anti-Volanesorsen | | | | | | | |
| | Bloc | Antibodies | | | Х | | Х | | |
| | | FSH (women only, if applicable) | | | | | | | |
| | | Serum Pregnancy Test <sup>d</sup> | | Χ | Χ | Χ | Χ | | |
| | | Archived Serum & | | | Х | | Х | | |
| | | Plasma Samples <sup>e</sup> | | | L^ | | L^`\ | | |
| | | Troponin I° | | <b>∵</b> m | <b>√</b> m | <b>√</b> m | .∠m | | |
| | | <br>nalysis <sup>c</sup><br>ndus Photography <sup>f</sup> | | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> | | |
| | Ger | netic testing for FCS | | | | | | | |
| | diag | gnosis (if not available in | | | | | | | |
| | med | dical history) <sup>g</sup> | | | | | | | |
| | | ekly Study Drug: SC | | | | | | | |
| | | ection<br>nptom Diary (weekly) | Х | Х | Х | Х | <u> </u> | | |
| | | ality of Life | | <del> ^</del> | X | <del> ^</del> | X | | |
| | | sessment(s) | | | <b>l</b> ^` | | `` | | |
| | Foo | od/Drink Diary | | | Х | | Х | | |
| | | arterly) <sup>h</sup> | | ., | ., | ., | \ | | |
| | | t/Alcohol Counseling <sup>i</sup><br>verse Events | Х | X | X | X | X | | |
| | | rerse Events comitant Medication | X | X | X | X | X | | |
| | | f needed, the post-treatme | | | | | | | |
| | | r needed, the post-treatme<br>ended (with patients moni | | | | | | | |
| | | C-III levels return to base | | | | - <i>,</i> and | | | |
| | | | | | | | | <u>!</u> | |

| Protocol Section | Protocol Section Description of Change | |
|---|---|---|
| 3.4.4 Post-<br>Treatment<br>6.1.5 Post-<br>Treatment Period | Treatment After completion of the Week-52 visit assessments, patients 6.1.5 Post- will enter the 13-week post-treatment evaluation period. This | |
| 6.2.4 ECG 6.2.6 Quality of Life A 6.2.8 Diet Monitoring 8.8.1 Follow-up Visits 8.8.2 Follow-up Visits 8.10.2 Concomitant F 9.4.1 Serious Advers 9.4.2 Non-Serious Advers | s for Early Termination from Treatment Period s for Early Termination from Post-Treatment Follow-up Period Procedures se Events | |
| 8.6.3 Stopping Rules for Platelet Count Results Table 2 Actions in Patients with Low Platelet Count | Was: Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm³. Recovery in platelet coumay be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et a 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). Is: Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm³. Recovery in platelet coumay be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et a 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potentia increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period. | patient safety regarding monitoring of triglyceride levels nt |

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | <ol> <li>Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or<br/>ISIS 304801-CS16 (index studies) with an acceptable safety profile, per<br/>Sponsor and Investigator judgement.</li> </ol> |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) by documentation of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for<br/>the ISIS 304801-CS16 index study<br/>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label<br/>study</li> </ul> |
| | 4. Able and willing to participate in a 78-week study |

#### Study Population Continued

#### Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### **Exclusion Criteria**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening\*
  - b. HbA1c ≥ 9.0% at Screening\*
  - Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening\* [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)
  - e. Current use of GLP-1 agonists
- Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening\*
- 4. History within 6 months of screening\* of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening\*

#### Study Population Continued

ISIS 304801-CS7

Protocol - France

#### Exclusion Criteria Continued

- Any of the following laboratory values at Screening\*
  - Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - $ALT > 2.0 \times ULN$
    - $AST > 2.0 \times UIN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests  $\geq$  1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- Cardiac Troponin I > ULN at Screening\* C.
- d. LDL-C > 130 mg/dL at Screening\*
- Any other laboratory abnormalities which, in the opinion of the e. Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm<sup>3</sup>) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening\*
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening\*, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to screening* and dose<br>and regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>screening*</li> </ul> |
| | <ul> <li>Systemic corticosteroids or anabolic steroids within 6 weeks prior to<br/>screening* unless approved by the Sponsor Medical Monitor</li> </ul> |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening* and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening* and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to screening* |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br>apixaban) unless on a stable dose for at least 4 weeks prior to<br>screening* and regular clinical monitoring is performed |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening* and dose and regimen expected to remain constant during the treatment period |
| | <ul> <li>Plasma apheresis within 4 weeks prior to screening* or planned<br/>during the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to<br/>screening* (Occasional or intermittent use of over-the-counter<br/>medications will be allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of screening* or of > 499 mL within 60 days of screening* |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| | *(Group 3) or Qualification (Groups 1 and 2) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or<br/>ISIS 304801-CS16 index study): A qualification period of up to<br/>2 weeks (unless approved by the Sponsor). Please refer to<br/>Section 4.1 and Appendix A</li> </ul> |
| | Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A |
| | All patients: |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | <ul> <li>An at least 26-week post-treatment evaluation period</li> </ul> |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. |

| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> <li>Echocardiography</li> </ul> |
| | <ul> <li>Electrocardiograms (ECGs)</li> <li>Use of concomitant medications</li> <li>MRIs</li> </ul> |
| | Efficacy Endpoints: |
| | Frequency and severity of patient reported abdominal pain during the treatment period |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | <ul> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> </ul> |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



Amendment 6

#### STUDY GLOSSARY

#### Abbreviation/Acronym **Definition**

anti-drug antibody ADA AΕ adverse Event

alkaline Phosphatase **ALP** alanine Aminotransferase ALT ANA antinuclear Antibody apolipoprotein A-1 apoA-1 apoB apolipoprotein B apoC-III apolipoprotein C-III apolipoprotein E apoE

activated partial thromboplastin time aPTT

antisense oligonucleotide **ASO AST** aspartate aminotransferase

area under the curve **AUC BMI** body mass index **CBC** complete blood count

 $C_{max}$ maximum observed drug concentration

**CRF** case report form

deoxyribonucleic Acid DNA

**DSMB** Data and Safety Monitoring Board

electrocardiogram **ECG** 

**eCRF** electronic Case Report Form **EDC** electronic data capture

ET early termination full analysis set FAS

**FCS** Familial Chylomicronemia Syndrome

**GCP** Good Clinical Practice GLP-1 glucagon-like peptide-1

GPIHBP1 Glycosylphosphatidylinositol-anchored HDL-binding Protein 1

Heritability and Phenotype Intervention **HAPI** 

Glycated Hemoglobin HbA1c **HDL** High-Density Lipoprotein

High-Density Lipoprotein-Cholesterol HDL-C hsCRP High-sensitivity C-reactive protein

**ICH** International Conference on Harmonization

**IDL** Intermediate density lipoprotein **IEC Independent Ethics Committee** 

IM immunogenicity

**Index Studies** ISIS 304801-CS6 and ISIS 304801-CS16 CONFIDENTIAL Amendment 6
16 September 2016

#### STUDY GLOSSARY Continued

Protocol - France

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. **OBJECTIVES**

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

## 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

## 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

## 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

### 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter an at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities.

## 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

## 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Oualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

#### 3.4.3 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.4 Post-Treatment

The post-treatment evaluation period is at least 26 weeks and consists of at least 6 Study Center visits on Weeks 54, 56, 58, 65, 71, and 78 (Weeks 54, 56, 58, and 71 may be conducted by a home healthcare nurse).

#### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

## 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

## 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
- c. Group 2: Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
  - Group 3: Fasting  $TG \ge 750 \text{ mg/dL}$  at Screening for this open-label study
- 4. Able and willing to participate in a 78-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative

medical cause <u>and</u> FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

- b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening\*
  - b. HbA1c  $\geq$  9.0% at Screening\*
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening\* [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening\*
- 4. History within 6 months of screening\* of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening\*
- 5. Any of the following laboratory values at Screening\*
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Screening\*
- d. LDL-C > 130 mg/dL at Screening\*
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening\*
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening\*, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening\* and dose and regimen expected to

- remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
- b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening\*
- c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening\* unless approved by the Sponsor Medical Monitor
- d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening\* and dose and regimen expected to remain stable throughout the study
- e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening\* and dose and regimen expected to remain constant during the treatment period
- f. Glybera gene therapy within 2 years prior to screening\*
- g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening\* and regular clinical monitoring is performed
- h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening\* and dose and regimen expected to remain constant during the treatment period
- i. Plasma apheresis within 4 weeks prior to screening\* or planned during the study
- j. Prior exposure to ISIS 304801
- k. Any other medication unless stable at least 4 weeks prior to screening\* (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening\* or of > 499 mL within 60 days of screening\*
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

<sup>\*(</sup>Group 3) or Qualification (Groups 1 and 2)

## 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

## 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

#### 6.1.3 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, and 50 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on

Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.5 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the at least 26-week post-treatment evaluation period or will participate in an expanded access program pending approval by the IRBs/IEC, and the appropriate regulatory authorities. The 26-week period consists of at least 6 Study Center visits on Weeks 54, 56, 58, 65, 71, and 78 (Weeks 54, 56, 58, and 71 may be conducted by a home healthcare nurse), as outlined in the Schedule of Procedures in Appendix A.

### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

## 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should

Amendment 6

always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

## 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

## 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

## 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, Week 65, and Week 78.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, Week 65, and Week 78.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.3 **Restriction on the Lifestyle of Patients**

#### 6.3.1 **Contraception Requirements**

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent; or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq$  55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

## For male patients:

Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception,

intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

- Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.
- \* Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.
- † Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

## 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

## 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.
# Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

# 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

## 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

# 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

Frequency of Repeat Measurements: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3.

Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation

parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

# 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

# 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

# 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

<u>All patients on insulin</u> will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

## 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

#### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c > 8 and < 9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\ge 2$  weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

# 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 2 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

#### Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)

- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Table 2 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1-week until stable* |
| 75K-100K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1-week |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

<sup>\*</sup> At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>

<sup>\*\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone). In order to reduce the unlikely but potential increased risk of pancreatitis during the period of corticosteroid therapy, triglyceride levels will be monitored weekly during corticosteroid treatment and the laboratory alert will be changed from an increase of 2,000 to 500 mg/dL during that period.

## 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 2 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

# 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 78 visit assessments) approximately 26 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

# 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 78, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent.
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

# **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

# **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 78 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### 8.11 Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

# 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

# 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 3 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the

study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

# 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 78 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 78 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

# 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

# 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### *9.4.3.2 Severity*

Protocol - France

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

# 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

# 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

# 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

# 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### **10.** STATISTICAL CONSIDERATIONS

#### 10.1 **Study Endpoints**

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

<u>Safety Set</u>: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

## 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

## 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

# 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification for Group 1 and 2 patients by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index studies had been on volunesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24hr</sub> /F<sub>0-24hr</sub>) will be calculated from  $CL_{0-24hr}/F_{0-24hr} = Actual Dose/AUC_{0-24hr}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be

listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged ( $T_{\rm first}$ , i.e., onset of ADA development), the last positive IM status observed ( $T_{\rm last}$ ), the duration of ADA response (number of days between  $T_{\rm first}$  and  $T_{\rm last}$ ) if appropriate, the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., %change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

# 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

# 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

# 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

# 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

Screen/Run In through Treatment Period

Post-Treatment Follow-up

Appendix A Schedule of Procedures – Screen/Run In through Treatment Period

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | Treatment Period | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | -2 to - | V | Wk | Wk | Wk | Wk | Wk | Wk | Mor | nth 3 | | | Wk<br>21 | Mor | Month 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 |
| | | -8 to -2 | 1 | 1 | | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | Wk<br>19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| Study Day | | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| | ormed Consent | Χ | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| | tpatient Visit | Х | Χ | Χ | X | X <sup>j</sup> | $X^{j}$ | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | X <sup>j</sup> | Χ | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | X <sup>j</sup> | Χ | X <sup>j</sup> | $X^{j}$ | X <sup>j</sup> | Χ | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | $X^{j}$ | Χ |
| | usion/Exclusion Criteria | Χ | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| | Vital Signs + body weight<br>(+ height on Day 1 only) | | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х |
| Phy | sical Examination | Χ | Χ | Χ | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| 12- | lead ECG (triplicate) | Χ | Х | | | | | | | | | Χ | | | | | Χ | | | | Х | | | | | X |
| MR | I (liver/spleen) | Х | _ | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> |
| Ech | nocardiography | Х | | | | | | | | | | | | | | | $X^k$ | | | | | | | | | $X^k$ |
| | Chemistry Panel | Χ | Х | Х | | | Х | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | Х | | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| | Serum Lipid Panel | Χ | Х | Х | | | Χ | | Χ | | Χ | Χ | | | | Χ | Χ | | | | Χ | | | | Χ | Х |
| <u>°</u> | Coagulation (aPTT, PT, INR) | Χ | Χ | | | | | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | X |
| (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | X <sup>n</sup> | X <sup>n</sup> | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Ę, | Sedimentation Rate | | | Х | | | | | | | | Χ | | | | | Χ | | | | | | | | | Χ |
| > | Complement (C5a, Bb) | | | Х | | | | | | | | Χ | | | | | Χ | | | | | | | | | Χ |
| Draw | Plasma PK - Volanesorsen | | | X | Х | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| l b | Anti-Volanesorsen Antibodies | | | Х | | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ |
| Blood | FSH (women only, if applicable) | Χ | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| В | Serum Pregnancy Test <sup>d</sup> | Χ | Χ | | | | Χ | | Х | | | Χ | | Χ | | | Χ | | Х | | Χ | | Χ | | | Χ |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | | Х | | | | | Х | | | Х | | | | | Х | | | | | | | | | Х |
| | Troponin I° | Х | Х | | | | | | | | | | | | | | | | | | | | | | | |

Appendix A Schedule of Procedures - Screen/Run In through Treatment Period Continued

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | Treatment Period | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -2 to - | w | lk | Wk | Wk | Wk | k Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 |
| Study Week | -8 to -2 | 1 | "1 | | 2.5 | 4 | | 8 | | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET |
| Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Urinalysis <sup>c</sup> | Х | Х | X <sup>m</sup> | | | Х | | Х | | | X <sup>m</sup> | | $X^{m}$ | | | X <sup>m</sup> | | $\mathbf{X}^{m}$ | | $\mathbf{X}^{m}$ | | X <sup>m</sup> | | | X <sup>m</sup> |
| Fundus Photography <sup>f</sup> | Х | • | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Symptom Diary (weekly) | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Χ | Х |
| Quality of Life Assessment(s) | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х |
| Diet/Alcohol Counseling | Х | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х |
| Adverse Events | Х | Х | Χ | | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Х | Χ | Х |
| Concomitant Medication | Х | Х | Χ | | Х | Χ | Χ | Χ | Χ | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ |

# Appendix A Schedule of Procedures – Post-Treatment Follow-up

| | Study Period | Post | Treat | ment | Follow | /-up <sup>p</sup> |
|---|---|---|---|---|---|---|
| | Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| | Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| | Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Informe | ed Consent | | | | | |
| | ient Visit | X <sup>j</sup> | $X^{j}$ | Χ | X <sup>j</sup> | Х |
| | on/Exclusion Criteria | | | | | |
| | gns + body weight | | | Х | | Χ |
| | ht on Day 1 only) | | | Х | | V |
| | al Examination | | | X | | X |
| | d ECG (triplicate) ver/spleen) | | | | | Λ |
| | ardiography | | | | | |
| ECHOCA | | | V | · · | · · | |
| | Chemistry Panel CBC with Differential <sup>D</sup> | Х | X | X | X | X |
| | Serum Lipid Panel | ^ | ^ | X | ^ | X |
| ° | Coagulation (aPTT, PT, INR) | | | ^ | | _^_ |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and | | | | | |
| ast | de-lipidated free glycerol | | | Х | | Х |
| F) | Sedimentation Rate | | | Х | | Χ |
| aw | Complement (C5a, Bb) | | | Χ | | Χ |
| ۵ | Plasma PK - Volanesorsen | | | Χ | | Χ |
| poo | Anti-Volanesorsen Antibodies | | | Χ | | Χ |
| Bic | FSH (women only, if applicable) | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | | Χ | Χ | Χ | Χ |
| | Archived Serum & Plasma Samples <sup>e</sup> | | | Χ | | Χ |
| | Troponin I° | | | | | |

# **Appendix A** Schedule of Procedures – Post-Treatment Follow-up *Continued*

| Study Period | Pos | st Trea | tment l | Follow- | up <sup>p</sup> |
|---|---|---|---|---|---|
| Study Week | Wk<br>54<br>&<br>56 | Wk<br>58 | Wk<br>65 | Wk<br>71 | Wk<br>78 |
| Study Day | 372<br>&<br>386 | 400 | 449 | 491 | 540 |
| Visit Window+/- Days | 2 | 7 | 7 | 7 | 7 |
| Urinalysis <sup>c</sup> | | X <sup>m</sup> | X <sup>m</sup> | X <sup>m</sup> | $X^{m}$ |
| Fundus Photography <sup>f</sup> | | | | | |
| Genetic testing for FCS diagnosis<br>(if not available in medical<br>history) <sup>9</sup> | | | | | |
| Weekly Study Drug: SC Injection | | | | | |
| Symptom Diary (weekly) | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | | Х | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | | Х | Х | Х | Х |
| Adverse Events | Х | Х | Х | Х | Х |
| Concomitant Medication | Χ | X | Χ | Χ | Χ |

#### Appendix A Schedule of Procedures Continued

- a Screening (Group 3) and Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. In the event of any platelet count less than 50,000/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor
- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- I Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)
- n HbA1c only
- o All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB
- p If needed, the post-treatment follow-up period will be extended (with patients monitored every 6 weeks) until apoC-III levels return to baseline values

# **Appendix B** List of Laboratory Analytes
# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | <b>Coagulation</b> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Chloride Bicarbonate Total protein Albumin Calcium Magnesium Phosphorus Glucose BUN Creatinine Uric Acid Total bilirubin Direct (conjugated) bilirubin Indirect (unconjugated bilirubin ALT AST Alkaline phosphatase | <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP | Urinalysis Color Appearance Specific gravity pH Protein Blood Ketones Urobilinogen Glucose Bilirubin Leukocyte esterase Nitrate Microscopic examination <sup>2</sup> Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin B2-microglobulin |
| 1 Plasma PK samples m | | <ul> <li>Sedimentation Rate</li> <li>C5a, Bb</li> <li>De-lipidated free glycerol</li> <li>HbA1c, FPG</li> </ul> | |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

# PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 | Wk<br>78 |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 | D540 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm <sup>3</sup> - 20,000/mm <sup>3</sup> | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160<br>mg/dL; Fasting glucose value >ULN -<br>8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L; hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>ī</td><td>&lt;130 mmol/L</td></lln> | ī | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td colspan="2">&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria<br>Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs;<br>Urine P/C (Protein/Creatinine) | Urinary protein ≥3.5 g/24 hrs; |
| Children | A constant at a state of a state | ratio 0.5 - 1.9 | Urine P/C >1.9 Gross hematuria; transfusion, IV medications or |
| Hematuria | Asymptomatic; clinical or diagnostic<br>observations only; intervention not<br>indicated | Symptomatic; urinary catheter or bladder irrigation indicated | hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





A subsidiary of Ionis Pharmaceuticals, Inc.

**Sponsor:** Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

# ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Protocol Amendment 5 - France – 19 August 2016** 

EudraCT No: 2015-003755-21

### ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 5 - France – 19 August 2016

# **Protocol History:**

Original Protocol:

28 August 2015

Protocol Amendment 1:

2 February 2016

Protocol Amendment 2:

22 April 2016

Protocol Amendment 3:

9 May 2016

Protocol Amendment 4:

6 June 2016

### Sponsor:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

MD, MBA

### **Ionis Protocol Number: ISIS 304801-CS7**

**Protocol Amendment 5 - France** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

# An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 19 August 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Vol<br>Patients with Familial Chylor | anesorsen Administered Subcutaneously to micronemia Syndrome (FCS) |
| Amendment: | Amendment 5 - France | |
| Date: | 19 August 2016 | |
| Open-Label Study of | Volanesorsen Administered S | nd the attached clinical protocol, entitled "Arabeutaneously to Patients with Familial ast 2016, and agree to conduct the study as |
| I agree to comply wi<br>Good Clinical Praction | | on Harmonization Tripartite Guideline on |
| any purpose other that | | ontained in this document will not be used fo<br>the clinical investigation without the prior |
| Investigator's Signar | ture | |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

# **TABLE OF CONTENTS**

| | Paş | _ |
|---|---|---|
| | T | |
| STUDY DESIGN AND TRE | ATMENT SCHEMA | <b>26</b> |
| STUDY GLOSSARY | | <b>27</b> |
| 2. BACKGROUND AND | RATIONALE | <b>29</b> |
| 2.1 Overview of Disease | | 29 |
| 2.2 Therapeutic Rational | e | 30 |
| 2.3 Volanesorsen | | 31 |
| 2.3.1 Mechanism of A | ection | 31 |
| 2.3.2 Chemistry | | 32 |
| 2.3.3 Preclinical Expe | rience | 33 |
| 2.3.4 Clinical Experie | nce | 34 |
| 2.4 Rationale for Dose a | nd Schedule of Administration | 35 |
| 3. EXPERIMENTAL PLA | N | 36 |
| 3.1 Study Design | | 36 |
| 3.2 Number of Study Ce | nters | 36 |
| 3.3 Number of Patients. | | 36 |
| 3.4 Overall Study Durati | on and Follow-up | 36 |
| | atients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 | |
| | palification | 36 |
| 3.4.2 Group 3 Patients | s (did not participate in an index study): Screening/Qualification3 | 36 |
| 3.4.3 Treatment | | 36 |
| 3.4.4 Post-Treatment | | 36 |
| 3.5 End-of-Study | | 37 |
| 3.6 Data and Safety Mor | itoring Board | 37 |
| 4. PATIENT ENROLLM | ENT. | <b>37</b> |
| 4.1 Screening/Qualificat | ion | 37 |
| 4.2 Enrollment | | 37 |
| 5. PATIENT ELIGIBILIT | Υ | 38 |
| 5.1 Inclusion Criteria | | 38 |
| 5.2 Exclusion Criteria | | 39 |
| | $\mathbf{S}$ | |
| • | roups 1 and 2) | |
| | Pualification (Group 3) | |
| | d | |
| | c (PK) Subgroup | |

| | 6.1.5 | Post-Treatment Period. | 43 |
|----|-------|----------------------------------------------|------------|
| | 6.2 | Additional Study Assessments | 43 |
| | 6.2.1 | Laboratory Assessments | 43 |
| | 6.2.2 | | |
| | 6.3 | 2.2.1 Eruptive Xanthoma | |
| | 6.3 | 2.2.2 Lipemia Retinalis | 44 |
| | 6.2.3 | Echocardiography | 44 |
| | 6.2.4 | ECG | 44 |
| | 6.2.5 | MRI | 44 |
| | 6.2.6 | Quality of Life Assessments | <b>4</b> 4 |
| | 6.2.7 | Disease Symptom Diary | 44 |
| | 6.2.8 | Diet Monitoring | 44 |
| | 6.2.9 | Family History | 45 |
| | 6.3 | Restriction on the Lifestyle of Patients | 45 |
| | 6.3.1 | Contraception Requirements | 45 |
| | 6.3.2 | Other Requirements | 46 |
| 7. | . STU | JDY DRUG | |
| | 7.1 | Volanesorsen Description | |
| | 7.2 | Packaging and Labeling | |
| | 7.3 | Study Drug Accountability | |
| 3. | | EATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5.1 | , c | |
| | 8.5.2 | | |
| | 8.5.3 | , | |
| | 8.5.4 | 7 8 | |
| | 8.5.5 | , | |
| | 8.5.6 | , , | |
| | 8.5.7 | , | |
| | 8.5.8 | | |
| | 8.5.9 | | |
| | 8.6 | Stopping Rules | |
| | 8.6.1 | 11 8 | |
| | 8.6.2 | 11 & | |
| | 8.6.3 | | |
| | 8.7 | Adjustment of Dose Frequency | 55 |

| | 8.8 | Dis | continuation of Study Treatment | 56 |
|---|---|---|---|---|
| | 8.8. | 1 | Follow-up Visits for Early Termination from Treatment Period | 56 |
| | 8.8.2 | 2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Per | |
| | 8.9 | Wit | thdrawal of Patients from the Study | |
| | 8.10 | | ncomitant Therapy and Procedures | |
| | 8.10 | ).1 | Concomitant Therapy | 57 |
| | 8.10 | ).2 | Concomitant Procedures. | 58 |
| | 8.11 | Tre | atment Compliance | 58 |
| 9. | SE) | | US AND NON-SERIOUS ADVERSE EVENT REPORTING | |
| | 9.1 | Spo | onsor Review of Safety Information | 58 |
| | 9.2 | Reg | gulatory Requirements | 58 |
| | 9.3 | Def | initions | 59 |
| | 9.3. | 1 | Adverse Event | 59 |
| | 9.3. | 2 | Adverse Reaction and Suspected Adverse Reaction | 59 |
| | 9.3. | 3 | Serious Adverse Event (SAE) | 60 |
| | 9.4 | Mo | nitoring and Recording Adverse Events | 60 |
| | 9.4. | 1 | Serious Adverse Events | 60 |
| | 9.4.2 | 2 | Non-Serious Adverse Events | 61 |
| | 9.4. | 3 | Evaluation of Adverse Events (Serious and Non-Serious) | 61 |
| | 9. | .4.3.1 | Relationship to the Study Drug | 61 |
| | 9. | .4.3.2 | 2 Severity | 61 |
| | 9. | .4.3.3 | 3 Action Taken with Volanesorsen | 62 |
| | 9. | .4.3.4 | Treatment Given for Adverse Event | 62 |
| | 9. | .4.3.5 | 5 Outcome of the Adverse Event | 62 |
| | 9.4.4 | 4 | Adjudication Committees | 63 |
| | 9.5 | Pro | cedures for Handling Special Situations | 63 |
| | 9.5. | 1 | Abnormalities of Laboratory Tests | 63 |
| | 9.5.2 | 2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 63 |
| | 9.5. | 3 | Dosing Errors | 64 |
| | 9.5.4 | 4 | Contraception and Pregnancy | 64 |
| 1( | ). ST | ATIS | STICAL CONSIDERATIONS | 65 |
| | 10.1 | Stu | dy Endpoints | |
| | 10.1 | 1 | Efficacy Endpoints | 65 |
| | 10.1 | .2 | Safety Endpoints | 65 |
| | 10.2 | San | nple Size | 65 |
| | 10.3 | - | oulations | |
| | 10.4 | | inition of Baseline | |
| | 10.5 | | erim Analysis | |
| | 10.6 | | nned Methods of Analysis | |
| | 10.6 | 5.1 | Demographic and Baseline Characteristics | 67 |

| 10.0 | 6.2 Safety Analysis | 67 |
|---|---|---|
| 10.0 | 6.3 Efficacy Analysis | 67 |
| 10.0 | 6.4 Pharmacokinetic and Immunogenicity Analysis | 68 |
| 1 | 0.6.4.1 Pharmacokinetic Analysis | 68 |
| 1 | 0.6.4.2 Immunogenicity Analysis | 68 |
| 11. IN | VESTIGATOR'S REGULATORY OBLIGATIONS | 69 |
| 11.1 | Informed Consent | 69 |
| 11.2 | Ethical Conduct of the Study | 70 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 70 |
| 11.4 | Patient Confidentiality | 70 |
| 12. AI | OMINISTRATIVE AND LEGAL OBLIGATIONS | 71 |
| 12.1 | Protocol Amendments | 71 |
| 12.2 | Study Termination | 71 |
| 12.3 | Study Documentation and Storage | 71 |
| 12.4 | Study Monitoring | 72 |
| 12.5 | Language | 72 |
| 12.6 | Compensation for Injury | 72 |
| 13. RF | EFERENCES | 73 |
| 14. AF | PPENDICES | 75 |
| Apper | ndix A Schedule of Procedures | 76 |
| Apper | ndix B List of Laboratory Analytes | |
| Apper | ndix C Pharmacokinetic Sampling Schedule | 82 |
| Apper | ndix D Grading Scale for Adverse Events Relating to Laboratory Abno | ormalities84 |
| | TABLE OF TABLES | |
| | | Page |
| | Volanesorsen (ISIS 304801) Characteristics | |
| Table 2 | Actions in Patients With Low Platelet Count | |
| Table 3 | Expected Event for the Protocol Defined Population by Preferred Term | |
| | the Expected Incidence | 59 |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | | sms 30 |
| Figure 2 | | 22 |
| Et a | (MOE-Gapmer). The sequence of volunesorsen is shown | |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesor | sen 34 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 5 - France

**Amendment Date:** 19 August 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 4 dated 6 June 2016:

1. To enroll FCS patients in this open-label study who did not participate in the ISIS 304801–CS6 or ISIS 304801–CS16 index studies.

For clarity, the protocol now specifies 3 patient groups, with assignment based on prior involvement in index studies of ISIS 304801:

Group 1: ISIS 304801-CS6 (index study) rollover FCS patients

Group 2: ISIS 304801-CS16 (index study) rollover FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

- 2. To remove language that indicates that lipoprotein lipase (LPL) activity can be measured if needed for study qualification for patients in Groups 2 and 3.
- 3. To add language to indicate that a second Study Drug rechallenge will not be allowed following a platelet count decrease below 75,000/mm<sup>3</sup>.
- 4. To provide clarifications to the platelet safety monitoring rules in Table 2.
- 5. To add language to indicate that patients who discontinue early from Study Drug, or the study, should be followed as per the platelet monitoring rules shown in Table 2 for the first 6 weeks after discontinuing Study Drug and the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.
- 6. Following guidance provided by the ANSM
  - a. Following guidance provided by the ANSM, the complete stop of Study Drug in patients whose platelet threshold is below 25,000/mm<sup>3</sup> will be changed to below 50.000/mm<sup>3</sup>

- b. To add a criteria for treatment discontinuation: patient participation to the trial must be stopped if a decrease in platelets greater than or equal to 50% between two consecutive assessments is observed, irrespective of the platelet level
- c. To add in the footnote to Appendix A that in the event of any platelet count less than 50,000/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently
- d. To add in the Exclusion Criteria patients that already had thrombocytopenia
- e. To add language to exclude patients that meet the Exclusion Criteria of their index study

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Title pages Signature page Protocol Synopsis: Title, Study Population, Rationale for Dose and Schedule Selection, Study Visit Schedule and Procedures, Statistical Considerations 5.1 Inclusion Criteria | "Extension" was removed from the study title. | To note that FCS patients who did not participate in an index study will also be enrolled. |
| Protocol Synopsis:<br>Study Design<br>3.1 Study Design | Was: This is a multi-center open-label extension study of ISIS 304801-CS6 and ISIS 304801-CS16 Is: This is a multi-center open-label study of: Group 1: ISIS 304801-CS6 (index study) roll over FCS patients Group 2: ISIS 304801-CS16 (index study) roll over FCS patients Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies | To distinguish patients who participated in an index study from those who did not. |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Population<br>5.1 Inclusion Criteria | <ul> <li>Inclusion Criteria</li> <li>Was:</li> <li>3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> <li>c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study</li> </ul> </li> </ul></li></ul> | To define the inclusion criteria for each Group of patients. LPL removed to avoid the production of heparin induced anti-platelet antibodies. |
| | <ul> <li>Is:</li> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study</li> <li>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label study</li> </ul> </li> </ul></li></ul> | |

| Protocol Section Description of Change Rationale |
|---|
| Protocol Synopsis: Study Population 5.2 Exclusion Criteria Was: 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) 1. Diabetes mellitus with any of the following: a. Newly diagnosed within 12 weeks of screening* b. HbA1c≥9.0% at Screening* c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening* with the exception of ± 10 units of insulin ) d. Anticipated need to change dose or type of medication during the treatment period of the Study [with the exception of ± 10 units of insulin e. Current use of GLP-1 agonists 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome 3. Active pancreatitis within 4 weeks prior to screening* 4. History within 6 months of screening* of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening* 5. Any of the following laboratory values at Screening* 5. Any of the following laboratory values at Screening* 6. ALT > 2.0 x ULN 6. AST > 2.0 x ULN 6. AST > 2.0 x ULN 6. Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs 9. Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs 9. Persistently positive (2 out of 3 consecutive tests ≥ trace positive) |

| 5.2 Exclusion Criteria Continued C. Cardiac Troponin 1 > OEN at Screening d. LDL-C > 130 mg/dL at Screening* e. Any other laboratory abnormalities which, in the opinion of the make | dofina tha |
|---|---|
| unsuitable for inclusion 6. Uncontrolled hypertension (BP > 160/100 mm Hg) 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening* 8. History of heart failure with NYHA greater than Class II | lusion eria for each up of ents and to ke the ibility criteria the Group 3 |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis: Study Population Continued 5.2 Exclusion Criteria Continued | Exclusion Criteria Is: Continued j. Prior exposure to ISIS 304801 k. Any other medication unless stable at least 4 weeks prior to screening* (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion) 15. Blood donation of 50 to 499 mL within 30 days of screening* or of > 499 mL within 60 days of screening* 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study *(Group 3) or Qualification (Groups 1 and 2) | To define the exclusion criteria for each Group of patients and to make the eligibility criteria for the Group 3 patients consistent with those for the Group 1 index study patients. |
| Protocol Synopsis: Study Visit Schedule and Procedures 3.4 Overall Study Duration and Follow-up Appendix A | <ul> <li>Was: <ul> <li>The study for an individual patient will generally consist of the following periods:</li> <li>A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.</li> <li>○ A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection</li> <li>○ A 13-week post-treatment evaluation period</li> </ul> </li> <li>Is: <ul> <li>The study for an individual patient will generally consist of the following periods:</li> <li>● Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.</li> <li>● Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A.</li> <li>All patients:</li></ul></li></ul> | To distinguish the Screening/ Qualification period for patients who participated in an index study from those who did not. |
| 4.1<br>Screening/Qualification | Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used | To define the enrollment criteria for patients who did not participate in an index study. |

| Protocol Section | | | Description of Chang | е | | Rationale |
|---|---|---|---|---|---|---|
| 6.1.2 Screening and Qualification (Group 3) | pa<br>pe<br>(s<br>ap<br>di<br>so<br>pe<br>de | Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes | | | To define the<br>Screening and<br>Qualification<br>procedures for<br>patients who did<br>not participate in<br>an index study. | |
| 8.6.3 Stopping Rules for Platelet Count Results | If 75 co parto to ex M lf 75 will so de M lf M lf T5 lf 75 l | Was: If after the first dosing rechallenge the platelet count again falls below 75,000/mm³, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm³. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be reexamined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above. If after the second rechallenge the platelet count falls below 75,000/mm³ and is subsequently confirmed (see Section 8.5), dosing with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor. Is: If after the first dosing rechallenge the platelet count again falls below 75,000/mm³, then dosing of the patient with Study Drug will be stopped permanently. | | | Text was removed as a second Study Drug rechallenge will not be allowed following a platelet count decrease below 75,000/mm <sup>3</sup> . | |
| 8.6.3 Stopping Rules for Platelet Count Results | | Platelet Count on Rx | Drug Dose | Monitoring | | To provide clarification to the platelet |
| Table 2 Actions in Patients with Low | | Normal range,<br>> 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks | | safety<br>monitoring rules. |
| Platelet Count | | 100K-<br>140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1-week <u>until</u> <u>stable*</u> | | Note: Changes<br>are reflected as<br>bold underlined<br>text. |
| | | 75K-100K/mm <sup>3</sup> | Permanently reduce<br>dose frequency to<br>300mg every 2 weeks<br>or reduce dose to<br>150 mg weekly | Closer observation<br>Monitor every<br>1-week | | ioni. |

| Protocol Section | | Description of Chang | e | Rationale |
|---|---|---|---|---|
| 8.6.3 Stopping Rules for Platelet Count Results Table 2 Actions in Patients with Low Platelet Count Continued | Platelet Count on Rx | Drug Dose | Monitoring | To provide clarification to the platelet |
| | 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. Dose pause When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication | safety<br>monitoring rules Note: Changes<br>are reflected as<br>bold underlined<br>text |
| | 25K-50K/mm³ or a rate of decline ≥ 50% between 2 consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2 3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/an ticoagulant medication while platelet count < 50K/mm³ if possible | |

| Protocol Section | | Description of Chang | e | Rationale |
|---|---|---|---|---|
| 8.6.3 Stopping Rules for Platelet Count Results Table 2 Actions in Patients with Low Platelet Count Continued | ** Recovery in pla<br>of high dose steroid<br>thrombocytopenia (<br>40 mg daily for 4 da<br>0.5-2 mg/kg/d for 2- | Permanently discontinue Study Drug secutive values measured remined by the Sponsor Management of the Sponsor Management o | ated by administration r immune nend Dexamethasone cycles; Prednis(ol)one chylprednisolone | To provide clarification to the platelet safety monitoring rules Note: Changes are reflected as bold underlined text |
| 8.8.1 Follow-up Visits | steroids after methy Was: | l prednisolone) | | To provide |
| for Early Termination<br>from Treatment Period | Any patient who dis be strongly encoura Weeks 2, 13, 25, 26 since Day 1) to colle assessments in acc Appendix A. Any pashould also be stron (Week 65 visit asse | continues early from the Traged to attend applicable la 5, and 51, 52 (calculated based fasting lipid panels and cordance with the schedule atient who discontinues treatingly encouraged to attend assments) approximately 13, in addition to the applicab | ndmark visits at ased on the time elapsed conduct safety of procedures in atment after Week 44 a final follow-up visit weeks after their last | guidance to the platelet safety monitoring rules for patients that discontinue early from the Treatment Period. |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| 8.8.1 Follow-up Visits for Early Termination from Treatment Period Continued | Is: Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits. | To provide guidance to the platelet safety monitoring rules for patients that discontinue early from the Treatment Period. |
| 8.8.2 Follow-up Visits<br>for Early Termination<br>from Post-Treatment<br>Follow-up Period | Was: The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study. Is: The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor medical monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study. | To provide guidance to the platelet safety monitoring rules for patients that discontinue early from the Post-Treatment Follow-up Period. |
| 8.6.3 Stopping Rules for Platelet Count Results Table 2 Actions in Patients with Low Platelet Count | Was: In the event of any platelet count less than 25,000/mm³, or a platelet count less than 75,000/mm³ that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week, then dosing of a patient with volanesorsen will be stopped permanently. Is: In the event of any platelet count less than 50,000/mm³, or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with volanesorsen will be stopped permanently. | To follow guidance provided by the ANSM to provide additional patient safety regarding platelet stopping rules. |
| Appendix A | Added to Footnote "b": In the event of any platelet count less than 50,000/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently. | To follow guidance provided by the ANSM to clarify the additional patient safety regarding platelet stopping rules in Appendix A. |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Population<br>5.2<br>Exclusion Criteria | Exclusion Criteria Was: Thistory of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening Is: History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening | To exclude patients with a history of thrombocytopeni a because it sometimes seems to be associated with patients suffering from hyperchylomicronemia |

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, Sponsor and Investigator judgement. |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) by documentation of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for<br/>the ISIS 304801-CS16 index study<br/>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label<br/>study</li> </ul> |
| | 4. Able and willing to participate in a 65-week study |

#### Study Population Continued

#### Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### Exclusion Criteria

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening\*
  - b. HbA1c ≥ 9.0% at Screening\*
  - Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening\* [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening\*
- 4. History within 6 months of screening\* of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening\*

#### Study Population Continued

#### Exclusion Criteria Continued

- Any of the following laboratory values at Screening\*
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Screening\*
- d. LDL-C > 130 mg/dL at Screening\*
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- History of thrombocytopenia (platelet count < 100,000/mm<sup>3</sup>) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening\*
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening\*, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)

| Study Population Continued | Exclusion Criteria Continued |
|---|---|
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to screening* and dose<br>and regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | <ul> <li>b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to<br/>screening*</li> </ul> |
| | <ul> <li>Systemic corticosteroids or anabolic steroids within 6 weeks prior to<br/>screening* unless approved by the Sponsor Medical Monitor</li> </ul> |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening* and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening* and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to screening* |
| | <ul> <li>g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br/>apixaban) unless on a stable dose for at least 4 weeks prior to<br/>screening* and regular clinical monitoring is performed</li> </ul> |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening* and dose and regimen expected to remain constant during the treatment period |
| | <ul> <li>Plasma apheresis within 4 weeks prior to screening* or planned<br/>during the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to<br/>screening* (Occasional or intermittent use of over-the-counter<br/>medications will be allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of screening* or of > 499 mL within 60 days of screening* |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| | *(Group 3) or Qualification (Groups 1 and 2) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or<br/>ISIS 304801-CS16 index study): A qualification period of up to<br/>2 weeks (unless approved by the Sponsor). Please refer to<br/>Section 4.1 and Appendix A</li> </ul> |
| | Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A |
| | All patients: |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | <ul> <li>A 13-week post-treatment evaluation period</li> </ul> |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an open-label study. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

### STUDY DESIGN AND TREATMENT SCHEMA



# STUDY GLOSSARY

**Index Studies** 

| Abbreviation/Acronym | <b>Definition</b> |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| T 1 0 11 | |

ISIS 304801-CS6 and ISIS 304801-CS16

#### STUDY GLOSSARY Continued

INR International Normalized Ratio IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time SAE serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V
(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

# 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Protocol - France

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

### 2.3 Volanesorsen

### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

## 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

## 2.3.3 Preclinical Experience

Protocol - France

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

## 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

## 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 **Study Design**

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volunesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 **Number of Study Centers**

This study will be conducted at multiple centers worldwide.

#### 3.3 **Number of Patients**

Up to approximately 70 patients will be dosed.

#### 3.4 **Overall Study Duration and Follow-up**

The Study will consist of the following periods:

### 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

#### 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

#### 3.4.3 **Treatment**

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.4 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

## 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

### 4. PATIENT ENROLLMENT

## 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 **Inclusion Criteria**

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement  $\geq 880 \text{ mg/dL} (10 \text{ mmol/L})$
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
- c. Group 2: Fasting  $TG \ge 750 \text{ mg/dL}$  (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
  - Group 3: Fasting  $TG \ge 750 \text{ mg/dL}$  at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq$  55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer

to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

\* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 **Exclusion Criteria**

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening\*
  - b.  $HbA1c \ge 9.0\%$  at Screening\*
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening\* [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening\*
- 4. History within 6 months of screening\* of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening\*
- 5. Any of the following laboratory values at Screening\*
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be  $\leq 3 \text{ mg/dL}$
    - $ALT > 2.0 \times ULN$
    - AST  $> 2.0 \times ULN$
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests  $\geq 1+$ ) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs

- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Screening\*
- d. LDL-C > 130 mg/dL at Screening\*
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of thrombocytopenia (platelet count < 100,000/mm³) or bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening\*
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated
- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening\*, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening\* and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening\*
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening\* unless approved by the Sponsor Medical Monitor

- d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening\* and dose and regimen expected to remain stable throughout the study
- e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening\* and dose and regimen expected to remain constant during the treatment period
- f. Glybera gene therapy within 2 years prior to screening\*
- g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening\* and regular clinical monitoring is performed
- h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening\* and dose and regimen expected to remain constant during the treatment period
- i. Plasma apheresis within 4 weeks prior to screening\* or planned during the study
- j. Prior exposure to ISIS 304801
- k. Any other medication unless stable at least 4 weeks prior to screening\* (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening\* or of > 499 mL within 60 days of screening\*
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, including new or worsening of existing condition, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study
- \*(Group 3) or Qualification (Groups 1 and 2)

## 6. STUDY PROCEDURES

## 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

# 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

## 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least

6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

### 6.1.3 Treatment Period

Protocol - France

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, and 50 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

## 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being

Amendment 5 Protocol - France 19 August 2016

withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### Post-Treatment Period 6.1.5

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 4 Study Center visits on Weeks 54, 56, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A.

#### **6.2 Additional Study Assessments**

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

## 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

## 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

# 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.3 **Restriction on the Lifestyle of Patients**

#### 6.3.1 **Contraception Requirements**

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent\* or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females  $\leq 55$  years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

## For male patients:

Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

## For female patients:

Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

# 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

### 7. STUDY DRUG

# 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

## 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

<sup>\*</sup>Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

<sup>\*</sup> Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 7.3 **Study Drug Accountability**

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### Volanesorsen Administration 8.1

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volunesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 **Other Protocol-Required Drugs**

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 **Other Protocol-Required Treatment Procedures**

There are no other protocol required treatment procedures for this study.

#### 8.4 **Treatment Precautions**

There are no specific treatment precautions required for this study.

#### 8.5 **Safety Monitoring Rules**

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

Amendment 5 19 August 2016 Protocol - France

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

Confirmation Guidance: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below must be confirmed by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest must be available prior to administering the next dose of volunesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### Safety Monitoring for Liver Chemistry Tests 8.5.1

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times 10^{-2} \times 10^{-2}$ value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

Frequency of Repeat Measurements: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

Further Investigation into Liver Chemistry Elevations: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3.

Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinicallyrelevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

The Investigator or delegate will review the glucometer reading or printout at every clinic visit to evaluate if fasting pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for Hyperglycemia below.

All diabetic patients will note any changes in their insulin dose and /or oral antidiabetic therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - o Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose  $\leq$  70 mg/dL ( $\leq$  3.9 mmol/L).
  - o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### **8.5.** 7 Safety Monitoring for Documented Severe Hypoglycemia

A documented severe hypoglycemic event is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level ≤ 70 mg/dL (≤ 3.9 mmol/L). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly. Protocol - France

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

## 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

## 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

## 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\ge 2$  weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

## 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5 µmol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 2 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than  $50,000/\text{mm}^3$ , or a rate of decline  $\geq 50\%$  between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone).

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

# <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

## <u>Definition of Clinically-Relevant, Non-Major Bleeding Events</u> (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Protocol - France

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1-week until stable* |
| 75K-100K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1-week |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level | Permanently discontinue Study Drug | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

<sup>\*</sup> At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>

## 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 2 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment

<sup>\*\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone)

schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

## 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

## 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

## 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.

Amendment 5 Protocol - France 19 August 2016

Patients should also be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 **Concomitant Therapy and Procedures**

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-thecounter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

## **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

## **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

## 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

## 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 3 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

### 9.3 Definitions

### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

## 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

Protocol - France

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

# 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

## 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's

follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- Related: There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

#### 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volanesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

## 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

## 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- **Persists (as non-serious AE):** Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)

- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 **Adjudication Committees**

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 **Procedures for Handling Special Situations**

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment

Amendment 5 Protocol - France 19 August 2016

The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 **Dosing Errors**

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volanesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

Should an overdose occur, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

### 10. STATISTICAL CONSIDERATIONS

## 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

## 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

## 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

## 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.
#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Protocol - France

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

Protocol - France

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification for Group 1 and 2 patients by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index studies had been on volunesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24hr</sub> /F<sub>0-24hr</sub>) will be calculated from  $CL_{0-24hr}/F_{0-24hr} = Actual Dose/AUC_{0-24hr}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be

listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 **Ethical Conduct of the Study**

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 **Independent Ethics Committee/Institutional Review Board**

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volunesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 **Patient Confidentiality**

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

Amendment 5 Protocol - France 19 August 2016

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 **Study Monitoring**

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 **Compensation for Injury**

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

### 14. APPENDICES

# **Appendix A** Schedule of Procedures

## **Appendix A** Schedule of Procedures

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | - | Γreatn | nent l | Period | | | | | | | | | | Post<br>Fo | Treat | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | -2 to - | w | ık | Wk | Wk | Wk | Wk | Wk | Mor | th 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| | Study Week | -8 to -2 | 1 | 1 1 | | 2.5 | | | 8 | 10 | Wk<br>12 | Wk<br>13 | Wk & | 19 | &<br>23 | Wk<br>25 | | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| | Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| Visit Window+/- Days | | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Informed Consent | | Χ | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Ou | patient Visit | Х | Х | Χ | $X_1$ | Χ <sup>J</sup> | $X_{l}$ | $X_1$ | $X_1$ | $X_{l}$ | $X_1$ | Χ | $X_1$ | $X_1$ | $X_{l}$ | X | Х | $X_{l}$ | $X_1$ | $X_1$ | Χ | $X_1$ | X <sub>l</sub> | $X_{l}$ | $X_1$ | Х | $X_1$ | $X_1$ | Х |
| | Inclusion/Exclusion Criteria | | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | Vital Signs + body weight (+ height on Day 1 only) | | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| Ph | sical Examination | Χ | Х | Χ | | | | | | | | Χ | | | | | Χ | | | | Χ | | | | | Χ | | | Х |
| 12- | lead ECG (triplicate) | Х | Х | | | | | | | | | Χ | | | | | Х | | | | Χ | | | | | Χ | | | X |
| MR | I (liver/spleen) | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> | | | |
| Ecl | ocardiography | X | | | | | | | | | | | | | | | $X^k$ | | | | | | | | | $X^k$ | | | |
| | Chemistry Panel | Х | Х | Χ | | | Х | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Х | | Х | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х |
| | Serum Lipid Panel | Χ | Χ | Χ | | | Χ | | Χ | | Χ | Χ | | | | Χ | Х | | | | Χ | | | | Χ | Χ | | | Х |
| ی | Coagulation (aPTT, PT, INR) | Х | Χ | | | | | | Χ | | | Χ | | | | | Х | | | | Χ | | | | | X | | | |
| (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | X <sup>n</sup> | $X^{n}$ | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Ήa | Sedimentation Rate | | | Χ | | | | | | | | Χ | | | | | Х | | | | | | | | | Χ | | | Х |
| | Complement (C5a, Bb) | | | Χ | | | | | | | | Χ | | | | | Х | | | | | | | | | Χ | | | Х |
| Draw | Plasma PK - Volanesorsen | | | Χ <sup>I</sup> | Χ | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ | | | Χ |
| ] p | Anti-Volanesorsen Antibodies | | | Χ | | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Χ | | | Χ |
| Blood | FSH (women only, if applicable) | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| В | Serum Pregnancy Test <sup>d</sup> | X | Χ | | | | Χ | | Χ | | | Χ | | Χ | | | Χ | | Χ | | Χ | | Χ | | | Χ | | Χ | Χ |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | | Χ | | | | | Х | | | X | | | | | Х | | | | | | | | | Х | | | Х |
| | Troponin I° | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |

## Appendix A Schedule of Procedures Continued

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | T | reatm | ent Pe | riod | | | | | | | | | | | Treatr<br>Ilow-u | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | -2 to - | w | /k | Wk | Wk | Wk | Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| Study Week | -8 to -2 | 1 | | 1 2.5 | | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | Х | $\mathbf{X}^{m}$ | | | Х | | Х | | | X <sup>m</sup> | | $X^{m}$ | | | X <sup>m</sup> | | $\mathbf{X}^{m}$ | | $X^{m}$ | | X <sup>m</sup> | | | X <sup>m</sup> | | X <sup>m</sup> | $X^{m}$ |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> | | | |
| Genetic testing for FCS<br>diagnosis (if not available in<br>medical history) <sup>g</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC<br>Injection | | | Х | | Х | Х | х | Х | х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | х | Х | Х | Х | х | Х | | | |
| Symptom Diary (weekly) | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life<br>Assessment(s) | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Food/Drink Diary (quarterly)h | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | Х | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | Х | Х |
| Adverse Events | Х | Х | Х | | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х | Х |
| Concomitant Medication | Х | Х | Χ | | Χ | Х | Х | Χ | Х | Χ | Х | Х | Х | Χ | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х |

- Screening (Group 3) and Qualification procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. In the event of any platelet count less than 50,000/mm³ or a rate of decline ≥ 50% between two consecutive assessments, irrespective of the platelet level, then dosing of a patient with Study Drug (ISIS 304801 or placebo) will be stopped permanently. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor

#### Appendix A Schedule of Procedures Continued

#### Legend Text Continued

- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)
- n HbA1c only
- All abnormal troponin samples will be rerun at the central laboratory and also analyzed for CK-MB

# **Appendix B** List of Laboratory Analytes

#### Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | <u>Coagulation</u> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| <ul> <li>Sodium</li> <li>Potassium</li> <li>Chloride</li> <li>Bicarbonate</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>Phosphorus</li> <li>Glucose</li> <li>BUN</li> <li>Creatinine</li> <li>Uric Acid</li> <li>Total bilirubin</li> <li>Direct (conjugated) bilirubin</li> <li>Indirect (unconjugated) bilirubin</li> <li>ALT</li> <li>AST</li> <li>Alkaline phosphatase</li> </ul> | aPTT (sec) PT (sec) INR Lipid Panel Total Cholesterol LDL-C HDL-C HDL-C Triglycerides Non-HDL-C VLDL-C apoA-1 apoB apoC-III | Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Monocytes Pharmacokinetics KImmunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>2</sup></li> </ul> Additional Measures for Expanded Urinalysis <ul> <li>Total protein (quantitative)</li> <li>Microalbumin</li> <li>β2-microglobulin</li> </ul> |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

#### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm <sup>3</sup> ;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria<br>Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine)<br>ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

A subsidiary of Isis Pharmaceuticals, Inc.

**Collaborator:** Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

#### ISIS 304801-CS7

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia **Syndrome (FCS)** 

Protocol Amendment 5 – 6 July 2016

EudraCT No: 2015-003755-21

#### ISIS 304801-CS7

# The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

## An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

## Protocol Amendment 5 – 6 July 2016

#### **Protocol History:**

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

Protocol Amendment 3: 9 May 2016

Protocol Amendment 4: 6 June 2016

#### **Sponsor:**

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010



**Protocol Amendment 5** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

## The APPROACH Open-Label Study

Volanesorsen (ISIS 304801)

An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia **Syndrome (FCS)** 

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Ph.D. **Key Sponsor Contact:** 

> 2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 6 July 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | An Open-Label Study of Volanesorsen Administered Subcutaneousle<br>Patients with Familial Chylomicronemia Syndrome (FCS) | |
| Amendment: | Amendment 5 | |
| Date: | 6 July 2016 | |
| Open-Label Study of | Volanesorsen Administered | rand the attached clinical protocol, entitled "An Subcutaneously to Patients with Familial 2016, and agree to conduct the study as |
| I agree to comply wi<br>Good Clinical Praction | | ce on Harmonization Tripartite Guideline on |
| any purpose other tha | | contained in this document will not be used for of the clinical investigation without the prior |
| Investigator's Signa | ture | <del>-</del> |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| PROTOCOL SYNOPSIS 18 STUDY DESIGN AND TREATMENT SCHEMA 24 STUDY GLOSSARY 25 1. OBJECTIVES 27 2. BACKGROUND AND RATIONALE 27 2.1 Overview of Disease 27 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): 35 Screening/Qualification 34 3.4.2 Freatment 34 3.4 PATIENT ELIGIBILITY 35 4. PATIENT ELIGIBILITY <t< th=""><th><b>DDOTO</b></th><th>COL AMENDMENT</th><th>Page</th></t<> | <b>DDOTO</b> | COL AMENDMENT | Page |
|---|---|---|---|
| STUDY DESIGN AND TREATMENT SCHEMA | | | |
| STUDY GLOSSARY 25 1. OBJECTIVES 27 2. BACKGROUND AND RATIONALE 27 2.1 Overview of Disease 27 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): 35 3.4.2 Forther Endit 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATTENT ENGLIMENT 35 4.1 Screening/Qualification 35 | | | |
| 1. OBJECTIVES 27 2. BACKGROUND AND RATIONALE 27 2.1 Overview of Disease 27 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5.1 Inclusion Criteria 36 5.2 Exclusion Crite | | | |
| 2. BACKGROUND AND RATIONALE 27 2.1 Overview of Disease 27 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) I | | | |
| 2.1 Overview of Disease 27 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.2 Froup 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.5. End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screenin | | | |
| 2.2 Therapeutic Rationale 28 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study); 34 3.4.2 Group 3 Ppgatients (did not participate in an index study); 35 3.4.2 Group 3 Ppgatients (did not participate in an index study); 35 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4.1 Screening/Qualification 35 4.2< | | | |
| 2.3 Volanesorsen 29 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 4.1 Screening/Qualification 35 4.2 Enrollment 36 5.1 In | | | |
| 2.3.1 Mechanism of Action 29 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): 35 3.4.2 Group 3 Ppgatients (did not participate in an index study): 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 | | 1 | |
| 2.3.2 Chemistry 30 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): 35 Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 | _ | | |
| 2.3.3 Preclinical Experience 31 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 5.2 Enrollment 35 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. | _ | | |
| 2.3.4 Clinical Experience 32 2.4 Rationale for Dose and Schedule of Administration 33 3.3 EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | _ | · | |
| 2.4 Rationale for Dose and Schedule of Administration 33 3.1 EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): 35 Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 3. EXPERIMENTAL PLAN 34 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | _ | • | |
| 3.1 Study Design 34 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 3.2 Number of Study Centers 34 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 3.3 Number of Patients 34 3.4 Overall Study Duration and Follow-up 34 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | 3.2 | • | |
| 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | 3.3 | • | |
| 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification 34 3.4.2 Group 3 Ppgatients (did not participate in an index study): Screening/Qualification 34 3.4.3 Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | 3.4 | Overall Study Duration and Follow-up | 34 |
| index study): Qualification | 3.4. | · | |
| Screening/Qualification 34 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | index study): Qualification | 34 |
| 3.4.3 Treatment 34 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) 1ndex Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | 3.4.2 | | |
| 3.4.4 Post-Treatment 34 3.5 End-of-Study 35 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 3.5 End-of-Study | | | |
| 3.6 Data and Safety Monitoring Board 35 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | _ | | |
| 4. PATIENT ENROLLMENT 35 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 4.1 Screening/Qualification 35 4.2 Enrollment 35 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 4.2 Enrollment .35 5. PATIENT ELIGIBILITY .36 5.1 Inclusion Criteria .36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) .37 6. STUDY PROCEDURES .40 6.1 Study Schedule .40 | | | |
| 5. PATIENT ELIGIBILITY 36 5.1 Inclusion Criteria 36 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 5.1 Inclusion Criteria | | | |
| 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients | | | |
| Index Study Roll-over Patients 37 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | | | |
| 6. STUDY PROCEDURES 40 6.1 Study Schedule 40 | 5.2 | | |
| 6.1 Study Schedule | C CTPI | • | |
| · | | | |
| | 6.1. | • | |
| 6.1.2 Screening and Qualification (Group 3) | | | |

| | 6.1. | 3 Treatment Period | 40 |
|----|------|--------------------------------------------------|----|
| | 6.1. | | |
| | 6.1. | | |
| | 6.2 | Additional Study Assessments | |
| | 6.2. | | |
| | 6.2. | · | |
| | _ | 2.2.1 Eruptive Xanthoma | |
| | 6 | 2.2.2 Lipemia Retinalis | |
| | 6.2. | 1 | |
| | 6.2. | | |
| | 6.2. | 5 MRI | 42 |
| | 6.2. | Quality of Life Assessments | 42 |
| | 6.2. | 7 Disease Symptom Diary | 42 |
| | 6.2. | 8 Diet Monitoring | 43 |
| | 6.2. | 9 Family History | 43 |
| | 6.3 | Restriction on the Lifestyle of Patients | 43 |
| | 6.3. | 1 Contraception Requirements | 43 |
| | 6.3. | 2 Other Requirements | 44 |
| 7. | ST. | UDY DRUG | 44 |
| | 7.1 | Volanesorsen Description | 44 |
| | 7.2 | Packaging and Labeling | 45 |
| | 7.3 | Study Drug Accountability | 45 |
| 8. | TR | EATMENT OF PATIENTS | 45 |
| | 8.1 | Volanesorsen Administration | 45 |
| | 8.2 | Other Protocol-Required Drugs | 45 |
| | 8.3 | Other Protocol-Required Treatment Procedures. | 46 |
| | 8.4 | Treatment Precautions | 46 |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | | |
| | 8.5. | , e | |
| | 8.5. | , | |
| | 8.5. | J 1 | |
| | 8.5. | , | |
| | 8.5. | ; · | |
| | 8.5. | 71 87 | |
| | 8.5. | | |
| | 8.5. | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | | |
| | 8.6. | 2 Stopping Rules for Renal Function Test Results | 51 |

| 8.6.3 | Stopping Rules for Platelet Count Results | 51 |
|---|---|---|
| | ustment of Dose Frequency | |
| • | continuation of Study Treatment | |
| 8.8.1 | Follow-up Visits for Early Termination from Treatment Period | |
| 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Pe | |
| | hdrawal of Patients from the Study | |
| | comitant Therapy and Procedures | |
| 8.10.1 | Concomitant Therapy | |
| 8.10.2 | Concomitant Procedures. | |
| | atment Compliance | |
| | US AND NON-SERIOUS ADVERSE EVENT REPORTING | |
| | nsor Review of Safety Information | |
| | ulatory Requirements | |
| _ | initions | |
| 9.3.1 | Adverse Event | |
| 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | |
| 9.3.3 | Serious Adverse Event (SAE) | |
| | nitoring and Recording Adverse Events | |
| 9.4.1 | Serious Adverse Events | |
| 9.4.2 | Non-Serious Adverse Events. | |
| 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | |
| 9.4.3.1 | | |
| 9.4.3.2 | | |
| 9.4.3.3 | Action Taken with Volanesorsen | 60 |
| 9.4.3.4 | Treatment Given for Adverse Event | 60 |
| 9.4.3.5 | Outcome of the Adverse Event | 60 |
| 9.4.4 | Adjudication Committees | 61 |
| 9.5 Proc | cedures for Handling Special Situations | 61 |
| 9.5.1 | Abnormalities of Laboratory Tests | |
| 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 61 |
| 9.5.3 | Dosing Errors | 62 |
| 9.5.4 | Contraception and Pregnancy | 62 |
| 10. STATIS | TICAL CONSIDERATIONS | 63 |
| 10.1 Stud | ly Endpoints | 63 |
| 10.1.1 | Efficacy Endpoints | 63 |
| 10.1.2 | Safety Endpoints | 63 |
| 10.2 Sam | ple Size | 63 |
| - | ulations | |
| | inition of Baseline | |
| 10.5 Inter | rim Analysis | 64 |

| 10.6 | Planned Methods of Analysis | 64 |
|---|---|---|
| 10.6 | • | |
| 10.6 | | |
| 10.6 | | |
| 10.6 | | |
| 1 | 0.6.4.1 Pharmacokinetic Analysis | |
| 1 | 0.6.4.2 Immunogenicity Analysis | |
| 11. IN | VESTIGATOR'S REGULATORY OBLIGATIONS | |
| 11.1 | Informed Consent | |
| 11.2 | Ethical Conduct of the Study | |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 68 |
| 11.4 | Patient Confidentiality | |
| 12. AD | OMINISTRATIVE AND LEGAL OBLIGATIONS | 68 |
| 12.1 | Protocol Amendments | |
| 12.2 | Study Termination | 69 |
| 12.3 | Study Documentation and Storage | |
| 12.4 | Study Monitoring | |
| 12.5 | Language | |
| 12.6 | Compensation for Injury | |
| 13. RE | EFERENCES | |
| | PPENDICES | |
| Apper | ndix A Schedule of Procedures | 74 |
| | ndix B List of Laboratory Analytes | 78 |
| | ndix C Pharmacokinetic Sampling Schedule | |
| | ndix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities. | |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | |
| Table 2 | Actions in Patients With Low Platelet Count | 53 |
| Table 3 Expected Event for the Protocol Defined Population by Preferred Term and | | 57 |
| | the Expected Incidence | 37 |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | _ |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volanesorsen is shown | |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 32 |

Protocol


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 5

**Amendment Date:** 6 July 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 4 dated 6 June 2016:

1. To enroll FCS patients in this open label study who did not participate in the ISIS 304801–CS6 or ISIS 304801–CS16 index studies.

For clarity, the protocol now specifies 3 patient groups, with assignment based on prior involvement in index studies of ISIS 304801:

Group 1: ISIS 304801-CS6 (index study) rollover FCS patients

Group 2: ISIS 304801-CS16 (index study) rollover FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

- 2. To remove language that indicates that lipoprotein lipase (LPL) activity can be measured if needed for study qualification for patients in Groups 2 and 3.
- 3. To add language to indicate that a second Study Drug rechallenge will not be allowed following a platelet count decrease below 75,000/mm<sup>3</sup>.
- 4. To provide clarifications to the platelet safety monitoring rules in Table 2.
- 5. To add language to indicate that patients who discontinue early from Study Drug, or the study, should be followed as per the platelet monitoring rules shown in Table 2 for the first 6 weeks after discontinuing Study Drug and the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.

Minor changes (not included in the list of changes below) have been made throughout the protocol to correct errors and/or to improve the overall clarity of the original protocol but these changes do not impact subject safety, exposure, or the overall study design.

The following table provides a summary list of major changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis: Study Population Continued 5.1 Inclusion Criteria Continued | <ul> <li>Is: Continued</li> <li>3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.</li> <li>Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> </li> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label study</li> </ul> </li> </ul> | To define the inclusion criteria for each Group of patients LPL removed to avoid the production of heparin induced anti-platelet antibodies Continued |
| Protocol Synopsis:<br>Study Population<br>5.2 Exclusion Criteria | <ul> <li>Was: <ul> <li>Exclusion Criteria</li> </ul> </li> <li>Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study</li> </ul> <li>Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)</li> <li>Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients</li> <li>Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study</li> <li>Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)</li> <li>Exclusion Criteria for Group 3 (patients who did not participate in an index study)</li> <li>Diabetes mellitus with any of the following: <ul> <li>Newly diagnosed within 12 weeks of screening</li> <li>Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of ± 10 units of insulin])</li> <li>Anticipated need to change dose or type of medication during the treatment period of the Study [with the exception of ± 10 units of insulin]</li> <li>Current use of GLP-1 agonists</li> </ul> </li> | To define the exclusion criteria for each Group of patients and to make the eligibility criteria for the Group 3 patients consistent with those for the Group 1 index study patients |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis:<br>Study Population | <u>Is:</u> Continued Exclusion Criteria for Group 3 (patients who did not participate in | To define the exclusion |
| Continued | an index study) | criteria for each |
| 5.2 Exclusion Criteria Continued | Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome | Group of patients and to make the |
| | Active pancreatitis within 4 weeks prior to screening | eligibility criteria |
| | History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening | for the Group 3<br>patients<br>consistent with<br>those for the<br>Group 1 index |
| | 5. Any of the following laboratory values at Screening | study patients |
| | a. Hepatic: | Continued |
| | <ul> <li>Total bilirubin &gt; upper limit of normal (ULN), unless prior<br/>diagnosis and documentation of Gilbert's syndrome in<br/>which case total bilirubin must be ≤ 3 mg/dL</li> </ul> | |
| | <ul> <li>ALT &gt; 2.0 x ULN</li> </ul> | |
| | <ul> <li>AST &gt; 2.0 x ULN</li> </ul> | |
| | b. Renal: | |
| | <ul> <li>Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of &lt; 500 mg/24 hrs</li> </ul> | |
| | <ul> <li>Persistently positive (2 out of 3 consecutive tests ≥ trace<br/>positive) for blood on urine dipstick. In the event of a<br/>positive test eligibility may be confirmed with urine<br/>microscopy showing ≤ 5 red blood cells per high power<br/>field</li> </ul> | |
| | <ul> <li>Estimated creatinine clearance calculated according to<br/>the formula of Cockcroft and Gault &lt; 50 mL/min (MDRD<br/>or CKD-EPI formulas can be used instead of Cockcroft-<br/>Gault for estimation of GFR in patients with low body<br/>weight after discussion with Sponsor Medical Monitor)</li> </ul> | |
| | c. Cardiac Troponin I > ULN at Screening | |
| | d. LDL-C > 130 mg/dL at Screening | |
| | Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion | |
| | 6. Uncontrolled hypertension (BP > 160/100 mm Hg) | |
| | History of bleeding diathesis or coagulopathy or clinically-<br>significant abnormality in coagulation parameters at Screening | |
| | 8. History of heart failure with NYHA greater than Class II | |
| | Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1 | |
| | Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B | |
| | Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma <i>in situ</i> of the cervix that has been successfully treated | |
| | 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer | |
| | 13. Unwilling to comply with lifestyle requirements (Section 6.3) | |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis: Study Population Continued 5.2 Exclusion Criteria Continued | Is: Continued Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued 14. Use of any of the following: a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period f. Glybera gene therapy within 2 years prior to screening g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period i. Plasma apheresis within 4 weeks prior to screening or planned during the study j. Prior exposure to ISIS 304801 k. Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion) 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening | Rationale To define the exclusion criteria for each Group of patients and to make the eligibility criteria for the Group 3 patients consistent with those for the Group 1 index study patients Continued |
| | <ul> <li>16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)</li> <li>17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study</li> </ul> | |
| Protocol Synopsis:<br>Study Visit Schedule<br>and Procedures<br>3.4 Overall Study<br>Duration and Follow-up<br>Appendix A | Was: The study for an individual patient will generally consist of the following periods: A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A. A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection A 13-week post-treatment evaluation period | To distinguish the Screening/ Qualification period for patients who participated in an index study from those who did not |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Protocol Synopsis: Study Visit Schedule and Procedures Continued 3.4 Overall Study Duration and Follow-up Continued Appendix A Continued | <ul> <li>Is: Continued The study for an individual patient will generally consist of the following periods: <ul> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.</li> </ul> </li> <li>Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor</li> </ul> | To distinguish the Screening/ Qualification period for patients who participated in an index study from those who did not Continued |
| | <ul> <li>approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A.</li> <li>All patients: <ul> <li>A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection</li> <li>A 13-week post-treatment evaluation period</li> </ul> </li> </ul> | |
| 4.1 Screening / Qualification | Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used | To define the enrollment criteria for patients who did not participate in an index study |
| 6.1.2 Screening and Qualification (Group 3) | Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes | To define the<br>Screening and<br>Qualification<br>procedures for<br>patients who did<br>not participate in<br>an index study |
| 8.6.3 Stopping Rules<br>for Platelet Count<br>Results | Was: If after the first dosing rechallenge the platelet count again falls below 75,000/mm³, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm³. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be reexamined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above. If after the second rechallenge the platelet count falls below 75,000/mm³ and is subsequently confirmed (see Section 8.5), dosing with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor. | Text was removed as a second Study Drug rechallenge will not be allowed following a platelet count decrease below 75,000/mm <sup>3</sup> |
| Protocol Section | Description of Change | | | Rationale |
|---|---|---|---|---|
| 8.6.3 Stopping Rules for Platelet Count Results <i>Continued</i> | Is: If after the first dosing rechallenge the platelet count again falls below 75,000/mm³, then dosing of the patient with Study Drug will be stopped permanently. | | | Text was removed as a second Study Drug rechallenge will not be allowed following a platelet count decrease below 75,000/mm <sup>3</sup> |
| 8.6.3 Stopping Rules for Platelet Count Results | Platelet Count on Rx | Drug Dose | Monitoring | To provide clarification to the platelet |
| Table 2 Actions in Patients with Low | Normal range,<br>> 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks | safety<br>monitoring rules |
| Platelet Count | 100K-<br>140K/mm <sup>3</sup> | No action | Closer observation<br>Monitor every<br>1-week <u>until</u><br><u>stable*</u> | Note: Changes<br>are reflected as<br>bold underlined |
| | 75K-100K/mm <sup>3</sup> | Permanently reduce<br>dose frequency to<br>300mg every 2 weeks<br>or reduce dose to<br>150 mg weekly | Closer observation<br>Monitor every<br>1-week | text |
| | 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. Dose pause When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication | |

| Protocol Section | | Description of Chang | е | Rationale |
|---|---|---|---|---|
| 8.6.3 Stopping Rules for Platelet Count Results | Platelet Count on Rx | Drug Dose | Monitoring | To provide clarification to the platelet |
| Table 2 Actions in Patients with Low Platelet Count Continued | 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2 3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/an ticoagulant medication while platelet count < 50K/mm³ if possible | safety monitoring rules Note: Changes are reflected as bold underlined text Continued |
| | < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/an ticoagulant medication while platelet count < 50K/mm³ if possible | |
| | ** Recovery in plate of high dose stee thrombocytoper Dexamethasone | telet count may be acceler<br>roids. Treatment guideling<br>iia (Provan et al. 2010) rec<br>e 40 mg daily for 4 days ev | rated by administration es for immune commend very 2-4 weeks for | |
| | or Methylpredni | lnis(oI)one 0.5-2 mg/kg/d f<br>solone 30 mg/kg/day for 7<br>h oral steroids after methyl | days (note: may require | |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| 8.8.1 Follow-up Visits for Early Termination from Treatment Period | Was: Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 2, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits. | To provide guidance to the platelet safety monitoring rules for patients that discontinue early from the Treatment Period |
| | Is: Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits. | |
| 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period | Was: The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study. Is: The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor medical monitor and > 100,000/mm³), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study. | To provide guidance to the platelet safety monitoring rules for patients that discontinue early from the Post-Treatment Follow-up Period |

# PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of dosing and extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center open-label study of: |
| | Group 1: ISIS 304801-CS6 (index study) roll over FCS patients |
| | Group 2: ISIS 304801-CS16 (index study) roll over FCS patients |
| | Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies |
| | All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. |
| | Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1<br/>Hyperlipoproteinemia) by documentation of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>c. Group 2: Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for<br/>the ISIS 304801-CS16 index study<br/>Group 3: Fasting TG ≥ 750 mg/dL at Screening for this open-label<br/>study</li> </ul> |
| | 4. Able and willing to participate in a 65-week study |

## Study Population Continued

Protocol

Inclusion Criteria: Continued

- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral ophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3)

 $\underline{\text{Exclusion Criteria for Group 3}} \text{ (patients who did not participate in an index study)}$ 

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b. HbA1c ≥ 9.0% at Screening
  - Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of ± 10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of ± 10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening

## Study Population Continued

Protocol

Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued

- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening
- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT > 2.0 x ULN
    - AST > 2.0 x ULN
  - b. Renal:
    - Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs</li>
    - Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
    - Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
  - c. Cardiac Troponin I > ULN at Screening
  - d. LDL-C > 130 mg/dL at Screening
  - e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
- Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer

# PROTOCOL SYNOPSIS Continued

| Study Population Continued | Exclusion Criteria for Group 3 (patients who did not participate in an index study) Continued |
|---|---|
| | 13. Unwilling to comply with lifestyle requirements (Section 6.3) |
| | 14. Use of any of the following: |
| | a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless<br>on a stable dose for at least 3 months prior to screening and dose and<br>regimen expected to remain constant during the treatment period.<br>Patients taking OTC omega-3 fatty acids should make every effort to<br>remain on the same brand throughout the study |
| | Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening |
| | c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor |
| | <ul> <li>d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study</li> </ul> |
| | Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period |
| | f. Glybera gene therapy within 2 years prior to screening |
| | g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and<br>apixaban) unless on a stable dose for at least 4 weeks prior to<br>screening and regular clinical monitoring is performed |
| | h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period |
| | <ul> <li>Plasma apheresis within 4 weeks prior to screening or planned during<br/>the study</li> </ul> |
| | j. Prior exposure to ISIS 304801 |
| | <ul> <li>k. Any other medication unless stable at least 4 weeks prior to screening<br/>(Occasional or intermittent use of over-the-counter medications will be<br/>allowed at Investigator's discretion)</li> </ul> |
| | 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening |
| | 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo) |
| | 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |

| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6 and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies (Section 2.4) which included a subset of patients with FCS. The same dose of 300 mg once weekly will be used in this open-label study of FCS patients. |
|---|---|
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>Group 1 and 2 patients (participated in ISIS 304801-CS6 or<br/>ISIS 304801-CS16 index study): A qualification period of up to<br/>2 weeks (unless approved by the Sponsor). Please refer to<br/>Section 4.1 and Appendix A</li> </ul> |
| | Group 3 patients (did not participate in an index study): An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening). Please refer to Section 6.1.2 and Appendix A |
| | All patients: |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

| de<br>ev<br>M/ | verall safety and tolerability of volanesorsen will be assessed by etermining the incidence and severity of adverse and serious adverse vents (including independently adjudicated events of acute pancreatitis and |
|---|---|
| | ACE), withdrawals due to adverse events, and changes in laboratory and her safety parameters. |
| Planned Analyses Sa | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| Ef | ficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | <ul> <li>Percent change from baseline in fasting total apolipoprotein C-III<br/>(apoC-III)</li> </ul> |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| vo<br>po<br>of<br>vo<br>pa | asma samples will be taken from all patients for the measurement of blanesorsen as follows: trough levels (pre-dose) throughout treatment and ost-treatment levels during the post-treatment follow-up period. In a subset patients, more frequent assessment of plasma concentrations of blanesorsen will be performed to determine volanesorsen pharmacokinetic arameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations No | o sample size calculations were performed as this is an open-label study. |
| Sponsor lor | nis Pharmaceuticals, Inc. |
| Collaborator Ak | ccea Therapeutics |

## STUDY DESIGN AND TREATMENT SCHEMA



# STUDY GLOSSARY

| STUDY GLOSSARY | |
|---|---|
| Abbreviation/Acronym | <u>Definition</u> |
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| ароЕ | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event Statistical Analysis Plan SAP

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of dosing and extended dosing with volunesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

## 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

## 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

## 2.3.3 Preclinical Experience

Protocol

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

## 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open-label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

## 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

## 3.1 Study Design

This is an open-label study of:

Group 1: ISIS 304801-CS6 (index study) roll over FCS patients

Group 2: ISIS 304801-CS16 (index study) roll over FCS patients

Group 3: FCS patients who did not participate in the ISIS 304801-CS6 or ISIS 304801-CS16 index studies

Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

## 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

## 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

# 3.4.1 Group 1 and 2 Patients (participated in ISIS 304801-CS6 or ISIS 304801-CS16 index study): Qualification

A period of up to 2 weeks (unless approved by the Sponsor) is given to complete qualification assessments outlined in the Schedule of Procedures. Please refer to Section 4.1 and Appendix A.

## 3.4.2 Group 3 Patients (did not participate in an index study): Screening/Qualification

An up to 8-week screening and qualification period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening. Please refer to Section 6.1.2 and Appendix A.

#### 3.4.3 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule of Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.4 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

#### 3.5 End-of-Study

The End-of-Study is last patient, last visit.

## 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

## 4.1 Screening/Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open-label study are performed.

Groups 1 and 2 (Qualification): During the qualification period, the eligibility of the patient to enroll in the open-label study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

Group 3 (Screening and Qualification): At the time of consent, the patient will be considered enrolled into the study and will be assigned a unique screening number before any study procedures, including screening procedures, are performed. At the time of enrollment, patients will be assigned a unique patient identification number. This number will be used to identify the patient throughout the trial and must be used on all study documentation related to that patient. The screening number and patient identification number must remain constant throughout the entire trial. In the event the patient is re-consented and re-screened the patient must be given a new screening number. Screening numbers and patient identification numbers, once assigned, will not be re-used.

#### 4.2 Enrollment

Patients will be enrolled into the treatment phase of the study after all Screening (Group3) and qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Groups 1 and 2: Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement.

Groups 2 and 3: Patients must also meet the following criteria in order to enter into the open-label Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
- c. Group 2: Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 index study
  - Group 3: Fasting  $TG \ge 750 \text{ mg/dL}$  at Screening for this open-label study
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

- b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

# 5.2 Exclusion Criteria for Group 1 (ISIS 304801-CS6) and Group 2 (ISIS 304801-CS16) Index Study Roll-over Patients

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

## Exclusion Criteria for Group 3 (patients who did not participate in an index study)

- 1. Diabetes mellitus with any of the following:
  - a. Newly diagnosed within 12 weeks of screening
  - b.  $HbA1c \ge 9.0\%$  at Screening
  - c. Recent change in anti-diabetic pharmacotherapy (change in dosage or addition of new medication within 12 weeks of screening [with the exception of  $\pm$  10 units of insulin])
  - d. Anticipated need to change dose or type of medication during the treatment period of the Study (with the exception of  $\pm$  10 units of insulin)
  - e. Current use of GLP-1 agonists
- 2. Severe hypertriglyceridemia other than due to familial chylomicronemia syndrome
- 3. Active pancreatitis within 4 weeks prior to screening
- 4. History within 6 months of screening of acute or unstable cardiac ischemia (myocardial infarction, acute coronary syndrome, new onset angina), stroke, transient ischemic attack or unstable congestive cardiac failure requiring a change in medication or major surgery within 3 months of screening

- 5. Any of the following laboratory values at Screening
  - a. Hepatic:
    - Total bilirubin > upper limit of normal (ULN), unless prior diagnosis and documentation of Gilbert's syndrome in which case total bilirubin must be ≤ 3 mg/dL
    - ALT  $> 2.0 \times ULN$
    - AST  $> 2.0 \times ULN$

#### b. Renal:

- Persistently positive (2 out of 3 consecutive tests ≥ 1+) for protein on urine dipstick. In the event of a positive test eligibility may be confirmed by a quantitative total urine protein measurement of < 500 mg/24 hrs
- Persistently positive (2 out of 3 consecutive tests ≥ trace positive) for blood on urine dipstick. In the event of a positive test eligibility may be confirmed with urine microscopy showing ≤ 5 red blood cells per high power field
- Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 50 mL/min (MDRD or CKD-EPI formulas can be used instead of Cockcroft-Gault for estimation of GFR in patients with low body weight after discussion with Sponsor Medical Monitor)
- c. Cardiac Troponin I > ULN at Screening
- d. LDL-C > 130 mg/dL at Screening
- e. Any other laboratory abnormalities which, in the opinion of the Investigator or the Sponsor, would make the patient unsuitable for inclusion
- 6. Uncontrolled hypertension (BP > 160/100 mm Hg)
- 7. History of bleeding diathesis or coagulopathy or clinically-significant abnormality in coagulation parameters at Screening
- 8. History of heart failure with NYHA greater than Class II
- 9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
- 10. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
- 11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma *in situ* of the cervix that has been successfully treated

- 12. Treatment with another investigational drug, biological agent, or device within 1-month of screening, or 5 half-lives of investigational agent, whichever is longer
- 13. Unwilling to comply with lifestyle requirements (Section 6.3)
- 14. Use of any of the following:
  - a. Statins, omega-3 fatty acids (prescription and OTC), or fibrates unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain constant during the treatment period. Patients taking OTC omega-3 fatty acids should make every effort to remain on the same brand throughout the study
  - b. Nicotinic acid or derivatives of nicotinic acid within 4 weeks prior to screening
  - c. Systemic corticosteroids or anabolic steroids within 6 weeks prior to screening unless approved by the Sponsor Medical Monitor
  - d. Atypical antipsychotic medications (e.g., olanzapine and clozapine) unless on a stable dose for at least 3 months prior to screening and dose and regimen expected to remain stable throughout the study
  - e. Antihypertensive medication unless on a stable dose for at least 4 weeks prior to screening and dose and regimen expected to remain constant during the treatment period
  - f. Glybera gene therapy within 2 years prior to screening
  - g. Oral anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, and apixaban) unless on a stable dose for at least 4 weeks prior to screening and regular clinical monitoring is performed
  - h. Tamoxifen, estrogens or progestins unless on a stable dose for at least 4 months prior to screening and dose and regimen expected to remain constant during the treatment period
  - i. Plasma apheresis within 4 weeks prior to screening or planned during the study
  - j. Prior exposure to ISIS 304801
  - k. Any other medication unless stable at least 4 weeks prior to screening (Occasional or intermittent use of over-the-counter medications will be allowed at Investigator's discretion)
- 15. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening
- 16. Known hypersensitivity to any of the excipients of the Study Drug (ISIS 304801 or placebo)
- 17. Have any other conditions, which, in the opinion of the Investigator or the Sponsor would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

#### 6. STUDY PROCEDURES

## 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

## 6.1.1 Qualification (Groups 1 and 2)

Please refer to Section 4.1 and Appendix A.

## 6.1.2 Screening and Qualification (Group 3)

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. An 8-week period, including a diet stabilization period of at least 6 weeks (screening and diet stabilization period may be reduced, per Sponsor approval, if the patient is following a diet for optimal control of TGs and disease management prior to screening) is given to perform the screening evaluations. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal screening results may be retested for review by the Study Medical Monitor for eligibility purposes

## 6.1.3 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the open-label study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, and 50 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

## 6.1.4 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.5 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 4 Study Center visits on Weeks 54, 56, and 58 (which may be conducted by a home healthcare nurse), and Week 65 as outlined in the Schedule of Procedures in Appendix A.

## 6.2 Additional Study Assessments

## 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

## 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should

always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

## 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

## 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

## 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

## 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

## 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

## 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

## 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

## 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

## 6.3 Restriction on the Lifestyle of Patients

## 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent\* or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use

effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

## For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

\* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

## 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

## 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

## Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

## 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

## 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or ISIS 304801-CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

## 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

## 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

## 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

## 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3.

Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

## 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

## 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

## 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

## 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

## 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level

 $\leq$  70 mg/dL ( $\leq$  3.9 mmol/L). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

## 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1-week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

## 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:
- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 2 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 25,000/mm<sup>3</sup>, or a platelet count less than 75,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one

0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (**note:** may require continuation with oral steroids after methylprednisolone).

In the event of a platelet count less than 75,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to> 100,000/mm<sup>3</sup>. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient with Study Drug will be stopped permanently.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

#### <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

## <u>Definition of Clinically-Relevant, Non-Major Bleeding Events</u> (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every 1-week until stable* |
| 75K-100K/mm <sup>3</sup> | Permanently reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every 1-week |
| 50K-75K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended** Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

<sup>\*</sup> At least 3 consecutive values measured weekly that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>

#### 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 2 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment

<sup>\*\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methyl prednisolone)

schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### 8.8 Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be followed as per the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug. Patients should also be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 50, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the Schedule of Procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to follow the platelet monitoring rules shown in Table 2 in Section 8.6.3 for the first 6 weeks after discontinuing Study Drug. Following this period, if the platelet count is stable (at least 3 consecutive values that are stable as determined by the Sponsor Medical Monitor and > 100,000/mm<sup>3</sup>), the next platelet count should be taken within at least 6 weeks so that patients are monitored for at least 12 weeks after discontinuing Study Drug.

Patients should also be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volanesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 3 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's

follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen, e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- Mild: The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- **Persists (as non-serious AE):** Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

## 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 50 (Day 344) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### 10.2 Sample Size

No sample size calculations were performed as this is an open-label study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

<u>Safety Set</u>: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient in Groups 1 and 2: Group 1 (ISIS 304801-CS6) or Group 2 (ISIS 304801-CS16) index study baseline and the baseline in this open-label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the open-label study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this open-label study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification for Group 1 and 2 patients by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open-label study from the intensive PK subgroup, following a single-dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies (Group 1 and 2 patients). On Week 1 Day 1 of the open-label study, patients who received placebo in the index study (and all patients in Group 3) will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index studies had been on volunesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL<sub>0-24hr</sub> /F<sub>0-24hr</sub>) will be calculated from  $CL_{0-24hr}/F_{0-24hr} = Actual Dose/AUC_{0-24hr}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be

listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 (Groups 1 and 2) and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject - peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 (Groups 1 and 2) and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies of pre-study documentation and all correspondence to and from the IEC/IRB and the Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia. N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

# ${\bf Appendix} \; {\bf A} \quad {\bf Schedule} \; {\bf of} \; {\bf Procedures}$

| | Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | | Γreatr | nent l | Period | I | | | | | | | | | | Trea | tment<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0.4- | | <i>n</i> - | \A/I- | Wk | \A/I- | \A/I- | \A/I- | Mor | nth 3 | Wk | \A/I- | Wk | Mor | nth 6 | Wk | \A/I- | Wk | VA/Is | Wk<br>40 | \A/I- | Wk | Мо | nth 12 | Wk | \A/I- | \A/I- |
| | Study Week | -8 to -2 | -2 to -<br>1 | <b>W</b> | | 2.5 | 4 | Wk<br>6 | Wk<br>8 | Wk<br>10 | Wk<br>12 | Wk<br>13 | 15<br>&<br>17 | Wk<br>19 | 21<br>&<br>23 | Wk<br>25 | Wk<br>26 | 28<br>&<br>30 | & 32 | 34<br>&<br>36 | Wk<br>38 | 40<br>&<br>42 | Wk<br>44 | 46<br>&<br>48 | Wk<br>50 | Wk 52<br>or ET | 54<br>&<br>56 | Wk<br>58 | Wk<br>65 |
| | Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Inf | rmed Consent | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Οι | patient Visit | Х | Х | Х | $\mathbf{X}^{\mathbf{j}}$ | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | Х | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | $X^{j}$ | Х | $X^{j}$ | X <sup>j</sup> | $X^{j}$ | Χ | $X^{j}$ | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | Х | X <sup>j</sup> | $X^{j}$ | Х |
| Inc | usion/Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | al Signs + body weight<br>neight on Day 1 only) | Х | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| Ph | sical Examination | Х | | Х | | | | | | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| 12 | lead ECG (triplicate) | Х | | | | | | | | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| MF | I (liver/spleen) | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> | | | |
| Ec | nocardiography | Х | | | | | | | | | | | | | | | X <sup>k</sup> | | | | | | | | | X <sup>k</sup> | | | |
| | Chemistry Panel | Х | Х | Х | | | Х | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | | Х | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | Χ | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ |
| | Serum Lipid Panel | Х | Χ | Χ | | | Х | | Х | | Χ | Х | | | | Х | Χ | | | | Х | | | | Х | Х | | | Χ |
| 3)c | Coagulation (aPTT, PT, INR) | Х | PG | | | | | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | |
| (Fasting) <sup>6</sup> | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | | | х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| <u>&gt;</u> | Sedimentation Rate | | | Х | | | | | | | | Х | | | | | Χ | | | | | | | | | Х | | | Χ |
| Draw | Complement (C5a, Bb) | | | Χ | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Χ |
| l pc | Plasma PK - Volanesorsen | | | X | Χ | | Χ | | Χ | | | Χ | | | | | Χ | | | | Χ | | | | | Х | | <u> </u> | Χ |
| Blood | Anti-Volanesorsen Antibodies | | | Χ | _ | | Χ | | Х | | | Х | | | | | Χ | | | | Х | | | | | Х | | <u> </u> | Χ |
| | FSH (women only, if applicable) | Х | | | <u> </u> | | | | | | | | | | | | | | | | | | | | | | | — | |
| | Serum Pregnancy Test <sup>d</sup> | Х | Х | | | | Χ | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | | Х | Χ |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | | Х | | | | | Х | | | Х | | | | | Х | | | | | | | | | Х | | | Х |

# Appendix A Schedule of Procedures Continued

| Study Period | Screen/<br>Run In <sup>a</sup> | Qual <sup>a</sup> | | | | | | | | | | | | Treatn | nent P | eriod | | | | | | | | | | Tre | Post<br>atme<br>low-u | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 245 | | n. | \A/I+ | \A/I+ | \A/I+ | \A/I+ | \A/I+ | Mor | nth 3 | Wk | \A/I+ | Wk | Mor | nth 6 | Wk | \A/I+ | Wk<br>34 | Wk | Wk | \A/I+ | Wk | Мо | nth 12 | Wk | \A/I+ | \A/I+ |
| Study Week | -8 to -2 | -2 to -<br>1 | N. | | 2.5 | 4 | Wk<br>6 | 8<br>8 | 10 | Wk<br>12 | Wk<br>13 | 15<br>&<br>17 | Wk<br>19 | 21<br>&<br>23 | Wk<br>25 | Wk<br>26 | 28<br>&<br>30 | Wk<br>32 | | 38 | 40<br>&<br>42 | Wk<br>44 | 46<br>&<br>48 | Wk<br>50 | Wk 52<br>or ET | 54<br>&<br>56 | 58 | k Wk<br>8 65 |
| Study Day | -56 to -<br>15 | -14 to<br>-7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | Х | X <sup>m</sup> | | | Х | | Х | | | X <sup>m</sup> | | X | | | X <sup>m</sup> | | X | | X | | X <sup>m</sup> | | | X <sup>m</sup> | | X | X |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | X <sup>k</sup> | | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC<br>Injection | | | х | | х | Х | х | х | х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | х | Х | Х | Х | Х | Х | | | |
| Symptom Diary (weekly) | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life<br>Assessment(s) | | | х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Food/Drink Diary (quarterly) <sup>h</sup> | | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Diet/Alcohol Counseling <sup>i</sup> | Х | Х | Х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | Х | Х |
| Adverse Events | Х | Х | Х | | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant Medication | Х | Х | Χ | | Х | Χ | Х | Х | Х | Χ | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ |

a Screening and Qualification (Group 3) procedures performed (Please refer to Sections 3.4, 4.1, and 6.1.2)

b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm³. Any case of a platelet count < 50,000/mm³ should be reported in an expedited fashion to the Sponsor

## **Appendix A** Schedule of Procedures Continued

#### Legend Text Continued

- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study qualification (Group 2 [ISIS 304801-CS16 rollover patients] and Group 3); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- i To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- j Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- k A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- Full or abbreviated PK profile (see Appendix C)
- m Expanded urinalysis (see Appendix B)

Amendment 5 6 July 2016

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| | Hematology | Uringlysis |
|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Potasium P | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | Urinalysis Color Appearance Specific gravity pH Protein Blood Ketones Urobilinogen Glucose Bilirubin Leukocyte esterase Nitrate Microscopic examination <sup>2</sup> Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin β2-microglobulin |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

# Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

# PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase >ULN - 3.0 x ULN increased | | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm <sup>3</sup> ;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria<br>Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine)<br>ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

A subsidiary of Isis Pharmaceuticals, Inc. **Collaborator:** Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

# ISIS 304801-CS7

# The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia **Syndrome (FCS)** 

Protocol Amendment 4 –6 June 2016

EudraCT No: 2015-003755-21
### ISIS 304801-CS7

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

# An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

#### Protocol Amendment 4 – 6 June 2016

#### **Protocol History:**

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

Protocol Amendment 3: 9 May 2016

#### **Sponsor:**

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010



M.D., M.B.A.

### **Ionis Protocol Number: ISIS 304801-CS7**

#### **Protocol Amendment 4**

**EudraCT No: 2015-003755-21** 

**Clinical Phase: 3** 

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

## An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 6 June 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

Investigator's Name (please print)

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 |
|---|---|
| Protocol Title: An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) | |
| Amendment: | Amendment 4 |
| Date: | 6 June 2016 |
| Open-Label Extension Familial Chylomicron as described herein. I agree to comply wit Good Clinical Praction I agree to ensure that any purpose other that | that I have read and understand the attached clinical protocol, entitled "An in Study of Volanesorsen Administered Subcutaneously to Patients with memia Syndrome (FCS)", dated 6 June 2016, and agree to conduct the study the International Conference on Harmonization Tripartite Guideline on the (E6). The confidential information contained in this document will not be used for an the evaluation or conduct of the clinical investigation without the prior mis Pharmaceuticals, Inc. |
| Investigator's Signat | ture |

Date (DD Month YYYY)

### **TABLE OF CONTENTS**

| | | Page |
|------|--------------------------------------|------|
| | OCOL AMENDMENT | |
| | OCOL SYNOPSIS | |
| | Y DESIGN AND TREATMENT SCHEMA | |
| | Y GLOSSARY | |
| | BJECTIVES | |
| | ACKGROUND AND RATIONALE | |
| 2.1 | Overview of Disease | |
| 2.2 | Therapeutic Rationale | |
| 2.3 | Volanesorsen | |
| | 3.1 Mechanism of Action | |
| | 3.2 Chemistry | |
| 2 | 3.3 Preclinical Experience | |
| 2 | 3.4 Clinical Experience | |
| 2.4 | | |
| 3. E | XPERIMENTAL PLAN | 26 |
| 3.1 | Study Design | 26 |
| 3.2 | Number of Study Centers | 26 |
| 3.3 | Number of Patients | 26 |
| 3.4 | Overall Study Duration and Follow-up | 26 |
| 3.4 | 4.1 Qualification | 26 |
| 3.4 | 4.2 Treatment | 26 |
| 3.4 | 4.3 Post-Treatment | 26 |
| 3.5 | End of Study | 26 |
| 3.6 | Data and Safety Monitoring Board | 27 |
| 4. P | ATIENT ENROLLMENT | 27 |
| 4.1 | Qualification | 27 |
| 4.2 | Enrollment | 27 |
| 5. P | ATIENT ELIGIBILITY | 27 |
| 5.1 | Inclusion Criteria | 27 |
| 5.2 | Exclusion Criteria | 28 |
| 6. S | TUDY PROCEDURES | |
| 6.1 | Study Schedule | |
| 6. | 1.1 Qualification | 29 |
| 6. | 1.2 Treatment Period | |
| | 1.3 Pharmacokinetic (PK) Subgroup | |
| | 1.4 Post-Treatment Period | |
| 6.2 | Additional Study Assessments | |
| | 2.1 Laboratory Assessments | |

| | 6.2.2 | Physical Exams and Vital Signs | 30 |
|---|---|---|---|
| | 6. | 2.2.1 Eruptive Xanthoma | 30 |
| | 6. | 2.2.2 Lipemia Retinalis | 31 |
| | 6.2.3 | B Echocardiography | 31 |
| | 6.2.4 | 4 ECG | 31 |
| | 6.2. | 5 MRI | 31 |
| | 6.2. | Quality of Life Assessments | 31 |
| | 6.2. | 7 Disease Symptom Diary | 31 |
| | 6.2. | B Diet Monitoring | 31 |
| | 6.2.9 | 9 Family History | 32 |
| | 6.2. | 10 Lipoprotein Lipase Activity Sample Collection | 32 |
| | 6.3 | Restriction on the Lifestyle of Patients. | 32 |
| | 6.3. | Contraception Requirements | 32 |
| | 6.3.2 | 2 Other Requirements | 33 |
| 7. | | UDY DRUG | |
| | 7.1 | Volanesorsen Description | |
| | 7.2 | Packaging and Labeling | 34 |
| | 7.3 | Study Drug Accountability | |
| 8 | | EATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , | |
| | 8.5.2 | , | |
| | 8.5. | | |
| | 8.5.4 | J 5 1 | |
| | 8.5. | | |
| | 8.5.0 | | |
| | 8.5. | 7 8 | |
| | 8.5. | | |
| | 8.5.9 | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | 11 8 | |
| | 8.6.2 | | |
| | 8.6.3 | | |
| | 8.7 | Adjustment of Dose Frequency | |
| | 8.8 | Discontinuation of Study Treatment | |
| | 8.8. | Follow-up Visits for Early Termination from Treatment Period | 43 |

| | 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Per | riod .43 |
|---|---|---|---|
| 8.9 Wit | | Withdrawal of Patients from the Study | 43 |
| | 8.10 | Concomitant Therapy and Procedures | 44 |
| | 8.10. | 1 Concomitant Therapy | 44 |
| | 8.10. | 2 Concomitant Procedures | 45 |
| | 8.11 | Treatment Compliance | 45 |
| 9. | . SEF | RIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 45 |
| | 9.1 | Sponsor Review of Safety Information | 45 |
| | 9.2 | Regulatory Requirements | 45 |
| | 9.3 | Definitions | 46 |
| | 9.3.1 | Adverse Event | 46 |
| | 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 46 |
| | 9.3.3 | Serious Adverse Event (SAE) | 46 |
| | 9.4 | Monitoring and Recording Adverse Events | 47 |
| | 9.4.1 | Serious Adverse Events | 47 |
| | 9.4.2 | Non-Serious Adverse Events | 47 |
| | 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | 48 |
| | 9.4 | 4.3.1 Relationship to the Study Drug | 48 |
| | 9.4 | 4.3.2 Severity | 48 |
| | 9.4 | 4.3.3 Action Taken with Volanesorsen | 48 |
| | 9.4 | 4.3.4 Treatment Given for Adverse Event | 49 |
| | 9.4 | 4.3.5 Outcome of the Adverse Event | 49 |
| | 9.4.4 | Adjudication Committees | 49 |
| | 9.5 | Procedures for Handling Special Situations | 50 |
| | 9.5.1 | Abnormalities of Laboratory Tests. | 50 |
| | 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 50 |
| | 9.5.3 | Dosing Errors | 50 |
| | 9.5.4 | Contraception and Pregnancy | 51 |
| 1 | 0. STA | ATISTICAL CONSIDERATIONS | 51 |
| | 10.1 | Study Endpoints | 51 |
| | 10.1. | 1 Efficacy Endpoints | 51 |
| | 10.1. | 2 Safety Endpoints | 52 |
| | 10.2 | Sample Size | 52 |
| | 10.3 | Populations | 52 |
| | 10.4 | Definition of Baseline | 53 |
| | 10.5 | Interim Analysis | 53 |
| | 10.6 | Planned Methods of Analysis | 53 |
| | 10.6. | 1 Demographic and Baseline Characteristics | 53 |
| | 10.6. | 2 Safety Analysis | 53 |
| | 10.6 | 3 Efficacy Analysis | 54 |

| 10.6 | 5.4 Pharmacokinetic and Immunogenicity Analysis | 54 |
|---|---|---|
| 1 | 0.6.4.1 Pharmacokinetic Analysis | |
| 1 | 0.6.4.2 Immunogenicity Analysis | |
| 11. IN | VESTIGATOR'S REGULATORY OBLIGATIONS | |
| 11.1 | Informed Consent | |
| 11.2 | Ethical Conduct of the Study | 56 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | |
| 11.4 | Patient Confidentiality | 57 |
| 12. AD | OMINISTRATIVE AND LEGAL OBLIGATIONS | 57 |
| 12.1 | Protocol Amendments | 57 |
| 12.2 | Study Termination | 57 |
| 12.3 | Study Documentation and Storage | 57 |
| 12.4 | Study Monitoring | 58 |
| 12.5 | Language | 59 |
| 12.6 | Compensation for Injury | 59 |
| 13. RE | FERENCES | 60 |
| 14. AP | PENDICES | 62 |
| Apper | ndix A Schedule of Procedures | 63 |
| Apper | ndix B List of Laboratory Analytes | 67 |
| Apper | ndix C Pharmacokinetic Sampling Schedule | 69 |
| Apper | ndix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities | 71 |
| | TABLE OF TABLES | |
| | ī | age |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 0 |
| Table 2 | Actions in Patients With Low Platelet Count | |
| Table 3 | Expected Event for the Protocol Defined Population by Preferred Term and | 12 |
| Tuoic 3 | the Expected Incidence | 46 |
| | TABLE OF FIGURES | |
| | I | age |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | _ |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| - | (MOE-Gapmer). The sequence of volunesorsen is shown | 22 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | 24 |

**CONFIDENTIAL** Amendment 4 Protocol 6 June 2016


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Extension Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 

**Amendment Date:** 6 June 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 3 dated 9 May 2016:

- 1. To add hematology blood draws so that platelet counts are measured every 2 weeks during the treatment period and every 2 weeks for the first 6 weeks after the last dose of Study Drug.
- 2. To update the platelet safety monitoring rules (shown in Table 2).
- 3. To add language to indicate that if there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.
- 4. To add language to indicate that all platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of  $75,000/\text{mm}^3$ .
- 5. To change the platelet dose pause/stopping rule from 50,000/mm<sup>3</sup> to 75,000/mm<sup>3</sup> and to add that when platelet count returns to  $\geq 100,000/\text{mm}^3$  dosing may be continued but at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week and only if approved by the Sponsor Medical Monitor.
- 6. To add language to indicate that in the event of any platelet count less than 25,000/mm<sup>3</sup>, or a platelet count less than 50,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg per week, then dosing of a patient with volunesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.
- 7. To add language to indicate that administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup> and to provide treatment guidelines for the administration of steroids.
- 8. To add a Table summarizing actions to be taken in the event of a low platelet count.

9. To add language to indicate that patients will receive a suitable dose or dose frequency of volanesorsen, when they enter this CS7 study, based on safety/tolerability or non-safety/tolerability dosing rules.

Minor administrative changes or corrections (not included in the list of changes) have been made throughout the protocol in order to improve the overall clarity of the protocol but these changes do not impact the study design.

The following table provides a summary list of changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Section 6.1.2<br>Treatment Period<br>Section 6.1.4 Post-<br>Treatment Period<br>Appendix A<br>Schedule of<br>Procedures | Hematology blood draws added to Weeks 2.5, 6, 10, 15, 17, 21, 23, 28, 30, 34, 36, 40, 42, 46, 48, 50, 54, 56 and removed from Weeks 16, 22, 29, 35, 41, 47 and 51. | To implement more frequent evaluation of platelet counts to assess platelet fluctuations during the course of the study and to increase platelet count monitoring for safety purposes |
| Section 8.5.2<br>Safety Monitoring<br>for Platelet Count<br>Results | Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3. | To increase platelet count monitoring for safety purposes |
| Section 6.2.1 Laboratory Assessments Section 8.6.3 Stopping Rules for Platelet Count Results Appendix A Schedule of Procedures | If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. | To increase platelet count monitoring and provide added patient safety regarding ISIS 304801 dose exposure |
| Section 6.2.1<br>Laboratory<br>Assessments<br>Appendix A<br>Schedule of<br>Procedures | All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm <sup>3</sup> . | To increase platelet count monitoring for safety purposes |
| Section 8.6.3<br>Stopping Rules for<br>Platelet Count<br>Results | Dose pause/ stopping rule changed from 50,000/mm³ to 75,000/mm³ and when platelet count returns to ≥ 100,000/mm³ dosing may be continued but at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week and only if approved by the Sponsor Medical Monitor. | To increase platelet count monitoring and provide added patient safety regarding ISIS 304801 dose exposure |

| Protocol Section | | Description of Change | | Rationale |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping Rules for<br>Platelet Count<br>Results | count less than 50,000/mm³ that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg per week, then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable. Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm³. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for | | To increase platelet count monitoring for safety purposes | |
| Section 8.6.3<br>Stopping Rules for<br>Platelet Count<br>Results | | | To provide added patient safety regarding platelet count reductions and treatment recommendations | |
| Section 8.6.3 | Table 2 Action | ns in Patients with Low Platelet | Count | To provide added |
| Stopping Rules for<br>Platelet Count<br>Results | Platelet<br>Count on<br>Rx | Drug Dose | Monitoring | patient safety<br>regarding platelet<br>count reductions,<br>ISIS 304801 dose |
| | Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every<br>2 weeks | exposure, and<br>treatment<br>recommendations |
| | 100K-<br>140K/mm <sup>3</sup> | No action | Closer observation<br>Monitor every one<br>week | |
| | 75K-<br>100K/mm <sup>3</sup> | Reduce dose frequency to<br>300mg every 2 weeks or<br>reduce dose to 150 mg weekly | Closer observation<br>Monitor every one<br>week | |
| | 50K-<br>75K/mm <sup>3</sup> | Dose pause When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/antic | |
| | 25K-<br>50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | oagulant medication Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/antic oagulant medication while platelet count < 50K/mm³ if possible | |

| Protocol Section | Description of Change | | Rationale | |
|---|---|---|---|---|
| Section 8.6.3<br>Stopping Rules for<br>Platelet Count<br>Results Continued | Table 2 Action < 25K/mm <sup>3</sup> | Permanently discontinue Study<br>Drug | Closer observation: Monitor daily until 2 successive values show improvement | |
| | | | then monitor every 2-3 days until platelet count stable. Steroids recommended* | |
| | | | Consider need for hospitalization and referral to hematologist | |
| | | | Discontinue antiplatelet agents/NSAIDS/antic oagulant medication while platelet count < 50K/mm³ if possible | |
| | high dose of<br>thrombocy<br>40 mg dail<br>0.5-2 mg/k<br>30 mg/kg/c | n platelet count may be accelerate steroids. Treatment guidelines for topenia (Provan et al. 2010) recony for 4 days every 2-4 weeks for 1-g/d for 2-4 weeks then taper; or May for 7 days (note: may require otter methylprednisolone) | immune<br>nmend Dexamethasone<br>-4 cycles; Prednis(ol)one<br>ethylprednisolone | |
| Section 8.1<br>Volanesorsen<br>Administration | frequency of St<br>in their index st<br>dose or dose fr<br>as outlined in S<br>having dose or<br>13 weeks of tre | ng this ISIS 304801-CS7 study on udy Drug (volanesorsen), for safet udy (ISIS 304801-CS6 or –CS16), equency of volanesorsen for continuections 8.5 and 8.6. Patients enter dose frequency reduced in the CS eatment, as outlined in CS16 America 300 mg once weekly dose of volant designs and the contract of | ry or tolerability reasons will receive a reduced nued safety or tolerability ering this CS7 study after adment 4 Section 8.7, | To allow patients to receive a suitable dose or dose frequency of volanesorsen, based on safety/ tolerability or non-safety/ tolerability dosing rules |

### PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Extension Study of Volanesorsen Administered<br>Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center, open-label extension study of ISIS 304801-CS6 and ISIS 304801-CS16. All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement<br/>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study |
| | 4. Able and willing to participate in a 65-week study |
| | 5. Satisfy 1 of the following: |
| | a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |

### PROTOCOL SYNOPSIS Continued

| Study Population Continued | Inclusion Criteria: Continued |
|---|---|
| | b. Males: Surgically sterile, abstinent* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |
| | * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception |
| | Exclusion Criteria: |
| | Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study |
| | Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule<br>Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6- and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies which included a subset of patients with FCS. This is an extension to the ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Only the subset of patients from ISIS 304801-CS16 with FCS diagnosis may enter the Extension Study. (Please refer to inclusion criteria #3, above) |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A. A 52-week<br/>treatment period during which volanesorsen will be administered as<br/>a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

### PROTOCOL SYNOPSIS Continued

| Planned Analyses Safety Endpoints: Adverse events including adjudicated events of acute pancreatitis and MACE Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (NLDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein | Safety and Tolerability Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|---|
| and MACE • Vital signs and weight • Physical examinations • Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) • Echocardiography • Electrocardiograms (ECGs) • Use of concomitant medications • MRIs Efficacy Endpoints: • Percent change and absolute change from baseline in fasting TG • Frequency and severity of patient reported abdominal pain during the treatment period • Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-I [apoA-I], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C • Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) • Quality of Life questionnaires (EQ-5D, SF-36) • Adjudicated acute pancreatitis event rate • Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen as follows: trough levels (pre-dose) throughout treatment and apost-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | Planned Analyses | Safety Endpoints: |
| Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-hDL-C), applipoprotein B [apoB], high-density lipoprotein-cholesterol (N-DL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (V-DL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | | |
| Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (hon-HDL-C), apolipoprotein B[apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (HDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | | Vital signs and weight |
| urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | | Physical examinations |
| Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-High-density lipoprotein-cholesterol (N-IDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | |
| Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment felvels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | Echocardiography |
| MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | Electrocardiograms (ECGs) |
| Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | Use of concomitant medications |
| Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLD-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | MRIs |
| Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Efficacy Endpoints: |
| the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein A-1 [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoB-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | Percent change and absolute change from baseline in fasting TG |
| measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C • Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) • Quality of Life questionnaires (EQ-5D, SF-36) • Adjudicated acute pancreatitis event rate • Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | |
| (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], |
| Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | |
| Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Quality of Life questionnaires (EQ-5D, SF-36) |
| Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Adjudicated acute pancreatitis event rate |
| volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Other symptoms: eruptive xanthoma, lipemia retinalis |
| the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | Pharmacokinetic Evaluations | volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A |
| | Statistical Considerations | the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 |
| Collaborator Akcea Therapeutics | Sponsor | Ionis Pharmaceuticals, Inc. |
| | Collaborator | Akcea Therapeutics |



#### STUDY GLOSSARY

IM

**Index Studies** 

| STUDY GLOSSARY | |
|---|---|
| Abbreviation/Acronym | <b>Definition</b> |
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| 70.5 | |

ISIS 304801-CS6 and ISIS 304801-CS16

immunogenicity

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OLE Open Label Extension

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 6 June 2016

#### 1. **OBJECTIVES**

The objective of the study is to evaluate the safety and efficacy of extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 **Overview of Disease**

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 Therapeutic Rationale

Protocol

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Protocol

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label extension to the Phase 3 study of volanesorsen in patients with FCS (ISIS 304801-CS6 or ISIS 304801-CS16). Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

- A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.
- A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection
- A 13-week post-treatment evaluation period

Please refer to the Schedule of Procedures in Appendix A.

#### 3.4.1 *Qualification*

A period of up to 2 weeks is given to complete qualification assessments outlined in the Schedule of Procedures (Appendix A).

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule or Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

#### 3.5 End of Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 **Qualification**

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open label study are performed. During the qualification period, the eligibility of the patient to continue in the extension study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are

enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of  $\leq 20\%$  of normal
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study.
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 Exclusion Criteria

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 2.5, 4, 6, 8, 10, 12, 15, 17, 19, 21, 23, 25, 28, 30, 32, 34, 36, 40, 42, 44, 46, 48, 50, 54, 56, and 58 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally should also be sent to the central laboratory for analysis whenever possible. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 4 Study Center visits on Weeks 54, 56, 58 and 65 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.2.10 Lipoprotein Lipase Activity Sample Collection

Lipoprotein lipase (LPL) activity will be measured in ISIS 304801-CS16 rollover patients if needed for study qualification. In brief, fasted patients will be given a low intravenous dose of heparin. A blood sample will be drawn prior to and at 10 or 15 minutes after the heparin administration for measurement of LPL activity as per instructions provided to the Investigator.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent\* or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

• Using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

\* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL 300 mg injection once weekly for Weeks 1-52. Patients entering this ISIS 304801-CS7 study on a reduced dose or dose frequency of Study Drug (volanesorsen), for safety or tolerability reasons in their index study (ISIS 304801-CS6 or –CS16), will receive a reduced dose or dose frequency of volanesorsen for continued safety or tolerability as outlined in Sections 8.5 and 8.6. Patients entering this CS7 study having dose or dose frequency reduced in the CS16 index study after 13 weeks of treatment, as outlined in CS16 Amendment 4 Section 8.7, can receive the 300 mg once weekly dose of volanesorsen.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

Protocol

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. Reduction in dose or dose frequency may also be initiated as noted in Section 8.7. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be dose paused or permanently discontinued (as described in the stopping criterion concerned) from further treatment with volanesorsen, and evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio

(INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

Actions to be taken in the event of reduced platelet count are shown in Table 2 in Section 8.6.3.

Additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Protocol

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for Hyperglycemia below.

<u>All diabetic patients</u> will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.
Protocol

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate

Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

6 June 2016

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 **Stopping Rules**

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volanesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed and total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

Protocol

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5 µmol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rules for Platelet Count Results

Actions to be taken in the event of a low platelet count are summarized in Table 2 below.

In the event of a platelet count less than 75,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of any platelet count less than 25,000/mm<sup>3</sup>, or a platelet count less than 50,000/mm<sup>3</sup> that occurs while the patient is on dosing at 300 mg every 2 weeks or 150 mg every week then dosing of a patient with volanesorsen will be stopped permanently. Platelet count will be monitored daily until 2 successive values show improvement then monitored every 2-3 days until platelet count is stable.

Administration of steroids is recommended for patients whose platelet count is less than 25,000/mm<sup>3</sup>. Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (note: may require continuation with oral steroids after methylprednisolone).

In the event of a platelet count less than 75,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to ≥ 100,000/mm³. If dosing is continued it should be at a reduced dose frequency of 300 mg every 2 weeks or a reduced dose of 150 mg per week (refer to Section 8.7). The suitability of the patient for continued dosing will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 75,000/mm<sup>3</sup>, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm<sup>3</sup>. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be re-examined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above.

If after the second rechallenge the platelet count falls below 75,000/mm<sup>3</sup> and is subsequently confirmed (see Section 8.5), dosing with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed.

#### <u>Definition of Major Bleeding Events</u> (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

#### <u>Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):</u>

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

Table 2 Actions in Patients with Low Platelet Count

| Platelet Count on Rx | Drug Dose | Monitoring |
|---|---|---|
| Normal range, > 140K/mm <sup>3</sup> | No action | Monitor every 2 weeks |
| 100K-140K/mm <sup>3</sup> | No action | Closer observation Monitor every one week |
| 75K-100K/mm <sup>3</sup> | Reduce dose frequency to 300 mg every 2 weeks or reduce dose to 150 mg weekly | Closer observation Monitor every one week |
| 50K-75K/mm <sup>3</sup> | Dose pause When platelet count returns to >100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor every 2-3 days until 2 successive values show improvement Consider discontinuation of antiplatelet agents/NSAIDS/ anticoagulant medication |
| 25K-50K/mm <sup>3</sup> | If occurs while on dose of 300 mg every 2 weeks or 150 mg every week then permanently discontinue Study Drug, otherwise dose pause. When platelet count returns to > 100K/mm³ restart dosing at dose frequency of 300 mg every 2 weeks or 150 mg weekly only if approved by Sponsor Medical Monitor | Closer observation Monitor daily until 2 successive values show improvement then monitor every 2-3 days until platelet count stable Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |
| < 25K/mm <sup>3</sup> | Permanently discontinue Study Drug | Closer observation: Monitor daily until two successive values show improvement then monitor every 2-3 days until platelet count stable Steroids recommended* Consider need for hospitalization and referral to hematologist Discontinue antiplatelet agents/NSAIDS/anticoagulant medication while platelet count < 50K/mm³ if possible |

<sup>\*</sup> Recovery in platelet count may be accelerated by administration of high dose steroids. Treatment guidelines for immune thrombocytopenia (Provan et al. 2010) recommend Dexamethasone 40 mg daily for 4 days every 2-4 weeks for 1-4 cycles; Prednis(ol)one 0.5-2 mg/kg/d for 2-4 weeks then taper; or Methylprednisolone 30 mg/kg/day for 7 days (**note:** may require continuation with oral steroids after methyl prednisolone)

#### 8.7 Adjustment of Dose Frequency

Dose adjustments for platelet count reduction must be made in accordance with Section 8.6.3 and Table 2 (above).

Other dose adjustments, including dose interruptions, and/or decreasing the dose or dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

• At the discretion of the Investigator for medical reasons

- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Amendment 4

6 June 2016

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

## 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### 8.11 Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 3 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen e.g., confirmation by positive rechallenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volunesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

#### *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volunesorsen was discontinued and not restarted

- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Protocol

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- Became Serious: The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- Recovered: Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 **Adjudication Committees**

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

Amendment 4 6 June 2016

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Protocol

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 **Study Endpoints**

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.

#### *10.1.1* Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period

- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### 10.2 Sample Size

No sample size calculations were performed as this is an extension study to the double-blind, placebo-controlled ISIS 304801-CS6 and ISIS 304801-CS16 studies. Approximately 70 patients may be eligible to enroll into this study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Protocol

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient: ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline and the baseline in this open label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the extension study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this OLE study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open label extension (OLE) study from the intensive PK subgroup, following a single dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies. On Week 1 Day 1 of the OLE study, patients who received placebo in the index study will receive the first treatment of volunesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration  $(CL_{0-24hr}/F_{0-24hr})$  will be calculated from  $CL_{0-24hr}/F_{0-24hr} = Actual Dose/AUC_{0-24hr}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events

occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed

consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Protocol

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

# 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev. Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Provan D, Stasi R, Newland AC, et al. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood 2010; 115: 168-186.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

## 14. APPENDICES

# **Appendix A** Schedule of Procedures

# ${\bf Appendix} \; {\bf A} \quad {\bf Schedule} \; {\bf of} \; {\bf Procedures}$

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | | Treatr | nent l | Period | d | | | | | | | | | Post Fol | Treatr | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | w | n. | Wk | Wk | Wk | Wk | Wk | Mor | nth 3 | Wk<br>15 | Wk | Wk<br>21 | Mor | nth 6 | Wk<br>28 | Wk | Wk<br>34 | Wk | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk54 | Wk | Wk |
| | Study Week | -2 to -1 | 1 | l<br>I | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | &<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | &<br>30 | 32 | &<br>36 | 38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| | Study Day | -14 to -<br>7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Inf | ormed Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Ou | tpatient Visit | Х | Х | $\mathbf{X}^{k}$ | $X^k$ | $X^k$ | $X^k$ | $X^k$ | $X^k$ | $X^k$ | Χ | $X^k$ | X <sup>k</sup> | $X^k$ | X <sup>k</sup> | Х | X <sup>k</sup> | X <sup>k</sup> | $X^k$ | Χ | $X^k$ | $X^k$ | $X^k$ | X <sup>k</sup> | Х | X <sup>k</sup> | X <sup>k</sup> | Х |
| Inc | lusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Vit<br>(+ | al Signs + body weight<br>neight on Day 1 only) | Х | х | | | Х | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Х |
| Ph | ysical Examination | | Х | | | | | | | | Х | | | | | Х | | | | Χ | | | | | Х | | | Х |
| 12 | lead ECG (triplicate) | | | | | | | | | | Х | | | | | Х | | | | Χ | | | | | Х | | | Х |
| MF | I (liver/spleen) | | | | | | | | | | | | | | | | | | | | | | | | X | | | |
| Ec | nocardiography | | | | | | | | | | | | | | | Χ <sup>l</sup> | | | | | | | | | XI | | | |
| | Chemistry Panel | Х | Х | | | Х | | Х | | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | | Х | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | Serum Lipid Panel | Х | Х | | | Χ | ĺ | Х | | Х | Х | | | | Х | Х | | | | Х | | | | Х | Х | | | Х |
| g) <sub>c</sub> | Coagulation (aPTT, PT, INR) | PG | | | | | | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | |
| (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and<br>de-lipidated free glycerol | | х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| <b>&gt;</b> | Sedimentation Rate | | Х | | | | | | | | Χ | | | | | Х | | | | | | | | | Χ | | | Х |
| Draw | Complement (C5a, Bb) | | Х | | | | | | | | Χ | | | | | Х | | | | | | | | | Х | | | Х |
| l po | Plasma PK - Volanesorsen | | $X^{m}$ | Χ | | Χ | | Х | | | Χ | | | | | Х | | | | Χ | | | | | Х | | | Х |
| Blood | Anti-Volanesorsen Antibodies | | Х | H | | Χ | - | Х | | | Х | | | | | Х | | | | Х | | | | | Х | | | Χ |
| 1 | FSH (women only, if applicable) | <b>.</b> | | $\vdash$ | | L. | | | | | | | | | | | | l | | | | | | | | | | 1 |
| | Serum Pregnancy Test <sup>d</sup> | Х | | | | Χ | | Х | | | Х | | Х | | | Х | | Χ | | Χ | | Х | | | Х | | Х | Х |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | Х | | | | | Х | | | Х | | | | | Х | | | | | | | | | Х | | | Х |

### Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | | | | | | | | | | | Treatm | ent P | eriod | | | | | | | | | | Tre | Post<br>eatme<br>llow-u | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 14 | ۷k | Wk | Wk | Wk | Wk | \A/I+ | Mor | ıth 3 | Wk | Wk | Wk<br>21 | | | Wk | Wk | Wk<br>34 | k Mile | Wk<br>40 | Wk | Wk<br>46 | Мо | nth 12 | Wk<br>54 | Wk | Wk |
| Study Week | -2 to -1 | | 7 K | 2.5 | 4 | 6 | 8 | 10 | Wk<br>12 | Wk<br>13 | 15<br>&<br>17 | 19 | &<br>23 | Wk<br>25 | Wk<br>26 | 28<br>&<br>30 | 32 | | Wk<br>38 | &<br>42 | 44 | &<br>48 | Wk<br>50 | Wk 52<br>or ET | &<br>56 | 58 | 65 |
| Study Day | -14 to -7 | 1 | 2 | 11 | 22 | 36 | 50 | 64 | 78 | 85 | 99<br>&<br>113 | 127 | 141<br>&<br>155 | 169 | 176 | 190<br>&<br>204 | 218 | 232<br>&<br>246 | 260 | 274<br>&<br>288 | 302 | 316<br>&<br>330 | 344 | 358 | 372<br>&<br>386 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | X <sup>n</sup> | | | Х | | Х | | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | | X <sup>n</sup> | X <sup>n</sup> |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | XI | | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>g</sup> | × | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Postheparin Lipoprotein<br>Lipase activity <sup>h</sup> | х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC<br>Injection | | Х | | х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | Х | х | Х | Х | | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Food/Drink Diary (quarterly) <sup>i</sup> | | Х | | | | | | | | Х | | | | | Х | | | | | | | | | Х | | | Х |
| Diet/Alcohol Counseling <sup>j</sup> | Х | Χ | | | Х | | Χ | | | Х | | | | | Х | | | | Χ | | | | | Χ | | Х | Х |
| Adverse Events | Х | Χ | | Х | Х | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Concomitant Medication | Х | Х | | Χ | Χ | Х | Х | Х | Χ | Χ | Х | Х | Х | Χ | Х | Χ | Χ | Х | Χ | Х | Χ | Х | Χ | Х | Χ | Χ | Х |

a Qualification procedures performed (Please refer to Section 4.1)

b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue. If there is no reportable platelet count within 14 days of the last platelet count, the Investigator will contact the patient to hold dosing until a new platelet count is obtained and reviewed. All platelet count results will be promptly reviewed by the Investigator to ensure that the count has not met the stopping rule and to determine whether the rate of decline is suggestive that the patient could be approaching the dose pause rule of 75,000/mm<sup>3</sup>. Any case of a platelet count < 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor

#### **Appendix A** Schedule of Procedures Continued

#### Legend Text Continued

- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (ISIS 304801-CS16 rollover patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study qualification (ISIS 304801-CS16 rollover patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h Post-heparin lipoprotein lipase activity can be conducted for study qualification (ISIS 304801-CS16 rollover patients; please refer to Section 6.2.10)
- i In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- j To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- k Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- I A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- m Full or abbreviated PK profile (see Appendix C)
- n Expanded urinalysis (see Appendix B)

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| | Hematology | Uringlysis |
|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Potasium P | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | Urinalysis Color Appearance Specific gravity pH Protein Blood Ketones Urobilinogen Glucose Bilirubin Leukocyte esterase Nitrate Microscopic examination <sup>2</sup> Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin β2-microglobulin |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

# Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

## PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td colspan="3">Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm <sup>3</sup> ;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase >ULN - 3.0 x ULN increased | | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td colspan="4">&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | | Urine | |
| Proteinuria<br>Adults | 1+ proteinuria; | 2+ proteinuria; | Urinary protein ≥3.5 g/24 hrs; |
| | urinary protein <1.0 g/24 hrs | urinary protein 1.0 - 3.4 g/24 hrs;<br>Urine P/C (Protein/Creatinine) | |
| Children | | ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** Ionis Pharmaceuticals, Inc.

2855 Gazelle Court
Carlsbad, CA 92010

A subsidiary of Isis Pharmaceuticals, Inc.

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

### ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 3 –9 May 2016

EudraCT No: 2015-003755-21

#### ISIS 304801-CS7

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

## An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

## Protocol Amendment 3 – 9 May 2016

#### **Protocol History:**

Original Protocol: 28 August 2015

Protocol Amendment 1: 2 February 2016

Protocol Amendment 2: 22 April 2016

#### **Sponsor:**

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

M.D., M.B.A.

#### Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 3** 

**EudraCT No: 2015-003755-21** 

Clinical Phase: 3

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

## An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 9 May 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | * | udy of Volanesorsen Administered ith Familial Chylomicronemia Syndrome |
| Amendment: | Amendment 3 | |
| Date: | 9 May 2016 | |
| Open-Label Extension | on Study of Volanesorsen Adm | and the attached clinical protocol, entitled "An inistered Subcutaneously to Patients with 19 May 2016, and agree to conduct the study |
| I agree to comply wi<br>Good Clinical Practi | | on Harmonization Tripartite Guideline on |
| any purpose other that | | ontained in this document will not be used for<br>the clinical investigation without the prior |
| Investigator's Signa | ture | |
| Investigator's Name | c (please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| | | Page |
|------|---------------------------------------------------|------|
| | OCOL AMENDMENT | |
| | OCOL SYNOPSIS | |
| | Y DESIGN AND TREATMENT SCHEMA | |
| STUD | Y GLOSSARY | 15 |
| | OBJECTIVES | |
| | ACKGROUND AND RATIONALE | |
| 2.1 | Overview of Disease | |
| 2.2 | Therapeutic Rationale | |
| 2.3 | Volanesorsen | 19 |
| 2 | 3.1 Mechanism of Action | 19 |
| 2 | 3.2 Chemistry | 20 |
| 2 | 3.3 Preclinical Experience | 21 |
| 2. | 3.4 Clinical Experience | |
| 2.4 | Rationale for Dose and Schedule of Administration | 23 |
| 3. E | XPERIMENTAL PLAN | 24 |
| 3.1 | Study Design | 24 |
| 3.2 | Number of Study Centers | 24 |
| 3.3 | Number of Patients | 24 |
| 3.4 | Overall Study Duration and Follow-up | 24 |
| 3. | 4.1 Qualification | 24 |
| 3. | 4.2 Treatment | 24 |
| 3. | 4.3 Post-Treatment | 24 |
| 3.5 | End of Study | 24 |
| 3.6 | Data and Safety Monitoring Board | 25 |
| 4. P | ATIENT ENROLLMENT | 25 |
| 4.1 | Qualification | 25 |
| 4.2 | Enrollment | 25 |
| 5. P | ATIENT ELIGIBILITY | 25 |
| 5.1 | Inclusion Criteria | 25 |
| 5.2 | Exclusion Criteria | 26 |
| 6. S | TUDY PROCEDURES | 27 |
| 6.1 | Study Schedule | 27 |
| 6. | 1.1 Qualification | 27 |
| 6. | 1.2 Treatment Period | |
| 6. | 1.3 Pharmacokinetic (PK) Subgroup | |
| 6. | 1.4 Post-Treatment Period | |
| 6.2 | Additional Study Assessments | |
| | 2.1 Laboratory Assessments | |

| | 6.2. | Physical Exams and Vital Signs | 28 |
|---|---|---|---|
| | 6 | 2.2.1 Eruptive Xanthoma | |
| | 6 | 2.2.2 Lipemia Retinalis | 28 |
| | 6.2. | 3 Echocardiography | 29 |
| | 6.2. | 4 ECG | 29 |
| | 6.2. | 5 MRI | 29 |
| | 6.2. | 6 Quality of Life Assessments | 29 |
| | 6.2. | 7 Disease Symptom Diary | 29 |
| | 6.2. | 8 Diet Monitoring | 29 |
| | 6.2. | 9 Family History | 29 |
| | 6.2. | 10 Lipoprotein Lipase Activity Sample Collection | 30 |
| | 6.3 | Restriction on the Lifestyle of Patients. | 30 |
| | 6.3. | 1 Contraception Requirements | 30 |
| | 6.3. | 2 Other Requirements | 31 |
| 7. | ST | UDY DRUG | 31 |
| | 7.1 | Volanesorsen Description | 31 |
| | 7.2 | Packaging and Labeling | 32 |
| | 7.3 | Study Drug Accountability | |
| 8. | | EATMENT OF PATIENTS | |
| | 8.1 | Volanesorsen Administration | |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | |
| | 8.4 | Treatment Precautions | |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , c | |
| | 8.5. | $\mathcal{E}$ | |
| | 8.5. | , | |
| | 8.5. | J 5 1 | |
| | 8.5. | | |
| | 8.5. | , | |
| | 8.5. | 7 0 | |
| | 8.5. | | |
| | 8.5. | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | 11 8 | |
| | 8.6. | 11 & | |
| | 8.6. | | |
| | 8.7 | Adjustment of Dose Frequency | |
| | 8.8 | Discontinuation of Study Treatment | |
| | 8.8. | 1 Follow-up Visits for Early Termination from Treatment Period | 40 |

| 8.8.2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Pe | riod .40 |
|---|---|---|
| 8.9 Wit | hdrawal of Patients from the Study | 40 |
| 8.10 Cor | acomitant Therapy and Procedures | 41 |
| 8.10.1 | Concomitant Therapy | 41 |
| 8.10.2 | Concomitant Procedures | 41 |
| 8.11 Tre | atment Compliance | 42 |
| 9. SERIO | US AND NON-SERIOUS ADVERSE EVENT REPORTING | 42 |
| 9.1 Spo | nsor Review of Safety Information | 42 |
| 9.2 Reg | rulatory Requirements | 42 |
| 9.3 Def | initions | 43 |
| 9.3.1 | Adverse Event | 43 |
| 9.3.2 | Adverse Reaction and Suspected Adverse Reaction | 43 |
| 9.3.3 | Serious Adverse Event (SAE) | 43 |
| 9.4 Mo | nitoring and Recording Adverse Events | 44 |
| 9.4.1 | Serious Adverse Events | 44 |
| 9.4.2 | Non-Serious Adverse Events | 44 |
| 9.4.3 | Evaluation of Adverse Events (Serious and Non-Serious) | 44 |
| 9.4.3.1 | Relationship to the Study Drug | 44 |
| 9.4.3.2 | 2 Severity | 45 |
| 9.4.3.3 | Action Taken with Volanesorsen | 45 |
| 9.4.3.4 | Treatment Given for Adverse Event | 45 |
| 9.4.3.5 | Outcome of the Adverse Event | 46 |
| 9.4.4 | Adjudication Committees | 46 |
| 9.5 Pro | cedures for Handling Special Situations | 46 |
| 9.5.1 | Abnormalities of Laboratory Tests | 46 |
| 9.5.2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 47 |
| 9.5.3 | Dosing Errors | 47 |
| 9.5.4 | Contraception and Pregnancy | 47 |
| 10. STATIS | STICAL CONSIDERATIONS | 48 |
| 10.1 Stud | dy Endpoints | 48 |
| 10.1.1 | Efficacy Endpoints | 48 |
| 10.1.2 | Safety Endpoints | 49 |
| 10.2 San | nple Size | 49 |
| 10.3 Pop | ulations | 49 |
| 10.4 Def | inition of Baseline | 49 |
| 10.5 Inte | rim Analysis | 50 |
| 10.6 Plan | nned Methods of Analysis | 50 |
| 10.6.1 | Demographic and Baseline Characteristics | 50 |
| 10.6.2 | Safety Analysis | |
| 10.6.3 | Efficacy Analysis | 51 |

| 10.0 | 6.4 Pharmacokinetic and Immunogenicity Analysis | 51 |
|---|---|---|
| 1 | 0.6.4.1 Pharmacokinetic Analysis | |
| 1 | 0.6.4.2 Immunogenicity Analysis | |
| 11. IN | VESTIGATOR'S REGULATORY OBLIGATIONS | |
| 11.1 | Informed Consent | |
| 11.2 | Ethical Conduct of the Study | 53 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | |
| 11.4 | Patient Confidentiality | |
| 12. AI | OMINISTRATIVE AND LEGAL OBLIGATIONS | 54 |
| 12.1 | Protocol Amendments | |
| 12.2 | Study Termination | 54 |
| 12.3 | Study Documentation and Storage | 54 |
| 12.4 | Study Monitoring | 55 |
| 12.5 | Language | 56 |
| 12.6 | Compensation for Injury | 56 |
| 13. RF | EFERENCES | |
| 14. AF | PPENDICES | 59 |
| Appei | ndix A Schedule of Procedures | 60 |
| Appei | ndix B List of Laboratory Analytes | 64 |
| Appei | ndix C Pharmacokinetic Sampling Schedule | 66 |
| Apper | ndix D Grading Scale for Adverse Events Relating to Laboratory Abnormaliti | |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | U |
| Table 2 | Expected Event for the Protocol Defined Population by Preferred Term | 32 |
| Table 2 | and the Expected Incidence | 42 |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | 18 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides | |
| | (MOE-Gapmer). The sequence of volunesorsen is shown | 20 |
| Figure 3 | Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Extension Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 3

**Amendment Date:** 9 May 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 2 dated 22 April 2016:

- 1. To add language that any case of a platelet count  $\leq 50,000/\text{mm}^3$  should be reported in an expedited fashion to the Sponsor.
- 2. To add language regarding the frequency of obtaining platelet counts after a Study Drug dose pause and subsequent rechallenge.
- 3. To add language that any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

Minor administrative changes or corrections (not included in the list of changes) have been made throughout the protocol in order to improve the overall clarity of the protocol but these changes do not impact the study design.

The following table provides a summary list of changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Section 6.2.1<br>Laboratory Assessments<br>Section 8.5.2<br>Safety Monitoring for<br>Platelet Count Results<br>Appendix A Schedule<br>of Procedures | Any case of a platelet count ≤ 50,000/mm <sup>3</sup> should<br>be reported in an expedited fashion to the<br>Sponsor | To ensure that Sponsor is aware in a timely fashion of platelet counts performed in local lab that have met the rule for dose pause |
| Section 8.6.3<br>Stopping Rules for Platelet<br>Count Results | Following a rechallenge platelet count should be tested every week until count is stable | To more closely monitor platelet levels following a rechallenge |
| Section 6.2.1 Laboratory Assessments Section 8.6.3 Stopping Rules for Platelet Count Results Appendix A Schedule of Procedures | Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue | To provide added patient safety regarding platelet stopping rules |

## PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center, open-label extension study of ISIS 304801-CS6 and ISIS 304801-CS16. All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | <ol> <li>Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16<br/>(index studies) with an acceptable safety profile, per Sponsor and<br/>Investigator judgement. Patients who are enrolled in ISIS 304801-CS16<br/>must also meet the following criteria in order to enter into the Extension<br/>Study:</li> </ol> |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following: </li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study |
| | 4. Able and willing to participate in a 65-week study |
| | 5. Satisfy 1 of the following: |
| | a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |

| Study Population Continued | Inclusion Criteria: Continued |
|---|---|
| otacy i opulation commutes | b. Males: Surgically sterile, abstinent* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |
| | * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception |
| | Exclusion Criteria: |
| | Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study |
| | Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6- and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies which included a subset of patients with FCS. This is an extension to the ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Only the subset of patients from ISIS 304801-CS16 with FCS diagnosis may enter the Extension Study. (Please refer to inclusion criteria #3, above) |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A. A 52-week<br/>treatment period during which volanesorsen will be administered as<br/>a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

## PROTOCOL SYNOPSIS Continued

| urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | Safety and Tolerability Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|---|
| and MACE Vital signs and weight Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (hDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-priord. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesoren pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | Planned Analyses | Safety Endpoints: |
| Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein Elapost), high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | |
| Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (Non-HDL-C), apolipoprotein [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (HDL-C), apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations Ionis Pharmaceuticals, Inc. | | Vital signs and weight |
| urinalysis) Echocardiography Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | Physical examinations |
| Electrocardiograms (ECGs) Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-high-density lipoprotein-cholesterol (non-high-density lipoprotein-cholesterol (non-high-density lipoprotein-cholesterol (NLDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation,<br/>urinalysis)</li> </ul> |
| Use of concomitant medications MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein B [apoB-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | Echocardiography |
| MRIs Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Electrocardiograms (ECGs) |
| Efficacy Endpoints: Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [appB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor | | Use of concomitant medications |
| Percent change and absolute change from baseline in fasting TG Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. | | • MRIs |
| Frequency and severity of patient reported abdominal pain during the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein B-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment fellow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Efficacy Endpoints: |
| the treatment period Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) Quality of Life questionnaires (EQ-5D, SF-36) Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Percent change and absolute change from baseline in fasting TG |
| measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1] very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C • Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) • Quality of Life questionnaires (EQ-5D, SF-36) • Adjudicated acute pancreatitis event rate • Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor lonis Pharmaceuticals, Inc. | | |
| (apoC-III) | | measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1], |
| Adjudicated acute pancreatitis event rate Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | |
| Other symptoms: eruptive xanthoma, lipemia retinalis Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | <ul> <li>Quality of Life questionnaires (EQ-5D, SF-36)</li> </ul> |
| Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Adjudicated acute pancreatitis event rate |
| volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. Statistical Considerations No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | | Other symptoms: eruptive xanthoma, lipemia retinalis |
| the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Sponsor Ionis Pharmaceuticals, Inc. | Pharmacokinetic Evaluations | volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A |
| · | Statistical Considerations | the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 |
| | Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator Akcea Therapeutics | Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



#### STUDY GLOSSARY

## Abbreviation/Acronym Definition

ADA anti-drug antibody AE adverse Event

ALP alkaline Phosphatase
ALT alanine Aminotransferase
ANA antinuclear Antibody
apoA-1 apolipoprotein A-1
apoB apoC-III apolipoprotein C-III
apoE apolipoprotein E

aPTT activated partial thromboplastin time

ASO antisense oligonucleotide AST aspartate aminotransferase

AUC area under the curve
BMI body mass index
CBC complete blood count

C<sub>max</sub> maximum observed drug concentration

CRF case report form

DNA deoxyribonucleic Acid

DSMB Data and Safety Monitoring Board

ECG electrocardiogram

eCRF electronic Case Report Form
EDC electronic data capture
ET early termination
FAS full analysis set

FCS Familial Chylomicronemia Syndrome

GCP Good Clinical Practice
GLP-1 glucagon-like peptide-1

GPIHBP1 Glycosylphosphatidylinositol-anchored HDL-binding Protein 1

HAPI Heritability and Phenotype Intervention

HbA1c Glycated Hemoglobin
HDL High-Density Lipoprotein

HDL-C High-Density Lipoprotein-Cholesterol hsCRP High-sensitivity C-reactive protein

ICH International Conference on Harmonization

IDL Intermediate density lipoprotein IEC Independent Ethics Committee

IM immunogenicity

Index Studies ISIS 304801-CS6 and ISIS 304801-CS16

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OLE Open Label Extension

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

Amendment 3 9 May 2016 Protocol

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



**ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** Figure 1

From Ooi et al. 2008: ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester. CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volunesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

Amendment 3

9 May 2016

The pharmacokinetics (PK) and toxicity of volunesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), in vitro and in vivo genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volunesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (in vitro and in vivo) and was non-genotoxic (in vitro and in vivo). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

Protocol

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label extension to the Phase 3 study of volanesorsen in patients with FCS (ISIS 304801-CS6 or ISIS 304801-CS16). Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

- A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.
- A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection
- A 13-week post-treatment evaluation period

Please refer to the Schedule of Procedures in Appendix A.

#### 3.4.1 Qualification

A period of up to 2 weeks is given to complete qualification assessments outlined in the Schedule of Procedures (Appendix A).

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule or Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

#### 3.5 End of Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 **Qualification**

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open label study are performed. During the qualification period, the eligibility of the patient to continue in the extension study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are

enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of  $\leq 20\%$  of normal
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study.
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 Exclusion Criteria

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 4, 8, 12, 16, 19, 22, 25, 29, 32, 35, 41, 44, 47, 51, and 58 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally must be sent to the central laboratory for analysis. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 2 Study Center visits on Weeks 58 and 65 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of these analytes is contained in Appendix B.

Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue.

Any case of a platelet count  $\leq$  50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 *MRI*

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.2.10 Lipoprotein Lipase Activity Sample Collection

Lipoprotein lipase (LPL) activity will be measured in ISIS 304801-CS16 rollover patients if needed for study qualification. In brief, fasted patients will be given a low intravenous dose of heparin. A blood sample will be drawn prior to and at 10 or 15 minutes after the heparin administration for measurement of LPL activity as per instructions provided to the Investigator.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent\* or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause <u>and</u> FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

• Using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine

contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) <u>together with spermicidal foam/gel/film/cream/suppository</u>.

- \*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.
- \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

#### Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL injection once weekly for Weeks 1-52.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be permanently discontinued from further treatment with volanesorsen, evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio

(INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become < 1.2 x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

In the event of any significant fall in platelet count, or if the absolute platelet count is 75,000/mm<sup>3</sup> or less, then the patient's platelet counts should be monitored more frequently. The frequency of monitoring and additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

Any case of a platelet count  $\leq 50,000/\text{mm}^3$  should be reported in an expedited fashion to the Sponsor (See also Stopping Rules Section 8.6.3).

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any <u>hypoglycemic</u> episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L).
  - Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.
If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

# 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate

• Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

Protocol

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5 µmol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault  $\leq$  40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

## 8.6.3 Stopping Rules for Platelet Count Results

In the event of a platelet count less than 50,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of a platelet count less than  $50,000/\text{mm}^3$ , and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to  $\geq 100,000/\text{mm}^3$ . The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing rechallenge the platelet count again falls below 50,000/mm<sup>3</sup>, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm<sup>3</sup>. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be re-examined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above.

If after the second rechallenge the platelet count falls below 50,000/mm<sup>3</sup> and is subsequently confirmed (see Section 8.5), dosing with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor.

Following a rechallenge platelet count should be tested every week until count is stable.

Any unreportable platelet count result must be rechecked and determined not to have met a stopping rule before dosing can continue.

# Definition of Major Bleeding Events (Schulman et al. 2005):

• Fatal bleeding, and/or

Protocol

- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

## Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

# 8.7 Adjustment of Dose Frequency

Dose adjustments, including dose interruptions, and/or decreasing the dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed for patients that are unable to tolerate the once weekly dose (for example if platelet counts fall below 50,000/mm³ as described in Section 8.6.3). If the patient remains stable after adjustment, they may be cautiously returned to the original once weekly regimen after consultation with the Study Medical Monitor.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment

• The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

# 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be

encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

# 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 2 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the

aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volunesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate

medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

• **Related:** There is clear evidence that the event is related to the use of volunesorsen e.g., confirmation by positive rechallenge test

- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volunesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

# *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volunesorsen

Action taken with volanesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- Temporarily Interrupted, restarted same dose: Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

## 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor

Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

# 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### 10.2 Sample Size

No sample size calculations were performed as this is an extension study to the double-blind, placebo-controlled ISIS 304801-CS6 and ISIS 304801-CS16 studies. Approximately 70 patients may be eligible to enroll into this study.

# 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volunesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volanesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient: ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline and the baseline in this open label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study

baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the extension study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this OLE study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

# 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

## 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volanesorsen will be carried out on each individual patient data set using data collected in the open label extension (OLE) study from the intensive PK subgroup, following a single dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies. On Week 1 Day 1 of the OLE study, patients who received placebo in the index study will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration ( $C_{max}$ ) and the time

taken to reach  $C_{max}$  ( $T_{max}$ ) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours ( $AUC_{0-24hr}$ ) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration ( $CL_{0-24hr}$ / $F_{0-24hr}$ ) will be calculated from  $CL_{0-24hr}$ / $F_{0-24hr}$  = Actual Dose/AUC<sub>0-24hr</sub>. Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr}$  =  $AUMC_{0-24hr}$ / $AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

# 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

# 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Amendment 3

9 May 2016

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with

Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

# 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev. Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

# ${\bf Appendix} \; {\bf A} \quad {\bf Schedule} \; {\bf of} \; {\bf Procedures}$

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | | | Trea | ost<br>tment<br>ow-up | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Mor | th 3 | | | | Month 6 | ith 6 | | | | | | | | Month 12 | | | |
| Study Week | | -2 to -1 | Y | /k<br>1 | Wk 4 8 | Wk<br>12 | Wk<br>13 | Wk<br>16 | Wk<br>19 | Wk Wk<br>19 22 | Wk<br>25 | Wk<br>26 | Wk<br>29 | Wk<br>32 | Wk<br>35 | Wk<br>38 | Wk<br>41 | Wk<br>44 | Wk<br>47 | Wk<br>51 | Wk 52<br>or ET | Wk<br>58 | Wk<br>65 | |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 106 | 127 | 148 | 169 | 176 | 197 | 218 | 239 | 260 | 281 | 302 | 323 | 351 | 358 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Inform | ned Consent | Х | | | | | | | | | | | | | | | | | | | | | | |
| Outpa | tient Visit | Х | Х | $X^k$ | $X^k$ | X <sup>k</sup> | X <sup>k</sup> | Х | $X^k$ | $X^k$ | X <sup>k</sup> | X <sup>k</sup> | Х | $X^k$ | X <sup>k</sup> | X <sup>k</sup> | Х | X <sup>k</sup> | $X^k$ | X <sup>k</sup> | $X^k$ | Х | $X^k$ | Х |
| Inclus | ion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | | | |
| | Signs + body weight<br>ght on Day 1 only) | Х | Х | | Х | Х | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| Physical Examination | | | Х | | | | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| 12- le | 12- lead ECG (triplicate) | | | | | | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| | iver/spleen) | | | | | | | | | | | | | | | | | | | | | XI | | |
| Echoo | cardiography | | | | | | | | | | | | XI | | | | | | | | | X <sup>I</sup> | | |
| | Chemistry Panel | Х | Х | | Х | Х | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | Х | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | Serum Lipid Panel | Х | Х | | Х | Х | Х | Х | | | | Х | Х | | | | Х | | | | Х | Х | | Х |
| رور | Coagulation (aPTT, PT, INR) | PG | | | | Х | | Х | | | | | Х | | | | Х | | | | | Х | | |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| )<br>WE | Sedimentation Rate | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| Dra | Complement (C5a, Bb) | | Х | | | | | Х | | | | | Χ | | | | | | | | | Х | | Х |
| poc | Plasma PK - Volanesorsen | | X <sup>m</sup> | Х | Х | Х | | Х | | | | | Χ | | | | Х | | | | | Х | | Χ |
| В | Anti-Volanesorsen Antibodies | | Х | | Х | Х | | Χ | | | | | Χ | | | | Х | | | | | X | | Х |
| | FSH (women only, if applicable) | | | | | | | | | | | | | | | | | | | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | Х | | | Х | Х | | Χ | | Χ | | | Х | | Х | | Х | | Х | | | X | Х | Х |
| | Archived Serum & Plasma Samples <sup>e</sup> | | Х | | | Χ | | Χ | | | | | Х | | | | | | | | | Х | | Х |

# Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | | Treatment Period Tre | | | | | | | | | | | | Trea | ost<br>tment<br>ow-up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ١٨ | II. | WL | Wk | Mor | nth 3 | Wk | Wk | Wk | Mor | nth 6 | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Мо | nth 12 | Wk | Wk |
| Study Week | -2 to -1 | Wk<br>1 | | Wk Wk<br>4 8 | Wk<br>12 | Wk<br>13 | 16 | | 22 | Wk<br>25 | Wk<br>26 | 29 | 32 | 35 | 38 | 41 | 44 | 47 | Wk<br>51 | Wk 52<br>or ET | | | |
| Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 106 | 127 | 148 | 169 | 176 | 197 | 218 | 239 | 260 | 281 | 302 | 323 | 351 | 358 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | X <sup>n</sup> | | Х | Х | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | XI | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |
| Postheparin Lipoprotein Lipase activity <sup>h</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>i</sup> | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| Diet/Alcohol Counseling <sup>j</sup> | Х | Х | | Х | Х | | Х | | | | | Х | | | | Х | | | | | Х | Х | Х |
| Adverse Events | Х | Χ | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Х |
| Concomitant Medication | Х | Х | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

- Qualification procedures performed (Please refer to Section 4.1)
- Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are unreportable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week and determined not to have met a stopping rule before dosing can continue. Any case of a platelet count ≤ 50,000/mm<sup>3</sup> should be reported in an expedited fashion to the Sponsor
- Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- Females of childbearing potential only
- Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen

# **Appendix A** Schedule of Procedures Continued

#### Legend Text Continued

- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (ISIS 304801-CS16 rollover patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)
- g Genetic testing can be conducted for study qualification (ISIS 304801-CS16 rollover patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h Post-heparin lipoprotein lipase activity can be conducted for study qualification (ISIS 304801-CS16 rollover patients; please refer to Section 6.2.10)
- i In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- j To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- k Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- I A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- m Full or abbreviated PK profile (see Appendix C)
- n Expanded urinalysis (see Appendix B)

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| | Hematology | Uringlysis |
|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Potasium P | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other Assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | Urinalysis Color Appearance Specific gravity pH Protein Blood Ketones Urobilinogen Glucose Bilirubin Leukocyte esterase Nitrate Microscopic examination <sup>2</sup> Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin β2-microglobulin |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

# Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

# PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional

Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td colspan="3">Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN; >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation on anticoagulation | | |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes<br>decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm <sup>3</sup> ;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm <sup>3</sup> ;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated | |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td colspan="4">&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td colspan="4">&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Urine | | | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)




**Sponsor:**Ionis Pharmaceuticals, Inc. 2855 Gazelle Court
Carlsbad, CA 92010

A subsidiary of Isis Pharmaceuticals, Inc.

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

## ISIS 304801-CS7

## The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 2 –22 April 2016

EudraCT No: 2015-003755-21

## ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 2 - 22 April 2016

#### **Protocol History:**

Original Protocol:

28 August 2015

Protocol Amendment 1:

2 February 2016

#### Sponsor:

Ionis Pharmaceuticals, Inc. 2855 Gazelle Court

Carlshad CA 92010

M.D., M.B.A.

## Ionis Protocol Number: ISIS 304801-CS7

**Protocol Amendment 2** 

**EudraCT No: 2015-003755-21** 

Clinical Phase: 3

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

## An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 22 April 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrom (FCS) | | • |
| Amendment: | Amendment 2 | |
| <b>Date:</b> 22 April 2016 | | |
| Open-Label Extension Familial Chylomicro study as described he | on Study of Volanesorsen Admonemia Syndrome (FCS)", date erein. | and the attached clinical protocol, entitled "An inistered Subcutaneously to Patients with d 22 April 2016, and agree to conduct the e on Harmonization Tripartite Guideline on |
| Good Clinical Practic | | e on Harmonization Tripartite Guideline on |
| any purpose other tha | | ontained in this document will not be used for the clinical investigation without the prior |
| Investigator's Signa | ture | |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| | | Page |
|------|---------------------------------------------------|------|
| | OCOL AMENDMENT | |
| | OCOL SYNOPSIS | |
| | Y DESIGN AND TREATMENT SCHEMA | |
| | Y GLOSSARY | |
| | OBJECTIVES | |
| | ACKGROUND AND RATIONALE | |
| 2.1 | Overview of Disease | |
| 2.2 | Therapeutic Rationale | |
| 2.3 | Volanesorsen | |
| 2 | 3.1 Mechanism of Action | 20 |
| 2. | 3.2 Chemistry | |
| 2 | 3.3 Preclinical Experience | 22 |
| 2 | 3.4 Clinical Experience | |
| 2.4 | Rationale for Dose and Schedule of Administration | 24 |
| 3. E | XPERIMENTAL PLAN | 25 |
| 3.1 | Study Design | 25 |
| 3.2 | Number of Study Centers | 25 |
| 3.3 | Number of Patients | 25 |
| 3.4 | Overall Study Duration and Follow-up | 25 |
| 3. | 4.1 Qualification | 25 |
| 3. | 4.2 Treatment | 25 |
| 3. | 4.3 Post-Treatment | 25 |
| 3.5 | End of Study | 25 |
| 3.6 | Data and Safety Monitoring Board | 26 |
| 4. P | ATIENT ENROLLMENT | 26 |
| 4.1 | Qualification | 26 |
| 4.2 | Enrollment | 26 |
| 5. P | ATIENT ELIGIBILITY | 26 |
| 5.1 | Inclusion Criteria | 26 |
| 5.2 | Exclusion Criteria | 27 |
| 6. S | TUDY PROCEDURES | 28 |
| 6.1 | Study Schedule | |
| 6. | 1.1 Qualification | 28 |
| | 1.2 Treatment Period | |
| | 1.3 Pharmacokinetic (PK) Subgroup | |
| _ | 1.4 Post-Treatment Period | |
| 6.2 | Additional Study Assessments | |
| | 2.1 Laboratory Assessments | |

| | 6.2. | Physical Exams and Vital Signs | 29 |
|---|---|---|---|
| | 6 | 2.2.1 Eruptive Xanthoma | |
| | 6 | .2.2.2 Lipemia Retinalis | 29 |
| | 6.2 | 3 Echocardiography | 29 |
| | 6.2. | 4 ECG | 30 |
| | 6.2. | 5 MRI | 30 |
| | 6.2. | 6 Quality of Life Assessments | 30 |
| | 6.2. | 7 Disease Symptom Diary | 30 |
| | 6.2. | 8 Diet Monitoring | 30 |
| | 6.2. | 9 Family History | 30 |
| | 6.2. | 10 Lipoprotein Lipase Activity Sample Collection | 30 |
| | 6.3 | Restriction on the Lifestyle of Patients | 31 |
| | 6.3. | 1 Contraception Requirements | 31 |
| | 6.3. | 2 Other Requirements | 32 |
| <b>7.</b> | ST | UDY DRUG | 32 |
| | 7.1 | Volanesorsen Description | 32 |
| | 7.2 | Packaging and Labeling | 32 |
| | 7.3 | Study Drug Accountability | 32 |
| 8. | TR | EATMENT OF PATIENTS | 33 |
| | 8.1 | Volanesorsen Administration | 33 |
| | 8.2 | Other Protocol-Required Drugs | 33 |
| | 8.3 | Other Protocol-Required Treatment Procedures | 33 |
| | 8.4 | Treatment Precautions | 33 |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | , , | |
| | 8.5. | , | |
| | 8.5. | , | |
| | 8.5. | | |
| | 8.5. | Safety Monitoring for LDL-C Elevations | 35 |
| | 8.5. | | |
| | 8.5. | , | |
| | 8.5. | | |
| | 8.5. | | |
| | 8.6 | Stopping Rules | |
| | 8.6. | 11 8 | |
| | 8.6. | 11 & | |
| | 8.6. | 11 6 | |
| | 8.7 | Adjustment of Dose Frequency | |
| | 8.8 | Discontinuation of Study Treatment | |
| | 8.8. | 1 Follow-up Visits for Early Termination from Treatment Period | 40 |

| | 8.8.2 | 2 Follow-up Visits for Early Termination from Post-Treatment Follow-up P | eriod .41 |
|---|---|---|---|
| | 8.9 | Withdrawal of Patients from the Study | 41 |
| | 8.10 | Concomitant Therapy and Procedures | 41 |
| | 8.10 | | |
| | 8.10 | 0.2 Concomitant Procedures | 42 |
| | 8.11 | Treatment Compliance | 42 |
| 9. | . SEI | RIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 42 |
| | 9.1 | Sponsor Review of Safety Information | 42 |
| | 9.2 | Regulatory Requirements | 42 |
| | 9.3 | Definitions | 43 |
| | 9.3.1 | 1 Adverse Event | 43 |
| | 9.3.2 | 2 Adverse Reaction and Suspected Adverse Reaction | 44 |
| | 9.3.3 | 3 Serious Adverse Event (SAE) | 44 |
| | 9.4 | Monitoring and Recording Adverse Events | 44 |
| | 9.4.1 | 1 Serious Adverse Events | 44 |
| | 9.4.2 | Non-Serious Adverse Events | 45 |
| | 9.4.3 | 3 Evaluation of Adverse Events (Serious and Non-Serious) | 45 |
| | 9. | .4.3.1 Relationship to the Study Drug | 45 |
| | 9. | .4.3.2 Severity | 46 |
| | 9. | .4.3.3 Action Taken with Volanesorsen | 46 |
| | 9. | .4.3.4 Treatment Given for Adverse Event | 46 |
| | 9. | .4.3.5 Outcome of the Adverse Event | 46 |
| | 9.4.4 | 4 Adjudication Committees | 47 |
| | 9.5 | Procedures for Handling Special Situations | 47 |
| | 9.5.1 | 1 Abnormalities of Laboratory Tests | 47 |
| | 9.5.2 | 2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments. | 47 |
| | 9.5.3 | 3 Dosing Errors | 48 |
| | 9.5.4 | | |
| 1 | 0. <b>ST</b> A | ATISTICAL CONSIDERATIONS | 49 |
| | 10.1 | Study Endpoints | 49 |
| | 10.1 | .1 Efficacy Endpoints | 49 |
| | 10.1 | .2 Safety Endpoints | 49 |
| | 10.2 | Sample Size. | 50 |
| | 10.3 | Populations | 50 |
| | 10.4 | Definition of Baseline | 50 |
| | 10.5 | Interim Analysis | 50 |
| | 10.6 | Planned Methods of Analysis | 50 |
| | 10.6 | 5.1 Demographic and Baseline Characteristics | 51 |
| | 10.6 | 5.2 Safety Analysis | 51 |
| | 10.6 | 5.3 Efficacy Analysis | 51 |

| 1515 504001 |
|-------------|
| Protocol |

| 10.6 | 5.4 Pharmacokinetic and Immunogenicity Analysis | 52 |
|---|---|---|
| 10 | 0.6.4.1 Pharmacokinetic Analysis | 52 |
| | 0.6.4.2 Immunogenicity Analysis | |
| 11. INV | VESTIGATOR'S REGULATORY OBLIGATIONS | 53 |
| 11.1 | Informed Consent | |
| 11.2 | Ethical Conduct of the Study | |
| 11.3 | Independent Ethics Committee/Institutional Review Board | |
| 11.4 | Patient Confidentiality | |
| 12. AD | MINISTRATIVE AND LEGAL OBLIGATIONS | 55 |
| 12.1 | Protocol Amendments | 55 |
| 12.2 | Study Termination | |
| 12.3 | Study Documentation and Storage | 55 |
| 12.4 | Study Monitoring | 56 |
| 12.5 | Language | |
| 12.6 | Compensation for Injury | |
| 13. RE | FERENCES | 57 |
| 14. AP | PENDICES | |
| Appen | | |
| Appen | | |
| Appen | · • | |
| Appen | dix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities | 68 |
| | TABLE OF TABLES | |
| | P | age |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | _ |
| Table 2 | Expected Event for the Protocol Defined Population by Preferred Term | , 52 |
| Table 2 | and the Expected Incidence | . 43 |
| | and the Expected metachee | , 15 |
| | TABLE OF FIGURES | |
| | n | 0.050 |
| Figure 1 | | age |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms | . 19 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volanesorsen is shown | 21 |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorsen | |
| 1 15410 3 | rading ringly certaes in radions with reservoir with voidinesorself | . 23 |


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Extension Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 2

**Amendment Date:** 22 April 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 Amendment 1 dated 02 February 2016:

- 1. To modify the clinical experience safety language to reflect updated blinded safety data from ongoing studies.
- 2. To indicate that the DSMB is independent.
- 3. To revise the contraceptive requirements to state that abstinence is only acceptable as true abstinence, i.e., when it is in line with the preferred and usual lifestyle of the patient.
- 4. To add lipoprotein lipase activity as a qualification assessment for ISIS 304801-CS16 rollover patients.
- 5. To add genetic testing as a qualification assessment for ISIS 304801-CS16 rollover patients.
- 6. To increase the frequency of the pregnancy testing.
- 7. To add hematology blood draws at Weeks 12, 16, 22, 25, 29, 35, 41, 47, and 51 to more frequently assess platelet counts.
- 8. To allow blood sampling at Weeks 4, 8, 12, 16, 19, 22, 25, 29, 32, 35, 41, 44, 47, 51, and 58 to be conducted by a home healthcare nurse.
- 9. To allow blood sampling at the 24-hour PK blood draw to be conducted by a home healthcare nurse.
- 10. To add language that each time a hematology lab is drawn and sent to the central laboratory for analysis, an additional sample should be collected in parallel and analyzed locally, to reduce the occurrence of unreportable hematology results.
- 11. To provide guidance that the length of fasting should preferably not be more than 12 hours.

- 12. To update platelet monitoring rule language to allow for more frequent monitoring as determined by the Sponsor Medical Monitor in consultation with the Investigator.
- 13. To add language to the safety monitoring for insulin, oral antidiabetic medication and glucose that all patients, including those not on insulin, who use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.
- 14. To clarify guidance on determining relatedness of a SUSAR.

Protocol

Minor administrative changes or corrections (not included in the list of changes) have been made throughout the protocol in order to improve the overall clarity of the protocol but these changes do not impact the study design.

The following table provides a summary list of changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Section 2.3.4 Clinical Experience | In the completed studies there have been no ISIS 304801 associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with ISIS 304801 administration that recovered in the post-treatment period and was not associated with platelet-related adverse events. In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing. | To modify the clinical experience safety language to reflect updated blinded safety data from ongoing studies |
| Section 3.6 Data and Safety Monitoring Board | Independent added before Data and Safety<br>Monitoring Board (DSMB) | To clarify that the DSMB is independent |
| Protocol Synopsis Study Population Section 5.1 Inclusion Criteria Section 6.3.1 Contraception Requirements | Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception | Per the MHRA's guidance to<br>state that only true<br>abstinence would be<br>acceptable, and that periodic<br>abstinence is not an<br>acceptable method of<br>contraception |
| Section 6.2.10 Lipoprotein<br>Lipase Activity Sample<br>Collection<br>Appendix A Schedule<br>of Procedures | Lipoprotein lipase (LPL) activity will be measured in ISIS 304801-CS16 rollover patients if needed for study qualification. In brief, fasted patients will be given a low intravenous dose of heparin. A blood sample will be drawn prior to and at 10 or 15 minutes after the heparin administration for measurement of LPL activity as per instructions provided to the Investigator. | Lipoprotein lipase activity<br>added as a qualification<br>assessment for<br>ISIS 304801-CS16 rollover<br>patients |
| | Post heparin lipoprotein lipase activity can be conducted for study qualification (ISIS 304801-CS16 rollover patients; please refer to Section 6.2.10) | |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Appendix A Schedule of Procedures | Genetic testing can be conducted for study qualification (ISIS 304801-CS16 rollover patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing | Genetic testing added as a qualification assessment for ISIS 304801-CS16 rollover patients |
| Appendix A Schedule of Procedures | Pregnancy testing was added at Weeks 4, 19, 32, 44, and 58 | To reduce the time period between pregnancy tests |
| Appendix A Schedule of Procedures | Hematology blood draws were added at Weeks 12, 16, 22, 25, 29, 35, 41, 47, and 51 | To implement more frequent evaluation of platelet counts to assess platelet fluctuations during the course of the study and to increase monitoring of platelet counts in patients for safety purposes |
| Section 6.1.2 Treatment<br>Period<br>Appendix A Schedule<br>of Procedures | Blood sampling at Weeks 4, 8, 12, 16, 19, 22, 25, 29, 32, 35, 41, 44, 47, 51, and 58 may be conducted by a home healthcare nurse | To decrease study burden on the patient by removing the requirement for a visit to the clinic or study center for blood draws |
| Section 6.1.3 Pharmacokinetic (PK) Subgroup Appendix A Schedule of Procedures | Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1 | To decrease study burden<br>on the patient by removing<br>the requirement for a visit to<br>the clinic or study center for<br>the 24-hour PK blood draw |
| Appendix A Schedule of Procedures | Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are uninterpretable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week. | To reduce the occurrence of unreportable hematology results (e.g., hemolyzed or clumped blood samples) |
| Section 6.3.2 Treatment<br>Period<br>Appendix A Schedule<br>of Procedures | Wording was added to note that fasting should preferably not be more than 12 hours | To provide guidance on the length of fasting |
| Section 8.5.2<br>Safety Monitoring for<br>Platelet Count Results | Addition to platelet monitoring rules that more frequent testing may also be required | To allow more frequent monitoring of platelets when appropriate |
| Section 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | In addition, patients who are not on insulin (e.g., patients with type 2 diabetes), but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit. | To implement that all patients, including those not on insulin, who use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit |
| Section 9.2 Regulatory<br>Requirements | In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR. | To clarify guidance on determining relatedness of a SUSAR |

## PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Extension Study of Volanesorsen Administered<br>Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center, open-label extension study of ISIS 304801-CS6 and ISIS 304801-CS16. All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13-week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law |
| | 2. Age ≥ 18 years at time of informed consent |
| | 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study |
| | 4. Able and willing to participate in a 65-week study |
| | 5. Satisfy 1 of the following: |
| | a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |

## PROTOCOL SYNOPSIS Continued

| Study Population Continued | Inclusion Criteria: Continued |
|---|---|
| | b. Males: Surgically sterile, abstinent* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |
| | * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception |
| | Exclusion Criteria: |
| | <ol> <li>Have any new condition or worsening of existing condition which in<br/>the opinion of the Investigator would make the patient unsuitable for<br/>enrollment, or could interfere with the patient participating in or<br/>completing the study</li> </ol> |
| | Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6- and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies which included a subset of patients with FCS. This is an extension to the ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Only the subset of patients from ISIS 304801-CS16 with FCS diagnosis may enter the Extension Study. (Please refer to inclusion criteria #3, above) |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A. A 52-week<br/>treatment period during which volanesorsen will be administered as<br/>a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

## PROTOCOL SYNOPSIS Continued

| Safety and Tolerability Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
|---|---|
| Planned Analyses | Safety Endpoints: |
| | <ul> <li>Adverse events including adjudicated events of acute pancreatitis and MACE</li> </ul> |
| | Vital signs and weight |
| | Physical examinations |
| | <ul> <li>Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)</li> </ul> |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | • MRIs |
| | Efficacy Endpoints: |
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during<br/>the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-<br/>density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| | Other symptoms: eruptive xanthoma, lipemia retinalis |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 and ISIS 304801-CS16 index studies. |
| Sponsor | Ionis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



## STUDY GLOSSARY

| Abbreviation/Acronym | Definition |
|---|---|
| ADD ACTORYM ADA | <u>Definition</u> anti-drug antibody |
| | adverse Event |
| ALD | |
| ALT | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OLE Open Label Extension

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, 1 hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

### 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index  $[BMI] = 24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

Amendment 2 22 April 2016

The hybridization (binding) of volunes or to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volanesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

In the completed studies there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin). In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs). In the blinded ongoing clinical trials of ISIS 304801, 2 patients of 142 dosed (as of February 29, 2016) had a decrease in platelet count to less than 50,000/mm³ in the absence of major bleeding or clinically-relevant non-major bleeding and had Study Drug paused as per the monitoring and stopping rules for platelet counts (Section 8.6.3). Platelet counts recovered following suspension of dosing.

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label extension to the Phase 3 study of volanesorsen in patients with FCS (ISIS 304801-CS6 or ISIS 304801-CS16). Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

- A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.
- A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection
- A 13-week post-treatment evaluation period

Please refer to the Schedule of Procedures in Appendix A.

#### 3.4.1 *Qualification*

A period of up to 2 weeks is given to complete qualification assessments outlined in the Schedule of Procedures (Appendix A).

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule or Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

#### 3.5 End of Study

The End-of-Study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

An independent Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 **Qualification**

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open label study are performed. During the qualification period, the eligibility of the patient to continue in the extension study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are

enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least 1 of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoC-II, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of  $\leq 20\%$  of normal
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study.
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy 1 of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent\*, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent\* or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - \* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 5.2 Exclusion Criteria

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 5 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling at Weeks 4, 8, 12, 16, 19, 22, 25, 29, 32, 35, 41, 44, 47, 51, and 58 may be conducted by a home healthcare nurse. Approval for study procedures to be conducted by a home healthcare nurse on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally must be sent to the central laboratory for analysis. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic, or by a home healthcare nurse, on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 2 Study Center visits on Weeks 58 and 65 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study.

A list of these analytes is contained in Appendix B.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug (for ISIS 304801-CS16 rollover patients) and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 1, Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.2.10 Lipoprotein Lipase Activity Sample Collection

Lipoprotein lipase (LPL) activity will be measured in ISIS 304801-CS16 rollover patients if needed for study qualification. In brief, fasted patients will be given a low intravenous dose of heparin. A blood sample will be drawn prior to and at 10 or 15 minutes after the heparin administration for measurement of LPL activity as per instructions provided to the Investigator.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and either be abstinent\* or, if engaged in sexual relations of child-bearing potential, practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet 1 of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

#### For female patients:

• Using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

\* Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours and preferably not more than 12 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

## 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### 8.1 Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL injection once weekly for Weeks 1-52.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be permanently discontinued from further treatment with volanesorsen, evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring for Platelet Count Results

In the event of any significant fall in platelet count, or if the absolute platelet count is 75,000/mm<sup>3</sup> or less, then the patient's platelet counts should be monitored more frequently. The frequency of monitoring and additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically-relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

All patients on insulin will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit. In addition, patients who are not on insulin (e.g., patients with type 2 diabetes), but use a glucometer should also bring their glucometer and/or glucometer log printout to every clinic visit.

• The Investigator or delegate will <u>review the glucometer</u> reading or printout at every clinic visit to evaluate if <u>fasting</u> pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for <u>Hyperglycemia</u> below.

All diabetic patients will note any changes in their <u>insulin dose</u> and /or <u>oral antidiabetic</u> therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - Ocumented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose ≤ 70 mg/dL (≤ 3.9 mmol/L.
  - o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### 8.5.7 Safety Monitoring for Documented Severe Hypoglycemia

A **documented severe hypoglycemic event** is defined as 1 in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level  $\leq 70 \text{ mg/dL}$  ( $\leq 3.9 \text{ mmol/L}$ ). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Coma could occur if blood sugar correction is not performed.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.
#### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within 1 week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control
- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the 3 criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3$  mg/dL (26.5  $\mu$ mol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rules for Platelet Count Results

In the event of a platelet count less than 50,000/mm<sup>3</sup> that is associated with major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of a platelet count less than 50,000/mm³, and in the absence of major bleeding or clinically-relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to ≥ 100,000/mm³. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing re-challenge the platelet count again falls below 50,000/mm<sup>3</sup>, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm<sup>3</sup>. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be re-examined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above.

If after the second re-challenge the platelet count falls below 50,000/mm<sup>3</sup> and is subsequently confirmed (see Section 8.5), dosing with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor.

Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

Definition of Clinically-Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)

- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

#### 8.7 Adjustment of Dose Frequency

Dose adjustments, including dose interruptions, and/or decreasing the dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed for patients that are unable to tolerate the once weekly dose (for example if platelet counts fall below 50,000/mm³ as described in Section 8.6.3). If the patient remains stable after adjustment, they may be cautiously returned to the original once weekly regimen after consultation with the Study Medical Monitor.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be

recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH

E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Independent DSMB will be notified of any SAE as specified in the DSMB charter.

In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an Investigator's decision it is not permissible to downgrade the Investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 2 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An adverse reaction is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee

within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by 1 of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen e.g., confirmation by positive re-challenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by 1 of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by 1 of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by 1 of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### **10.2** Sample Size

No sample size calculations were performed as this is an extension study to the double-blind, placebo-controlled ISIS 304801-CS6 and ISIS 304801-CS16 studies. Approximately 70 patients may be eligible to enroll into this study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least 1 dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least 1 dose of volunesorsen, and have at least 1 evaluable PK sample collected, analyzed, and reported.

#### 10.4 Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient: ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline and the baseline in this open label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.5 Interim Analysis

An interim analysis may be conducted after the last patient's Week 13 visit of the extension study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this OLE study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values

will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

#### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open label extension (OLE) study from the intensive PK subgroup, following a single dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies. On Week 1 Day 1 of the OLE study, patients who received placebo in the index study will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration (C<sub>max</sub>) and the time taken to reach C<sub>max</sub> (T<sub>max</sub>) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration  $(CL_{0-24hr}/F_{0-24hr})$  will be calculated from  $CL_{0-24hr}/F_{0-24hr} = Actual Dose/AUC_{0-24hr}$ . Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev. Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

#### 14. APPENDICES

## **Appendix A** Schedule of Procedures

**Appendix A** Schedule of Procedures

| | Study Period | Qual <sup>a</sup> | | | | | | | | | | Trea | tment | Period | | | | | | | | | Trea | ost<br>atment<br>ow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | v | Vk | 14/14 | Vk Wk | Mor | ith 3 | Wk | Wk Wk | Wk | Month 6 | | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Month 12 | | 2<br>Wk | Wk |
| | Study Week | -2 to -1 | _ | 1 | 4 | 8 | Wk<br>12 | Wk<br>13 | 16 | 19 | 22 | Wk<br>25 | Wk<br>26 | 29 | 32 | 35 | 38 | 41 | 44 | 47 | Wk<br>51 | Wk 52<br>or ET | 58 | |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 106 | 127 | 148 | 169 | 176 | 197 | 218 | 239 | 260 | 281 | 302 | 323 | 351 | 358 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Inform | ned Consent | Χ | | | | | | | | | | | | | | | | | | | | | | |
| Outpa | tient Visit | Х | Х | $X^k$ | $X^k$ | $X^k$ | $X^k$ | Х | $X^k$ | $X^k$ | $X^k$ | X <sup>k</sup> | Х | $X^k$ | $X^k$ | $X^k$ | Х | X <sup>k</sup> | $X^k$ | $X^k$ | $X^k$ | Х | $X^k$ | Х |
| Inclus | ion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | | | | | | | |
| | Signs + body weight<br>ght on Day 1 only) | Х | Х | | х | х | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| Physic | cal Examination | | Х | | | | | Χ | | | | | Х | | | | Х | | | | | Х | | Х |
| 12- le | ad ECG (triplicate) | | | | | | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| MRI ( | iver/spleen) | | | | | | | | | | | | | | | | | | | | | XI | | |
| Echod | cardiography | | | | | | | | | | | | Χ <sup>I</sup> | | | | | | | | | XI | | |
| | Chemistry Panel | Х | Х | | Х | Х | | Х | | Х | | | Х | | Х | | Х | | Х | | | Х | Х | Х |
| | CBC with Differential <sup>b</sup> | Х | Х | | Х | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| | Serum Lipid Panel | Х | Х | | Х | Х | Х | Х | | | | X | Х | | | | Х | | | | Х | Х | | Х |
| ) <sub>c</sub> | Coagulation (aPTT, PT, INR) | | | | | Χ | | Х | | | | | Х | | | | Х | | | | | Х | | |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-lipidated free glycerol | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| × | Sedimentation Rate | | Х | | | | | Х | | | | | Х | | | | | | | | | Χ | | Х |
| Dra | Complement (C5a, Bb) | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| pool | Plasma PK - Volanesorsen | | $\boldsymbol{X}^{m}$ | Х | Х | Х | | Х | | | | | Х | | | | Х | | | | | Х | | Х |
| В | Anti-Volanesorsen Antibodies | | Х | | Х | Х | | Χ | | | | | Х | | | | Х | | | | | Х | | Х |
| | FSH (women only, if applicable) | | | | | | | | | | | | | | | | | | | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | Χ | | | Х | Х | | Χ | | Χ | | | Χ | | Х | | Χ | | Χ | | | Х | Х | Х |
| | Archived Serum & Plasma Samples <sup>e</sup> | | Χ | | | Х | | Х | | | | | Х | | | | | | | | | X | | Х |

Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | | | | | | | | | | | | | Post<br>Treatment<br>Follow-up | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | W | /k | Wk | Wk | | nth 3 | Wk | Wk | Wk | Mor | nth 6 | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Мо | nth 12 | Wk | Wk |
| Study Week | -2 to -1 | , | 1 | 4 | 8 | Wk<br>12 | Wk<br>13 | 16 | 19 | 22 | Wk<br>25 | Wk<br>26 | 29 | | 35 | 38 | 41 | 44 | 47 | Wk<br>51 | Wk 52<br>or ET | | 65 |
| Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 106 | 127 | 148 | 169 | 176 | 197 | 218 | 239 | 260 | 281 | 302 | 323 | 351 | 358 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | X <sup>n</sup> | | Х | Х | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | X <sup>n</sup> | | | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> |
| Fundus Photography <sup>f</sup> | Х | | | | | | | | | | | | | | | | | | | | XI | | |
| Genetic testing for FCS diagnosis (if not available in medical history) <sup>9</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |
| Postheparin Lipoprotein Lipase activity <sup>h</sup> | Х | | | | | | | | | | | | | | | | | | | | | | |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>i</sup> | | Х | | | | | Х | | | | | Х | | | | | | | | | Х | | Х |
| Diet/Alcohol Counseling <sup>j</sup> | Х | Х | | Х | Х | | Х | | | | | Х | | | | Х | | | | | Х | Х | Х |
| Adverse Events | Х | Χ | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х |
| Concomitant Medication | Х | Χ | _ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

- a Qualification procedures performed (Please refer to Section 4.1)
- b Each time a hematology lab is drawn and sent to the central laboratory for analysis an additional sample should be collected in parallel and analyzed locally. In the event that both the central and local sample are uninterpretable (e.g., due to hemolyzed or clumped blood samples) another sample must be repeated within 1-week
- c Blood samples to be collected after an overnight fast of at least 10 hours and preferably not more than 12 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f If possible, fundus photography should be completed prior to administration of the first dose of Study Drug (ISIS 304801-CS16 rollover patients) and repeated at Week 52 (Please refer to Section 6.2.2.2)

#### **Appendix A** Schedule of Procedures Continued

#### Legend Text Continued

- g Genetic testing can be conducted for study qualification (ISIS 304801-CS16 rollover patients); genetic testing will only be conducted if allowed in the geographic region and only after the patient has given specific written informed consent for genetic testing
- h Post-heparin lipoprotein lipase activity can be conducted for study qualification (ISIS 304801-CS16 rollover patients; please refer to Section 6.2.10)
- i In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- j To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- k Assessments and procedures to be conducted by either a home healthcare nurse, or the Study Center as arranged by the Study Center personnel
- I A ± 7-day window is allowed for MRI, echocardiography procedures and fundus photography
- m Full or abbreviated PK profile (see Appendix C)
- n Expanded urinalysis (see Appendix B)

## **Appendix B** List of Laboratory Analytes

#### Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | <u>Coagulation</u> | Hematology | <u>Urinalysis</u> |
|---|---|---|---|
| <ul> <li>Sodium</li> <li>Potassium</li> <li>Chloride</li> <li>Bicarbonate</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>Phosphorus</li> <li>Glucose</li> <li>BUN</li> <li>Creatinine</li> <li>Uric Acid</li> <li>Total bilirubin</li> </ul> | <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | <ul> <li>Red blood cells</li> <li>Hemoglobin</li> <li>Hematocrit</li> <li>MCV, MCH, MCHC</li> <li>Platelets</li> <li>White blood cells</li> <li>WBC Differential (% and absolute)</li> <li>Neutrophils</li> <li>Eosinophils</li> <li>Basophils</li> <li>Lymphocytes</li> <li>Monocytes</li> </ul> Pharmacokinetics¹ | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>2</sup></li> </ul> |
| Direct (conjugated) bilirubin Indirect (unconjugated) bilirubin ALT AST Alkaline phosphatase | | Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol HbA1c, FPG | Additional Measures for Expanded Urinalysis Total protein (quantitative) Microalbumin β2-microglobulin |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

2 Will be performed on abnormal findings unless otherwise specified

### **Appendix C** Pharmacokinetic Sampling Schedule

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

#### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional.

## Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event Mild | | Moderate | Severe |
|---|---|---|---|
| | Hem | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 - 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation | |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm <sup>3</sup> ;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | emistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as define by the manufacturer |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160<br>mg/dL; Fasting glucose value >ULN -<br>8.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated | |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic consequences | - | >ULN - 10 mg/dL (0.59<br>mmol/L) with physiologic<br>consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td colspan="3">&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 -<br/>7.0 mg/dL; &lt;2.0 - 1.75 mmol/L;<br/>lonized calcium &lt;1.0 - 0.9<br/>mmol/L; symptomatic</td><td colspan="3">Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 -<br>7.0 mg/dL; <2.0 - 1.75 mmol/L;<br>lonized calcium <1.0 - 0.9<br>mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | ypoglycemia <lln -="" 55="" <3.0="" <55="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>t</sup></td></lln> | | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>t</sup> |
| Hypokalemia | emia <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" symptomatic="" td=""><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 0.4="" 0.5="" 0.9="" 1.2="" <0.5="" <1.2="" <1.ln="" dl;="" l="" l<="" mg="" mmol="" td=""><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln> | | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td colspan="4">&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Urine | | | |
| Proteinuria | 1 | The second second | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 A subsidiary of Isis Pharmaceuticals, Inc.

Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

#### ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Supplement 1 - UK - 15 April 2016

EudraCT No: 2015-003755-21
## ISIS 304801-CS7

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Supplement 1 - UK - 15 April 2016

#### Sponsor:

Ionis Pharmaceuticals, Inc.
2855 Gazelle Court
Carlshad CA 920

M.D., M.B.A.

## **Protocol Supplement Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | udy of Volanesorsen Administered<br>vith Familial Chylomicronemia Syndrome | |
| Supplement: | 1 - UK | |
| Date: | 15 April 2016 | |
| for the protocol entit. Subcutaneously to Pa 15 April 2016, and a I agree to comply wire Good Clinical Practical Practical Agree to ensure that any purpose other that | led "An Open-Label Extension atients with Familial Chylomic gree to conduct the study as deth the International Conference (E6). The confidential information can the evaluation or conduct of nis Pharmaceuticals, Inc. | nd the attached clinical protocol supplement Study of Volanesorsen Administered ronemia Syndrome (FCS)", dated scribed herein. on Harmonization Tripartite Guideline on ontained in this document will not be used for the clinical investigation without the prior |
| Investigator's Name | (please print) | Date (DD Month YYYY) |

## PROTOCOL SUPPLEMENT - UK

**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Extension Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia Syndrome

(FCS)

**Supplement:** 1 - UK

**Date:** 15 April 2016

The purpose of this supplement (to the global study protocol) is to fulfill MHRA requirements.

The following changes will be made to the protocol:

- 1. To indicate that the DSMB is independent.
- 2. To revise the contraceptive requirements to state that abstinence is only acceptable as true abstinence, i.e., when it is in line with the preferred and usual lifestyle of the patient.
- 3. To increase the frequency of the pregnancy testing.
- 4. To clarify guidance on determining relatedness of a SUSAR.

The following table provides a summary list of the modifications to the protocol.

## LIST OF PROTOCOL MODIFICATIONS

| Section | Modification | Rationale |
|---|---|---|
| Section 3.6 Data and Safety Monitoring Board | Was: The Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP). | To clarify that the<br>DSMB is independent |
| | Is: An independent Data and Safety Monitoring Board (DSMB) will be assembled to review safety, tolerability and efficacy (as needed) data collected on ISIS 304801 during this study. Based on its ongoing assessment of the safety and tolerability of ISIS 304801, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review, meeting schedules and controlled access to unblinded data are outlined in the DSMB Charter and/or the statistical analysis plan (SAP). | |
| Section 5.1<br>Inclusion Criteria<br>Section 6.3.1<br>Contraception<br>Requirements | New: * Abstinence is only acceptable as true abstinence, i.e., when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial and withdrawal are not acceptable methods of contraception | Per the MHRA's guidance to state that only true abstinence would be acceptable, and that periodic abstinence is not an acceptable method of contraception |
| Appendix A<br>Schedule of<br>Procedures | Pregnancy testing added at Weeks 4, 19, 32, 44, and 58 (See Appendix A below) | To reduce the time period between pregnancy tests |
| Section 9.2<br>Regulatory<br>Requirements | Was: The Sponsor or designee will evaluate the available information and decide if there is a reasonable possibility that volanesorsen caused the AE and, therefore, meets the definition of a SUSAR. Is: | To clarify guidance on determining relatedness of a SUSAR |
| | In addition to the Investigator's assessment of relatedness, the Sponsor or designee will evaluate the available information and perform an independent assessment of relatedness. While the Sponsor may upgrade an investigator's decision it is not permissible to downgrade the investigator's opinion for the purposes of determining whether the SAE meets the definition of a SUSAR. | |

## ${\bf Appendix} \; {\bf A} \quad {\bf Schedule} \; {\bf of} \; {\bf Procedures}$

| | Study Period | Qual <sup>a</sup> | Treatment Period F | | | | | | | Post Tre | eatment<br>w-up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| , | | | V | //v | Wk | Wk | Mor | nth 3 | Wk | Mo | nth 6 | Wk | Wk | Wk | Мо | nth 12 | Wk | Wk |
| | Study Week | -2 to -1 | Wk<br>1 | | 4 | 8 | Wk Wk<br>12 13 | | 19 | Wk Wk<br>25 26 | | 32 | 38 | 44 | Wk<br>51 | Wk 52<br>or ET | 58 | 65 |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Inf | ormed Consent | Х | | | | | | | | | | | | | | | | |
| Οι | ıtpatient Visit | Х | Х | Х | Χ | Х | $X^h$ | Х | $X^h$ | $X^h$ | Χ | $X^h$ | Χ | $X^h$ | $X^h$ | Х | $X^h$ | Х |
| Ind | clusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | |
| | al Signs + body weight (+ height on y 1 only) | Х | Х | | Х | Х | | Х | | | Х | | Х | | | Х | | Х |
| Ph | ysical Examination | | Х | | | | | Χ | | | Х | | Х | | | Х | | Х |
| 12 | - lead ECG (triplicate) | | | | | | | Χ | | | Χ | | Х | | | Х | | Х |
| МІ | RI (liver/spleen) | | | | | | | | | | | | | | | X <sup>i</sup> | | |
| Ed | hocardiography | | | | | | | | | | X <sup>i</sup> | | | | | X <sup>i</sup> | X <sup>i</sup> | |
| Fυ | ndus Photography <sup>b</sup> | Х | | | | | | | | | | | | | | X <sup>i</sup> | | |
| | Chemistry Panel | Х | Х | | Х | Х | | Х | X <sup>h</sup> | | Х | $X^h$ | Х | $X^h$ | | Х | X <sup>h</sup> | Х |
| | CBC with Differential | Х | Х | | Х | Х | | Х | $X^h$ | | Х | $X^h$ | Х | X <sup>h</sup> | | Х | X <sup>h</sup> | Х |
| | Serum Lipid Panel | Х | Χ | | Х | Χ | X <sup>h</sup> | Χ | | X <sup>h</sup> | Χ | | Χ | | X <sup>h</sup> | Χ | | Χ |
| رد | Coagulation (aPTT, PT, INR) | | | | | Х | | Χ | | | Χ | | Χ | | | Χ | | |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-<br>lipidated free glycerol | | Х | | | | | х | | | х | | | | | Х | | Х |
| × (F | Sedimentation Rate | | Х | | | | | Χ | | | Χ | | | | | Х | | Х |
| )rav | Complement (C5a, Bb) | | Х | | | | | Χ | | | Χ | | | | | Х | | Х |
| Ĭğ | Plasma PK - Volanesorsen | | X <sup>k</sup> | Х | Х | Х | | Χ | | | Χ | | Х | | | Х | | Х |
| 360 | Anti-Volanesorsen Antibodies | | Х | | Х | Х | | Х | | | Χ | | Χ | | | X | | X |
| ٦ | FSH (women only, if applicable) | | | | | | | | | | | | | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | Х | | | Х | Х | | Х | Х | | Χ | Χ | Χ | Х | | X | Х | X |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | Х | | | Х | | X | | | Х | | | | | Х | | Х |

#### Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | | | | | | Trea | tmen | t Perio | d | | | | | Post Treatment Follow-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 04 1 1144 1 | 0.14 | W | Wk | | Wk | Мо | nth 3 | Wk | Mor | nth 6 | Wk | Wk | Wk | Мо | nth 12 | Wk | Wk |
| Study Week | -2 to -1 | 1 | | 4 | 4 8 | Wk<br>12 | Wk<br>13 | 19 | Wk<br>25 | Wk<br>26 | 32 | | 44 | Wk<br>51 | Wk 52<br>or ET | 58 | 65 |
| Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | $X^{j}$ | | Х | Х | | $X^{j}$ | $X^{j,h}$ | | $X^{j}$ | $X^{j,h}$ | $X^{j}$ | $X^{j,h}$ | | $X^{j}$ | $X^{j,h}$ | $X^{j}$ |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | Х | | | | | Х | | | Х | | | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>f</sup> | | Х | | | | | Х | | | Х | | | | | Х | | Х |
| Diet/Alcohol Counseling <sup>g</sup> | Х | Χ | | Х | Х | | Χ | | | Χ | | Χ | | | Х | Х | Х |
| Adverse Events | Х | Χ | | Х | Х | | Х | | | Х | | Χ | | | Х | | Х |
| Concomitant Medication | Х | Х | | Х | Х | | Х | | | Х | | Х | | | Х | | Х |

- a Qualification procedures performed (Please refer to Section 4.1)
- b If possible, prior to administration of the first dose of Study Drug and repeated at Week 52 (Please refer to Section 6.2.2.2)
- c Blood samples to be collected after an overnight fast of at least 10 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- g To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- h To be collected by either a clinical service, or Study Center as arranged by the Study Center personnel. Approval for study procedures to be conducted by a clinical service on other outpatient visit days will require prior approval by the Sponsor.
- i A ± 7 day window is allowed for MRI, echocardiography procedures and fundus photography
- j Expanded urinalysis (see Appendix B)
- k Full or abbreviated PK profile (see Appendix C)





A subsidiary of Isis Pharmaceuticals, Inc.

Collaborator:
Akcea Therapeutics
55 Cambridge Parkway, Suite 100
Cambridge, MA 02142

**Sponsor:**Ionis Pharmaceuticals, Inc. 2855 Gazelle Court
Carlsbad, CA 92010

### ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 1 –2 February 2016

EudraCT No: 2015-003755-21

#### ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Protocol Amendment 1 – 2 February 2016

#### **Protocol History:**

Original Protocol:

28 August 2015

#### Sponsor:



#### Ionis Protocol Number: ISIS 304801-CS7

#### **Protocol Amendment 1**

EudraCT No: 2015-003755-21

**Clinical Phase: 3** 

## The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

## An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Ionis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010 Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 2 February 2016

#### **Confidentiality Statement**

This document contains confidential information of Ionis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Ionis Pharmaceuticals, Inc.

## **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | | udy of Volanesorsen Administered ith Familial Chylomicronemia Syndrome |
| Amendment: | Amendment 1 | |
| Date: | 2 February 2016 | |
| Open-Label Extension<br>Familial Chylomicro<br>study as described he | on Study of Volanesorsen Admonemia Syndrome (FCS)", dated erein. | and the attached clinical protocol, entitled "An inistered Subcutaneously to Patients with 12 February 2016, and agree to conduct the |
| I agree to comply wi<br>Good Clinical Praction | | on Harmonization Tripartite Guideline on |
| any purpose other tha | | ontained in this document will not be used for<br>the clinical investigation without the prior |
| Investigator's Signa | ture | |
| Investigator's Name | c (please print) | Date (DD Month YYYY) |

## **TABLE OF CONTENTS**

| | | Page |
|------------------|---------------------------------------------------|------|
| PROTO | COL AMENDMENT | 9 |
| <b>PROTO</b> | COL SYNOPSIS | 12 |
| <b>STUDY</b> | DESIGN AND TREATMENT SCHEMA | 15 |
| | GLOSSARY | |
| | BJECTIVES | |
| | ACKGROUND AND RATIONALE | |
| 2.1 | Overview of Disease | |
| 2.2 | Therapeutic Rationale | |
| 2.3 | Volanesorsen | |
| 2.3. | | |
| 2.3. | <b>5</b> | |
| 2.3. | - I | |
| 2.3. | 1 | |
| 2.4 | Rationale for Dose and Schedule of Administration | |
| | XPERIMENTAL PLAN | |
| 3.1 | Study Design. | |
| 3.2 | Number of Study Centers | |
| 3.3 | Number of Patients | |
| 3.4 | Overall Study Duration and Follow-up | |
| 3.4. | | |
| 3.4. | | |
| 3.4. | | |
| 3.5 | End of Study | |
| 3.6 | Data and Safety Monitoring Board | |
| <b>4. PA</b> 4.1 | TIENT ENROLLMENT | |
| 4.1 | Qualification | |
| | TIENT ELIGIBILITY | |
| 5. FA | Inclusion Criteria | |
| 5.2 | Exclusion Criteria | |
| | UDY PROCEDURES | |
| 6.1 | Study Schedule | |
| 6.1. | • | |
| 6.1. | | |
| 6.1. | | |
| 6.1. | | |
| | Additional Study Assessments. | |

| | 6.2. | Laboratory Assessments | 29 |
|---|---|---|---|
| | 6.2.2 | Physical Exams and Vital Signs | 29 |
| | 6. | 2.2.1 Eruptive Xanthoma | 29 |
| | 6. | 2.2.2 Lipemia Retinalis | 29 |
| | 6.2 | B Echocardiography | 29 |
| | 6.2.4 | FCG | 29 |
| | 6.2. | 5 MRI | 29 |
| | 6.2. | Quality of Life Assessments | 30 |
| | 6.2. | 7 Disease Symptom Diary | 30 |
| | 6.2. | B Diet Monitoring | 30 |
| | 6.2.9 | Family History | 30 |
| | 6.3 | Restriction on the Lifestyle of Patients | 30 |
| | 6.3. | Contraception Requirements | 30 |
| | 6.3.2 | 2 Other Requirements | 31 |
| <b>7.</b> | ST | UDY DRUG | 31 |
| | 7.1 | Volanesorsen Description | 31 |
| | 7.2 | Packaging and Labeling | 32 |
| | 7.3 | Study Drug Accountability | 32 |
| 8. | TR | EATMENT OF PATIENTS | 32 |
| | 8.1 | Volanesorsen Administration | 32 |
| | 8.2 | Other Protocol-Required Drugs | |
| | 8.3 | Other Protocol-Required Treatment Procedures | 32 |
| | 8.4 | Treatment Precautions | 33 |
| | 8.5 | Safety Monitoring Rules | |
| | 8.5. | Safety Monitoring Rules for Liver Chemistry Tests | 33 |
| | 8.5.2 | , 5 | |
| | 8.5. | | |
| | 8.5.4 | J 5 1 | |
| | 8.5. | Safety Monitoring for LDL-C Elevations | 35 |
| | 8.5.0 | Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose | 35 |
| | 8.5. | Safety Monitoring Rule for Documented Severe Hypoglycemia | 35 |
| | 8.5. | Safety Monitoring for Hyperglycemia | 36 |
| | 8.5.9 | Acute Pancreatitis | 37 |
| | 8.6 | Stopping Rules | |
| | 8.6. | Stopping Rules for Liver Chemistry Elevations | 37 |
| | 8.6.2 | Stopping Rules for Renal Function Test Results | 38 |
| | 8.6. | | |
| | 8.7 | Adjustment of Dose Frequency | 39 |
| | 8.8 | Discontinuation of Study Treatment | 39 |
| | 8.8. | Follow-up Visits for Early Termination from Treatment Period | 40 |

| | 8.8. | 2 | Follow-up Visits for Early Termination from Post-Treatment Follow-up Pe | riod .40 |
|---|---|---|---|---|
| | 8.9 | Wit | hdrawal of Patients from the Study | 40 |
| | 8.10 | Cor | ncomitant Therapy and Procedures | 41 |
| | 8.10 | ).1 | Concomitant Therapy | 41 |
| | 8.10 | ).2 | Concomitant Procedures | 41 |
| | 8.11 | Tre | atment Compliance | 41 |
| 9. | SE | RIO | US AND NON-SERIOUS ADVERSE EVENT REPORTING | 42 |
| | 9.1 | Spo | nsor Review of Safety Information | 42 |
| | 9.2 | Reg | gulatory Requirements | 42 |
| | 9.3 | Def | initions | 43 |
| | 9.3. | 1 | Adverse Event | 43 |
| | 9.3. | 2 | Adverse Reaction and Suspected Adverse Reaction | 43 |
| | 9.3. | 3 | Serious Adverse Event (SAE) | 43 |
| | 9.4 | Mo | nitoring and Recording Adverse Events | 44 |
| | 9.4. | 1 | Serious Adverse Events | 44 |
| | 9.4. | 2 | Non-Serious Adverse Events | 44 |
| | 9.4. | 3 | Evaluation of Adverse Events (Serious and Non-Serious) | 44 |
| | 9 | .4.3.1 | Relationship to the Study Drug | 44 |
| | 9 | .4.3.2 | 2 Severity | 45 |
| | 9 | .4.3.3 | 3 Action Taken with Volanesorsen | 45 |
| | 9 | .4.3.4 | Treatment Given for Adverse Event | 45 |
| | 9 | .4.3.5 | Outcome of the Adverse Event | 45 |
| | 9.4. | 4 | Adjudication Committees | 46 |
| | 9.5 | Pro | cedures for Handling Special Situations | 46 |
| | 9.5. | 1 | Abnormalities of Laboratory Tests | 46 |
| | 9.5. | 2 | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 47 |
| | 9.5. | 3 | Dosing Errors | 47 |
| | 9.5. | | Contraception and Pregnancy | |
| 1( | 0. ST. | ATIS | STICAL CONSIDERATIONS | 48 |
| | 10.1 | Stu | dy Endpoints | 48 |
| | 10.1 | .1 | Efficacy Endpoints | 48 |
| | 10.1 | .2 | Safety Endpoints | 48 |
| | 10.2 | San | nple Size | 49 |
| | 10.3 | Pop | ulations | 49 |
| | 10.4 | Def | inition of Baseline | 49 |
| | 10.5 | Inte | rim Analysis | 50 |
| | 10.6 | Plan | nned Methods of Analysis | 50 |
| | 10.6 | 5.1 | Demographic and Baseline Characteristics | 50 |
| | 10.6 | 5.2 | Safety Analysis | 50 |
| | 10.6 | . 3 | Efficacy Analysis | 51 |

| 10.6 | 7.4 Pharmacokinetic and Immunogenicity Analysis | 51 |
|---|---|---|
| 10 | 0.6.4.1 Pharmacokinetic Analysis | 51 |
| 10 | 0.6.4.2 Immunogenicity Analysis | 52 |
| 11. INV | VESTIGATOR'S REGULATORY OBLIGATIONS | 52 |
| 11.1 | Informed Consent | 52 |
| 11.2 | Ethical Conduct of the Study | 53 |
| 11.3 | Independent Ethics Committee/Institutional Review Board | 53 |
| 11.4 | Patient Confidentiality | 53 |
| 12. AD | MINISTRATIVE AND LEGAL OBLIGATIONS | 54 |
| 12.1 | Protocol Amendments. | 54 |
| 12.2 | Study Termination | 54 |
| 12.3 | Study Documentation and Storage | 54 |
| 12.4 | Study Monitoring | 55 |
| 12.5 | Language | 56 |
| 12.6 | Compensation for Injury | 56 |
| 13. RE | FERENCES | 57 |
| 14. AP | PENDICES | 59 |
| Appen | dix A Schedule of Procedures | 60 |
| Appen | | |
| Appen | dix C Pharmacokinetic Sampling Schedule | 65 |
| Appen | | malities6/ |
| | TABLE OF TABLES | Родо |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 32 |
| Table 2 | Expected Event for the Protocol Defined Population by Preferred Te | |
| | and the Expected Incidence | 42 |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanism | ns19 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown | |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volanesorse | |

CONFIDENTIAL Amendment 1 2 February 2016


**Protocol Number:** ISIS 304801-CS7

**Protocol Title:** An Open-Label Extension Study of Volanesorsen Administered

Subcutaneously to Patients with Familial Chylomicronemia

Syndrome (FCS)

**Amendment Number:** 1

Protocol

**Amendment Date:** 2 February 2016

The purpose of this protocol amendment is to implement the following modifications to Protocol ISIS 304801-CS7 dated 28 August 2015:

- 1. To update the approximate anticipated number of patients that may enroll into the study (now approximately 70 patients) so that the number of patients is reflective of the estimated number of qualified patients from the ISIS 304801-CS6 and ISIS 304801-CS16 index studies.
- 2. To define the specific patient population from ISIS 304801-CS16 who will be allowed to enter the Open Label Extension Study.
- 3. Clarification of when final assessments from the ISIS 304801-CS6 and ISIS 304801-CS16 index studies may be used for enrollment into ISIS 304801-CS7.
- 4. Clarification of how food and alcohol will be monitored during the study.
- 5. An addition to the platelet monitoring rule language to allow for more frequent monitoring has been included.
- 6. To provide guidance to Investigators with enrolled FCS patients who also have T2DM. Specific glucose monitoring rules are provided for patients on insulin and oral antidiabetic medications. The definition of documented severe hypoglycemia is included and safety monitoring rules have been defined. Also, specific monitoring rules are incorporated into the protocol for hyperglycemic events.

Minor administrative changes or corrections (not included in the list of changes below) have been made throughout the protocol in order to improve the overall clarity of the protocol but these changes do not impact the study design.

The following table provides a summary list of changes to the protocol:

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Synopsis Section 3: Experimental Plan Section 10.2: Sample Size | Up to approximately 50 patients dosed has been changed to up to approximately 70 patients dosed. | Reflective of the updated patient numbers in the ISIS 304801-CS6 study and the addition of ISIS 304801-CS16 patients - with a diagnosis of FCS who will be allowed to enter the Extension Study after successful completion of ISIS 304801-CS16. |
| Synopsis Study Population: Inclusion Criteria #3 Section 5.1: Inclusion Criteria #3 | <ul> <li>3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study: <ul> <li>a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)</li> <li>b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least one (1) of the following: <ul> <li>Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoCII, GPIHBP1, or LMF1)</li> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> </ul> </li> <li>c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study</li> </ul></li></ul> | Inclusion of the specific criteria that must be met in order for patients who successfully complete ISIS 304801-CS16 to enter into the Open Label Extension Study. |
| Section 4.1:<br>Qualification | Eligibility requirements provided for enrollment into the extension study. | Clarification of when final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 study may be used for qualification. |
| Section 6.1.1<br>Qualification<br>Appendix A | Please refer to Section 4.1 and Appendix A. | Deletion of repetitive information in Section 6.1.1 of when final assessments from ISIS 304801-CS6 or ISIS 304801-CS16 can be used for qualification. Qualification assessments explained in Section 4.1 |
| Section 6.1.2<br>Study Procedures | Approval for study procedures to be conducted by a clinical service on other outpatient visit days will require prior approval by the Sponsor. | Blood sampling for lipid panels at Weeks 12, 25, and 51 may be conducted by a clinical service if more convenient for the patient. Patient must get prior approval from the Sponsor for study procedures to be conducted by a clinical service on days not listed above |

| Protocol Section | Description of Change | Rationale |
|---|---|---|
| Section 6.2.2.1<br>Eruptive Xanthoma<br>Section 6.2.2.2<br>Lipemia Retinalis<br>Section 10.1.1<br>Efficacy Endpoints | Inquiries into the number and duration of Eruptive Xanthoma by study staff will occur at each clinic visit. Fundus photography will be performed prior to Day 1 Study Drug administration and at Week 52 | Eruptive Xanthoma and Lipemia<br>Retinalis included as efficacy<br>endpoints to obtain additional clinical<br>endpoint data. |
| Section 6.2.8:<br>Diet Monitoring | Explanation of how food/alcohol will be monitored throughout the course of the study. | Clarification of how and when food/alcohol will be monitored by the patient, dietician or qualified study personnel. |
| Section 8.5.2:<br>Safety Monitoring<br>Rules for Platelet<br>Count Results | Addition to platelet monitoring rules that more frequent testing may be required. | More frequent monitoring of platelets may be warranted if a patient is experiencing a significant decline in platelet count. |
| Section 8.5.6<br>Section 8.5.7<br>Section 8.5.8<br>Glucose Monitoring<br>in T2DM | Addition of monitoring rules for patients with T2DM. Monitoring rules established for patients on insulin and oral antidiabetic medications. Also included are monitoring rules for documented hypoglycemia and hyperglycemia. | Added sections to enhance safety monitoring for 52-week study in diabetic patients with FCS. |
| Appendix A<br>Footnote "j" | A ±7 day window is allowed for MRI and echocardiography | Window expanded from 2 days to 7 days for scheduling flexibility and patient convenience. |

## PROTOCOL SYNOPSIS

| Protocol Title | An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) |
|---|---|
| Study Phase | 3 |
| Indication | Familial Chylomicronemia Syndrome |
| Study Objectives | To evaluate the safety and efficacy of extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS |
| Study Design | This is a multi-center, open-label extension study of ISIS 304801-CS6 and ISIS 304801-CS16. All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13 week post-treatment evaluation period. |
| Number of Patients | Up to approximately 70 patients dosed |
| Study Population | Inclusion Criteria: |
| | <ol> <li>Must give written informed consent to participate in the study (signed and<br/>dated) and any authorizations required by law</li> </ol> |
| | <ol> <li>Age ≥ 18 years at time of informed consent</li> </ol> |
| | 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study: |
| | <ul> <li>a. History of chylomicronemia as evidenced by documentation of<br/>lactescent serum (a creamy top layer after ultracentrifugation of a<br/>fasting blood sample) or documentation of fasting TG measurement</li> <li>≥ 880 mg/dL (10 mmol/L)</li> </ul> |
| | <ul> <li>A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least one (1) of the following:</li> </ul> |
| | <ul> <li>Confirmed homozygote, compound heterozygote or double<br/>heterozygote for known loss-of-function mutations in Type 1-<br/>causing genes (such as LPL, apoCII, GPIHBP1, or LMF1)</li> </ul> |
| | <ul> <li>Post heparin plasma LPL activity of ≤ 20% of normal</li> </ul> |
| | c. Fasting TG ≥ 750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study |
| | 4. Able and willing to participate in a 65-week study |
| | 5. Satisfy one (1) of the following: |
| | a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration |

| Study Population Continued | Inclusion Criteria: Continued |
|---|---|
| | <ul> <li>Males: Surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration</li> </ul> |
| | Exclusion Criteria: |
| | <ul> <li>Have any new condition or worsening of existing condition which in<br/>the opinion of the Investigator would make the patient unsuitable for<br/>enrollment, or could interfere with the patient participating in or<br/>completing the study</li> </ul> |
| | Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) |
| Treatment Group | Volanesorsen 300 mg once per week |
| Study Drug Administration | Volanesorsen will be administered as subcutaneous (SC) injections. |
| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
| Rationale for Dose and Schedule Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index studies (ISIS 304801-CS6- and ISIS 304801-CS16) based on the pharmacodynamic and safety analysis of the Phase 2 studies which included a subset of patients with FCS. This is an extension to the ISIS 304801-CS6 and ISIS 304801-CS16 index studies. Only the subset of patients from ISIS 304801-CS16 with FCS diagnosis may enter the Extension Study. (Please refer to inclusion criteria #3, above) |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor). Please refer to Section 4.1 and Appendix A. A 52-week<br/>treatment period during which volanesorsen will be administered as<br/>a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |

## PROTOCOL SYNOPSIS Continued

| Planned Analyses Safety Endpoints: Adverse events including adjudicated events of acute pancreal MACE Vital signs and weight Physical examinations Clinical laboratory tests (serum chemistry, hematology, coagulurinalysis) Echocardiography | |
|---|---|
| <ul> <li>MACE</li> <li>Vital signs and weight</li> <li>Physical examinations</li> <li>Clinical laboratory tests (serum chemistry, hematology, coaguurinalysis)</li> </ul> | |
| <ul> <li>Physical examinations</li> <li>Clinical laboratory tests (serum chemistry, hematology, coaguurinalysis)</li> </ul> | lation, |
| Clinical laboratory tests (serum chemistry, hematology, coagu urinalysis) | lation, |
| urinalysis) | lation, |
| Echocardiography | |
| Electrocardiograms (ECGs) | |
| Use of concomitant medications | |
| • MRIs | |
| Efficacy Endpoints: | |
| Percent change and absolute change from baseline in fasting | TG |
| Frequency and severity of patient reported abdominal pain du treatment period | ring the |
| Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-high-density lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [approximately lipoprotein-cholesterol (VLDL-C), and LDL-C). | high-<br>ooA-1], |
| Percent change from baseline in fasting total apolipoprotein C (apoC-III) | :-III |
| Quality of Life questionnaires (EQ-5D, SF-36) | |
| Adjudicated acute pancreatitis event rate | |
| Other symptoms: eruptive xanthoma, lipemia retinalis | |
| Pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement volanesorsen as follows: trough levels (pre-dose) throughout treatment post-treatment levels during the post-treatment follow-up period. In of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement volanesorsen in the post-treatment follow-up period. In of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic Evaluations Plasma samples will be taken from all patients for the measurement volanesorsen as follows: trough levels (pre-dose) throughout treatment post-treatment follow-up period. In of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic patients. | ent and<br>a subset<br>cokinetic |
| Statistical Considerations No sample size calculations were performed as this is an extension the double-blind placebo controlled ISIS 304801-CS6 and ISIS 3048 index studies. | |
| Sponsor Ionis Pharmaceuticals, Inc. | |
| Collaborator Akcea Therapeutics | |

#### STUDY DESIGN AND TREATMENT SCHEMA



#### STUDY GLOSSARY

| Abbreviation/Acronym | <u>Definition</u> |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse Event |
| ALP | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Studies | ISIS 304801-CS6 and ISIS 304801-CS16 |

|-----------------|-----------------|
| Protocol | 2 February 2016 |

INR International Normalized Ratio IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically-significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OLE Open Label Extension

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic PK pharmacokinetic **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment-emergent occurring after first dose of Study Drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride WMA World Medical Association

Amendment 1 2 February 2016

#### 1. OBJECTIVES

Protocol

The objective of the study is to evaluate the safety and efficacy of extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/L probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, one (1) hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include:

ISIS 304801-CS7 Amendment 1 Protocol 2 February 2016

apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V (APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009): glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 **Therapeutic Rationale**

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 **ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms** 

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, **CETP** = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

ISIS 304801-CS7 Amendment 1 Protocol 2 February 2016

The hybridization (binding) of volunes or to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

ISIS 304801-CS7

#### 2.3.3 Preclinical Experience

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volanesorsen can be found in the volanesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, 3 patients with FCS were treated with 300 mg/wk volanesorsen in an open label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all 3 patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

In clinical studies conducted to date volunesorsen has been well-tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

To date, there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin) despite many patients in the Phase 2 clinical trials receiving concomitant medications that are known to be associated with elevations in hepatic enzymes, such as fibrates and statins. In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs).

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well-tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label extension to the Phase 3 study of volanesorsen in patients with FCS (ISIS 304801-CS6 or ISIS 304801-CS16). Up to approximately 70 patients will receive 300 mg once weekly volanesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 70 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

- A qualification period of up to 2 weeks (unless approved by the Sponsor). Please refer to Section 4.1 and Appendix A.
- A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection
- A 13-week post-treatment evaluation period

Please refer to the Schedule of Procedures in Appendix A.

#### 3.4.1 Qualification

A period of up to 2 weeks is given to complete qualification assessments outlined in the Schedule of Procedures (Appendix A).

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule or Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of 2 Study Center visits on Weeks 58 and 65.

#### 3.5 End of Study

The end of study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

The Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 **Qualification**

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open label study are performed. During the qualification period, the eligibility of the patient to continue in the extension study will be determined. Final assessments from the ISIS 304801-CS6 or ISIS 304801-CS16 studies may be used for qualification. A period of up to 2 weeks after completion of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the ISIS 304801-CS6 or ISIS 304801-CS16 index studies. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Satisfactory completion of ISIS 304801-CS6 or ISIS 304801-CS16 (index studies) with an acceptable safety profile, per Sponsor and Investigator judgement. Patients who are

enrolled in ISIS 304801-CS16 must also meet the following criteria in order to enter into the Extension Study:

- a. History of chylomicronemia as evidenced by documentation of lactescent serum (a creamy top layer after ultracentrifugation of a fasting blood sample) or documentation of fasting TG measurement ≥ 880 mg/dL (10 mmol/L)
- b. A diagnosis of Familial Chylomicronemia Syndrome (Type 1 Hyperlipoproteinemia) by documentation of at least one (1) of the following:
  - Confirmed homozygote, compound heterozygote or double heterozygote for known loss-of-function mutations in Type 1-causing genes (such as LPL, apoCII, GPIHBP1, or LMF1)
  - Post heparin plasma LPL activity of ≤ 20% of normal
- c. Fasting TG  $\geq$  750 mg/dL (8.4 mmol/L) at Screening for the ISIS 304801-CS16 study.
- 4. Able and willing to participate in a 65-week study
- 5. Satisfy one (1) of the following:
  - a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
  - b. Males: Surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

#### 5.2 Exclusion Criteria

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

Amendment 1 2 February 2016

#### 6.1.1 Qualification

Protocol

Please refer to Section 4.1 and Appendix A.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database locks for the ISIS 304801-CS6 and ISIS 304801-CS16 index studies become available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 10 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs, concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling for lipid panels at Weeks 12, 25, and 51 may be conducted by a clinical service if more convenient for the patient. Approval for study procedures to be conducted by a clinical service on other outpatient visit days will require prior approval by the Sponsor. Patients must be fasted prior to drawing all blood samples and samples drawn locally must be sent to the central laboratory for analysis. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volunesorsen. Patients in this subgroup will have an additional visit to the clinic on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of 2 Study Center visits on Weeks 58 and 65 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study.

A list of these analytes is contained in Appendix B.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.2.1 Eruptive Xanthoma

At each visit, patients will be asked whether they have had any episodes of eruptive xanthoma since their last visit and the number/duration of the events will be recorded. Physical exams should also include skin examination for presence/resolution of eruptive xanthomas. If a patient experiences an episode of eruptive xanthoma during the study, photos of the area should be taken, if possible.

#### 6.2.2.2 Lipemia Retinalis

If possible, lipemia retinalis will be assessed by fundus photography prior to administration of the first dose of Study Drug and repeated at Week 52. Images will be evaluated by an independent assessor, blinded to the patient's treatment assignment.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment-emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 13, Week 26, Week 52, and Week 65.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

The diets of patients enrolled in the study will be monitored as follows:

- 1. All patients will be required to maintain a 7-day food diary prior to Week 1, Week 13, Week 26, Week 52, and Week 65.
- 2. Patients will receive diet/alcohol counseling by qualified study personnel at clinic visits throughout the course of the study. Qualified study personnel will telephone the patient to provide diet/alcohol counseling for visits that are conducted by a clinical service.
- 3. In addition to the 7-day food diary and the diet /alcohol counseling during clinic visits, telephone calls from a dietitian or qualified study personnel to assess as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does <u>not</u> meet one (1) of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy
Amendment 1 2 February 2016 Protocol

For the purposes of the study, effective contraception is defined as follows:

### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/ cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the Study Drug.

### For female patients:

• Using one (1) or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 **Volanesorsen Description**

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at  $2^{\circ}$  to  $8^{\circ}$  C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volunesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### **8.1** Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL injection once weekly for Weeks 1-52.

Patients should receive one (1) dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

Amendment 1 2 February 2016

#### **8.4** Treatment Precautions

Protocol

There are no specific treatment precautions required for this study.

### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from the final visits of ISIS 304801-CS6 and ISIS 304801-CS16 index studies if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be permanently discontinued from further treatment with volanesorsen, evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring Rules for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is  $> 3 \times ULN$  (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

### 8.5.2 Safety Monitoring Rules for Platelet Count Results

If a patient's platelet count falls by 30% or greater from baseline <u>and</u> the absolute platelet count is 75,000/mm<sup>3</sup> or less, then the patient's platelet counts should be monitored more frequently. In the event of any significant fall in platelet count, the frequency of monitoring and additional lab tests will be determined by the Sponsor Medical Monitor or designee in consultation with the Investigator.

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

# 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on 2 consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Safety Monitoring for Insulin, Oral Antidiabetic Medication and Glucose

<u>Patients on insulin</u> will monitor their glucose levels with a glucometer as per standard practice guidelines and bring their glucometer or glucometer log printout to every clinic visit.

The Investigator or delegate will review the glucometer reading or printout at every clinic visit to evaluate if fasting pre-breakfast self-monitored plasma glucose values exceed threshold values as per the Safety Monitoring Rules for Hyperglycemia below.

All diabetic patients will note any changes in their insulin dose and /or oral antidiabetic therapy, as well as any hypoglycemic episode they may experience.

- The Investigator or delegate will ask patients at every clinic visit if they made changes in their insulin dose or oral antidiabetic therapy, and if they experienced a hypoglycemic episode.
  - o Patients will be instructed on the monitoring and management of hypoglycemic episodes at each visit.
  - o Documented symptomatic hypoglycemic episodes should be captured as adverse events in the adverse event CRF. Documented symptomatic hypoglycemia is defined as typical hypoglycemia symptoms accompanied by measured plasma glucose  $\leq$  70 mg/dL ( $\leq$  3.9 mmol/L.
  - o Any changes in insulin dose or oral antidiabetic therapy should be captured into the Concomitant Medication CRF.

#### **8.5.** 7 Safety Monitoring Rule for Documented Severe Hypoglycemia

A documented severe hypoglycemic event is defined as one (1) in which the patient requires assistance of another person to obtain treatment for the event and has a plasma glucose level ≤ 70 mg/dL (≤ 3.9 mmol/L). The rescue treatment of hypoglycemia may include IV glucose or buccal or intramuscular glucagon.

The definition of severe symptomatic hypoglycemia includes all episodes in which neurological impairment was severe enough to prevent self-treatment and which were thus thought to place patients at risk for injury to themselves or others. Note that "requires assistance" means that the patient could not help himself or herself. Someone being kind that assists spontaneously the patient when not necessary does not qualify as "requires assistance."

Severe hypoglycemia will be qualified as a SAE only if it fulfills SAE criteria.

If a patient presents with symptoms of hypoglycemia, the Investigator will need to take immediate action to confirm the patient's glucose level and treat the patient accordingly.

The experience of hypoglycemia may vary greatly from patient to patient. However, there are certain classical signs and symptoms, of which patients should be aware as a clue that their blood glucose may be low. Common symptoms include headache, heart pounding, confusion, disorientation, numbness or tingling, pale skin, shakiness or tremulousness, increased appetite, anxiousness or nervousness, lightheadedness or dizziness, sweating, and weakness. Many of these symptoms are listed in the diary provided to patients. These diaries will be used only to assist the Investigator in assessing the event. Appropriate source documentation should capture the necessary information on the event with the aid of the diaries. Patients must be given adequate instructions on the use of the diaries.

If patients suspect they might be having a hypoglycemia reaction, they should check their blood glucose using their meters as soon as possible, before treatment if possible, provided they feel it is safe to do so. If there is doubt about safety they should treat the event first, using some sugar, milk, or juice for example, then obtain and record a blood glucose value as soon as possible thereafter. The time and nature of treatment should be noted, and especially if any blood glucose result was before or after treatment. It would be helpful for the patient to note if a contributory factor (e.g., missed or reduced meals, unaccustomed physical activity) occurred earlier in the day of the event.

### 8.5.8 Safety Monitoring for Hyperglycemia

Upward dose titration and/or addition of any other anti-hyperglycemic agent(s) will not be allowed during the course of the study, unless specific threshold values are met at Week 13 or later and confirmed on subsequent testing (ideally within one (1) week of the initial test).

HbA1c is monitored every 3 months throughout the study. In addition, patients on insulin should self-monitor their plasma glucose (SMPG) routinely on a glucometer as per practice guidelines. If a <u>fasting</u> pre-breakfast SMPG value exceeds the specific glycemic limit, the patient should check it again on the following 2 days. If all the <u>fasting</u> pre-breakfast values on 3 consecutive days exceed the specific limit, the patient should contact the Investigator and an unscheduled central laboratory FPG measurement and HbA1c should be performed.

The threshold values are defined as:

- FPG > 270 mg/dL (15.0 mmol/L)
- HbA1c > 9% (for patients with baseline HbA1c < 8% and HbA1c increase of more than 1% from baseline (for patients with baseline HbA1c  $\geq$  8 and  $\leq$  9%)

In case of confirmed FPG/HbA1c above the threshold value, the Investigator should ensure that no reasonable explanation exists for insufficient glucose control and in particular that:

- Plasma glucose was actually measured in the fasting condition (i.e., after at least 10 hours fast)
- Absence of intercurrent disease which may jeopardize glycemic control. In case of an emergency (e.g., surgery, infection), the Investigator can take appropriate measures for glycemic control

- Compliance to treatment is appropriate
- Compliance to diet and lifestyle is appropriate

If any of the above can reasonably explain the insufficient glycemic control, the Investigator should consider the following:

- Investigation and treatment of intercurrent disease (to be reported in adverse event (AE)/concomitant medication parts of the e-CRF)
- Stress on the absolute need to be compliant to treatment
- Organize a specific interview with a Registered Dietician or other qualified nutrition professional and stress on the absolute need to be compliant to diet and lifestyle recommendations

A FPG/HbA1c follow-up assessment should be arranged after appropriate action has been taken. If none from the above-mentioned reasons can be found, or if appropriate action fails to decrease FPG/HbA1c under the threshold values, additional medication may be introduced at the Investigator's discretion and according to local guidelines after discussion with the Sponsor Medical Monitor.

#### 8.5.9 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with Study Drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

## 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for any of the three criteria below, dosing of a patient with volunesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$ (26.5  $\mu$ mol/L) and  $\geq$  40% above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24-hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault ≤ 40 mL/min that is confirmed by a 24-hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rule for Platelet Count Results

In the event of a platelet count less than 50,000/mm<sup>3</sup> that is associated with major bleeding or clinically relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of a platelet count less than 50,000/mm<sup>3</sup>, and in the absence of major bleeding or clinically relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to  $\geq 100,000/\text{mm}^3$ . The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing re-challenge the platelet count again falls below 50,000/mm<sup>3</sup>, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm<sup>3</sup>. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be re-examined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above.

If after the second re-challenge the platelet count falls below 50,000/mm<sup>3</sup> and is subsequently confirmed (see Section 8.5), dosing with volunesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor.

Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of 2 or more units of whole or red cells

Definition of Clinically Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

### 8.7 Adjustment of Dose Frequency

Dose adjustments, including dose interruptions, and/or decreasing the dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to 2 adjustments in the treatment schedule may be allowed for patients that are unable to tolerate the once weekly dose (for example if platelet counts fall below 50,000/mm<sup>3</sup> as described in Section 8.6.3). If the patient remains stable after adjustment, they may be cautiously returned to the original once weekly regimen after consultation with the Study Medical Monitor.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

### Amendment 1 2 February 2016

### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

# **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), -glucagon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Data and Safety Monitoring Board (DSMB) will be notified of any SAE as specified in the DSMB charter.

The Sponsor or designee will evaluate the available information and decide if there is a reasonable possibility that volunesorsen caused the AE and, therefore, meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 2 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse

### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

### 9.4.1 Serious Adverse Events

Protocol

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by one (1) of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen e.g., confirmation by positive re-challenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volunesorsen administration

- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)
- **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volanesorsen

#### 9.4.3.2 Severity

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- Mild: The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by one (1) of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by one (1) of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- **Recovered:** Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by one (1) of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

# 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically-significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically-significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically-significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study
- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 **Dosing Errors**

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volanesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

Should an overdose occur, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

Female patients: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

Male patients: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 **Study Endpoints**

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 **Efficacy Endpoints**

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 (apoA-1), VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate
- Other symptoms: eruptive xanthoma, lipemia retinalis

#### Safety Endpoints 10.1.2

• Adverse events including adjudicated events of pancreatitis and MACE

- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

### 10.2 Sample Size

No sample size calculations were performed as this is an extension study to the double-blind, placebo-controlled ISIS 304801-CS6 and ISIS 304801-CS16 studies. Approximately 70 patients may be eligible to enroll into this study.

### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least one (1) dose of volunesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least one (1) dose of volanesorsen, and have at least one (1) evaluable PK sample collected, analyzed, and reported.

#### **10.4** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, 2 baselines are defined for each patient: ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline and the baseline in this open label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the ISIS 304801-CS6 or ISIS 304801-CS16 index studies if used for qualification).

For other measurements, baseline for patients on active treatment in the ISIS 304801-CS6 or ISIS 304801-CS16 index study will be the ISIS 304801-CS6 or ISIS 304801-CS16 index study baseline. For patients on placebo in the ISIS 304801-CS6 or ISIS 304801-CS16 index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

Amendment 1 2 February 2016

#### 10.5 Interim Analysis

Protocol

An interim analysis may be conducted after the last patient's Week 13 visit of the extension study or after the database of the ISIS 304801-CS6 and ISIS 304801-CS16 index studies are locked and unblinded. Both safety and efficacy information from this OLE study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.6 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

## 10.6.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index studies. All patients enrolled will be included in a summary of patient disposition.

### 10.6.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index studies.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index studies. Narratives of treatment-emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment-emergent AEs, all treatment-emergent AEs potentially related to Study Drug, all treatment-emergent serious AEs, and all treatment-emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index studies, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index studies.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index studies.

These safety variables will also be presented as change and percent change from baseline over time after Study Drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index studies.

#### 10.6.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index studies. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index studies for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, quality of life assessments, and comparison of other symptoms including eruptive xanthomas and lipemia retinalis will be summarized by treatment group of the index studies.

Additional details of the analyses to be conducted will be provided in the SAP.

## 10.6.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.6.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801 CS16 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volanesorsen will be carried out on each individual patient data set using data collected in the open label extension (OLE) study from the intensive PK subgroup, following a single dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index studies. On Week 1 Day 1 of the OLE study, patients who received placebo in the index study will receive the first treatment of volanesorsen (single-dose PK), while patients who received volanesorsen in the index studies had been on volanesorsen treatment for 12 months (ISIS 304801-CS6) or 6 months (ISIS 304801-CS16), thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration ( $C_{max}$ ) and the time taken to reach  $C_{max}$  ( $T_{max}$ ) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours ( $AUC_{0-24hr}$ ) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration ( $CL_{0-24hr}$ / $F_{0-24hr}$ ) will be calculated from  $CL_{0-24hr}$ / $F_{0-24hr}$  will be calculated from  $CL_{0-24hr}$ / $F_{0-24hr}$  and  $CL_{0-24hr}$ . Mean

residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where  $AUMC_{0-24hr}$  is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.6.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with Study Drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in study ISIS 304801-CS6 or ISIS 304801-CS16 and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject peak titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16 study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6 and ISIS 304801-CS16. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase 2 and 3 studies and reported separately.

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### **Informed Consent** 11.1

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 **Ethical Conduct of the Study**

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

#### 11.3 **Independent Ethics Committee/Institutional Review Board**

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volunesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 **Patient Confidentiality**

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

• Patient files containing completed CRFs, informed consents, and supporting copies of source documentation

- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, et al. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev. Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, et al. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, et al. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, et al. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase  $C-\alpha$  expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, et al. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, et al. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

# 14. APPENDICES

# **Appendix A** Schedule of Procedures

Appendix A Schedule of Procedures

| | Study Period | Qual <sup>a</sup> | Treatment Period | | | | | | | | | Post Tre | eatment<br>w-up | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | 100 | | Wk | Wk | Month 3 | | Wk | Mo | nth 6 | Wk | Wk | Wk | Month 12 | | Wk | Wk |
| | | -2 to -1 | | Wk Wk<br>1 4 | | 8 | Wk<br>12 | Wk<br>13 | 19 | Wk<br>25 | Wk<br>26 | 32 | 38 | 44 | Wk<br>51 | Wk 52<br>or ET | 58 | 65 |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Inf | ormed Consent | X | | | | | | | | | | | | | | | | |
| Οι | utpatient Visit | Х | Х | Х | Х | Х | $X^h$ | Х | $X^h$ | $X^h$ | Х | $X^h$ | Χ | $X^h$ | $X^h$ | X | $X^h$ | Х |
| Ind | clusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | |
| | tal Signs + body weight (+ height on ay 1 only) | Х | Х | | Х | Х | | Х | | | Х | | Х | | | Х | | Х |
| Pł | nysical Examination | | Х | | | | | Χ | | | Х | | Х | | | Х | | Х |
| 12 | - lead ECG (triplicate) | | | | | | | Χ | | | Х | | Χ | | | Х | | Х |
| М | RI (liver/spleen) | | | | | | | | | | | | | | | X <sup>i</sup> | | |
| Ed | hocardiography | | | | | | | | | | X <sup>i</sup> | | | | | X <sup>i</sup> | | |
| Fι | ındus Photography <sup>b</sup> | Х | | | | | | | | | | | | | | X <sup>i</sup> | | |
| | Chemistry Panel | Х | Х | | Х | Х | | Х | X <sup>h</sup> | | Х | $X^h$ | Χ | $X^h$ | | Х | X <sup>h</sup> | Х |
| | CBC with Differential | Х | Х | | Х | Х | | Х | X <sup>h</sup> | | Х | $X^h$ | Χ | $X^h$ | | Х | X <sup>h</sup> | Х |
| | Serum Lipid Panel | Х | Χ | | Х | Х | X <sup>h</sup> | Х | | X <sup>h</sup> | Х | | Χ | | X <sup>h</sup> | Х | | Х |
| ) <sub>C</sub> | Coagulation (aPTT, PT, INR) | | | | | Χ | | Χ | | | Χ | | Χ | | | Х | | |
| Blood Draw (Fasting) <sup>c</sup> | hsCRP, HbA1c, FPG, and de-<br>lipidated free glycerol | | х | | | | | Х | | | Х | | | | | Х | | Х |
| V (F | Sedimentation Rate | | Χ | | | | | Χ | | | Χ | | | | | Х | | Х |
| )rav | Complement (C5a, Bb) | | Χ | | | | | Х | | | Χ | | | | | X | | X |
| ] pc | Plasma PK - Volanesorsen | | X <sup>k</sup> | Χ | Χ | Χ | | Х | | | Χ | | Χ | | | Х | | Х |
| Bloc | Anti-Volanesorsen Antibodies | | Χ | | Х | Х | | Χ | | | Χ | | Χ | | | Х | | Х |
| ľ | FSH (women only, if applicable) | | | | | | | | | | | | | | | | | |
| | Serum Pregnancy Test <sup>d</sup> | Х | | | | Χ | | Χ | | | Χ | | Χ | | | X | | Х |
| | Archived Serum & Plasma<br>Samples <sup>e</sup> | | х | | | х | | Х | | | Х | | | | | Х | | Х |

Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | Treatment Period | | | | | | | | | | | Post Treatment<br>Follow-up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | -2 to -1 | Wk | | Wk | Wk | | | Wk | | | Wk | Wk | Wk | _ | nth 12 | Wk | Wk |
| | -2 (0 -1 | , | 1 | 4 8 | Wk<br>12 | Wk<br>13 | 19 | Wk Wk<br>25 26 | | 32 | 38 | 44 | Wk<br>51 | Wk 52<br>or ET | 58 | 65 | |
| Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Urinalysis <sup>c</sup> | Х | $X^{j}$ | | Х | Х | | $X^{j}$ | $X^{j,h}$ | | $X^{j}$ | $X^{j,h}$ | $X^{j}$ | $X^{j,h}$ | | X <sup>j</sup> | $X^{j,h}$ | $X^{j}$ |
| Weekly Study Drug: SC Injection | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality of Life Assessment(s) | | Х | | | | | Х | | | Х | | | | | Х | | Х |
| Food/Drink Diary (quarterly) <sup>f</sup> | | Х | | | | | Х | | | Х | | | | | Х | | Х |
| Diet/Alcohol Counseling <sup>9</sup> | Х | Х | | Х | Х | | Χ | | | Х | | Х | | | Х | Х | Х |
| Adverse Events | Х | Χ | | Χ | Х | | Χ | | | Χ | | Х | | | Х | | Х |
| Concomitant Medication | Х | Х | | Χ | Х | | Χ | | | Х | | Χ | | | Х | | Х |

- a Qualification procedures performed (Please refer to Section 4.1)
- b If possible, prior to administration of the first dose of Study Drug and repeated at Week 52 (Please refer to Section 6.2.2.2)
- c Blood samples to be collected after an overnight fast of at least 10 hours. During treatment period urine and blood samples will be collected prior to Study Drug administration. Does not apply to 24-hour PK blood draw
- d Females of childbearing potential only
- e Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- f In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits
- g To reinforce compliance to the diet and alcohol restrictions. Random diet/alcohol assessments (phone visits) will also be performed by dietician or study personnel
- h To be collected by either a clinical service, or Study Center as arranged by the Study Center personnel. Approval for study procedures to be conducted by a clinical service on other outpatient visit days will require prior approval by the Sponsor.
- i A ± 7 day window is allowed for MRI, echocardiography procedures and fundus photography
- j Expanded urinalysis (see Appendix B)
- k Full or abbreviated PK profile (see Appendix C)

# **Appendix B** List of Laboratory Analytes

# Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| Clinical Chemistry Panel | <b>Coagulation</b> | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|---|
| Clinical Chemistry Panel Sodium Potassium Chloride Bicarbonate Total protein Albumin Calcium Magnesium Phosphorus Glucose BUN Creatinine Uric Acid Total bilirubin Indirect (unconjugated) bilirubin | <ul> <li>aPTT (sec)</li> <li>PT (sec)</li> <li>INR</li> </ul> Lipid Panel <ul> <li>Total Cholesterol</li> <li>LDL-C</li> <li>HDL-C</li> <li>Triglycerides</li> <li>Non-HDL-C</li> <li>VLDL-C</li> <li>apoA-1</li> <li>apoB</li> <li>apoC-III</li> </ul> | Hematology Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen | <ul> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>2</sup></li> </ul> Additional Measures for Expanded Urinalysis <ul> <li>Total protein</li> </ul> |
| <ul><li>ALT</li><li>AST</li><li>Alkaline phosphatase</li></ul> | | Other assessments • hsCRP • Sedimentation Rate | <ul><li>(quantitative)</li><li>Microalbumin</li><li>β2-microglobulin</li></ul> |
| | | <ul> <li>C5a, Bb</li> <li>De-lipidated free glycerol</li> <li>HbA1c, FPG</li> </ul> | |

<sup>1</sup> Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

# **Appendix C** Pharmacokinetic Sampling Schedule

# **Appendix C** Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

Amendment 1

2 February 2016

# PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

# PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional.
# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hema | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 – 1,500 cell/mm³ | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or<br>above baseline if baseline is above<br>ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm <sup>3</sup> ;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm³;<br=""><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm³;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm³;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Chemistry | | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T increased | Levels above the upper limit of normal and below the level of myocardial infarction as defined by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm³;<br=""><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160 mg/dL; Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L) without physiologic consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75 mmol/L; lonized calcium &lt;1.0 - 0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 mg/dL; &lt;1.75 mmol/L; lonized calcium &lt;0.9 mmol/L; hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 - 7.0 mg/dL; <2.0 - 1.75 mmol/L; lonized calcium <1.0 - 0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 mg/dL; <1.75 mmol/L; lonized calcium <0.9 mmol/L; hospitalization indicated |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 mg/dL;<br/>&lt;3.0 mmol/L</td><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>‡</sup></td></lln></lln> | <55 mg/dL;<br><3.0 mmol/L | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>‡</sup> |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln></td><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" p="" symptomatic;=""></lln> | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | U | rine | |
| Proteinuria | | | |
| Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | - | Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion,<br>IV medications or<br>hospitalization indicated;<br>elective endoscopic, radiologic<br>or operative intervention<br>indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)





**Sponsor:** 

Isis Pharmaceuticals, Inc. 2855 Gazelle Court Carlsbad, CA 92010

### Collaborator:

Akcea Therapeutics 55 Cambridge Parkway, Suite 100 Cambridge, MA 02142

#### ISIS 304801-CS7

# The APPROACH Open Label Extension Study Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

**Original Protocol – 28 August 2015** 

EudraCT No: 2015-003755-21

#### ISIS 304801-CS7

# The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Original Protocol – 28 August 2015

#### **Sponsor:**

Isis Pharmaceuticals, Inc.
2855 Gazelle Court
Carlsbad, CA 92010

M.D., M.B.A.

#### Isis Protocol Number: ISIS 304801-CS7

**Original Protocol** 

EudraCT No: 2015-003755-21

Clinical Phase: 3

# The APPROACH Open Label Extension Study

Volanesorsen (ISIS 304801)

# An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS)

Trial Sponsor: Isis Pharmaceuticals, Inc.

2855 Gazelle Court Carlsbad, CA 92010

Phone: + 01 760 931 9200

Fax:

Key Sponsor Contact: Ph.D.

2855 Gazelle Court Carlsbad, CA 92010

Phone:

Collaborator: Akcea Therapeutics

55 Cambridge Parkway, Suite 100

Cambridge, MA 02142

Date: 28 August 2015

#### **Confidentiality Statement**

This document contains confidential information of Isis Pharmaceuticals, Inc., that must not be disclosed to anyone other than the recipient study staff and members of the independent ethics committee, institutional review board, or authorized regulatory agencies. This information cannot be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Isis Pharmaceuticals, Inc.

# **Protocol Signature Page**

| Protocol Number: | ISIS 304801-CS7 | |
|---|---|---|
| Protocol Title: | ol Title: An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndron (FCS) | |
| Date: | 28 August 2015 | |
| Open-Label Extension | on Study of Volanesorsen Admonemia Syndrome (FCS)", date | and the attached clinical protocol, entitled "An inistered Subcutaneously to Patients with d 28 August 2015, and agree to conduct the |
| I agree to comply wi<br>Good Clinical Practi | | e on Harmonization Tripartite Guideline on |
| any purpose other that | | contained in this document will not be used for f the clinical investigation without the prior |
| Investigator's Signa | ture | • |
| Investigator's Name | e (please print) | Date (DD Month YYYY) |

# **TABLE OF CONTENTS**

| | | Page |
|-------------|---------------------------------------|------|
| PROT | TOCOL SYNOPSIS | 9 |
| <b>STUD</b> | OY DESIGN AND TREATMENT SCHEMA | 12 |
| <b>STUD</b> | OY GLOSSARY | 13 |
| 1. ( | OBJECTIVES | 15 |
| 2. I | BACKGROUND AND RATIONALE | 15 |
| 2.1 | Overview of Disease | |
| 2.2 | Therapeutic Rationale | 16 |
| 2.3 | Volanesorsen | |
| 2. | .3.1 Mechanism of Action | 17 |
| | .3.2 Chemistry | |
| 2. | .3.3 Preclinical Experience | |
| | .3.4 Clinical Experience | |
| 2.4 | | |
| 3. I | EXPERIMENTAL PLAN | |
| 3.1 | Study Design | |
| 3.2 | Number of Study Centers | |
| 3.3 | Number of Patients | |
| 3.4 | Overall Study Duration and Follow-up | |
| | .4.1 Qualification | |
| | .4.2 Treatment | |
| _ | .4.3 Post-Treatment | |
| 3.5 | End of Study | |
| 3.6 | Data and Safety Monitoring Board | |
| | PATIENT ENROLLMENT | |
| 4.1 | Qualification | |
| 4.2 | Enrollment | |
| | PATIENT ELIGIBILITY | |
| 5.1 | Inclusion Criteria | |
| 5.2 | Exclusion Criteria | |
| | STUDY PROCEDURES | |
| 6.1 | Study Schedule | |
| _ | .1.1 Qualification | |
| | .1.2 Treatment Period | |
| | .1.3 Pharmacokinetic (PK) Subgroup | |
| | .1.4 Post-Treatment Period | |
| 6.2 | · | |
| 6. | 2.1 Laboratory Assessments | 25 |

8.11

| Protocol | | 28 August 2015 |
|---|---|---|
| 6.2. | .2 Physical Exams and Vital Signs | 25 |
| 6.2. | | |
| 6.2 | | |
| 6.2 | .5 MRI | 26 |
| 6.2. | .6 Quality of Life Assessments | 26 |
| 6.2. | .7 Disease Symptom Diary | 26 |
| 6.2. | • • | |
| 6.2. | .9 Family History | 26 |
| 6.3 | Restriction on the Lifestyle of Patients | 26 |
| 6.3 | .1 Contraception Requirements | 26 |
| 6.3 | | |
| 7. ST | TUDY DRUG | 28 |
| 7.1 | Volanesorsen Description | 28 |
| 7.2 | Packaging and Labeling | |
| 7.3 | Study Drug Accountability | 28 |
| 8. TF | REATMENT OF PATIENTS | 28 |
| 8.1 | Volanesorsen Administration | 28 |
| 8.2 | Other Protocol-Required Drugs | 29 |
| 8.3 | Other Protocol-Required Treatment Procedures | |
| 8.4 | Treatment Precautions | 29 |
| 8.5 | Safety Monitoring Rules | 29 |
| 8.5 | .1 Safety Monitoring Rules for Liver Chemistry Tests | 30 |
| 8.5 | .2 Safety Monitoring Rules for Platelet Count Results | 30 |
| 8.5 | .3 Safety Monitoring for Minor Bleeding Events | 30 |
| 8.5 | .4 Safety Monitoring for Constitutional Symptoms | 31 |
| 8.5 | .5 Safety Monitoring for LDL-C Elevations | 31 |
| 8.5 | .6 Acute Pancreatitis | 31 |
| 8.6 | Stopping Rules | 31 |
| 8.6 | .1 Stopping Rules for Liver Chemistry Elevations | 31 |
| 8.6 | .2 Stopping Rules for Renal Function Test Results | 32 |
| 8.6 | .3 Stopping Rule for Platelet Count Results | 32 |
| 8.7 | Adjustment of Dose Frequency | 33 |
| 8.8 | Discontinuation of Study Treatment | 33 |
| 8.8 | .1 Follow-up Visits for Early Termination from Treatment Period | 34 |
| 8.8 | .2 Follow-up Visits for Early Termination from Post-Treatment Follow- | -up Period .34 |
| 8.9 | Withdrawal of Patients from the Study | _ |
| 8.10 | Concomitant Therapy and Procedures | 35 |
| 8.10 | | |

| 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 36 |
|---|---|
| 9.1 Sponsor Review of Safety Information | 36 |
| 9.2 Regulatory Requirements | 36 |
| 9.3 Definitions | 37 |
| 9.3.1 Adverse Event | 37 |
| 9.3.2 Adverse Reaction and Suspected Adverse Reaction | 37 |
| 9.3.3 Serious Adverse Event (SAE) | 37 |
| 9.4 Monitoring and Recording Adverse Events | 38 |
| 9.4.1 Serious Adverse Events | 38 |
| 9.4.2 Non-Serious Adverse Events | 38 |
| 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious) | 38 |
| 9.4.3.1 Relationship to the Study Drug | 38 |
| 9.4.3.2 Severity | 39 |
| 9.4.3.3 Action Taken with Volanesorsen | 39 |
| 9.4.3.4 Treatment Given for Adverse Event | 39 |
| 9.4.3.5 Outcome of the Adverse Event | 39 |
| 9.4.4 Adjudication Committees | 40 |
| 9.5 Procedures for Handling Special Situations | 40 |
| 9.5.1 Abnormalities of Laboratory Tests | 40 |
| 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treats | nents40 |
| 9.5.3 Dosing Errors | 41 |
| 9.5.4 Contraception and Pregnancy | 41 |
| 10. STATISTICAL CONSIDERATIONS | 42 |
| 10.1 Study Endpoints | 42 |
| 10.1.1 Efficacy Endpoints | 42 |
| 10.1.2 Safety Endpoints | 42 |
| 10.2 Sample Size | 43 |
| 10.3 Populations | 43 |
| 10.3 Definition of Baseline | 43 |
| 10.4 Interim Analysis | 43 |
| 10.5 Planned Methods of Analysis | 43 |
| 10.5.1 Demographic and Baseline Characteristics | 44 |
| 10.5.2 Safety Analysis | 44 |
| 10.5.3 Efficacy Analysis | 44 |
| 10.5.4 Pharmacokinetic and Immunogenicity Analysis | 45 |
| 10.5.4.1 Pharmacokinetic Analysis | 45 |
| 10.5.4.2 Immunogenicity Analysis | 45 |
| 11. INVESTIGATOR'S REGULATORY OBLIGATIONS | 46 |
| 11.1 Informed Consent | 46 |
| 11.2 Ethical Conduct of the Study | 46 |

| Protocol | | 28 August 2015 |
|---|---|---|
| 11.3 | Independent Ethics Committee/Institutional Review Board | 47 |
| 11.4 | Patient Confidentiality | |
| | OMINISTRATIVE AND LEGAL OBLIGATIONS | |
| 12.1 | Protocol Amendments | |
| 12.2 | Study Termination | |
| 12.3 | Study Documentation and Storage | 48 |
| 12.4 | Study Monitoring | 48 |
| 12.5 | Language | 49 |
| 12.6 | Compensation for Injury | 49 |
| 13. RF | FERENCES | 50 |
| 14. AF | PENDICES | 52 |
| Apper | ndix A Schedule of Procedures | 53 |
| Apper | ndix B List of Laboratory Analytes | 56 |
| Apper | ndix C Pharmacokinetic Sampling Schedule | |
| Apper | ndix D Grading Scale for Adverse Events Relating to Laboratory A | bnormalities60 |
| | TABLE OF TABLES | |
| | | Page |
| Table 1 | Volanesorsen (ISIS 304801) Characteristics | 28 |
| Table 2 | Expected Event for the Protocol Defined Population by Preferre | |
| | and the Expected Incidence | |
| | TABLE OF FIGURES | |
| | | Page |
| Figure 1 | ApoC-III Regulates Lipoprotein Metabolism by Multiple Mech | anisms16 |
| Figure 2 | Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotide | |
| _ | (MOE-Gapmer). The sequence of volunesorsen is shown | |
| Figure 3 | Fasting Triglycerides in Patients with FCS Treated with Volane | sorsen 20 |

#### **Protocol Title** An Open-Label Extension Study of Volanesorsen Administered Subcutaneously to Patients with Familial Chylomicronemia Syndrome (FCS) **Study Phase** 3 Indication Familial Chylomicronemia Syndrome **Study Objectives** To evaluate the safety and efficacy of extended dosing with volanesorsen (volanesorsen sodium 300 mg) in patients with FCS Study Design This is a multi-center, open-label extension study of ISIS 304801-CS6. All patients will receive volanesorsen 300 mg once per week for 52 weeks. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period. Following the Week 52 visit, patients will enter a 13 week post-treatment evaluation period. **Number of Patients** Up to approximately 50 patients dosed **Study Population** Inclusion Criteria: Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law Age ≥ 18 years at time of informed consent Satisfactory completion of ISIS 304801-CS6 (index study) with an acceptable safety profile, per Sponsor and Investigator judgment Able and willing to participate in a 65-week study 5. Satisfy one of the following: a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years. 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration Males: Surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration **Exclusion Criteria:** Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3) **Treatment Group** Volanesorsen 300 mg once per week Study Drug Administration Volanesorsen will be administered as subcutaneous (SC) injections.

## PROTOCOL SYNOPSIS Continued

| Dose Adjustments | Dose adjustments, including dose interruptions and/or decreasing the dose frequency will be allowed for safety or tolerability after consultation with the Sponsor Medical Monitor. |
|---|---|
| Rationale for Dose and Schedule<br>Selection | The dose of 300 mg once weekly was chosen for the double-blinded placebo-controlled Phase 3 index study (ISIS 304801-CS6) based on the pharmacodynamic and safety analysis of the Phase 2 studies which included a subset of patients with FCS. This is an extension to the ISIS 304801-CS6 study. |
| Study Visit Schedule and Procedures | The study for an individual patient will generally consist of the following periods: |
| | <ul> <li>A qualification period of up to 2 weeks (unless approved by the<br/>Sponsor)</li> </ul> |
| | <ul> <li>A 52-week treatment period during which volanesorsen will be<br/>administered as a once weekly SC injection</li> </ul> |
| | A 13-week post-treatment evaluation period |
| | The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the extension study or until results from the database lock for the index study (ISIS 304801-CS6) becomes available, whichever comes first. |
| | Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), adverse events (AE), concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen magnetic resonance imaging (MRI), ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Dietary counseling will be repeated at intervals throughout the treatment and follow-up period and a daily food/drink diary will be completed for the week prior to each quarterly visit by each patient. Following the Week 52 visit, patients will enter the 13-week post-treatment evaluation period. |
| Safety and Tolerability<br>Evaluations | Overall safety and tolerability of volanesorsen will be assessed by determining the incidence and severity of adverse and serious adverse events (including independently adjudicated events of acute pancreatitis and MACE), withdrawals due to adverse events, and changes in laboratory and other safety parameters. |
| Planned Analyses | Safety Endpoints: |
| | Adverse events including adjudicated events of acute pancreatitis and MACE |
| | Vital signs and weight |
| | Physical examinations |
| | Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis) |
| | Echocardiography |
| | Electrocardiograms (ECGs) |
| | Use of concomitant medications |
| | MRIs |

# PROTOCOL SYNOPSIS Continued

| Planned Analyses Continued | Efficacy Endpoints: |
|---|---|
| | Percent change and absolute change from baseline in fasting TG |
| | <ul> <li>Frequency and severity of patient reported abdominal pain during the treatment period</li> </ul> |
| | <ul> <li>Percent change and change from baseline in other fasting lipid<br/>measurements including total cholesterol, non-high-density<br/>lipoprotein-cholesterol (non-HDL-C), apolipoprotein B [apoB], high-density lipoprotein-cholesterol (HDL-C), apolipoprotein A-1 [apoA-1],<br/>very-low-density lipoprotein-cholesterol (VLDL-C), and LDL-C</li> </ul> |
| | Percent change from baseline in fasting total apolipoprotein C-III (apoC-III) |
| | Quality of Life questionnaires (EQ-5D, SF-36) |
| | Adjudicated acute pancreatitis event rate |
| Pharmacokinetic Evaluations | Plasma samples will be taken from all patients for the measurement of volanesorsen as follows: trough levels (pre-dose) throughout treatment and post-treatment levels during the post-treatment follow-up period. In a subset of patients, more frequent assessment of plasma concentrations of volanesorsen will be performed to determine volanesorsen pharmacokinetic parameters. Plasma sample collection time points are detailed in Appendix A and Appendix C. |
| Statistical Considerations | No sample size calculations were performed as this is an extension study to the double-blind placebo controlled ISIS 304801-CS6 study. |
| Sponsor | Isis Pharmaceuticals, Inc. |
| Collaborator | Akcea Therapeutics |

#### STUDY DESIGN AND TREATMENT SCHEMA



### STUDY GLOSSARY

| Abbreviation/Acronym | Definition |
|---|---|
| ADD ACTORYM ADA | <u>Definition</u> anti-drug antibody |
| ADA<br>AE | adverse Event |
| ALP | |
| | alkaline Phosphatase |
| ALT | alanine Aminotransferase |
| ANA | antinuclear Antibody |
| apoA-1 | apolipoprotein A-1 |
| apoB | apolipoprotein B |
| apoC-III | apolipoprotein C-III |
| apoE | apolipoprotein E |
| aPTT | activated partial thromboplastin time |
| ASO | antisense oligonucleotide |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BMI | body mass index |
| CBC | complete blood count |
| $C_{max}$ | maximum observed drug concentration |
| CRF | case report form |
| DNA | deoxyribonucleic Acid |
| DSMB | Data and Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| ET | early termination |
| FAS | full analysis set |
| FCS | Familial Chylomicronemia Syndrome |
| GCP | Good Clinical Practice |
| GLP-1 | glucagon-like peptide-1 |
| GPIHBP1 | Glycosylphosphatidylinositol-anchored HDL-binding Protein 1 |
| HAPI | Heritability and Phenotype Intervention |
| HbA1c | Glycated Hemoglobin |
| HDL | High-Density Lipoprotein |
| HDL-C | High-Density Lipoprotein-Cholesterol |
| hsCRP | High-sensitivity C-reactive protein |
| ICH | International Conference on Harmonization |
| IDL | Intermediate density lipoprotein |
| IEC | Independent Ethics Committee |
| IM | immunogenicity |
| Index Study | ISIS 304801-CS6 |
| - | |

INR International Normalized Ratio
IRB Institutional Review Board

IXRS Interactive Voice/Web-Response System

LDL Low-Density Lipoprotein

LDL-C Low-Density Lipoprotein-Cholesterol

LMF1 Lipase Maturation Factor 1

LPL Lipoprotein Lipase

MACE Major Acute Cardiovascular Event

MOE 2'-*O*-(2-methoxyethyl)

MRI magnetic resonance imaging mRNA messenger ribonucleic acid NCS not clinically significant

NOAEL No-Observed-Adverse-Effect Level

non-HDL-C Non-High-Density Lipoprotein-Cholesterol

OLE Open Label Extension

OTC over the counter **PFS** prefilled syringe PD pharmacodynamic pharmacokinetic PK **PPS** per protocol set PT prothrombin time **SAE** serious adverse event SAP Statistical Analysis Plan

SC subcutaneous

SUSAR suspected unexpected serious adverse reaction

T2DM type 2 diabetes mellitus

T<sub>max</sub> time to maximal concentration

TG triglycerides

Treatment emergent occurring after first dose of study drug

TRL Triglyceride-Rich Lipoproteins

ULN upper limit of normal

VLDL Very-Low-Density Lipoprotein

VLDL-C Very-Low-Density Lipoprotein-Cholesterol

VLDL-TG Lipoprotein-Triglyceride
WMA World Medical Association

#### 1. OBJECTIVES

The objective of the study is to evaluate the safety and efficacy of extended dosing with volanesorsen in patients with familial chylomicronemia syndrome.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Overview of Disease

Familial Chylomicronemia Syndrome (FCS) is an inherited disease characterized by severe hypertriglyceridemia and chylomicronemia, and risk or history of pancreatitis. It is a rare autosomal recessive disease that can be diagnosed either in childhood or adulthood.

Fasting plasma triglyceride (TG) levels in FCS patients are typically 10-fold to 100-fold above normal (1,500 to 15,000 mg/dL), despite extreme dietary fat restriction (20 g or approximately 15-20% of daily calorie intake) (Brunzell 1999-2011). Patients with FCS often present in infancy or childhood with frequent and severe abdominal pain, repetitive colicky pain, repeated episodes of potentially fatal acute pancreatitis, and failure to thrive (Brunzell 1999-2011; Tremblay et al. 2011). Physical examination frequently reveals eruptive xanthomas, lipemia retinalis and hepatosplenomegaly, and plasma from patients appears lactescent, interfering with determination of other laboratory parameters (Tremblay et al. 2011).

Patients with fasting triglyceride levels > 10 mmol/l probably have a component of chylomicronemia. Clinical diagnosis would include evidence of clinical features of chylomicronemia syndrome and secondary causes such as uncontrolled type 1 or type 2 diabetes mellitus (T2DM), hypothyroidism, poor diet, alcohol use, nephrotic syndrome or use of associated medications should be ruled out. The diagnosis of FCS may be made more specifically by genotyping or confirmation of very low or absent lipoprotein lipase (LPL) enzyme activity in post heparin plasma (Brunzell 1999-2011).

Patients with FCS carry a heavy burden of medical complications, the most serious, as described above, being an extreme risk of recurrent and potentially fatal pancreatitis. Due to the recurrent episodes of acute pancreatitis, these patients may also develop chronic pancreatitis and signs of exocrine or endocrine pancreatic insufficiency, including diabetes mellitus (Gaudet et al. 2013). While the pathophysiology underlying chylomicron-related pancreatitis has not been completely elucidated, one hypothesis is that large chylomicrons lodged in pancreatic capillaries are exposed to pancreatic lipase, with the subsequent release of free fatty acids through the hydrolysis of chylomicron-associated TGs. High concentrations of free fatty acids are thought to damage pancreatic cells leading to emergent pancreatitis (Yang et al. 2009; Berglund et al. 2012).

The etiology of extreme hypertriglyceridemia in FCS is considered to be ineffective triglyceride clearance, due to an extremely low level of LPL activity. LPL normally functions to hydrolyze triglycerides (TG) in chylomicrons along the luminal surface of capillaries, mainly in heart, skeletal muscle, and adipose tissue, promoting triglyceride clearance from the circulation. LPL is regulated by a number of key genes, and loss-of-function mutations in one of these genes, or the LPL gene itself, results in FCS (Surendran et al. 2012). In addition to loss of function mutations, null mutations, and nonsense mutations in the LPL gene, other genes currently identified in FCS patients, and known to directly influence LPL activity include: apolipoprotein C-II (APOC2) a cofactor for LPL (Schuster et al. 2011); apolipoprotein A-V

(APOA5) an enhancer of LPL activity (Schaap et al. 2004); lipase maturation Factor 1 (LMF1), a transmembrane protein involved in LPL maturation (Doolittle et al. 2009); glycosylphosphatidylinositol-anchored HDL-binding protein 1 (GPIHBP1), a capillary endothelial cell protein that provides a platform for LPL-mediated processing of chylomicrons (Beigneux et al. 2007).

#### 2.2 Therapeutic Rationale

Apolipoprotein C-III (ApoC-III), a key regulator of plasma triglyceride levels, is a 79 amino acid glycoprotein synthesized principally in the liver (Ooi et al. 2008; Figure 1). ApoC-III is a major regulator of lipoprotein metabolism and plays a pivotal role in regulating plasma TG levels (Chan et al. 2008). It is a component of triglyceride-rich lipoproteins (TRLs) and a potent inhibitor of LPL (Lemieux et al. 2003). At higher concentrations apoC-III also inhibits hepatic lipase activity (Kinnunen and Ehnolm 1976), an enzyme which plays an important role in the conversion of dense very-low-density lipoprotein (VLDL) to intermediate density lipoprotein (IDL) and to LDL (Mendivil et al. 2010), as well as in the remodeling of HDL (Brown et al. 2010). In addition, increased apoC-III content adversely affects apoE-mediated hepatic uptake of TG-rich remnants (Mann et al. 1997). Thus, elevated plasma apoC-III levels are associated with impaired hydrolysis and retarded clearance of TG-rich particles, resulting in the accumulation of lipoprotein-triglyceride (VLDL-TG) and chylomicrons in plasma and the development of hypertriglyceridemia (Ito et al. 1990).



Figure 1 ApoC-III Regulates Lipoprotein Metabolism by Multiple Mechanisms

From Ooi et al. 2008; ABCA1 = ATP-binding cassette A1, apo = apolipoprotein, CE = cholesterol ester, CETP = cholesterol ester transfer protein, FC = free cholesterol, HDL = high-density lipoprotein, HL = hepatic lipase, IDL = intermediate-density lipoprotein, LCAT = lecithin cholesterol acyltransferase, LDL = low-density lipoprotein, LDLr = LDL receptor, LPL = lipoprotein lipase, LSR = lipolysis-stimulated receptor, SR-B1 = scavenger receptor B-1, TG = triglyceride, VLDL = very low-density lipoprotein.

Mechanistically, FCS is primarily a consequence of ineffective clearance of TRL. ApoC-III is a prominent component of TRL (e.g., VLDL and chylomicrons). In addition to its role in inhibiting LPL, apoC-III inhibits TRL remnant (TG-depleted remnant lipoprotein) uptake by hepatic lipoprotein receptors by steric inhibition of the interaction of apoE with these receptors.

Human genetic data have demonstrated positive phenotypic associations with loss (e.g., null or nonsense mutations) and negative effects with gain of function mutations (Atzmon et al. 2006; Pollin et al. 2008; Petersen et al. 2010). A novel nonsense mutation in the apoC-III gene was identified in the heritability and phenotype intervention (HAPI) heart study in Old Order Amish that results in lower plasma apoC-III and TG levels and lower LDL-C, increased HDL-C and reduced atherosclerosis (Pollin et al. 2008). In another study involving a group of 214 Ashkenazi Jews of advanced age (had passed or nearly reached 100 years of age), genotype analysis revealed a polymorphism in the apoC-III gene (APOC3-641CC genotype) with a clear pattern of age-dependent frequency that was associated with significantly lower levels of apoC-III protein, a favorable lipoprotein profile and increased longevity (Atzmon et al. 2006). In contrast to the Amish and Ashkenazi apoC-III polymorphisms associated with lower plasma TG, apoC-III polymorphisms associated with higher plasma TG have also been recently described (Petersen et al. 2010). In a cohort of lean (mean body mass index [BMI] =  $24.7 \pm 3.6 \text{ kg/m}^2$ ) Asian Indians, carriers of apoC-III variant alleles (C-482T, T-455C, or both) were noted to have significantly higher plasma apoC-III and TG levels, and decreased ability to clear postprandial plasma TG from the circulation. Taken together, the available data strongly support the development of a therapy that reduces plasma apoC-III levels in order to reduce the very high circulating triglyceride and chylomicron levels that are accompanied by increasing risk for acute pancreatitis.

Given the profound reductions in TGs observed with volanesorsen treatment in FCS patients who have no detectable LPL activity (See Section 2.3.4), and the mechanistic data available to date on apoC-III function, potential mechanisms that explain how apoC-III inhibition results in triglyceride reduction in FCS patients include: (1) enhancing the very small residual amounts of LPL activity that these patients may have, below the limit of detection of the assay in many cases (2) potentially enhanced activity of other lipases also involved in the metabolism and breakdown of TGs, such as hepatic lipase or endothelial lipase (Kinnunen and Ehnolm 1976), and (3) apoC-III interaction with Apolipoprotein E (apoE), an important factor in liver reuptake of lipid particles by blocking apoE-mediated uptake of lipid particles in the liver (Breyer et al. 1999), and therefore, reducing apoC-III might enhance apoE-mediated uptake of lipid particles. Volanesorsen-mediated reduction of apoC-III could be contributing to one or all of these mechanisms resulting in the observed potent and sustained reductions in TG.

Through a novel apoC-III lowering mechanism of action, volunesorsen may provide the potential to manage triglyceride levels in FCS patients.

#### 2.3 Volanesorsen

#### 2.3.1 Mechanism of Action

Volanesorsen is a second-generation antisense oligonucleotide (ASO) drug targeted to human apoC-III. It is complementary to a region within the 3' untranslated region of the apoC-III messenger ribonucleic acid (mRNA) and binds to the mRNA by Watson and Crick base pairing.

The hybridization (binding) of volanesorsen to the cognate mRNA, results in the RNase H1-mediated degradation of the apoC-III mRNA, thus preventing production of the apoC-III protein. Maximal antisense-mediated reduction of target mRNA levels is typically greater than 90% of control levels in sensitive tissues (Crooke and Bennett 1996; Zhang et al. 2010). Furthermore, reduction in target mRNA levels using this approach correlates directly with a subsequent reduction in target protein levels.

#### 2.3.2 Chemistry

Chemically, volanesorsen is a synthetic oligomer of 20 nucleotides (i.e., a 20-mer) that are connected sequentially by phosphorothioate linkages. The nucleotide sequence of volunesorsen (Figure 2) is complementary to a 20-nucleotide stretch within the 3' untranslated region of the apoC-III mRNA transcript at base position 489-508. Structurally, the oligonucleotide has 3 regions. Two (2) of them, the 5 nucleotides at the 5' end and the 5 nucleotides at the 3' end, are composed of 2'-O-(2-methoxyethyl) (MOE)-modified ribonucleotides. These MOE-modified nucleotides confer (1) increased affinity to the target mRNA (Altmann et al. 1996; McKay et al. 1999), (2) increased resistance to exonucleases and endonucleases (thereby increasing stability in tissue) (Geary et al. 2003), and (3) amelioration of some of the high dose toxicities thereby resulting in an improved safety profile compared to first generation antisense drugs containing phosphorothioate modified oligodeoxynucleotides (DNA) (Henry et al. 2000). The third region, the central portion of the oligonucleotide, is composed of 10 oligodeoxynucleotides. This chimeric design is called a MOE-Gapmer, and volunesorsen employs this chimeric structure to enable use of the RNase H1-mechanism for antisense activity. This is because while the 2'-MOE modification confers increased stability and affinity, it does not support RNase H1 catalysis of RNA hybridized to 2'-MOE-modified nucleotides (McKay et al. 1999). This is caused by conformational changes induced in the heteroduplex by 2'-alkoxy:RNA hybrids that are not recognized by RNase H1 enzymes (Inoue et al. 1987; Monia et al. 1993). By limiting the 2'-MOE modification to nucleotides flanking the phosphorothioate oligodeoxynucleotide core, the beneficial attributes of the 2'-MOE chemistry are preserved while also retaining RNase H1 recognition.



Figure 2 Design of Chimeric 2'-MOE Phosphorothioate Oligonucleotides (MOE-Gapmer). The sequence of volunesorsen is shown

Original 28 August 2015

#### 2.3.3 Preclinical Experience

Protocol

Inhibition of apoC-III using volanesorsen has been shown to potently reduce hepatic apoC-III mRNA as well as plasma apoC-III protein and TG in a dose- and time-dependent fashion in several species, including human apoC-III transgenic mice, and other rodent and monkey models. Treatment with volanesorsen also resulted in reduced VLDL and chylomicron TG and reduced postprandial TG in hypertriglyceridemic monkeys (Graham et al. 2013).

The pharmacokinetics (PK) and toxicity of volanesorsen have been assessed in mice, rats, and cynomolgus monkeys. General toxicity studies with volanesorsen for up to 39 weeks of treatment followed by up to a 20-week recovery period are complete. The preclinical toxicology program for volanesorsen consists of single dose safety pharmacology studies in the monkey (cardiovascular) and mouse (neurobehavioral and pulmonary assessment studies), *in vitro* and *in vivo* genetic toxicity assessment, repeat dose fertility and/or developmental reproductive toxicology studies in the mouse and rabbit and evaluation in the *in vitro* human Ether-á-go-go-related gene (hERG) assay.

Volanesorsen treatment-related findings in mice and monkeys were generally consistent with those expected for the 2'-MOE-class of ASOs. Treatment-related findings included effects consistent with drug accumulation in tissues in rodents and monkeys, species-dependent proinflammatory response in rodents and monkeys and complement activation and reductions in platelet counts in the monkey. In the mouse and monkey general toxicity studies, reduction of hepatic apoC-III mRNA (> 75%) was not associated with any findings that could be considered related to the pharmacologic inhibition of apoC-III for up to 39 weeks of treatment.

The long-term, chronic toxicology studies in rodents with volanesorsen produced a significant proinflammatory response that led to subsequent effects on the heart at high doses. The rodent species are most sensitive to the proinflammatory effects of antisense molecules. Importantly, these effects on the heart were not observed in the monkey chronic toxicity studies even at the highest doses tested where drug exposure was higher than that in rodents.

Because these changes were not observed in monkeys, the findings in the heart are considered to be rodent-specific and not relevant to humans. Nevertheless, such effects will be monitored by measurement of echocardiograms that will be included in this clinical study.

Volanesorsen caused no untoward effects in safety pharmacology studies (*in vitro* and *in vivo*) and was non-genotoxic (*in vitro* and *in vivo*). Volanesorsen had no effects on fertility or embryo/fetal development in the mouse or rabbit reproductive toxicity studies. In these studies, volanesorsen was detected in placental tissue but not in fetal tissue indicating that little, if any, drug was able to cross the placenta to reach the fetus. Reduction of apoC-III mRNA (64% in males and 47% in females) also did not affect fertility or cause untoward effects on embryo/fetal development in mice.

Detailed information concerning the preclinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure.

#### 2.3.4 Clinical Experience

Detailed information concerning the clinical studies conducted with volunesorsen can be found in the volunesorsen Investigator's Brochure. A summary is included below.

Volanesorsen has been evaluated in one Phase 1 study and two Phase 2 studies, all double blinded and placebo controlled. The total exposures comprise 99 patients and healthy volunteers administered volanesorsen from 50 to 400 mg subcutaneously up to 3 months (compared to 37 administered placebo).

All clinical trials of volanesorsen have shown large and clinically meaningful reductions in fasting plasma apoC-III and TG (~80% and 70%, respectively, mean reduction from baseline with 300 mg dose) with a very high degree of consistency of response between the different patient groups. This includes healthy volunteers, patients with moderate to severe hypertriglyceridemia not on background TG-lowering therapy, patients with moderate to severe hypertriglyceridemia on a background stable fibrate therapy (Gaudet et al. 2015), patients with FCS, and patients with T2DM.

In a Phase 2 study, three patients with FCS were treated with 300 mg/wk volanesorsen in an open label fashion. These patients had a mean baseline fasting TG level of 1,844 mg/dL and all three patients achieved TG levels below or close to 500 mg/dL during the dosing period out to Day 92 (Figure 3). Two (2) of the FCS patients had an absolute reduction in fasting TG in excess of 1,500 mg/dL (Gaudet et al. 2014).



Figure 3 Fasting Triglycerides in Patients with FCS Treated with Volanesorsen

Original

In clinical studies conducted to date volunesorsen has been well tolerated and has shown a favorable safety profile. There has been no clinical or laboratory evidence of drug-drug interactions.

To date, there have been no volanesorsen associated laboratory abnormalities suggestive of an effect on the renal (serum creatinine, proteinuria) or hepatic systems (alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin) despite many patients in the Phase 2 clinical trials receiving concomitant medications that are known to be associated with elevations in hepatic enzymes, such as fibrates and statins. In Phase 2 studies, there was a mild decrease of platelet count associated with volanesorsen administration that recovered in the post-treatment period and was not associated with platelet-related adverse events (AEs).

The most frequently observed AEs with volanesorsen were local reactions at the injection site. Local cutaneous reactions at the injection site defined as those events presenting as either pain, tenderness, erythema, pruritus or swelling occurring on the day of injection and persisting for at least 2 days were infrequent (~15% of injections), were almost always mild, resolved spontaneously, were non-progressive, and were not associated with systemic sequelae.

#### 2.4 Rationale for Dose and Schedule of Administration

The dose and schedule selected for this study is 300 mg per week for 52 weeks. The dose of 300 mg per week is supported by both the cumulative nonclinical data available to date and the Phase 2 clinical data. In nonclinical studies, volanesorsen treatment-related effects in rodents and monkeys were consistent with drug accumulation in tissues and also include species-specific proinflammatory responses. In the monkey, the No-Observed-Adverse-Effect Level (NOAEL) was defined by the cumulative clinical pathology results and histopathology data which provide an adequate clinical margin. No nonclinical findings were considered to be related to the pharmacologic inhibition of apoC-III.

The safety data to date suggest that volanesorsen has been well tolerated at dose levels up to 300 mg in patients with high triglycerides (including type 2 diabetes patients and administration in combination with fibrates and statins) with the most common AEs being local to the injection site and predominantly mild. A pooled analysis of safety for the Phase 2 studies did not demonstrate any clear difference in safety or tolerability between the different doses tested (100 mg, 200 mg, and 300 mg per week for 13 weeks).

Analysis of the cohorts in which volanesorsen was studied at different doses demonstrates dose-dependent pharmacology with respect to pharmacodynamic (PD) effect on the target, apoC-III, with a clear difference in the TG-lowering effect between the different doses in the 100 mg to 300 mg dose range as compared to placebo.

In addition to the nonclinical and clinical experience of volanesorsen, the dose and schedule of administration is supported by the preclinical and clinical safety experience of several other 2'-MOE-modified ASOs that have been safely administered intravenously and subcutaneously in multiple clinical studies at doses up to 1000 mg and for treatment durations that exceed 24 months (Santos et al. 2015).

#### 3. EXPERIMENTAL PLAN

#### 3.1 Study Design

This is an open-label extension to the Phase 3 study of volunesorsen in patients with FCS (ISIS 304801-CS6). Up to approximately 50 patients will receive 300 mg once weekly volunesorsen for 52 weeks.

Following the Week 52 visit, patients enter a 13-week post-treatment evaluation period.

#### 3.2 Number of Study Centers

This study will be conducted at multiple centers worldwide.

#### 3.3 Number of Patients

Up to approximately 50 patients will be dosed.

#### 3.4 Overall Study Duration and Follow-up

The Study will consist of the following periods:

- A qualification period of up to 2 weeks (unless approved by the Sponsor)
- A 52-week treatment period during which volanesorsen will be administered as a once weekly SC injection
- A 13-week post-treatment evaluation period

Please refer to the Schedule of Procedures in Appendix A.

#### 3.4.1 Qualification

A period of up to 2 weeks is given to complete qualification assessments outlined in the Schedule of Procedures (Appendix A).

#### 3.4.2 Treatment

The treatment period is 52 weeks. Eligible patients will report to the Study Center for assessments at specified intervals throughout the 52-week treatment period as detailed in the Schedule or Procedures (Appendix A). During the treatment period, volunesorsen is administered by SC injection once weekly.

#### 3.4.3 Post-Treatment

The post-treatment evaluation period is 13 weeks and consists of two Study Center visits on Weeks 58 and 65.

#### 3.5 End of Study

The end of study is last patient, last visit.

#### 3.6 Data and Safety Monitoring Board

The Data and Safety Monitoring Board (DSMB) will review (as needed) safety, tolerability and efficacy data collected on volanesorsen during this study. Based on its ongoing assessment of

the safety and tolerability of volanesorsen, the DSMB will provide recommendations to the Sponsor for modifying, stopping or continuing the study as planned. Details on the safety assessments, frequency of review and meeting schedules are outlined in the DSMB Charter and/or the statistical analysis plan (SAP).

#### 4. PATIENT ENROLLMENT

#### 4.1 Qualification

Before patients may be enrolled into the study, the Sponsor requires a copy of the Study Center's written independent ethics committee/institutional review board (IEC/IRB) approval of the protocol, informed consent form, and all other patient information.

Final assessments from the index study may be used for qualification as long as they were conducted within 4 weeks of the qualification period. Patients or their legally acceptable representatives must sign the consent form before any study-specific procedures or evaluations related to this open label study are performed. During the qualification period, the eligibility of the patient to continue in the extension study will be determined. A period of up to 2 weeks after completion of the index study (unless approved by the Sponsor) is given to complete qualification. Qualified patients will retain the unique patient identification number that was assigned to them during the index study. The patient identification number will be used to identify the patient throughout the extension trial and must be used on all study documentation related to that patient. The patient identification number must remain constant throughout the extension trial.

#### 4.2 Enrollment

Patients will be enrolled after all qualification assessments have been completed and after the Investigator has verified that they are eligible per criteria in Sections 5.1 and 5.2. No patient may begin treatment prior to enrollment.

Eligible patients will be enrolled using an Interactive Voice/Web-Response System (IXRS).

#### 5. PATIENT ELIGIBILITY

To be eligible to participate in this study candidates must meet the following eligibility criteria within 2 weeks of Study Day 1, or at the time point specified in the individual eligibility criterion listed.

#### 5.1 Inclusion Criteria

- 1. Must give written informed consent to participate in the study (signed and dated) and any authorizations required by law
- 2. Age  $\geq$  18 years at time of informed consent
- 3. Satisfactory completion of ISIS 304801-CS6 (index study) with an acceptable safety profile, per Sponsor and Investigator judgment
- 4. Able and willing to participate in a 65-week study

#### 5. Satisfy one of the following:

- a. Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, patient is using an acceptable contraceptive method (refer to Section 6.3.1) from time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.
- b. Males: Surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, patient is utilizing an acceptable contraceptive method (refer to Section 6.3.1) from the time of signing the informed consent form until 13 weeks after the last dose of Study Drug administration.

#### 5.2 Exclusion Criteria

- 1. Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.
- 2. Unwilling to comply with lifestyle requirements for the duration of the study (Section 6.3).

#### 6. STUDY PROCEDURES

#### 6.1 Study Schedule

All required study procedures are outlined in Appendices A, B, C, and D.

#### 6.1.1 Qualification

Before any study-specific procedures or evaluations are initiated, patients must sign and date the informed consent form. A 2-week period is given after the index study to complete the qualification assessments. The qualification assessments will be performed at Week -2 to -1, ideally after patient eligibility has been determined, and on Study Day 1. Abnormal results may be retested for review by the Study Medical Monitor for eligibility purposes. Final assessments from the index study may be used for qualification as long as they were conducted within 4 weeks of the qualification period.

#### 6.1.2 Treatment Period

The patients, Investigators, study staff, and the Sponsor will remain blinded to lipid data through the last patient's Week 13 visit of the index study or until results from database lock for the index study becomes available, whichever comes first.

During the treatment period, patients will report to the study center for clinic visits a minimum of 10 times during Weeks 1-52 (see Schedule of Procedures in Appendix A). Study Drug will be administered once weekly (Section 8.1). Collection and measurement of vital signs, clinical laboratory parameters (including hematology, serum chemistry, and urinalysis), AEs,

concomitant medication/procedure information, lipid panel, volanesorsen plasma concentrations, immunogenicity (IM) testing, liver/spleen MRI, ECGs, echocardiograms and quality of life assessments will be performed according to the schedule of procedures in Appendix A. Adverse events at the injection site should be collected as adverse events. Dietary counseling will be reinforced at intervals throughout the treatment and follow-up period and all patients will complete a daily food diary for one week prior to their quarterly visit. All blood and urine samples should be collected prior to volanesorsen administration. Blood sampling for lipid panels at Weeks 12, 25 and 51 may be conducted by a home healthcare nurse if more convenient for the patient. Patients must be fasted prior to drawing all blood samples and samples drawn locally must be sent to the central laboratory for analysis. Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit. Dosing instructions and training will be provided to the patient where applicable.

All visits have a visit window of at least  $\pm 2$  days. All reasonable attempts should be made to ensure compliance with the visit schedule as outlined in Appendix A. However, in the event that a visit does not occur or is delayed, all subsequent visits should be calculated based on the time elapsed since Day 1 rather than from the date of the previous visit.

#### 6.1.3 Pharmacokinetic (PK) Subgroup

A subgroup of patients will participate in an extended PK collection. Patients in this subgroup will have more frequent PK sampling over a 24-hour period following the first dose on Study Day 1 in order to evaluate the plasma PK parameters of volanesorsen. Patients in this subgroup will have an additional visit to the clinic on Day 2 to collect a 24-hour post-dose blood draw after dosing on Day 1. The detailed PK sampling schedules are outlined in Appendix C.

Participation in the PK subgroup is optional for sites and patients, and consent may be withdrawn for the subgroup-specific procedures (e.g., multiple blood draws for PK) without being withdrawn from the study. If a patient withdraws consent from the subgroup procedures, he/she should remain on study and continue to follow all the non-subgroup assessments and procedures as outlined in Appendix A.

#### 6.1.4 Post-Treatment Period

After completion of the Week 52 visit assessments, patients will enter the 13-week post-treatment evaluation period. This period consists of two Study Center visits on Weeks 58 and 65 as outlined in the Schedule of Procedures in Appendix A.

#### 6.2 Additional Study Assessments

#### 6.2.1 Laboratory Assessments

Laboratory analyte samples will be collected throughout the study.

A list of these analytes is contained in Appendix B.

#### 6.2.2 Physical Exams and Vital Signs

Physical exams and vital signs will be performed as indicated in the Schedule of Procedures (Appendix A). Vital signs should include weight, blood pressure, pulse rate, respiratory rate and body temperature. Blood pressure and pulse rate will be recorded after the patient has been in a

sitting position for at least 5 minutes. Semi-supine systolic and diastolic blood pressure should always be measured on the same arm (preferentially on the left arm). Height will be measured at the Day 1 visit.

#### 6.2.3 Echocardiography

Echocardiography for assessment of left and right ventricular function and mitral and aortic valve function will be conducted at Week 26 and Week 52 in all patients. For the purpose of assessment of treatment emergent changes, all echocardiograms will be evaluated on an ongoing basis by an independent central reader. Results will be provided to the DSMB for their review.

#### 6.2.4 ECG

The ECG will be recorded after the patient has been resting in a supine position for at least 5 minutes. ECGs will be performed in triplicate at Week 13, Week 26, Week 38, Week 52, and Week 65.

#### 6.2.5 MRI

MRI of the liver and spleen will be conducted at Week 52 for all patients for whom MRI is not contraindicated, e.g., patients having metal implants.

MRIs will be conducted using standardized procedures and settings. MRIs will be read by an independent central reader to assess liver fat and liver and spleen size.

#### 6.2.6 Quality of Life Assessments

All patients will complete Quality of Life Questionnaires (EQ-5D and SF-36) at Week 13, Week 26 and Week 52.

#### 6.2.7 Disease Symptom Diary

All patients will complete a symptom questionnaire once a week starting at the beginning of the qualification period and continuing to the end of the post-treatment follow-up period.

#### 6.2.8 Diet Monitoring

All patients will be required to maintain a 7-day food diary at Week 1, Week 13, Week 26, and Week 52. Inquiries from a dietitian as to how each patient is maintaining their diet will be conducted randomly during the treatment and post treatment follow-up periods. Counseling will also be provided at home visits.

#### 6.2.9 Family History

Family history of hypertriglyceridemia and pancreatitis will be collected for each patient.

#### 6.3 Restriction on the Lifestyle of Patients

#### 6.3.1 Contraception Requirements

All male patients and women of childbearing potential must refrain from sperm/egg donation and practice effective contraception from the time of signing the informed consent form until at least 13 weeks after their last dose of study treatment.

Original

Protocol

Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 13 weeks after the subject's last dose of study treatment.

For the purposes of this Study, women of childbearing potential are defined as any female who has experienced menarche, and who does not meet one of the following conditions:

- Postmenopausal: 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved
- 6 weeks after surgical bilateral oophorectomy with or without hysterectomy
- Post hysterectomy

For the purposes of the study, effective contraception is defined as follows:

#### For male patients:

• Effective male contraception includes a vasectomy with negative semen analysis at follow-up, or the use of condoms together with spermicidal foam/gel/film/cream/suppository. Male patients must also encourage their female partner to use effective contraception from the time of signing the informed consent until 3 months after the patient's last dose of study treatment. Effective contraceptive for the female partner includes: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or barrier methods (female condom\*, diaphragm, sponge, cervical cap) together with spermicidal foam/gel/film/cream/suppository. Male patients with partners that are pregnant must use condoms to ensure that the fetus is not exposed to the study drug.

#### For female patients:

• Using 1 or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, intrauterine contraception/device, or any 2 barrier methods (a combination of male or female condom\* with diaphragm, sponge, or cervical cap) together with spermicidal foam/gel/film/cream/suppository.

\*Note: A female condom and a male condom should not be used together as friction between the two can result in either product failing.

#### 6.3.2 Other Requirements

All patients will be required to fast for at least 10 hours before visits requiring fasted blood sampling.

All patients will be encouraged to follow a diet comprising  $\leq 20$  g fat per day during the study.

Alcohol should not be consumed during the study.

All patients will be given an instruction card that must be presented to the treating physician if a suspected case of pancreatitis occurs. The card will explain that the patient is in a clinical trial and that serum lipase and/or amylase measures should be done in order to adjudicate the event, based on Atlanta Classification (Banks et al. 2013). If serum or amylase activity is less than 3 x upper limit of normal (ULN), imaging, preferably contrast-enhanced computed tomography, should be considered to confirm the diagnosis of acute pancreatitis per the Atlanta Criteria.

#### 7. STUDY DRUG

#### 7.1 Volanesorsen Description

Volanesorsen drug product (ISIS 304801) characteristics are listed in Table 1.

Volanesorsen (ISIS 304801) is contained in glass prefilled syringes (PFS). Volanesorsen and its storage and preparation instructions will be provided by the Sponsor or designee. Volanesorsen must be stored securely at 2° to 8° C and be protected from light.

Table 1 Volanesorsen (ISIS 304801) Characteristics

| Strength | 200 mg/mL |
|-------------------------|-------------------------|
| Volume/Formulation | 1.5 mL solution per PFS |
| Dose | 300 mg once weekly |
| Route of Administration | SC |

#### 7.2 Packaging and Labeling

The Sponsor will provide the Investigator with packaged volanesorsen labeled (ISIS 304801) in accordance with specific country regulatory requirements.

#### 7.3 Study Drug Accountability

The study staff is required to document the receipt, dispensing, and return/destruction of volanesorsen provided by the Sponsor. The Study Center must return all unused volanesorsen to the Sponsor or designee. All used syringes must be disposed of as per the site's hazardous waste destruction policy.

#### 8. TREATMENT OF PATIENTS

#### **8.1** Volanesorsen Administration

For each individual patient, volanesorsen will be administered subcutaneously as a single 1.5 mL injection once weekly for Weeks 1-52.

Patients should receive 1 dose per week, with weeks always defined relative to Study Day 1. For example if a patient receives the first dose on a Monday, subsequent doses should be given on Mondays, if possible. If a patient misses an injection, or if dosing on the usual day is not

possible, the patient can reschedule the injection provided that 2 doses are administered at least 2 days apart.

Every effort should be made to ensure the previous week's dose is given 7 days prior to a scheduled clinic visit.

Please refer to the Study Drug Manual provided by the Sponsor for more detailed instructions for volanesorsen preparation and administration.

#### 8.2 Other Protocol-Required Drugs

There are no other protocol-required drugs (Section 6.2.5).

#### 8.3 Other Protocol-Required Treatment Procedures

There are no other protocol required treatment procedures for this study.

#### **8.4** Treatment Precautions

There are no specific treatment precautions required for this study.

#### 8.5 Safety Monitoring Rules

Please refer also to the 'Guidance for Investigator' section of the Investigator's Brochure.

For the purposes of safety monitoring baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the index study if used for qualification).

In addition to the standard monitoring of clinical safety parameters, the following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study (Treatment or Post-Treatment Periods), the initial clinical laboratory results meeting the safety monitoring or stopping criteria presented below **must be confirmed** by performing measurements (ideally in the same laboratory that performed the initial measurement) on new specimens. All new specimen collections should take place as soon as possible (ideally within 3 days of the initial collection). For stopping rules, if the initial laboratory result is observed during the Treatment Period, the results from the retest **must be available** prior to administering the next dose of volanesorsen.

In addition to the safety monitoring parameters listed below, the Sponsor may request confirmation of additional lab values.

Re-dosing Guidance: Patients with initial laboratory test values that reach a stopping rule must not be re-dosed until the re-test results are available. In general, patients who do not meet the stopping rules based upon retest may continue dosing. However, the Investigator and the Sponsor Medical Monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the patient is appropriate. If any of the stopping criteria described below (refer to Sections 8.6.1 to 8.6.3) are met, the patient will be permanently discontinued from further treatment with volanesorsen, evaluated fully as outlined below and in consultation with the Sponsor Medical Monitor or appropriately qualified designee, and will be followed up in accordance with Section 8.8 of the protocol.

#### 8.5.1 Safety Monitoring Rules for Liver Chemistry Tests

The following rules are adapted from the draft guidance for industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation," issued by the U.S. Department of Health and Human Services, Food and Drug Administration, July 2009. For a definition of Baseline please refer to guidance in Section 8.5 above.

In the event of an ALT or AST measurement that is > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) at any time during the study (Treatment or Post-Treatment Period), the initial measurement(s) should be confirmed as described above. Additional confirmatory measurements should also be performed if ALT or AST levels increase to 5 x ULN.

<u>Frequency of Repeat Measurements</u>: Patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN) should have their liver chemistry tests (ALT, AST, alkaline phosphatase (ALP), international normalized ratio (INR) and total bilirubin) retested at least once-weekly until ALT and AST levels become  $\le 1.2$  x ULN or 1.2 x baseline value if the baseline value was > ULN.

<u>Further Investigation into Liver Chemistry Elevations</u>: For patients with confirmed ALT or AST levels > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), the following evaluations should be performed:

- 1. Obtain a more detailed history of symptoms and prior and concurrent diseases
- 2. Obtain further history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- 3. Obtain a history for exposure to environmental chemical agents and travel
- 4. Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel)
- 5. Serology for autoimmune hepatitis (e.g., antinuclear antibody [ANA])

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the Investigator, in consultation with the Sponsor Medical Monitor. Repetition of the above evaluations should be considered if a patient's ALT and/or AST levels reach 5 x ULN.

#### 8.5.2 Safety Monitoring Rules for Platelet Count Results

If a patient's platelet count falls by 30% or greater from baseline <u>and</u> the absolute platelet count is 75,000/mm<sup>3</sup> or less, then the patient's platelet counts should be monitored more frequently. The frequency of monitoring and additional lab tests will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.5.3 Safety Monitoring for Minor Bleeding Events

Minor bleeding events are those that do not fulfill the criteria for major bleeding or clinically relevant, non-major bleeding events (which are defined in Section 8.6.3), for example excess

bruising, petechiae, gingival bleeding on brushing teeth. If a minor bleeding event occurs, the Investigator must notify the Sponsor Medical Monitor and additional testing of coagulation parameters activated partial thromboplastin time (aPTT), prothrombin time (PT), INR and platelet count should be performed.

#### 8.5.4 Safety Monitoring for Constitutional Symptoms

Patients will be instructed to promptly report any signs of symptoms of fever or constitutional symptoms that may arise during the study and the Investigator should closely evaluate all potential causes, including concomitant illness. Patients that experience persistent constitutional symptoms should be discussed with the Sponsor Medical Monitor or designee to determine whether additional monitoring or laboratory tests are required.

#### 8.5.5 Safety Monitoring for LDL-C Elevations

Beginning at Week 13, laboratory alerts will be in place to notify the Investigator if a patient has a low-density lipoprotein-cholesterol (LDL-C) > 160 mg/dL (> 130 mg/dL for patients with T2DM) on two consecutive visits. If this occurs, LDL-C values for this patient will be unblinded for the remainder of the study and the Investigator will be encouraged to initiate/adjust treatment to lower LDL-C according to country-specific guidelines (e.g., initiate statin therapy or increase the statin dose for patients who are already on treatment).

#### 8.5.6 Acute Pancreatitis

If a patient has an episode of acute pancreatitis, dosing with study drug should be suspended temporarily until the patient is clinically stable. The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor.

#### 8.6 Stopping Rules

For the purposes of stopping rules baseline is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1.

#### 8.6.1 Stopping Rules for Liver Chemistry Elevations

In the event of laboratory results meeting the following criteria, and the event is without an alternative explanation as discussed with the Sponsor Medical Monitor, dosing of a patient with volunesorsen will be stopped permanently; values that are not confirmed due to failure to retest or missing lab values will be presumed confirmed:

- 1. ALT or AST > 8 x ULN, which is confirmed
- 2. ALT or AST > 5 x ULN, which is confirmed and persists for  $\geq$  2 weeks
- 3. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed **and** total bilirubin > 2 x ULN or INR > 1.5
- 4. ALT or AST > 3 x ULN (or the greater of 2 x baseline value or 3 x ULN if the baseline value was > ULN), which is confirmed, and the new appearance (i.e., onset coincides with the changes in hepatic enzymes) of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (> ULN) felt by the Investigator to be potentially related to hepatic inflammation

Protocol

28 August 2015

Original

#### 8.6.2 Stopping Rules for Renal Function Test Results

In the event of a persistent elevation that is observed over 2 consecutive weeks, for <u>any</u> of the three criteria below, dosing of a patient with volanesorsen may be stopped temporarily:

- 1. Serum creatinine increase that fulfill all of the following criteria:  $\geq 0.3 \text{ mg/dL}$  (26.5 µmol/L) and  $\geq 40\%$  above baseline creatinine values and > ULN
- 2. Proteinuria, dipstick 2 + (confirmed by dipstick retest and then further confirmed by a quantitative total urine protein measurement of > 1.0 g/24 hour)
- 3. Estimated creatinine clearance calculated according to the formula of Cockcroft and Gault < 40 mL/min that is confirmed by a 24 hour urine collection

The possible dosing re-initiation or follow-up schedule for any events meeting either of these criteria will be determined by the Investigator in consultation with the Sponsor Medical Monitor or designee.

#### 8.6.3 Stopping Rule for Platelet Count Results

In the event of a platelet count less than 50,000/mm<sup>3</sup> that is associated with major bleeding or clinically relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volunesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Sponsor Medical Monitor.

In the event of a platelet count less than  $50,000/\text{mm}^3$ , and in the absence of major bleeding or clinically relevant non-major bleeding (defined below; Schulman et al. 2005), dosing of a patient with volanesorsen should be suspended temporarily until the platelet count has recovered to  $\geq 100,000/\text{mm}^3$ . The suitability of the patient for continued dosing and the need for any modification to treatment schedule (refer to Section 8.7) will be determined by the Investigator in consultation with the Study Medical Monitor and will be based on factors such as the original rate of decline in the patient's platelet count, whether any bleeding events were experienced by the patient, and the speed of recovery of platelet count upon holding of dosing.

If after the first dosing re-challenge the platelet count again falls below 50,000/mm<sup>3</sup>, then dosing of the patient must be held until the platelet count again returns to at least 100,000/mm<sup>3</sup>. The suitability of the patient for continued dosing and the need for any further modification to treatment schedule or dose (refer to Section 8.7) will be re-examined by the Investigator in consultation with the Study Medical Monitor based on (at least) the factors mentioned above.

If after the second re-challenge the platelet count falls below 50,000/mm<sup>3</sup> and is subsequently confirmed (see Section 8.5), dosing with volunesorsen will be stopped permanently. The follow-up schedule for any events meeting this stopping criterion will be determined by the Investigator in consultation with the Study Medical Monitor.
Definition of Major Bleeding Events (Schulman et al. 2005):

- Fatal bleeding, and/or
- Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarterial or pericardial, or intramuscular with compartment syndrome, and/or
- Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more within 24 hours, or leading to transfusion of two or more units of whole or red cells

Definition of Clinically Relevant, Non-Major Bleeding Events (Schulman et al. 2005):

- 1. Multiple-source bleeding
- 2. Spontaneous hematoma  $> 25 \text{ cm}^2$
- 3. Excessive wound hematoma (not injection site related)
- 4. Macroscopic hematuria (spontaneous or lasting > 24 hours if associated with an intervention)
- 5. Spontaneous rectal bleeding; epitasis, gingival bleeding, hemoptysis, hematemesis
- 6. Bleeding after venipuncture for > 5 minutes

#### 8.7 Adjustment of Dose Frequency

Dose adjustments, including dose interruptions, and/or decreasing the dose frequency will be allowed for safety and tolerability. Any proposed adjustment to treatment schedule must be discussed with, and approved by, the Study Medical Monitor prior to initiation. Up to two adjustments in the treatment schedule may be allowed for patients that are unable to tolerate the once weekly dose (for example if platelet counts fall below 50,000/mm<sup>3</sup> as described in Section 8.6.3). If the patient remains stable after adjustment, they may be cautiously returned to the original once weekly regimen after consultation with the Study Medical Monitor.

Patients may be dose paused in response to AEs after consultation with Study Medical Monitor.

#### **8.8** Discontinuation of Study Treatment

A patient must permanently discontinue study treatment for any of the following:

- The patient becomes pregnant. Report the pregnancy according to instructions in Section 9.5.4
- The patient withdraws consent
- The patient experiences an AE that necessitates permanent discontinuation of study treatment
- The patient develops laboratory test abnormalities that meet any of the stopping rules listed in Section 8.6

The reason for discontinuation of study treatment must be recorded in the CRF and source documentation.

#### 8.8.1 Follow-up Visits for Early Termination from Treatment Period

Any patient who discontinues early from the Treatment Period should be strongly encouraged to attend applicable landmark visits at Weeks 12, 13, 25, 26, and 51, 52 (calculated based on the time elapsed since Day 1) to collect fasting lipid panels and conduct safety assessments in accordance with the schedule of procedures in Appendix A. Any patient who discontinues treatment after Week 44 should also be strongly encouraged to attend a final follow-up visit (Week 65 visit assessments) approximately 13 weeks after their last dose of Study Drug, in addition to the applicable landmark visits.

If the patient declines or is unable to participate in the above, an early termination (ET) visit (Week 52 visit assessments) should be performed at the time of withdrawal, at a minimum, and ideally within 2 weeks from the last dose of Study Drug.

#### 8.8.2 Follow-up Visits for Early Termination from Post-Treatment Follow-up Period

The patient who requests to withdraw from the study during the Post-Treatment Follow-up Period should be encouraged to undergo a final follow-up visit (Week 65, see Appendix A) prior to leaving the study.

If a patient withdraws due to an AE at any time during the study, the Investigator should arrange for the patient to have appropriate follow-up until the AE has resolved or stabilized.

#### 8.9 Withdrawal of Patients from the Study

Patients must be withdrawn from the study for any of the following:

- Withdrawal of consent
- The patient is unwilling or unable to comply with the protocol

Other reasons for withdrawal of patients from the study might include:

- At the discretion of the Investigator for medical reasons
- At the discretion of the Investigator or Sponsor for noncompliance
- Significant protocol deviation

All efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information, including the reason for withdrawal from Study, must be recorded in the CRF.

Any patient who withdraws consent to participate in the study will be removed from further treatment and study observation immediately upon the date of request. These patients should be encouraged to complete the ET study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

For patients withdrawn for reasons other than withdrawal of consent every effort should be made to complete the early termination study procedures and observations at the time of withdrawal (see Section 8.8 and Appendix A).

#### 8.10 Concomitant Therapy and Procedures

The use of concomitant therapies or procedures defined below must be recorded on the patient's CRF. AEs related to administration of these therapies or procedures must also be documented on the appropriate CRF.

#### 8.10.1 Concomitant Therapy

A concomitant therapy is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered between signing informed consent and completion of the post-treatment follow-up period. All concomitant medications/treatments and significant non-drug therapies (including supplements and assistive devices) received by a patient, including changes in the patient's current medications, must be recorded in the patient's source documents and CRF. Patients taking over the counter (OTC) omega-3 fatty acids should make every effort to remain on the same brand throughout the study.

#### **Allowed Concomitant Therapy**

Any medications deemed necessary by the Investigator are allowed except those listed in the disallowed concomitant therapy.

#### **Disallowed Concomitant Therapy**

No lipid lowering therapies (e.g., fibrates, niacin, fish oil or other products containing omega-3 fatty acids [including OTC preparations]), glucacon-like peptide-1 (GLP-1) agonists, Glybera, or systemic corticosteroids may be started or adjusted after baseline qualification. Doses of existing oral anti-diabetic medication, oral contraceptives, hormone replacement therapy, anticoagulants, or drugs or dietary supplements with potential lipid-altering effects should not be adjusted. Study patients are prohibited from receiving other experimental agents during the study. This includes marketed agents at experimental dosages that are being tested for the treatment of hypertriglyceridemia.

Patients should consult with the Site Investigator or designee prior to initiating any new medication, including non-prescription or herbal compounds or any other non-drug therapy.

#### 8.10.2 Concomitant Procedures

A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between signing of informed consent and Week 65 visit.

#### **Disallowed Concomitant Procedure**

Plasma apheresis is not allowed during the study.

#### **8.11** Treatment Compliance

Compliance with treatment dosing is to be monitored and recorded by Study Center staff. The Study Center staff is required to document the receipt, dispensing, and return/destruction of volunesorsen. Patients that are self-administering volunesorsen at home must record treatment in a dosing diary that will be reviewed periodically by Study Center staff and the Clinical Monitor.

#### 9. SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

#### 9.1 Sponsor Review of Safety Information

Safety information will be collected, reviewed, and evaluated by the Sponsor in accordance with the Safety Management Plan throughout the conduct of the clinical trial.

#### 9.2 Regulatory Requirements

The Sponsor is responsible for regulatory submissions and reporting to the Investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonization (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

Institutional Review Boards (IRB)/Independent Ethics Committees (IEC) will be notified of any SAE according to applicable regulations. The Data and Safety Monitoring Board (DSMB) will be notified of any SAE as specified in the DSMB charter.

The Sponsor or designee will evaluate the available information and decide if there is a reasonable possibility that volunesorsen caused the AE and, therefore, meets the definition of a SUSAR.

The following table identifies the SAEs that the Sponsor or designee will not report on an individual basis in an expedited manner because they are anticipated to occur in the study population independent of volunesorsen exposure. The Investigator still has the responsibility to report all SAEs to the Sponsor as described in Sections 9.4.1 to 9.4.3.5.

Table 2 Expected Event for the Protocol Defined Population by Preferred Term and the Expected Incidence

| Preferred Term | Expected Incidence in the Protocol Defined Population (Gaudet et al. 2010 and 2013) |
|---|---|
| Pancreatitis associated events including the PTs of hereditary pancreatitis, pancreatitis, pancreatitis acute, pancreatitis chronic, pancreatitis necrotizing, pancreatitis relapsing | 0.2-0.35 events per patient-year |

Fatal pancreatitis associated events will be considered as unexpected and are reportable. The Sponsor and DSMB will monitor non-fatal pancreatitis associated SAEs using the incidence rate of the event compared to the rate expected in a non-volanesorsen exposed population. If the aggregate analysis indicates that an event is occurring significantly more frequently or at a greater severity than expected, then the event will be reported.

SAEs not specified in the table will be evaluated on case by case basis to determine whether there is a reasonable possibility that the drug caused the event. If the event is considered by the Sponsor or designee to meet the definition of a SUSAR the event will be reported.

#### 9.3 Definitions

#### 9.3.1 Adverse Event

An <u>adverse event</u> is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

#### 9.3.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by volanesorsen.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that volanesorsen drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

#### 9.3.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the Investigator or Sponsor, meets any of the following criteria:

- Results in death
- Is life threatening: that is, poses an immediate risk of death at the time of the event

An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and does not always qualify as an AE
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly or birth defect in the offspring of the patient (whether the patient is male or female)
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

#### 9.4 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a patient prior to the start of the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. The Investigator should always group signs and symptoms into a single term that constitutes a **single unifying diagnosis** if possible.

#### 9.4.1 Serious Adverse Events

In the interest of patient safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to volanesorsen) should be reported to the Sponsor or designee within 24 hours of the Study Center's first knowledge of the event. The collection of SAEs will begin after the patient signs the informed consent form and stop at the end of the patient's follow-up period which is defined as the Week 65 visit. When the Investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An Initial Serious Adverse Event Form should be completed and a copy should be faxed to the Sponsor or designee.

Detailed information should be actively sought and included on Follow-Up Serious Adverse Event Forms as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the patient's last protocol-specified follow-up visit will be evaluated by the Investigator and Sponsor. If the Investigator and Sponsor agree the patient's condition is unlikely to resolve, the Investigator and Sponsor will determine the follow-up requirement.

#### 9.4.2 Non-Serious Adverse Events

The recording of non-serious AEs will begin after the patient signs the informed consent form and will stop at the end of the patient's follow-up period, which is defined as the Week 65 visit. The Investigator will monitor each patient closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 9.4.3 Evaluation of Adverse Events (Serious and Non-Serious)

The Investigator's opinion of the following should be documented on the Adverse Event Case Report Form:

#### 9.4.3.1 Relationship to the Study Drug

The event's relationship to volunesorsen is characterized by one of the following:

- **Related:** There is clear evidence that the event is related to the use of volunesorsen e.g., confirmation by positive re-challenge test
- **Possible:** The event cannot be explained by the patient's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and volanesorsen administration
- Unlikely/Remote: An event for which an alternative explanation is more likely (e.g., concomitant medications or ongoing medical conditions) or the temporal relationship to volanesorsen administration and/or exposure suggests that a causal relationship is unlikely (For reporting purposes, Unlikely/Remote will be grouped together with Not Related)

• **Not Related:** The event can be readily explained by the patient's underlying medical condition, concomitant therapy, or other causes, and therefore, the Investigator believes no relationship exists between the event and volunesorsen

#### *9.4.3.2 Severity*

The severity of AEs and SAEs will be graded based on criteria from the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010 (refer to Appendix D). Any AE not listed in Appendix D will be graded as follows:

- **Mild:** The event is easily tolerated by the patient and does not affect the patient's usual daily activities
- **Moderate:** The event causes the patient more discomfort and interrupts the patient's usual daily activities
- **Severe:** The event is incapacitating and causes considerable interference with the patient's usual daily activities

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 9.3.3).

#### 9.4.3.3 Action Taken with Volanesorsen

Action taken with volunesorsen due to the event is characterized by one of the following:

- None: No changes were made to volunesorsen administration and dose
- Permanently Discontinued: Volanesorsen was discontinued and not restarted
- **Temporarily Interrupted, restarted same dose:** Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose
- Reduced schedule: Dosing frequency was reduced

#### 9.4.3.4 Treatment Given for Adverse Event

Any treatment (e.g., medications or procedures) given for the AE should be recorded on the Adverse Event Case Report Form (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 9.4.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by one of the following:

- AE Persists: Patient terminates from the trial and the AE continues
- Recovered: Patient recovered completely from the AE
- **Became Serious:** The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE)
- Change in Severity (if applicable): AE severity changed

If the event is a SAE then the event's outcome is characterized by one of the following:

- Ongoing: SAE continuing
- Persists (as non-serious AE): Patient has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE)
- **Recovered:** Patient recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date)
- Fatal: Patient died (the date of death should be entered as the SAE resolution date)

#### 9.4.4 Adjudication Committees

All SAEs that occur during the study that are consistent with a major acute cardiovascular event (MACE) will be adjudicated by a blinded, independent committee as outlined in the MACE Adjudication Charter.

All AEs and SAEs that occur during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis (Banks et al. 2013) and as outlined in the Pancreatitis Adjudication Charter. In addition, data for prior episodes of acute pancreatitis or suspected pancreatitis will be collected by review of each patient's medical chart and these events will also be adjudicated.

#### 9.5 Procedures for Handling Special Situations

#### 9.5.1 Abnormalities of Laboratory Tests

Clinically significant abnormal laboratory test results may, in the opinion of the Investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment, e.g., bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia. Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically significant abnormalities will be monitored by the Investigator until the parameter returns to its baseline value or until agreement is reached between the Investigator and Sponsor Medical Monitor. Laboratory abnormalities deemed not clinically significant (NCS) by the Investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the Investigator should not be deemed NCS on the laboratory sheet.

The Investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents and should include the Investigator's assessment of clinical significance of out of range/abnormal laboratory values.

#### 9.5.2 Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the patient is hospitalized; the Study Center must document all of the following:

• The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the patient's consent to participate in the study

Original 28 August 2015

- The condition that required the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the patient's consent to participate in the study and the timing of the procedure or treatment
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission

#### 9.5.3 Dosing Errors

Volanesorsen dosing errors should be documented as Protocol Deviations. A brief description should be provided in the deviation, including whether the patient was symptomatic (list symptoms) or asymptomatic, and the event accidental or intentional.

Dosing details should be captured on the Dosing Case Report Form. If the patient takes a dose of volunesorsen that exceeds protocol specifications and the patient is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 9.4.

**Should an overdose occur**, the Investigator or designee should refer to the Guidance to Investigator's section of the Investigator's Brochure and contact the Sponsor or designee within 24 hours.

#### 9.5.4 Contraception and Pregnancy

Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity, as described in Section 6.3.1.

If a patient becomes pregnant or a pregnancy is suspected, or if a male patient makes or believes that he has made someone pregnant during the study, then the Study Center staff must be informed immediately. An Initial Pregnancy Form should be submitted to the Sponsor or designee **within 24 hours** of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination is reported on Follow-up Pregnancy Forms and reported within 24 hours.

Payment for all aspects of obstetrical care, child or related care will be the patient's responsibility.

<u>Female patients</u>: If a suspected pregnancy occurs while on the study (including follow-up), a pregnancy test will be performed. The patient with a confirmed pregnancy will be immediately withdrawn from treatment with volanesorsen. However, the patient will be encouraged to complete the post-treatment follow-up portion of the study to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the patient in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and

Sponsor may require access to the mother and infant's medical records for an additional 8 weeks after birth.

<u>Male patients</u>: The progress of the pregnancy in a male patient's partner should be followed until the outcome of the pregnancy is known (i.e., delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the Study Center and Sponsor may request access to the mother and infant's medical records for an additional 8 weeks after birth. Follow-up will be performed to the extent permitted by applicable regulations and privacy considerations.

#### 10. STATISTICAL CONSIDERATIONS

#### 10.1 Study Endpoints

For fasting lipid measurements, the values at Month 3 analysis time point are defined as the average of Week 12 (Day 78) and Week 13 (Day 85) fasting assessments, the values of Month 6 analysis time point is at the end of Month 6 are defined as the average of Week 25 (Day 169) and Week 26 (Day 176) fasting assessments, and the values at the Month 12 analysis time point are defined as the average of Week 51 (Day 351) and Week 52 (Day 358) fasting assessments.

#### 10.1.1 Efficacy Endpoints

- Percent change and absolute change from baseline in fasting TG
- Frequency and severity of patient reported abdominal pain during the treatment period
- Percent change and change from baseline in other fasting lipid measurements including total cholesterol, non-HDL-C, apoB, HDL-C, apolipoprotein A-1 [apoA-1], VLDL-C, and LDL-C
- Percent change from baseline in fasting total apolipoprotein C-III
- Quality of Life questionnaires (EQ-5D, SF-36)
- Adjudicated acute pancreatitis event rate

#### 10.1.2 Safety Endpoints

- Adverse events including adjudicated events of pancreatitis and MACE
- Vital signs and weight
- Physical examinations
- Clinical laboratory tests (serum chemistry, hematology, coagulation, urinalysis)
- Echocardiography
- Electrocardiograms (ECGs)
- Use of concomitant medications
- MRIs

#### **10.2** Sample Size

No sample size calculations were performed as this is an extension study to the double-blind, placebo-controlled ISIS 304801-CS6 study. Approximately 50 patients may be eligible to enroll into this study.

#### 10.3 Populations

<u>Full Analysis Set (FAS)</u>: All patients who are enrolled and have a baseline TG assessment. The FAS represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9.

<u>Per Protocol Set (PPS)</u>: Subset of the FAS who received 9 of first 13 scheduled doses of volanesorsen and with no significant protocol deviations that would be expected to affect efficacy and PD assessments. The detailed criteria will be specified and finalized prior to the final database lock.

Safety Set: All patients who are enrolled and receive at least one dose of volanesorsen.

<u>PK Population</u>: All patients who are enrolled, receive at least one dose of volanesorsen, and have at least one evaluable PK sample collected, analyzed, and reported.

#### **10.3** Definition of Baseline

Definitions of baseline are given below for the purposes of the final analysis.

For fasting lipid measurements, two baselines are defined for each patient: index study baseline and the baseline in this open label study, which is defined as the average of Day 1 pre-dose assessment and the last measurement prior to Day 1 (e.g., qualification assessments or assessments from final visit of the index study if used for qualification).

For other measurements, baseline for patients on active treatment in the index study will be the index study baseline. For patients on placebo in the index study, baseline for safety will be the last non-missing assessment prior to the first dose of Study Drug.

#### 10.4 Interim Analysis

An interim analysis may be conducted after the database of index study is locked and unblinded. Both safety and efficacy information from this study may be summarized during this interim analysis. Efficacy analyses will be detailed in the SAP.

#### 10.5 Planned Methods of Analysis

All eCRF data, lab data transfers, as well as any outcomes derived from the data, will be provided in the patient data listings. Patient data listings will be presented for all patients enrolled into the study. Descriptive summary statistics including n, mean, median, standard deviation, standard error, interquartile range (25th percentile, 75th percentile), and range (minimum, maximum) for continuous variables, and counts and percentages for categorical variables will be used to summarize most data by treatment group. Where appropriate, p-values will be reported. All statistical tests will be conducted using 2-sided tests with 5% Type I error rates unless otherwise stated.

All efficacy endpoints will be assessed in the FAS and PPS. All safety assessments will be performed on the Safety Set. PK endpoints will be assessed in the PK Set as applicable.

#### 10.5.1 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized using descriptive statistics by treatment group. The patient disposition will be summarized by treatment group of the index study. All patients enrolled will be included in a summary of patient disposition.

#### 10.5.2 Safety Analysis

Treatment duration and amount of Study Drug received will be summarized by treatment group of the index study.

Patient incidence rates of AEs will be tabulated by MedDRA system organ class, MedDRA preferred term, and treatment group of the index study. Narratives of treatment emergent deaths, serious and significant AEs, including early withdrawals due to AEs, will also be provided.

All treatment emergent AEs, all treatment emergent AEs potentially related to Study Drug, all treatment emergent serious AEs, and all treatment emergent serious AEs potentially related to Study Drug will be summarized.

Injection Site Reactions (ISRs) will be summarized by treatment group of the index study, MedDRA preferred term and severity.

Independently adjudicated events of MACE and pancreatitis will be summarized by treatment group of the index study.

Laboratory tests to ensure patient safety including chemistry panel, complete blood count (CBC) with differential, coagulation panel, IM, complement etc., will be summarized by study visits by treatment group of the index study. These safety variables will also be presented as change and percent change from baseline over time after study drug administration, as appropriate.

Vital signs, weight, ECG measures, echocardiography assessments, and MRI assessments will be tabulated by treatment group of the index study.

#### 10.5.3 Efficacy Analysis

Percent change and change from baseline to Month 3, Month 6, and Month 12 in fasting TG will be summarized by treatment group of the index study. Response rate of patients with fasting plasma TG < 750 mg/dL or achieving fasting  $TG \ge 40\%$  reduction from baseline at Month 3, Month 6, and Month 12 will be summarized. Response analysis will also be conducted using a range of fasting plasma TG thresholds for determination of responder status.

Percent change and change from baseline to Month 3, Month 6, and Month 12 will also be summarized by treatment group of the index study for other fasting lipid measures including non-HDL-C, apoB, HDL-C, apoA-1, VLDL-C, and LDL-C, total cholesterol, and fasting total apoC-III.

The incremental effects of volanesorsen on lipid measures will be explored and the association between changes in lipid parameters and total amount of drug received will be examined, as appropriate.

Frequency and severity of patient reported abdominal pain, adjudicated acute pancreatitis event rate, and quality of life assessments will be summarized by treatment group of the index study.

Additional details of the analyses to be conducted will be provided in the SAP.

#### 10.5.4 Pharmacokinetic and Immunogenicity Analysis

#### 10.5.4.1 Pharmacokinetic Analysis

For all patients, pre-dose and post-treatment volanesorsen plasma concentrations will be summarized using descriptive statistics, with stratification by their prior treatment in Study ISIS 304801-CS6 and IM status.

For patients in the PK subgroup only, non-compartmental PK analysis of volunesorsen will be carried out on each individual patient data set using data collected in the open label extension (OLE) study from the intensive PK subgroup, following a single dose (i.e., single-dose PK) or multiple doses (i.e., steady-state PK), depending on their earlier treatment in the index study. On Week 1 Day 1 of the OLE study, patients who received placebo in the index study will receive the first treatment of volunesorsen (single-dose PK), while patients who received volunesorsen in the index study had been on volanesorsen treatment for twelve months, thus the PK data collected from these patients reflect steady-state PK. The maximum observed drug concentration ( $C_{max}$ ) and the time taken to reach  $C_{max}$  ( $T_{max}$ ) will be obtained directly from the concentration-time data. Area under the plasma concentration-time curve from time zero to 24 hours (AUC<sub>0-24hr</sub>) will be calculated using the linear trapezoidal rule. Apparent systemic (plasma) clearance after SC administration (CL/ $F_{0-24hr}$ ) will be calculated from CL/ $F_{0-24hr}$  = Actual Dose/AUC<sub>0-24hr</sub>. Mean residence time (MRT) from time zero to 24 hours after the SC administration will be calculated from the equation,  $MRT_{0-24hr} = AUMC_{0-24hr}/AUC_{0-24hr}$ , where AUMC<sub>0-24hr</sub> is the area under the moment plasma concentration-time curve from time zero to 24 hours after the SC administration. Other PK parameters, as appropriate, may be determined or calculated at the discretion of the PK scientist.

Plasma PK parameters will be summarized using descriptive statistics, with and without stratification by their prior treatment in Study ISIS 304801-CS6 and IM status. Additional details regarding the PK analysis will be described in the SAP.

Population PK, PK/PD, and covariate analysis may be performed if deemed appropriate, and results will be reported separately.

#### 10.5.4.2 Immunogenicity Analysis

Immunogenicity (IM) results (screen positive/negative, confirmed positive/negative or not evaluable, and when applicable, titer of anti-volanesorsen antibodies) before, during, and after treatment with study drug (volanesorsen) (i.e., sample [anti-drug antibody] ADA status) will be listed by their prior treatment in Study ISIS 304801-CS6 and study day. Subject ADA status (positive/negative or not evaluable) for all evaluable patients, along with the study day associated

with the first positive IM status emerged (T<sub>first</sub>, i.e., onset of ADA development), the last positive IM status observed (T<sub>last</sub>), the duration of ADA response (number of days between T<sub>first</sub> and T<sub>last</sub>) if appropriate, the last ADA sample collection day, and subject maximum titer if applicable, will be listed by their prior treatment in Study ISIS 304801-CS6 and study day. Subjects with positive anti-volanesorsen antibody status may be further classified (when applicable) as being either 'persistent', 'transient', or 'not determinable', if deemed appropriate.

Additionally, the sample and subject IM incidence (number) and incidence rate (percent) will be summarized as the total number and percent of evaluated subjects with antibody negative, positive, and unknown status by their prior treatment in Study ISIS 304801-CS6. Furthermore, onset, duration, and titer of the ADA response, if applicable, will be summarized as median, quartiles (25% and 75%), and range.

Additional details regarding the IM data analysis will be described in the SAP.

Potential relationships between immunogenicity results (e.g., IM status) and selected efficacy (e.g., % change in fasting TG from baseline at 3-, 6-, and 12-month endpoints), safety, and PK (e.g., C<sub>trough</sub>) measures will be evaluated using graphical analysis and statistical analysis. These analyses will be either conducted and included in the study report, or data pooled and analyzed from all available Phase II and III studies and reported separately

#### 11. INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 11.1 Informed Consent

The written informed consent document should be prepared in the language(s) of the potential patient population, based on an English version provided by the Sponsor.

Before a patient's participation in the trial, the Investigator is responsible for obtaining written informed consent from the patient after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study and before any protocol-specific qualification procedures or any Study Drug are administered. The patient must be given sufficient time to consider whether to participate in the study.

The acquisition of informed consent and the patient's agreement or refusal to notify his/her primary care physician should be documented in the patient's medical records and the informed consent form should be signed and personally dated by the patient and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed informed consent form should be retained in the Study Master File and in any other locations required by institutional policy, and a copy of the signed consent form should be provided to the patient.

#### 11.2 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2002 the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

Protocol

Original 28 August 2015

#### 11.3 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent form, other written patient information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent form must be received by the Sponsor before recruitment of patients into the study and shipment of volanesorsen. A copy of the written approval of any other items/materials that must be approved by the Study Center or IEC/IRB must also be received by the Sponsor before recruitment of patients into the study and shipment of Study Drug. The Investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The Investigator must submit to and, where necessary, obtain approval from the IEC/IRB, for all subsequent protocol amendments and changes to the informed consent document. The Investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The Investigator should also notify the IEC/IRB of serious adverse events occurring at the Study Center and other adverse event reports received from the Sponsor, in accordance with local procedures.

The Investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the Investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the Sponsor.

#### 11.4 Patient Confidentiality

The Investigator must ensure that the patient's confidentiality is maintained. On the case report forms (CRF) or other documents submitted to the Sponsor, patients should be identified by unique initials and a patient study number only. Documents that are not for submission to the Sponsor (e.g., signed informed consent forms) should be kept in strict confidence by the Investigator.

In compliance with Federal and local regulations/ICH GCP Guidelines, it is required that the Investigator and institution permit authorized representatives of the company, of the regulatory agency(s), and the IEC/IRB direct access to review the patient's original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The Investigator is obligated to inform and obtain the consent of the patient to permit named representatives to have access to his/her study-related records without violating the confidentiality of the patient.

#### 12. ADMINISTRATIVE AND LEGAL OBLIGATIONS

#### 12.1 Protocol Amendments

Protocol amendments must be made only with the prior approval of the Sponsor. Agreement from the Investigator must be obtained for all protocol amendments and amendments to the informed consent document. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the patients or the conduct of the trial. The Investigator **must** send a copy of the approval letter from the IEC/IRB to the Sponsor.

#### 12.2 Study Termination

The Sponsor reserves the right to terminate the study according to the terms of the site contract. The Investigator reserves the right to terminate their participation in the study, according to the terms of the site contract. The Investigator/Sponsor should notify the IEC/IRB in writing of the trial's completion or early termination and send a copy of the notification to the Sponsor.

#### 12.3 Study Documentation and Storage

An electronic case report form (eCRF) utilizing an Electronic Data Capture (EDC) application will be used for this study.

The Investigator should ensure that all appropriately qualified persons to whom he/she has delegated trial duties are recorded on a Sponsor-approved Delegation of Site Responsibilities Form.

Source documents are original documents, data, and records from which the patient's CRF data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. In this study, CRFs may not be used as source documents.

The Investigator and Study Center staffs are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the Sponsor and/or applicable regulatory authorities. Elements should include:

- Patient files containing completed CRFs, informed consents, and supporting copies of source documentation
- Study files containing the protocol with all amendments, Investigator's Brochure, copies
  of pre-study documentation and all correspondence to and from the IEC/IRB and the
  Sponsor
- If volanesorsen supplies are maintained at the Study Center, proof of receipt, volanesorsen Accountability Record, Return of volanesorsen for Destruction, final study volanesorsen reconciliation, and all volanesorsen-related correspondence

In addition, all original source documents supporting entries in the CRFs must be maintained and be readily available.

No study document should be destroyed without prior written agreement between the Sponsor or and the Investigator. Should the Investigator wish to assign the study records to another party or move them to another location, he/she must notify the Sponsor.

#### 12.4 Study Monitoring

The Sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the Investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the trial (e.g., CRFs and other pertinent data) provided that patient confidentiality is respected.

The Sponsor monitor is responsible for inspecting the CRFs at regular intervals throughout the study to verify adherence to the protocol; completeness, accuracy, and consistency of the data; and adherence to local regulations on the conduct of clinical research. The monitor should have access to patient medical records and other study-related records needed to verify the entries on the CRFs.

The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits, including delays in completing CRFs, are resolved.

In accordance with ICH GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from the Sponsor's Clinical Quality Assurance Department. Inspection of Study Center facilities (e.g., pharmacy, drug storage areas, laboratories) and review of study-related records will occur to evaluate the trial conduct and compliance with the protocol, ICH GCP, and applicable regulatory requirements.

To ensure the quality of clinical data a clinical data management review will be performed on patient data received by the Sponsor. During this review, patient data will be checked for consistency, omissions, and any apparent discrepancies. In addition, the data will be reviewed for adherence to the protocol and GCP. To resolve any questions arising from the clinical data management review process, data queries and/or Study Center notifications will be sent to the Study Center for completion and return to Sponsor.

The Principal Investigator will sign and date the indicated places on the CRF. These signatures will indicate that the principal Investigator inspected or reviewed the data on the CRF, the data queries, and the Study Center notifications, and agrees with the content.

#### 12.5 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by patients and investigative staff must use vocabulary and language that are clearly understood.

#### 12.6 Compensation for Injury

The Sponsor maintains appropriate insurance coverage for clinical trials and will follow applicable local compensation laws. Patients will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Compensation for Injury section of the Informed Consent document.

#### 13. REFERENCES

Altmann KH, Fabbrot D, Dean NM, et al. Second generation of antisense oligonucleotides: from nuclease resistance to biological efficacy in animals. Chimia 1996; 50: 168-176.

Atzmon G, Rincon M, Schechter CB, et al. Lipoprotein genotype and conserve pathway for exceptional longevity in humans. PLoS Biol 2006; 4: e113.

Banks P, Bollen T, Dervenis C, et al; and Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis – 2012: revision of the Atlanta classification and definitions by international consensus. Gut 2013; 62: 102-111.

Beigneux AP, Davies BS, Gin P, et al. Glycosylphosphatidylinositol-anchored high-density lipoprotein-binding protein 1 plays a critical role in the lipolytic processing of chylomicrons. Cell Metab 2007 Apr; 5(4): 279-291.

Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: An endocrine society clinical practice guideline. J Clin Endocrinol Metab 2012; 97: 2969-2989.

Breyer ED, Le N-A, Li X, Martinson D, Brown WV. Apolipoprotein C-III displacement of apolipoprotein E from VLDAL: Effect of particle size. J Lipid Res 1999; 40: 1875-1882.

Brown RJ, Lagor WR, Sankaranaravanan S, et al. Impact of combined deficiency of hepatic lipase and endothelial lipase on the metabolism of both high-density lipoproteins and apolipoprotein B-containing lipoproteins. Circ Res 2010; 107: 357-364.

Brunzell JD. Familial lipoprotein lipase deficiency. In Pagon RA, Adam MP, Bird TD, et al. editors. GeneReviews [Internet], Seattle, WA, University of Washington, Seattle; 1999-2011.

Chan DC, Chen MM, Ooi MM, Watts GF. An ABC of apolipoprotein C-III: a clinically useful new cardiovascular risk factor? Int J Clin Pract 2008; 62 (5): 799-809.

Crooke ST and Bennett CF. Progress in antisense oligonucleotide therapeutics. Ann Rev. Pharmacol Toxicol 1996; 36: 107-129.

Doolittle MH, Neher SB, Ben-Zeev O, et al. Lipase maturation factor 1 (LMF1): Membrane topology and interaction with lipase proteins in the endoplasmic reticulum. J of Biological Chemistry 2009; 1-19.

Gaudet D, de Wal J, Tremblay K, et al. Review of the clinical development of alipogene tiparvovec gene therapy for lipoprotein lipase deficiency. Atherosclerosis Suppl 2010; 11: 55-56.

Gaudet D, Méthot T, Déry S, et al. Efficacy and long-term safety of alipogene tiparvovec (AAV1-LPLS447X) gene therapy for lipoprotein lipase deficiency: An open-label trial. Gene Therapy 2013; 20: 361-369.

Gaudet D, Brisson, D Tremblay K, et al. Targeting APOC3 in the Familial Chylomicronemia Syndrome. N Engl J Med 371; 23 Dec, 2014; 2200-2206.

Gaudet D, Alexander V, Baker BF, et al. Antisense Inhibition of Apolipoprotein C-III in Patients with Hypertriglyceridemia N Engl J Med 2015; 373(5): 438-447.

Geary RS, Yu RZ, Watanabe T, et al. Pharmacokinetics of a tumor necrosis factor-alpha phosphorothiate 2'-O-(2-methoxyethyl) modified antisense oligonucleotide: comparison across species. Drug Metab Dispos 2003; 31: 1419-1428.

Graham MJ, Lee RG, Bell TA, et al. Antisense oligonucleotide inhibition of apolipoprotein C-III reduces plasma triglycerides in rodents, nonhuman primates, and humans. Circ Res 2013 May 24; 112(11): 1479-1490.

Henry S, Stecker K, Brooks D, Monteith D, Conklin B, Bennett CF. Chemically modified oligonucleotides exhibit decreased immune stimulation in mice. J Pharmacol Exp Ther 2000; 292: 468-479.

Inoue H, Hayase Y, Iwai S, Ohtsuka E. Sequence-dependent hydrolysis of RNA using modified oligonucleotide splints and RNase H. Federation of European Biochemical Societies 1987; 215: 327-330.

Ito Y, Azrolan N, O'Connell A, Walsh A, Breslow JL. Hypertriglyceridemia as a result of human apo CIII gene expression in transgenic mice. Science 1990 Aug 17; 249: 790-793.

Kinnunen PK and Ehnolm C. Effect of serum and C-apoproteins from very low density lipoproteins on human postheparin plasma hepatic lipase. FEBS Lett 1976; 65: 354–357.

Lemieux I, Salomon H, Després JP. Contribution of apo CIII reduction to the greater effect of 12-week micronized fenofibrate than atorvastatin therapy on triglyceride levels and LDL size in dyslipidemic patients. Ann Med 2003; 35: 442-448.

Mann CJ, Troussard AA, Yen FT, et al. Inhibitory effects of specific apolipoprotein C-III isoforms on the binding of triglyceride-rich lipoproteins to the lipolysis-stimulated receptor. J Biol Chem 1997; 272: 31348-31354.

McKay RA, Miraglia LJ, Cummins LL, Owens SR, Samor H, Dean NM. Characterization of a potent and specific class of antisense oligonucleotide inhibitor of human protein kinase C-alpha expression. J Biol Chem 1999; 274: 1715-1722.

Mendivil CO, Zheng C, Furtado J, Lel J, Sacks FM. Metabolism of very-low-density lipoprotein and low-density lipoprotein containing apolipoprotein C-III and not other small apolipoproteins. Arterioscler Thromb Vasc Biol 2010; 30: 239-245.

Monia BP, Lesnik EA, Gonzalez C, et al. Evaluation of 2'-modified oligonucleotides containing 2'-deoxy gaps as antisense inhibitors of gene expression. J Biol Chem 1993; 268: 14514-14522.

Ooi EMM, Barrett PHR, Chan DC, Watts GF. Apolipoprotein C-III: Understanding an emerging cardiovascular risk factor. Clin Sci (Lond) 2008; 114: 611-624.

Petersen KF, Dufour S, Hariri A, et al. Apolipoprotein C3 gene variants in nonalcoholic fatty liver disease. N Engl J Med 2010; 362: 1082-1089.

Pollin TI, Damcott CM, Shen H, et al. A null mutation in human APOC3 confers a favorable plasma lipid profile and apparent cardioprotection. Science 2008; 322: 1702-1705.

Santos RD, Duell PB, East C, et al. Long-term efficacy and safety of mipomersen in patients with familial hypercholesterolaemia: 2-year interim results of an open-label extension. Eur Heart J 2015 Mar; 36(9): 566-575. ePub 2013 Dec 23: doi: 10.1093/eurheartj/eht549.

Schaap FG, Resen PCN, Voshol, et al. ApoAV reduces plasma triglycerides by inhibiting very low density lipoprotein-triglyceride (VLDL-TG) production and stimulating lipoprotein lipase-mediated VLDL-TG hydrolysis. J Biol Chem 2004; 279: 27941-27947.

Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medical products in non-surgical patients. J Thromb Haemost 2005; 3(4): 692-694.

Schuster KB, Wilfert W, Evans D, Thiery J, Teupser D. Identification of mutations in the lipoprotein lipase (LPL) and apolipoprotein C-II (APOC2) genes using denaturing high performance liquid chromatography (DHPLC). Clinica Chimia Acta 2011; 412: 240-244.

Surendran RP, Visser ME, Heemelaar S, et al. Mutations in LPL, APOC2, APOA5, GPIHBP1 and LMF1 in patients with severe hypertriglyceridaemia. J Internal Med 2012; 272: 185-196.

Tremblay K, Méthot J, Brisson D, Gaudet D. Etiology and risk of lactescent plasma and severe hypertriglyceridemia. J Clin Lipidol 2011; 5: 37-44.

Yang F, Wang Y, Sternfeld L, et al. The role of free fatty acids, pancreatic lipase and Ca2+ signalling in injury of isolated acinar cells and pancreatitis model in lipoprotein lipase-deficient mice. Acta Physiologica 2009; 195: 13-28.

Zhang H, Lowenberg EC, Crosby JR, et al. Inhibition of the intrinsic coagulation pathway Factor XI by antisense oligonucleotides: a novel antithrombotic strategy with lowered bleed risk. Blood 2010; 116: 4684-4692.

### 14. APPENDICES

## **Appendix A** Schedule of Procedures

ISIS 304801-CS7

### ${\bf Appendix} \; {\bf A} \quad {\bf Schedule} \; {\bf of} \; {\bf Procedures}$

| | Study Period | Qual <sup>a</sup> | | | | | | | Trea | tment | t Perio | d | | | | | Post Tre | eatment<br>w-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Wk | | Wk | Wk | Mont | th 3 | | Mor | nth 6 | Wk | Wk | Wk | Month 12 | | Wk | Wk |
| | Study Week | -2 to -1 | | l<br>I | 4 | 8 | Wk<br>12 | Wk<br>13 | 19 | Wk<br>25 | Wk<br>26 | 32 | 38 | 44 | Wk<br>51 | Wk 52<br>or ET | 58 | 65 |
| | Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| | Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Inf | ormed Consent | Х | | | | | | | | | | | | | | | | |
| Οι | tpatient Visit | Х | Х | Х | Х | Х | X <sup>g</sup> | Х | | X <sup>g</sup> | Χ | | Χ | | Xg | Х | | Х |
| Ind | clusion/Exclusion Criteria | Х | | | | | | | | | | | | | | | | |
| | al Signs + body weight (+ height on y 1 only) | Х | Х | | Х | Х | | Х | | | Х | | Х | | | Х | | Х |
| Physical Examination | | | Х | | | | | Х | | | Х | | Χ | | | Х | | Х |
| 12 | 12- lead ECG (triplicate) | | | | | | | Х | | | Χ | | Х | | | Х | | Х |
| MF | RI (liver/spleen) | | | | | | | | | | | | | | | Х | | |
| Ec | hocardiography | | | | | | | | | | Х | | | | | Х | | |
| Ur | nalysis <sup>b</sup> | Х | Xe | | Х | Х | | Xe | Xe | | Xe | Xe | Xe | Xe | | X <sup>e</sup> | Xe | X <sup>e</sup> |
| | Chemistry Panel | Х | Х | | Х | Х | | Х | X <sup>g</sup> | | Х | X <sup>g</sup> | Χ | X <sup>g</sup> | | Х | X <sup>g</sup> | Х |
| | CBC with Differential | Х | Х | | Х | Х | | Х | X <sup>g</sup> | | Х | X <sup>g</sup> | Χ | X <sup>g</sup> | | Х | X <sup>g</sup> | Х |
| | Serum Lipid Panel | Х | Χ | | Х | Х | X <sup>g</sup> | Х | | X <sup>g</sup> | Х | | Χ | | X <sup>g</sup> | Х | | Х |
| g) <sup>b</sup> | Coagulation (aPTT, PT, INR) | | | | | Χ | | Χ | | | Χ | | Χ | | | X | | |
| stin | hsCRP, HbA1c, FPG | | Χ | | | | | Χ | | | Χ | | | | | Χ | | Χ |
| (Fasting) <sup>b</sup> | Sedimentation Rate | | Χ | | | | | Χ | | | Χ | | | | | Χ | | Χ |
| Draw | Complement (C5a, Bb) | | Χ | | | | | Χ | | | Χ | | | | | Χ | | Χ |
| ے | Plasma PK - Volanesorsen | | X <sup>h</sup> | Χ | Х | Χ | | Χ | | | Χ | | X | | | Х | | Χ |
| Blood | Anti-Volanesorsen Antibodies | | Χ | | Х | Χ | | Χ | | | Χ | | Χ | | | Х | | Х |
| B | FSH (women only, if applicable) | | | | | | | | | | | | | | | | | |
| | Serum Pregnancy Test <sup>c</sup> | Х | | | | Х | | Χ | | | Х | | Χ | | | Х | | Х |
| | Archived Serum & Plasma<br>Samples <sup>f</sup> | | Х | | | Х | | Х | | | Х | | | | | Х | | Х |

#### Appendix A Schedule of Procedures Continued

| Study Period | Qual <sup>a</sup> | | Treatment Period | | | | | | | | | Post Treatment<br>Follow-up | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | , | \ <i>I</i> I. | \A/I+ | \A/Iz | Mon | th 3 | \A/I. | Moi | nth 6 | \A/I+ | \A/I+ | \A/Is | Мо | nth 12 | \A/I+ | \A/Iz |
| Study Week | -2 to -1 | v | Vk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>13 | 19 | Wk<br>25 | Wk<br>26 | Wk<br>32 | Wk<br>38 | Wk<br>44 | Wk<br>51 | Wk 52<br>or ET | - Wk<br>58 | Wk<br>65 |
| Study Day | -14 to -7 | 1 | 2 | 22 | 50 | 78 | 85 | 127 | 169 | 176 | 218 | 260 | 302 | 351 | 358 | 400 | 449 |
| Visit Window+/- Days | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 7 | 7 |
| Weekly Study Drug: SC Injection | | Χ | | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Х | | |
| Symptom Diary (weekly) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х |
| Food/Drink Diary (quarterly) <sup>i</sup> | | Х | | | | | Х | | | Χ | | | | | Х | | Х |
| Quality of Life Assessment(s) | | Х | | | | | Х | | | Χ | | | | | Х | | Х |
| Diet/Alcohol Counseling <sup>d</sup> | Х | Х | | Х | Χ | | Х | | | Χ | | Χ | | | Х | Х | Х |
| Adverse Events | Х | Х | | Χ | Χ | | Χ | | | Х | | Χ | | | Х | | Х |
| Concomitant Medication | Х | Х | | Х | Χ | | Х | | | Χ | | Х | | | Х | | Х |

- a Qualification procedures performed and the patient continues the symptom diary. Assessments from the Week 52 visit of the index study may be used for qualification purposes
- b Blood samples to be collected after an overnight fast of at least 10 hours. During treatment period urine and blood samples will be collected prior to study drug administration. Does not apply to 24 hour PK blood draw
- c Females of childbearing potential only
- d To reinforce compliance to the diet and alcohol restrictions
- e Expanded urinalysis (see Appendix B)
- f Serum and plasma samples will be collected and stored for follow-up exploration of laboratory findings and/or adverse events (e.g., measurement of cytokine and/or chemokine levels, measurement of additional markers of kidney function, measurement of antibodies, etc.) in this or subsequent clinical studies of volanesorsen
- g To be collected by either a clinical service, or Study Center as arranged by the Study Center personnel
- h Full or abbreviated PK profile (see Appendix C)
- i In addition to diary, patients will be contacted at random times during the study to review their current eating and drinking habits

## **Appendix B** List of Laboratory Analytes

#### Appendix B List of Laboratory Analytes

Based on emerging data from this or future studies, additional tests not listed below may be performed on stored samples to better characterize the profile of volunesorsen or other similar oligonucleotides.

| | <b>Hematology</b> | <u>Urinalysis</u> |
|---|---|---|
| <ul> <li>Sodium</li> <li>Potassium</li> <li>PT (sec)</li> <li>Chloride</li> <li>INR</li> <li>Bicarbonate</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>HDL-C</li> <li>Phosphorus</li> <li>Glucose</li> <li>BUN</li> <li>Creatinine</li> <li>Uric Acid</li> <li>Total bilirubin</li> <li>Indirect (unconjugated) bilirubin</li> <li>ALT</li> <li>AST</li> <li>Alkaline phosphatase</li> </ul> | Red blood cells Hemoglobin Hematocrit MCV, MCH, MCHC Platelets White blood cells WBC Differential (% and absolute) Neutrophils Eosinophils Basophils Lymphocytes Monocytes Pharmacokinetics¹ & Immunogenicity Volanesorsen levels in plasma Anti-volanesorsen antibodies in plasma Other assessments hsCRP Sedimentation Rate C5a, Bb De-lipidated free glycerol | <ul> <li>Urinalysis</li> <li>Color</li> <li>Appearance</li> <li>Specific gravity</li> <li>pH</li> <li>Protein</li> <li>Blood</li> <li>Ketones</li> <li>Urobilinogen</li> <li>Glucose</li> <li>Bilirubin</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Microscopic examination<sup>2</sup></li> </ul> Additional Measures for Expanded Urinalysis <ul> <li>Total protein (quantitative)</li> <li>Microalbumin</li> <li>β2-microglobulin</li> </ul> |

Plasma PK samples may also be used for profiling of drug binding proteins, bioanalytical method validation purposes, stability assessments, metabolite assessments, IM testing (or possibly for purposes of IM assay development and/or validation), or to assess other actions of volanesorsen with plasma constituents

<sup>2</sup> Will be performed on abnormal findings unless otherwise specified

Protocol

#### Appendix C Pharmacokinetic Sampling Schedule

Blood samples for the determination of plasma volanesorsen concentrations will be collected prior to dosing, and at various times throughout the dosing and post-treatment follow-up period as noted in the tables below.

#### PK Sampling Schedule (All Patients except PK Subgroup)

| Week | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Pre-dose | Anytime |

#### PK Sampling Schedule (PK Subgroup only\*)

| Week | Wk<br>1 | Wk<br>1 | Wk<br>4 | Wk<br>8 | Wk<br>13 | Wk<br>26 | Wk<br>38 | Wk<br>52 | Wk<br>65 |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | D1 | D2 | D22 | D50 | D85 | D176 | D260 | D358 | D449 |
| Visit Window<br>+/- Days | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 2 | 7 |
| Time Point | Pre-dose,<br>1, 2, 3, 4,<br>6, 8, and<br>12 hrs<br>post-dose | 24 hrs<br>post-dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Pre-<br>dose | Anytime |

<sup>\*</sup> Patients at selected sites will be asked to participate in the extended 24-hour PK profile beginning on Study Day 1. Participation is optional.

# The following grading recommendations for adverse events relating to lab test abnormalities are based upon the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, June 2010

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| | Hem | atology | |
| aPTT prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage |
| Eosinophils increased <sup>†</sup> | 650 - 1,500 cell/mm <sup>3</sup> | 1,501 - 5,000 cell/mm <sup>3</sup> | >5,000 cell/mm <sup>3</sup> |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 x LLN or ≥50% decrease from baseline |
| Hemoglobin decreased (Anemia) | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L; &lt;80 g/L;<br/>transfusion indicated</td></lln></lln> | Hgb <10.0 - 8.0 g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L; <80 g/L;<br>transfusion indicated |
| Hemoglobin increased | Increase in >0 - 2 g/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 g/dL above<br>ULN or above baseline if baseline<br>is above ULN | Increase in >4 g/dL above ULN or above baseline if baseline is above ULN |
| INR increased | >1 - 1.5 x ULN;<br>>1 - 1.5 times above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN;<br>>1.5 - 2.5 times above baseline if<br>on anticoagulation | >2.5 x ULN;<br>>2.5 times above baseline if on<br>anticoagulation |
| Lymphocyte count decreased | <lln -="" 800="" mm<sup="">3;<br/><lln -="" 0.8="" 10<sup="" x="">9/L</lln></lln> | <800 - 500/mm³;<br><0.8 - 0.5 x 10 <sup>9</sup> /L | <500 /mm³;<br><0.5 x 10 <sup>9</sup> /L |
| Lymphocyte count increased | - | >4000/mm³ - 20,000/mm³ | >20,000/mm <sup>3</sup> |
| Neutrophil count decreased | <lln -="" 1500="" mm<sup="">3;<br/><lln -="" 1.5="" 10<sup="" x="">9 /L</lln></lln> | <1500 - 1000/mm³;<br><1.5 - 1.0 x 10 <sup>9</sup> /L | <1000/mm³;<br><1.0 x 10 <sup>9</sup> /L |
| Platelet count<br>decreased | <lln -="" 75,000="" mm³;<br=""><lln -="" 10<sup="" 75.0="" x="">9 /L</lln></lln> | <75,000 - 50,000/mm³;<br><75.0 - 50.0 x 10 <sup>9</sup> /L | <50,000/mm <sup>3</sup> ;<br><50.0 x 10 <sup>9</sup> /L |
| White blood cell<br>decreased | <lln -="" 3000="" mm<sup="">3;<br/><lln -="" 10<sup="" 3.0="" x="">9 /L</lln></lln> | <3000 - 2000/mm <sup>3</sup> ;<br><3.0 - 2.0 x 10 <sup>9</sup> /L | <2000/mm³;<br><2.0 x 10 <sup>9</sup> /L |
| | Che | mistry | |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 |
| Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Alkalosis | pH >normal, but ≤7.5 | - | pH >7.5 |
| Aspartate aminotransferase >ULN - 3.0 x ULN ncreased | | >3.0 - 5.0 x ULN | >5.0 x ULN |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 x ULN |
| Cardiac troponin I<br>increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |

# Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

Original

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Cardiac troponin T<br>increased | Levels above the upper limit of normal<br>and below the level of myocardial<br>infarction as defined by the<br>manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer |
| CD4 lymphocytes decreased | <lln -="" 500="" mm<sup="">3;<br/><lln -="" 0.5="" 10<sup="" x="">9 /L</lln></lln> | <500 - 200/mm³;<br><0.5 - 0.2 x 10 <sup>9</sup> /L | <200/mm³;<br><0.2 x 10 <sup>9</sup> /L |
| CPK increased* | >ULN - <6 ULN | 6 - 10 x ULN | >10 x ULN |
| Creatinine increased | >1 - 1,5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x baseline;<br>>1.5 - 3.0 x ULN | >3.0 x baseline;<br>>3.0 x ULN |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 x ULN |
| Hypercalcemia | Corrected serum calcium of >ULN -<br>11.5 mg/dL; >ULN - 2.9 mmol/L;<br>lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; lonized calcium >1.6 mmol/L; hospitalization indicated |
| Hyperglycemia | Fasting glucose value >ULN - 160<br>mg/dL; Fasting glucose value >ULN -<br>8.9 mmol/L | Fasting glucose value >160 - 250 mg/dL; Fasting glucose value >8.9 - 13.9 mmol/L | >250 mg/dL; >13.9 mmol/L;<br>hospitalization indicated |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0; hospitalization indicated |
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | - | >3.0 mg/dL;<br>>1.23 mmol/L |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 mmol/L; hospitalization indicated |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic consequences | - | >ULN - 10 mg/dL (0.59<br>mmol/L) with physiologic<br>consequences |
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL;<br/>&lt;30 - 20 g/L</td><td colspan="3">&lt;2 g/dL;<br/>&lt;20 g/L</td></lln></lln> | <3 - 2 g/dL;<br><30 - 20 g/L | <2 g/dL;<br><20 g/L |
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" l;="" l<="" lonized="" mg="" mmol="" td=""><td>Corrected serum calcium of &lt;8.0 -<br/>7.0 mg/dL; &lt;2.0 - 1.75 mmol/L;<br/>lonized calcium &lt;1.0 - 0.9<br/>mmol/L; symptomatic</td><td>Corrected serum calcium of<br/>&lt;7.0 mg/dL; &lt;1.75 mmol/L;<br/>lonized calcium &lt;0.9 mmol/L;<br/>hospitalization indicated</td></lln> | Corrected serum calcium of <8.0 -<br>7.0 mg/dL; <2.0 - 1.75 mmol/L;<br>lonized calcium <1.0 - 0.9<br>mmol/L; symptomatic | Corrected serum calcium of<br><7.0 mg/dL; <1.75 mmol/L;<br>lonized calcium <0.9 mmol/L;<br>hospitalization indicated |
| Hypoglycemia | ypoglycemia <lln -="" 55="" <3.0="" <55="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;40 mg/dL (&lt;2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions<sup>†</sup></td></lln> | | <40 mg/dL (<2.2 mmol/L) AND requires assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions <sup>†</sup> |
| Hypokalemia | <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" symp="" td=""><td>&lt;3.0 mmol/L; hospitalization indicated</td></lln> | | <3.0 mmol/L; hospitalization indicated |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td colspan="3">&lt;0.9 mg/dL;<br/>&lt;0.4 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 mg/dL;<br><0.4 mmol/L |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 mmol/L</td></lln> | - | <130 mmol/L |
| Hypophosphatemia | <lln -="" 2.5="" dl;<br="" mg=""><lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6 mmol/L</td><td colspan="3">&lt;2.0 mg/dL;<br/>&lt;0.6 mmol/L</td></lln></lln> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6 mmol/L | <2.0 mg/dL;<br><0.6 mmol/L |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 x ULN |

#### Appendix D Grading Scale for Adverse Events Relating to Laboratory Abnormalities Continued

| Adverse Event | Mild | Moderate | Severe |
|---|---|---|---|
| Urine | | | |
| Proteinuria<br>Adults | 1+ proteinuria;<br>urinary protein <1.0 g/24 hrs | 2+ proteinuria;<br>urinary protein 1.0 - 3.4 g/24 hrs; | Urinary protein ≥3.5 g/24 hrs; |
| Children | | Urine P/C (Protein/Creatinine)<br>ratio 0.5 - 1.9 | Urine P/C >1.9 |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated |

<sup>&</sup>lt;sup>†</sup>Grading for this parameter is derived from the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, Sept 2007

<sup>\*</sup>Grading for this parameter is derived from the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, Nov 2014

<sup>&</sup>lt;sup>‡</sup>Modified for consistency with the ADA and Endocrine Society Guidelines (Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and Diabetes: A Report of a Workgroup of the American Diabetes Association and The Endocrine Society. Diabetes Care 2013;36:1384-95)